Protocol No: IVACFLU-S-0203 497 Dated: 12 March 2018


Version: 4.0 Dated 09/02/2017

Page i

# MINISTRY OF HEALTH

### RESEARCH PROTOCOL OF VACCINE CLINICAL TRIAL

A PHASE 2 / 3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF A SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

> **Protocol Number:** IVACFLU-S-0203 Vietnam MOH Reference: VX.2016.06

> > **PATH 051**

Version Number: 4.0 Date: 09/02/2017

SUMMARY NAME: SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE CLINICAL TRIAL (IVACFLU-S) – PHASE 2/3

Principal Investigator: Dr. Phan Cong Hung

**Investigator's Institution:** Pasteur Institute, Ho Chi Minh City, Vietnam **Sponsor:** Institute of Vaccines and Medical Biologicals (IVAC), Vietnam

Manufacturer: Institute of Vaccines and Medical Biologicals (IVAC), Vietnam

**Authority Agency:** Ministry of Health, Vietnam **Planned time:** March 2017 to October 2017

Total budget: VND 8.9 billion

In which: from Government budget for Science and Technology VND 0

Other source: funded by PATH VND 8.9 billion

Version 1.0 498

IVACFLU-S, Phase 2/3

Protocol No: IVACFLU-S-0203


Dated: 12 March 2018

Page ii

### STATEMENT OF COMPLIANCE

I am Dr. Phan Cong Hung, principal investigator of the study "A Phase 2/3 Double Blinded, Randomized, Placebo-Controlled Study in Adult Volunteers (age 18-60) in Vietnam to Examine the Safety and Immunogenicity of a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine (IVACFLU-S) Produced by IVAC". By signing below to ensure that the study will be carried out on schedule, content of approved protocol, and in accordance with Good Clinical Practice (GCP) as required by applicable rules of Vietnam: Decision No. 799/2008/QD-BYT, on "Guidance on Good Clinical Practice," Circular No. 03/2012/TT-BYT on "Guidance on Clinical Trial" and Decision No.22/2009/TT-BYT on "Medical Product Registration," Decision 1248/QD BYT on the National Guidelines on ethical issues in biomedical research; Decision 111/QD BYT on the guidelines on organizational and operational principles for IRBs; and Dispatch 6586/BYT-K2DT on the guidelines on recording/reporting SAE in clinical trial.

The study informed consent documents will embody the elements of consent as described in the Declaration of Helsinki, 2013.

All key personnel (those responsible for the design and conduct of this study) will have completed Human Subjects Protection Training prior to interaction with any participants or to have access to their confidential study data.

> Ho Chi Minh City, date 09 month 02 year 2017 Principal Investigator

> > Phan Cong Hung, MD Pasteur Institute in Ho Chi Minh City 167 Pasteur, Ward No 8, District No 3, Ho Chi Minh City, Vietnam

delMu)

Protocol No: IVACFLU-S-0203 499

IVACFLU-S, Phase 2/3


Page iii

# **TABLE OF CONTENTS**

| 1 | Ke | y Roles for Individuals and Institutions Involved | 1 |
|---|---|---|---|
| 2 | Ва | ckground Information and Scientific Rationale | 4 |
| | 2.1 E<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.1.5<br>2.1.6 | Background Information Overview of Influenza disease Seasonal Influenza in Vietnam Treatment and Prevention (vaccine, biological) Summary results of related preclinical trials Results of Clinical Trial Data on Clinical Trials from Seasonal Vaccines Similar to IVACFLU-S Flucelvax – Seqirus, Inc Fluzone® – Sanofi Pasteur Fluarix – GSK | 4<br>5<br>8<br>9<br>15<br>15 |
| | 2.3 F | Rationale of Current Study | 19 |
| | 2.4 | Oose Rationale | 20 |
| | 2.5.1 | Potential Risks and Benefits of Inactivated, split Influenza Vaccine Potential Risks Potential Benefits | 20 |
| 3 | Stı | udy Objectives and Endpoints | <b>21</b> |
| | 3.1 S<br>3.1.1<br>3.1.2<br>3.1.3 | Primary Objectives, Phase 2 Primary Objectives, Phase 3 Secondary Objective, Phase 3 | 21<br>21 |
| | 3.2 S<br>3.2.1<br>3.2.2 | Study Outcome Measures (Endpoints) | 21 |
| 4 | Stu | udy Design | 23 |
| | 4.1 8 | Study Design | 23 |
| | 4.2 C | Design Rational | <b>26</b> |
| | 4.3 | Study sites | 26 |
| 5 | Stı | udy Enrollment and Withdrawal | 27 |
| | 5.1 C | Description of Participants, Source of Participants | 27 |
| | 5.2 F | Participant Inclusion Criteria | 28 |

IVACFLU-S, Phase 2/3

IVACFLU-S Version 1.0

500 Protocol No: IVACFLU-S-0203


Dated: 12 March 2018

# Page iv

| | 5.3 | Participant Exclusion Criteria | 28 |
|---|---|---|---|
| | 5.4<br>5.4.1 | Treatment Assignment Procedures | |
| | 5.4.2 | Blinding and Unblinding Procedures | 30 |
| | 5.4.3 | Reasons for Withdrawal | 30 |
| | 5.4.4 | | |
| | 5.4.5 | Strategies to Maintain and Recruit Additional Participants | 30 |
| 6 | To | ermination of the Trial | 31 |
| | 6.1 | Termination According to the Protocol | 31 |
| | 6.2 | Suspension and/or Premature Termination of the Trial | 31 |
| 7 | S | tudy Products | 31 |
| | 7.1 | Study Product Descriptions | 31 |
| | 7.1.1 | Acquisition | 31 |
| | 7.1.2 | Promulation, Packaging and Labeling (Seasonal influenza vaccine, IVACFLU-S) | 32 |
| | 7.1.3 | | |
| | 7.1.4 | Lot number, Expiry date, Quality control results of study vaccine lots | 34 |
| | 7.2 | Dosage, Preparation and Administration of Study Products | 35 |
| | 7.2.1 | | |
| | 7.2.2 | | |
| | 7.2.3 | _ | |
| | 7.3 | Modification of Study Product for a Participant | 36 |
| | 7.4 | Accountability Procedures for Study Product | 36 |
| | 7.5 | Assessment of Compliance with Use of the Study Products | 37 |
| | 7.6 | Concomitant Medications/Treatment | 37 |
| | 7.7 | Unauthorized Products | 37 |
| 8 | S | tudy Schedule; Description of Visits | 38 |
| | 8.1 | Screening | 38 |
| | 8.1.1 | • | |
| | 8.2 | Follow-up Periods | 40 |
| | 8.2.1 | • | |
| | 8.2.2 | | |
| | 8.2.3 | | |
| | 8.2.4 | | |
| | 8.2.5 | | |
| | 8.3 | Early Termination Visit | 42 |

IVACFLU-S, Phase 2/3


Dated: 12 March 2018

# Page v

| 8.4 | Unscheduled Visits | . 42 |
|---|---|---|
| 9 8 | Study Evaluations | 42 |
| 9.1<br>9.1.<br>9.1.<br>9.1. | Medical History | 42<br>42<br>43 |
| 9.2<br>9.2.<br>9.2.<br>9.2. | 2 Special Assays | 44<br>44 |
| 10 A | Assessment of Safety and Adverse Events | 46 |
| 10.1<br>10.1<br>10.1 | I.1 Solicited Local and Systemic Adverse Events | 46 |
| 10.2 | Serious Adverse Events | . 47 |
| 10.3 | AE/SAE Reporting Period and Parameter | . 48 |
| 10.4 | Severity of Event | . 48 |
| 10.5 | Relationship to Study Vaccines | . 49 |
| 10.6 | Follow up of AE | . 50 |
| 10.7 | General Guidelines for Recording AEs | . 50 |
| 10.8 | Unexpected Allergic Reaction | . 51 |
| 10.9<br>10.9<br>10.9<br>10.9<br>10.9 | 9.2 Reporting of AEs | 51<br>52 |
| 11 S | Safety Oversight | 52 |
| 11.1<br>11.1<br>11.1 | I.2 Study Safety Pauses | 53<br>53 |
| 11.2 | Data Safety Monitoring Board | |
| | Monitoring and Auditing | |
| 12.1 | Monitoring Plan | . 53 |


IVACFLU-S, Phase 2/3


# Page vi

502

| 12.2 | Set-up Visit (Site Initiation) | . 54 |
|---------|-----------------------------------------------|------|
| 12.3 | Routine Monitoring Visits | . 54 |
| 12.4 | Close-out Visit | . 55 |
| 12.5 | Audits and Inspections | . 55 |
| 13 S | Statistical Considerations | 55 |
| 13.1 | Study Hypothesis | . 55 |
| 13.2 | Sample Size Considerations | . 56 |
| 13.3 | Safety | . 56 |
| 13.4 | Immunogenicity | . 57 |
| 13.4 | , | |
| 13.4 | | |
| 13.5 | Data Analysis | |
| 13.6 | Definition of Analysis Sets | |
| 13.7 | Analysis of Safety Endpoints | |
| 13.8 | Analysis of Immunogenicity Endpoints | . 60 |
| 13.9 In | terim Analysis | 61 |
| 14 [ | Data Management | 62 |
| 14.1 | Case Report Form (CRF) | . 62 |
| 14.2 | Source Documents and Source Document Access | . 63 |
| 14.3 | Database Management and Analysis Software | . 63 |
| 14.4 | Entering, Cleaning and Management of Database | . 63 |
| 14.5 | Source Data Verification | . 63 |
| 14.6 | Database Locking Procedures | . 64 |
| 14.7 | Study Record Retention | . 64 |
| 15 ( | Quality Control and Quality Assurance | 64 |
| 15.1 | General Considerations | . 64 |
| 15.2 | Trainings | . 64 |
| 16 E | thics/Protection of Human Subjects | 65 |
| 16.1 | Ethical Standard | . 65 |

IVACFLU-S Protocol No: IVACFLU-S-0203 Version 1.0 503 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page vii

| 16.2 Financing and Insurance | 65 |
|---|---|
| 16.3 Assurance of Emergency Medical Care and Care for other Adverse Events | 65 |
| 16.4 Institutional Review Boards and Independent Ethics Committee | 66 |
| 16.5 Media Planning for Participant and Community Engagement | 66 |
| 16.6 Informed Consent Process | 67 |
| 16.7 Inclusion of Women, Minorities, and Children | 68 |
| 16.8 Participant Confidentiality: | 69 |
| 16.8.1 Confidentiality of Data | |
| 16.8.2 Confidentiality of Participant Records | 69 |
| 16.9 Sharing of Study Results | 70 |
| 16.9.1 Sharing of Study Results with the Participant | |
| 16.9.2 Incidental Health Findings | |
| 16.9.3 Sharing of Study Results with the Community | |
| 16.10 Study Discontinuation | 70 |
| 16.11 Future Use of Stored Specimens | 70 |
| 16.12 Potential Risks and How They are Addressed | 71 |
| 16.13 Benefits to Study Participants | 72 |
| 17 Noncompliance and Unanticipated Problems | 72 |
| 18 Human Resource for the Study | <b>7</b> 3 |
| 18.1 Human Resource for the Study | <b>7</b> 3 |
| 18.2 Training Plan | <b>7</b> 3 |
| 19 Clinical Study Report and Publication Policy | <b>7</b> 3 |
| 19.1 Clinical Study Report | |
| 19.2 Publication Policy | 74 |
| APPENDIX A: Table of Grading Severity | |
| APPENDIX B: Roles and responsibilities matrix | |
| APPENDIX C: Template of interim study report of the phase 2/3 | |
| APPENDIX D: Assessment of Understanding | |
| APPENDIX E: Quality Certification by NICBV for study product lots | 90 |

Protocol No: IVACFLU-S-0203 504 Dated: 12 March 2018

Dated 09/02/2017

Page viii

### LIST OF ABBREVIATIONS

AE Adverse Event

BARDA Biomedical Advanced Research and Development Authority

CI Confidence Interval

cm Centimeter

CRF Case Report Form

°C Degrees Celsius

D Day

DSMB Data and Safety Monitoring Board

EIA Enzyme Immunoassay

GCP Good Clinical Practice

GMFRs Geometric Mean Fold Rises

GMT Geometric Mean Titer

HA Hemagglutinin

HAI Hemagglutination Inhibition

hCG Human Chorionic Gonadotropin

ICF Informed Consent Form

ICH International Conference on Harmonization

ICMJE International Committee of Medical Journal Editors

IEC Independent Ethics Committee

IP Investigational Product

IRB Institutional Review Board

IVAC Institute of Vaccines and Medical Biologicals

L Liter

MDCK Madin-Darby Canine Kidney

Mcg Microgram

Protocol No: IVACFLU-S-0203 505 Dated: 12 March 2018

Dated 09/02/2017

Page ix

mL Milliliter

Mm Millimeter

MNT Microneutralization test

MOH Ministry of Health

N number (typically refers to number of participants)

NA Neuraminidase

PI Principal Investigator

PBS Phosphate buffered saline

PSRT Protocol Safety Review Team

RBC Red Blood Cell

SAE Serious Adverse Event

SOP Standard Operating Procedure

SRID Single Radiation Immunodiffusion

TBD To Be Designated

TCID Tissue Culture Infectious Dose

US United States

WHO World Health Organization

Protocol No: IVACFLU-S-0203 506 Dated: 12 March 2018


Page x

# **PROTOCOL SUMMARY**

| Title: | A Phase 2/3 Double Blinded, Randomized, Placebo- |
|---|---|
| | Controlled Study in Healthy Adult Volunteers in Vietnam to |
| | Examine the Safety and Immunogenicity of a Seasonal |
| | Trivalent Inactivated Split Virion Influenza Vaccine (IVACFLU-S) produced by IVAC |
| | This is a phase 2/3, double-blind, placebo-controlled trial of |
| Description of Study | 888 adults, ages 18 to 60 years old randomized to receive |
| Description of Study Design: | vaccine or placebo according to schema below. Phase 2 will |
| | be conducted at 1 site of Long An (252 subjects). Following |
| | a determination of safety of vaccine in phase 2 study by Protocol Safety Review Team (PSRT) review and with |
| | approval from Vietnam Ministry of Health (MOH), Phase 3 |
| | enrollment will commence at 2 sites, Long An (252 subjects, |
| | including 210 vaccine recipients and 42 placebo recipients) |
| | and Dong Nai (384 subjects, including 320 vaccine recipients |
| | and 64 placebo recipients). |
| | Safety will be assessed in all Phase 2 and 3 participants |
| | through Day 91. Safety data till Day 8 post-vaccination from |
| | the phase 2 study will be presented to Protocol Safety Review Team (PSRT) for evaluation and an interim report will be filed |
| | with local institutional review board (IRB) and MOH. |
| | Immunogenicity will be assessed only in Phase 3 |
| | participants. Blood samples will be collected in a subset of |
| | 252 individuals (210 vaccine recipients and 42 placebo recipients) randomized at one of the study sites to get |
| | evaluable samples from at least 200 vaccine recipients (100 |
| | each from both age groups) and 40 placebo recipients (20 |
| | each from both age groups) 21 days after vaccination. |
| | Approximate participant distribution based on age, study arm |
| | and study will be as follows: |

Protocol No: IVACFLU-S-0203 507 Dated: 12 March 2018


Page xi

| Age<br>group | IVACFLU-S | Placebo | Total |
|---|---|---|---|
| | Phase | 2 | |
| 18 - 45 | 105 | 21 | 126 |
| 46 - 60 | 105 | 21 | 126 |
| | Phase | Phase 3 | |
| 18 - 45 | 265 | 53 | 318 |
| 46 - 60 | 265 | 53 | 318 |
| | group 18 - 45 46 - 60 18 - 45 | Phase 18 - 45 | group IVACELU-S Placebo Phase 2 18 - 45 105 21 46 - 60 105 21 Phase 3 265 53 |

# Safety:

A single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) will be safe and well tolerated in adults 18 to 60 years of age.

# Immunogenicity:

A single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) will induce immune responses to each of the three vaccine antigens to meet one or both age group specific Vietnam Ministry of Health (MOH) licensure requirements.

| Criteria | 18 – 45 year<br>old | 46 – 60 year<br>old |
|----------------------------|---------------------|---------------------|
| Seroprotection (HAI ≥1:40) | ≥70% | ≥60% |
| Seroconversion | ≥40% | ≥30% |
| HAI GMT increase | ≥2.5 times | ≥2.0 times |

Protocol No: IVACFLU-S-0203 508 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page xii

| Study Objectives, Phase 2: | Primary |
|---|---|
| olddy Objectives, i nase 2. | Safety: To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults, 18 to 60 years of age. |
| Study Objectives, Phase 3: | Primary |
| | <b>Safety:</b> To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults, 18 to 60 years of age. |
| | Immunogenicity: To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single intramuscular dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults, 18 to 45 and 46 to 60 years of age. |
| | Secondary |
| | To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults with and without pre-existing Hemaglutination Inhibition (HAI) antibody |
| Study Endpoints: | Primary Safety Endpoints, Phase 2 and 3 |
| | The number and proportion of participants reporting the following events: |
| | A. Solicited local adverse events, including redness / erythema, swelling / induration, pain within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination. |
| | B. Solicited systemic adverse events, including fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting and headache within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination. |

Protocol No: IVACFLU-S-0203 509 Dated: 12 March 2018

Dated 09/02/2017

Page xiii

- C. Unsolicited Adverse Events (AEs) occurring within 21 days post vaccination.
- D. Serious Adverse Events (SAE) occurring during the entire study period (Days 1-91).

# **Primary Immunogenicity Endpoint, Phase 3**

- A. Number and percentage of participants by age groups (18-45, 46-60) with seroconversion against each of the 3 vaccine antigens post-vaccination. Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
- Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or
- Pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 22
- B. Number and percentage of participants by age groups (18-45, 46-60) with a HAI antibody titer ≥1:40 to each of the 3 vaccine antigens measured on Day 22 post vaccination
- C. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens
- D. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/pre-vaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens

### Secondary Immunogenicity Endpoints, Phase 3

- A. Number and percentage of participants by age groups (18-45, 46-60) who develop at least a four-fold increase in HAI antibody titer to each of the vaccine antigen post vaccination measured on Day 22 by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.
- B. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups

Protocol No: IVACFLU-S-0203 510 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page xiv

(18-45, 46-60) for each of the 3 vaccine antigens by prevaccination HAI antibody titer of <1:10 or ≥1:10.

C. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/pre-vaccination) by age groups (18-45, 46-60) for each of the 3 vaccine by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.

### **Participant Eligibility**

### Inclusion criteria

All participants must meet all of the following criteria to be considered eligible to participate in the study:

- Aged 18 through 60 years on the day of screening/enrollment.
- Literate (by self-report) and willing to provide written informed consent.
- Able to attend all scheduled visits and to comply with all trial procedures.
- Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable under controlled or unchanged for the past 3 months. If medication is used to treat the condition, the medication dose must have been stable for at least 1 month preceding vaccination.

### For females participants:

 Not breastfeeding or pregnant (based on negative urine pregnancy test) or plan to become pregnant up to Day 22.
 Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than 1 year must have negative pregnancy test and, be willing to utilize reliable birth control measures (intrauterine device, hormonal contraception, condom or diaphragm with spermicide) through the Day 22 visit.

### **Exclusion Criteria**

Participants meeting any of the following criteria will be excluded from participation:

- Current or recent (within two weeks of enrollment) acute severe illness with or without fever.
- Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.

Protocol No: IVACFLU-S-0203 511 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page xv

- Receipt of any non-study vaccine within 4 weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 22 visit.
- Received seasonal influenza vaccine in last 6 months Receipt of immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 22 visit.
- Known or suspected congenital or acquired immunodeficiency.
- Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressant or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, ≥ 0.5 mg per kg per day; topical steroids are allowed.)
- Unstable illness by history or physical examination that in the opinion of the investigator, might interfere with the conduct or results of the study or pose additional risk to the participant.
- Hypersensitivity after previous administration of any vaccine.
- Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein, and rubber (from the vaccine vial stoppers).
- Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion.
- Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
- Current alcohol or drug addiction that in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
- History of Guillain-Barré Syndrome
- Neoplastic disease or any hematologic malignancy.
- Any condition that, in the opinion of the investigator, would increase the health risk to the participant if he/she

Protocol No: IVACFLU-S-0203 512 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page xvi

| Statistical Consideration The sample size for this study was selected for primary safet and immunogenicity analysis to satisfy the MOH licensur requirement for influenza vaccine in adults from age 1sthrough 60. Total sample size for the Phase 2 is approximately 252 participants (to have at least 20 randomized to vaccine and 40 randomized to placebo at the end of the study). Phase 3 sample size is approximately 63 participants (to have at least 500 randomized to vaccine and 100 randomized to placebo at the end of the study). So a least 700 evaluable participants will be randomized to IVACFLU-S arm in the phase 2/3 study. There are two type of immunogenicity measurements against each of the vaccine antigens, percentages of subjects with immunices ponse and Geometric Mean Titers (GMT) that will be used to evaluate this study objective. For each percentage subjects with the defined immune responses, the percentage and its corresponding 2-sided exact (Clopper-Pearson binomial 95% confidence interval (95% CI) around the percentage will be computed for each treatment group and by age group. GMT along with the corresponding two-side 95% CIs, by exponentiating the corresponding log transformed means and their 95% CIs, will be summarize by treatment group on Day1 and Day 22. The same approact will be used to summarize GMFR of Day 22/Day1 separated by treatment group and age group. For the solicited local and systemic/general adverse events, Fisher's exact test for two proportions or the Cochran-Mantel-Haenszel test for severiting grade categories at 2-sided 0.05 alpha will be used to compare the treatment groups. No formal hypothesis testing with multiplicity adjustment will be performed. Furthermore no statistical testing will be performed for unsolicited AE including SAEs. | | participates in the study, or would interfere with the evaluation of the study objectives. |
|---|---|---|
| Study Population: Approximately 888 male and female adults, 18 to 60 years of | Statistical Consideration | The sample size for this study was selected for primary safety and immunogenicity analysis to satisfy the MOH licensure requirement for influenza vaccine in adults from age 18 through 60. Total sample size for the Phase 2 is approximately 252 participants (to have at least 200 randomized to vaccine and 40 randomized to placebo at the end of the study). Phase 3 sample size is approximately 636 participants (to have at least 500 randomized to vaccine and 100 randomized to placebo at the end of the study). So at least 700 evaluable participants will be randomized to IVACFLU-S arm in the phase 2/3 study. There are two types of immunogenicity measurements against each of the 3 vaccine antigens, percentages of subjects with immune response and Geometric Mean Titers (GMT) that will be used to evaluate this study objective. For each percentage of subjects with the defined immune responses, the percentage and its corresponding 2-sided exact (Clopper-Pearson) binomial 95% confidence interval (95% CI) around the percentage will be computed for each treatment group and by age group. GMT along with the corresponding two-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs, will be summarized by treatment group on Day1 and Day 22. The same approach will be used to summarize GMFR of Day 22/Day1 separately by treatment group and age group. For the solicited local and systemic/general adverse events, Fisher's exact test for two proportions or the Cochran-Mantel-Haenszel test for severity grade categories at 2-sided 0.05 alpha will be used to compare the treatment groups. No formal hypothesis testing with multiplicity adjustment will be performed. Furthermore, no statistical testing will be performed for unsolicited AEs |
| age at the time of enrollment | Study Population: | Approximately 888 male and female adults, 18 to 60 years of age at the time of enrollment |
| <b>Phase:</b> 2/3 | Phase: | 2/3 |
| | Number of Sites: | Study is multicenter with Phase 2 conducted at 1 site of Long<br>An and Phase 3 conducted at 2 sites, Long An and Dong Nai: |

Protocol No: IVACFLU-S-0203 513 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 CONFIDENTIAL Version: 4.0 Dated 09/02/2017

Page xvii

| Study Duration: | The total duration for this study is approximately 22 months; with approximately 12 months (Sep 2016 to Sep 2017) for preparation and implementation of both phases of the study; and approximately 10 months for data analysis, CSR completion and review, approval by local IRBs and Ministry of Health. |
|---|---|
| Participation Duration: | Approximately 3 months |
| Description of Agent or Intervention: | Seasonal trivalent inactivated influenza vaccine (TIV), inactivated split virion, purified by sucrose gradient ultracentrifugation (IVAC, NhaTrang, Vietnam), or placebo (IVAC, Nha Trang, Vietnam). The vaccine will be produced in embryonated chicken eggs, and inactivated with formaldehyde. The dose of the vaccine to be tested is 15 mcg of each of the three components per 0.5 mL. The vaccine strains are |
| | NYMC BX-35 reassortant of B/Brisbane/60/2008 (B) |
| | NYMC X-179A reassortant of A/California/7/2009 (H1N1) |
| | NYMC X-263B reassortant of H3/A/Hong<br>Kong/4801/2014 (H3N2) |
| | Placebo is PBS with pH 7.2; 0.5 ml/per dose |
| Estimated Time to Complete Enrollment: | Approximate enrollment duration will be 3 weeks for phase 2 and 5 weeks for phase 3 study |

Protocol No: IVACFLU-S-0203 514 Dated: 12 March 2018

Version 1.0

Version: 4.0 Date: 09/02/2017


Page xviii

| Table 1: Sch | edule of events | 5 | | | | |
|---|---|---|---|---|---|---|
| Study Activities | Study Day (# days from D1) | | | | | |
| | S1/D1*<br>(up to -4/<br>D1<br>Clinic Visit | D1 to<br>D7 | D8<br>(+/- 1)<br>Clinic<br>Visit | D9 to<br>D21 | D22<br>(+/- 1)<br>Clinic<br>Visit | D91<br>(+/- 7)<br>Telephonic<br>contact |
| Information process and written informed consent | X | | | | | |
| Collect baseline demographic data | X | | | | | |
| Collect/review medical history | X | | | | | |
| Perform screening physical examination | X | | | | | |
| Perform vital signs & targeted physical examination (symptom based & reactogenicity only) | X* | | X | | | |
| Perform urine pregnancy check (women) | X* | | | | | |
| Check/confirm inclusion/exclusion criteria | X* | | | | | |
| Randomization | X | | | | | |
| Collect serum for influenza serology | X** | | | | X | |
| Administer one dose of study product (vaccine or placebo) | Х | | | | | |
| Observe for 30 Minutes; record and manage immediate reactions | X | | | | | |
| Instruct participant on use of Dairy card | Х | | | | | |
| Participant records solicited reactogenicity and unsolicited AEs in Dairy cards | Х | Х | | | | |
| Clinical staff reviews interim AEs/SAEs with participant; records in CRF | | | Х | | X | SAE only |
| Report SAEs to Sponsor, IRBs and regulatory authorities | Х | Χ | Х | X | X | Х |
| Participant completion of study | | | | | | X |

<sup>\*</sup>If Day 1 is conducted on a different day from S1, eligibility must be confirmed again on Day of Injection (D1); including Targeted physical examination (PE); inclusion/exclusion; urine pregnancy test.

<sup>\*\*</sup> Sera samples will be collected prior to vaccination in phase 3 study at one site (Ben Luc).

Version: 4.0

Date: 09/02/2017

Protocol No: IVACFLU-S-0203 515 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# **RESEARCH PROTOCOL**

# 1 Key Roles for Individuals and Institutions Involved

| Principal Investigator: | Dr. Phan Cong Hung |
|---|---|
| Co-Principal<br>Investigator | Dr. Nguyen Trong Toan |
| Investigator's Institution: | Pasteur Institute, Ho Chi Minh City, Vietnam |
| Institutional Review Boards: | Pasteur Institute IRB; WHO ERC and EC, MOH, Vietnam |
| Manufacturer | Institute of Vaccines and Medical Biologicals (IVAC) 9 Pasteur, Nha Trang, Vietnam Contact: Le Van Be, MD, PhD, Director phone: (+84 90) 3501529 fax: (+84 58) 3823815 email: ivaclevabe@dng.vnn.vn or ivaclevanbe@gmail.com |
| Sponsor | Institute of Vaccines and Medical Biologicals (IVAC) 9 Pasteur, Nha Trang, Vietnam Contact: Le Van Be, MD, PhD, Director phone: (+84 90) 3501529 fax: (+84 58) 3823815 email: ivaclevabe@dng.vnn.vn or ivaclevanbe@gmail.com |
| Contract Research<br>Organization | QuintilesIMS Plaza Building 4820 Emperor Boulevard Durham, North Carolina 27703 Phone: (+1 919) 998 2000 |
| Clinical Site,<br>Phase 2 | Only one site at District Health Center of Ben Luc district, Long An province where study activities (including screening, vaccinations, and follow-up visits as well as data entry) will be conducted. CRFs will be kept in the District Health Center and Pasteur Institute HCM city during study implementation, long term CRF storage will be at.IVAC |
| Clinical Sites,<br>Phase 3 | <ul> <li>Phase 3 will be conducted at 2 sites:</li> <li>District Health Center of Ben Luc district, Long An province</li> <li>District Health Center of Long Thanh district, Dong Nai province</li> <li>All study activities (including screening, blood draws (Ben Luc only),</li> </ul> |
| | vaccinations, and follow-up visits as well as data entry) will be |

Protocol No: IVACFLU-S-0203 516 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


V04


| | conducted at these district health centers. CRFs will be kept in the |
|---|---|
| | District Health Centers and Pasteur Institute HCM city during study |
| | implementation, long term CRF storage will be at IVAC. |
| | VisMederi srl |
| | Strada del Petriccio e Belriguardo, 35 |
| | 53100 Siena, Italia |
| Clinical and | phone +39 0577 381253 – 55 |
| Specialty | fax: +39 0577 381258 |
| Laboratories: | info@vismederi.com |
| | vismederi@pec.it |
| | Attn: Elisa Llorente Pastor |
| | Email: <u>llorentepastor@vismederiresearch.com</u> |
| | Le Van Be, MD, PhD, Director |
| Sponsor Medical | phone: (+84 90) 3501529 |
| Monitor: | fax: (+84 58) 3823815 |
| | email: ivaclevabe@dng.vnn.vn or ivaclevanbe@gmail.com |
| CRO Medical<br>Monitor: | TBD |
| | Tushar Tewari, MD |
| | Senior Medical Officer, Clinical and Regulatory Affairs |
| | Vaccine Development Global Program—PATH |
| | 2201 Westlake Avenue, Suite 200 |
| | Seattle, WA 98121 USA |
| PATH Medical | ocatile, ************************************ |
| Officer(s): | Tran Cong Thang, MD |
| | PATH Vietnam |
| | 11th Floor, Hanoi Towers, |
| | 49 Hai Ba Trung Street |
| | Hanoi 10000 Vietnam |
| | Tidilot 10000 Violitatii |
| | QuintilesIMS |
| Data Management | Quintilestivio |
| Organization: | |
| | Renee Holt, RN, JD, MPH |
| PATH Clinical | Clinical Operations Specialist |
| Operations | Vaccine Development Global Program—PATH |
| Specialists: | 2201 Westlake Avenue, Suite 200 |
| | Seattle, WA 98121 USA |
| | ı · |

Protocol No: IVACFLU-S-0203 517 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | PATH Vietnam office |
|-------------------|----------------------------------|
| | 11th Floor, Hanoi Towers |
| | 49 Hai Ba Trung |
| Other information | Hoan Kiem District |
| (Funders) | Hanoi, Vietnam |
| | PATH US office |
| | 2201 Westlake Avenue, Suite 200. |
| | Seattle, WA 98121, USA |
| | PATH Vietnam office |
| | 11th Floor, Hanoi Towers |
| | 49 Hai Ba Trung |
| | Hoan Kiem District |
| Technical support | Hanoi, Vietnam |
| | PATH US office |
| | 2201 Westlake Avenue, Suite 200. |
| | Seattle, WA 98121, USA |

Protocol No: IVACFLU-S-0203 518 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017


### 2 Background Information and Scientific Rationale

### 2.1 Background Information

#### 2.1.1 Overview of Influenza disease

Influenza is one of the major infectious disease threats to the human population due to both the adverse health impact of annual influenza epidemics and the detrimental global consequences of influenza pandemics [1,2]. The effects of an influenza are likely to be greatest in resource-limited countries where individuals may be more susceptible to severe outcomes of influenza due to underlying nutritional deficiencies and concomitant illness, limited access to health care, and the lack of widespread use of vaccines against common causes of bacterial pneumonia.

Influenza virus affects individuals of all ages, causes repeated infections throughout life, and is responsible for annual worldwide epidemics. While influenza leads to a self-limited respiratory disease in the majority of individuals, it can be deadly in others. The seriousness of influenza in young children, older adults, and persons of all ages with certain underlying medical conditions is the reason why many countries have recommendations to vaccinate such individuals and their close contacts every year.

A distinct feature of influenza virus is its ability to mutate, leading to antigenic changes that require the introduction of new vaccine strains each year. Seasonal changes in the surface glycoproteins enable the viruses to evade immunity induced by strains circulating previously. For this reason, natural infection or vaccination are generally only protective against infection for one influenza season. Evolutionary pressures lead to the emergence of new influenza strains to which there is decreased immunity in the population.

### 2.1.2 Seasonal Influenza

Seasonal influenza viruses circulate widely and cause disease in humans every year. The circulation of influenza virus is detected globally in various geographies of North America, Europe, Asia, Oceania and South America. In temperate climates, disease tends to occur seasonally in the winter months, spreading from person-to-person through sneezing, coughing, or touching contaminated surfaces. Seasonal influenza viruses can cause mild to severe illness and even death, particularly in some high-risk individuals. Persons at increased risk for severe disease include pregnant women, the very young and very old, immune-compromised people, and people with chronic underlying medical conditions. As mentioned above seasonal influenza viruses evolve continuously, which means that people can get infected multiple times throughout their lives. Therefore the components of seasonal influenza vaccines are reviewed frequently (currently biannually) and updated periodically to ensure continued effectiveness of the vaccines.

There are three large groupings or types of seasonal influenza viruses, labeled A, B, and C. Type A influenza viruses are further divided into subtypes according to the specific variety and combinations of two proteins that occur on the surface of the virus, the hemagglutinin or "H"

Protocol No: IVACFLU-S-0203 519 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0


protein and the neuraminidase or "N" protein. Type C influenza causes milder infections and is associated with sporadic cases and minor localized outbreaks. As influenza C poses much less of a disease burden than influenza A (A/H1N1 and A/H3N2 subtypes) and B, only the latter two are included in seasonal influenza vaccines.

### 2.1.3 Seasonal Influenza in Vietnam

The WHO's Global Influenza Programme (GIP) is involved in world-wide influenza surveillance. Global Influenza Programme (GIP) collects and analyzes virological and epidemiological influenza surveillance data from around the world [3]. The regular sharing of quality influenza surveillance and monitoring data by countries allows WHO to:

- provide information about pattern of influenza transmission globally to allow countries to better prepare for upcoming seasons;
- describe critical features of influenza epidemiology including risk groups, transmission characteristics, and impact;
- · monitor global trends in influenza transmission; and
- support the selection of influenza strains for vaccine production.

Vietnam has also been a part of this surveillance network. Surveillance data of influenza in Vietnam indicated that, of 29,499 specimens tested from 2006 to 2011, 5241 (17.8%) were positive for influenza infection [4]. Analysis of monthly data showed year-round circulation (Fig. 1 and Fig. 2), and some peak activity in July to August (Fig. 2). Subtype A H1N1 and type B viruses were the most frequently reported in 2006 (43.5 and 53.7%, respectively) and 2008 (40.8 and 41.3%, respectively), whereas A H3N2 subtype (73.9%) and type B viruses (25.1%) were the ones most frequently reported in 2007. Influenza A(H1N1)pdm09 emerged (46.6%) in mid-2009 and persisted in 2010 (28.0%), when it co-circulated with subtype A H3 (71.5%) viruses. In 2011, A(H1N1)pdm09 was the influenza virus most frequently reported (74.1%), followed by type B viruses (22.1%, Fig. 3) [4].

IVACFLU-S, Phase 2/3


520

Fig. 1. Monthly distribution of samples testing positive for influenza virus or viral nucleic acid by year in Vietnam, 2006–2011



<sup>&</sup>lt;sup>1</sup> This represents the samples testing positive on any given month, as a percentage of all the samples that tested positive during the year.

Fig. 2. Monthly patterns of influenza trends in samples testing positive to influenza virus or viral nucleic acid in Vietnam, 2006-2011



<sup>&</sup>lt;sup>1</sup> This represents the mean value for the samples testing positive on any given month from 2006 to 2011 as a percentage of all the samples that tested positive during each year.


Fig. 3. Influenza virus types and subtypes identified, by year in Vietnam, 2006–2011



The latest information from end of year 2015 (week 43-53) and 2016 (Week1-39) from the WHO for seasonal influenza in Vietnam is available. The figure 4 shows for 2015 A(H3) predominating in weeks 43-53, with some specimens positive for B and A (H1N1. For 2016, A(H1N1) continues to be the predominant strain from weeks 9 - 24 with B strain of undetermined lineage accounting for one third to half of all the specimens reported for the same period [5]. From week 26-39 A (H3) is the predominant subtype identified with B strain of undetermined lineage and A(H1N1)pdm09 also identified during this period.

Fig. 4. Influenza viruses surveillance in Vietnam, 2015-2016



Protocol No: IVACFLU-S-0203 522 Dated: 12 March 2018


#### 2.1.4 Treatment and Prevention (vaccine, biological)

Multiple manufacturers around the globe have developed various seasonal trivalent influenza vaccines and have tested these candidates in many trials in healthy adults and used them yearly before the influenza season. The choice of strains to include in the vaccine is guided by the "WHO Global Action Plan", an initiative to support development of new influenza vaccines, increase demand for seasonal vaccines, and enhance influenza vaccine production capacity [3]. With support from international donors, including the US Department of Health and Human Services, the WHO leads a program to support influenza vaccine manufacturers in developing countries that is crucial to increasing overall manufacturing capacity as well as to enhancing regional access to vaccines. In the first phase of the plan, the WHO provided funding and assistance to manufacturers in six countries, including Vietnam, to establish influenza vaccine production capacity.

Since 2008, IVAC has received technical assistance from PATH and WHO to develop and produce vaccines for A/H1N1/09, A/H5N1, A/H7N9 and seasonal flu vaccines under the guidance from the MOH.

### 2.1.5 Summary results of related preclinical trials

Three clinical lots of trivalent split inactivated seasonal vaccine formulated with the strains recommended for the 2016-2017 season were successfully manufactured, tested and released by IVAC in the late fourth quarter of 2016. WHO recommends that influenza vaccines for use in the 2016-2017 northern hemisphere influenza season contain the following viruses:

- NYMC BX-35 reassortant of B/Brisbane/60/2008 (B)
- NYMC X-179A reassortant of A/California/7/2009 (H1N1)
- NYMC X-263B reassortant of H3/A/Hong Kong/4801/2014 (H3N2)

Among circulating influenza B viruses, there are two distinct lineages. The B/Brisbane/60/2008-like viruses are from the influenza B/Victoria lineage and represent the predominant circulating influenza B virus [6].

The Preclinical evaluation was conducted with all three lots of seasonal vaccine used in the phase 1 study. The vaccine demonstrated good immunogenicity in mouse studies (quantitated by hemagglutination inhibition comparable to that induced by a comparator vaccine), and an acceptable safety profile in general safety and toxicology studies in experimental animals (rabbit, mice and guinea pig)..

The trivalent split inactivated seasonal vaccine lots which were produced by IVAC with strains recommended for the flu season of 2016-2017 and that will be used for the phase 2/3 study, IVAC has only conducted an additional pre-clinical study (September, 2016) of 3 bulk lots (with all 3 strains) for evaluation of safety and immunogenicity. The result showed the vaccine was well tolerated, safe and immunogenic in experimental animals with intramuscular administration.

Protocol No: IVACFLU-S-0203 523 Dated: 12 March 2018


#### 2.1.6 Results of Clinical Trial

A phase 1 clinical trial of the IVAC inactivated split virion influenza vaccine was conducted in 60 healthy adults, 18 through 45 years of age, in Hung Ha District, Thai Binh Province, Vietnam in 2015 [7]. Participants were randomized to either placebo or vaccine containing 15  $\mu$ g of HAI antigen from the following 3 viral strains:

- NYMC BX-51B reassortant of B/Massachusetts/2/2012 (B)
- NYMC X-179A reassortant of A/California/7/2009 (H1N1) and
- NYMC X-223 A reassortant of H3/A/Texas/50/2012 (H3N2).

Table 2 summarizes the demographic and baseline characteristic of the study population.

**Table 2 Summary of Demographics and Baseline Characteristics** 

| | Vaccine (N=30) | | Placebo | o (N-30) |
|-------------------|----------------|------|---------|----------|
| Characteristics | n | % | n | % |
| Gender | | | | |
| Male | 3 | 10 | 9 | 30 |
| Female | 27 | 90 | 21 | 70 |
| Age | | | | |
| Mean | 37 | 7.7 | 37.8 | |
| Minimum / Maximum | 27 | / 45 | 21 / 45 | |

### Safety Results of Phase 1 IVACFLU-S Seasonal Flu Vaccine Trial

The safety results can be summarized as follows:

No local or systemic solicited AEs were reported within 30 minutes after vaccination. All participants were observed to have oral temperature with in normal range (<37.7°C; Grade 0) Overall, 20 participants (66.7 %) on vaccine and 8 participants (26.7%) on placebo, reported at least 1 local solicited AE on Day 1. Among vaccine recipients who experienced local reactions, pain and tenderness at the injection site were the most common reaction (Table 3). Majority were assessed as mild and resolved spontaneously within 24-48 hours and. By day 7, only 1 participant (3.3%) on placebo reported at least 1 local solicited AE. In contrast no participant on vaccine reported any local solicited AE beyond day 4 [7].

Protocol No: IVACFLU-S-0203 524 Dated: 12 March 2018


No participant reported fever (oral temperature >37.7°C). Overall, the number of participants who reported any systemic solicited AEs at Day 1 and their severity were similar across vaccine and placebo groups (8 participants [26.7%] on vaccine and 7 participants [23.3%] on placebo). The majority of systemic solicited AEs reported by participants on vaccine were mild (Table 3) and none lasted beyond 6 days. In contrast in the group randomized to placebo, 2 participants reported severe reactions (fatigue and joint ache) and 3 participants reported multiple solicited systemic adverse events up to Day 7 (Figure 5).

There were no deaths, SAEs, or discontinuation due to AEs reported in the study. There were no clinically significant abnormalities observed in the clinical laboratory results or product-related trends based on a review of the mean and median laboratory values at each scheduled evaluation, vital signs, and physical examination evaluations during the study (data not shown). The incidence of unsolicited AEs (Table 4) were similar across vaccine and placebo groups (7 participants [23.3%] each). All unsolicited AEs reported in the study were mild in intensity and were considered to be not related to the investigational product by the Principal Investigator.

Overall the vaccine was safe and well tolerated with a safety profile similar to licensed seasonal influenza vaccine.

Table 3: Summary of Solicited Local and Systemic Adverse Events for Vaccine and placebo Recipients Occurring from Day 1-7 After Vaccination Based on Most Severe Symptom Reported

| | V | Vaccine (N=30) | | | Placebo (N=30) | |
|---|---|---|---|---|---|---|
| Solicited Adverse Event | Mild | Moderate | Severe | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Injection site | | <u> </u> | | | <u> </u> | |
| Pain | 17 (56.7) | 2 (6.7) | 0 | 5 (16.7) | 0 | 0 |
| Tenderness | 16 (53.3) | 1 (3.3) | 0 | 9 (30.0) | 0 | 0 |
| Hardness | 0 | 1 (3.3) | 0 | 0 | 0 | 0 |
| Swelling | 0 | 1 (3.3) | 0 | 0 | 0 | 0 |
| Systemic symptoms | | | | | <u> </u> | |
| Headache | 6 (20.0) | 1 (3.3) | 0 | 8 (26.7) | 1 (3.3) | 0 |
| Tiredness/discomfort | 5 (16.7) | 2 (6.7) | 0 | 6 (20.0) | 1 (3.3) | 1 (3.3) |
| Chills | 2 (6.7) | 0 | 0 | 3 (10.0) | 1 (3.3) | 0 |
| Muscle Aches | 3 (10.0) | 0 | 0 | 4 (13.3) | 1 (3.3) | 0 |
| Vomiting | 1 (3.3) | 0 | 0 | 1 (3.3) | 0 | 0 |
| Joint Aches | 0 | 1 (3.3) | 0 | 1 (3.3) | 0 | 1 (3.3) |
| Nausea | 0 | 0 | 0 | 3 (10.0) | 0 | 0 |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 525 Dated: 12 March 2018

 IVACFLU-S, Phase 2/3

 Date: 09/02/2017


Figure 5: Number of Participants Reporting Any Solicited Systemic Adverse Events Day 1 to 7 Following Vaccination



Overall, 14 subjects (23.3%) reported at least 1 unsolicited AE: 7 subjects (23.3%) each on vaccine and placebo. The overall summary of unsolicited AEs are presented in Table 4.

Table 4: Summary of unsolicited events

| Unsolicited event | Vaccine<br>(N=30)<br>n (%) | Placebo<br>(N=30)<br>n (%) | Total<br>(N=60)<br>n (%) |
|---|---|---|---|
| Total number of unsolicited AEs | 7 | 7 | 14 |
| Subjects with at least one unsolicited AE | 7 (23.3) | 7 (23.3) | 14 (23.3) |
| At least one vaccine related unsolicited AE | 0 | 0 | 0 |
| At least one severe unsolicited AE | 0 | 0 | 0 |
| Subjects requiring treatment during the study | 5 (16.7) | 3 (10.0) | 8 (13.3) |
| Number of subjects died | 0 | 0 | 0 |

N– Total number of subjects in each group; n – Total number of subjects meeting the event.

Any solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Protocol No: IVACFLU-S-0203 526 Dated: 12 March 2018


Overall, the most frequently reported AEs were in the System Organ Class of infections and infestations (6 subjects [10.0%]); respiratory thoracic and mediastinal disorders (4 subjects [6.7%]); and general disorders and administration site conditions (Table 5).

Table 5: Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term

| System Organ Class/ Preferred term | Vaccine<br>(N=30)<br>n (%) | Placebo<br>(N=30)<br>n (%) | Total<br>(N=60)<br>n (%) |
|---|---|---|---|
| Number of Subjects with at least one AE | 7 (23.3) | 7 (23.3) | 14 (23.3) |
| Infections and infestations | 5 (16.7) | 1 (3.3) | 6 (10.0) |
| Herpes zoster | 1 (3.3) | 0 | 1 (1.7) |
| Influenza | 1 (3.3) | 0 | 1 (1.7) |
| Nasopharyngitis | 1 (3.3) | 0 | 1 (1.7) |
| Pharyngitis | 1 (3.3) | 0 | 1 (1.7) |
| Upper respiratory tract infection | 0 | 1 (3.3) | 1 (1.7) |
| Urinary tract infection | 1 (3.3) | 0 | 1 (1.7) |
| Respiratory, thoracic and mediastinal disorders | 1 (3.3) | 3 (10.0) | 4 (6.7) |
| Oropharyngeal pain | 0 | 2 (6.7) | 2 (3.3) |
| Rhinorrhea | 1 (3.3) | 1 (3.3) | 2 (3.3) |
| General disorders and administration site conditions | 0 | 2 (6.7) | 2 (3.3) |
| Fatigue | 0 | 1 (3.3) | 1 (1.7) |
| Non-cardiac chest pain | 0 | 1 (3.3) | 1 (1.7) |
| Musculoskeletal and connective tissue disorders | 1 (3.3) | 0 | 1 (1.7) |
| Arthralgia | 1 (3.3) | 0 | 1 (1.7) |
| Nervous system disorders | 0 | 1 (3.3) | 1 (1.7) |
| Headache | 0 | 1 (3.3) | 1 (1.7) |

N– Total number of subjects in each group; n – Total number of subjects meeting the event. Percentages were based on the total number of subjects under each vaccine group (N).

### Immunogenicity Results of Phase 1 IVACFLU-S Seasonal Flu Vaccine Trial

Immune responses were measured at baseline and 21 days after vaccination. Approximately 50% of the participants had antibody titer  $\geq$ 1:40 baseline by HAI and Microneutralization Test (MNT) to A/H3N2 (Table 6). Nevertheless, the proportion of participants achieving a  $\geq$  4-fold rise in HAI and MNT titer against all three viral strains was high (Table 7A). Of the 16 participants with HAI

Adverse Event terms were coded by System Organ Class and Preferred Term using MedDRA version 18.1. Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories.

Any solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Protocol No: IVACFLU-S-0203 527 Dated: 12 March 2018


titer ≥1:40 at baseline to A/H3N2, 12 developed 4 fold or greater rise in HAI antibody following vaccination. No placebo participants developed a 4 fold rise in HAI and MNT antibody following vaccination. The vaccine also induced strong HAI seroprotection response (Table 7B), well above 90% for all three viral strains.

Table 6: Baseline titer ≥1:40 by HAI and MNT for vaccine and placebo recipients

| Vaccine | HAI | | M | NT |
|---------|-----------|--------------|-----------------------|--------------|
| N=30 | HAI | 95%CI | MNT | 95%CI |
| A/H1N1 | 5 (16.7) | (5.6, 34.7) | 4 (13.3) | (3.8, 30.7) |
| A/H3N2 | 16 (53.3) | (34.3, 71.7) | 16 (53.3) | (34.3, 71.7) |
| В | 3 (10.0) | (2.1, 26.5) | (2.1, 26.5) 11 (36.7) | |
| Placebo | | | | |
| N=30 | HAI | 95%CI | 95%CI MNT | |
| A/H1N1 | 6 (20.0) | (7.7, 38.6) | 5 (16.7) | (5.6, 34.7) |
| A/H3N2 | 16 (53.3) | (34.3, 71.7) | 15 (50.0) | (31.3, 68.7) |
| В | 0 (0.0) | (0.0, 11.6) | 9 (30.0) | (14.7, 49.4) |

### Table 7:

# A. Seroconversion rates by HAI and MNT for vaccine and placebo recipients 21 days after vaccination

| Vaccine | HAI | | N | INT |
|---------|-----------|--------------|-----------|--------------|
| N=30 | n=30 (%) | 95% CI | n=30 (%) | 95% CI |
| A/H1N1 | 28 (93.3) | (77.9, 99.2) | 28 (93.3) | (77.9, 99.2) |
| A/H3N2 | 25 (83.3) | (65.3, 94.4) | 25 (83.3) | (65.3, 94.4) |
| В | 23 (76.7) | (57.7, 90.1) | 21 (70.0) | (50.6, 85.3) |
| Placebo | | | | |
| N=30 | n=30 (%) | 95% CI | n=30 (%) | 95% CI |
| A/H1N1 | 0 (0.0) | (0.0, 11.6) | 0 (0.0) | (0.0, 11.6) |
| A/H3N2 | 0 (0.0) | (0.0, 11.6) | 0 (0.0) | (0.0, 11.6) |
| В | 0 (0.0) | (0.0, 11.6) | 0 (0.0) | (0.0, 11.6) |

Seroconversion is defined as a serum HAI titer meeting the following criteria:

- pre-vaccination titer <1:10 and a post-vaccination titer ≥ 1:40 or</li>
- pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination measured on Day 22

# B. Seroprotection rates (Titer ≥1:40) by HAI and MNT for vaccine and placebo recipients 21 days after vaccination

| Vaccine | HAI | MNT |
|---------|-----|-----|

Dated: 12 March 2018


| N=30 | N, % | 95% CI | N, % | 95% CI |
|---------|-----------|--------------|-----------|--------------|
| A/H1N1 | 29 (96.7) | (82.8, 99.9) | 29 (96.7) | (82.8, 99.9) |
| A/H3N2 | 29 (96.7) | (82.8, 99.9) | 29 (96.7) | (82.8, 99.9) |
| В | 28 (93.3) | (77.9, 99.2) | 26 (86.7) | (69.3, 96.2) |
| Placebo | | | | |
| N=30 | N, % | 95% CI | N, % | 95% CI |
| A/H1N1 | 6 (20.0) | (7.7, 38.6) | 5 (16.7) | (5.6, 34.7) |
| A/H3N2 | 16 (53.3) | (34.3, 71.7) | 14 (46.7) | (28.3, 65.7) |
| В | 0 (0.0) | (0.0, 11.6) | 9 (30.0) | (14.7, 49.4) |

Seroprotection: Number and percentage of subjects with a serum Hemagglutination Inhibition (HAI) antibody titer ≥ 1:40 to each of the 3 vaccine components measured on Day 22 post-vaccination

Geometric mean titer (GMT) responses by HAI and MNT showed a strong response to all 3 viral strains, H1N1>H3N2>B, post-vaccination (Table 8). GMT at baseline was low and there was no rise in antibodies among placebo participants. For participants randomized to vaccine HAI GMT rose to 37.2 (A/H1N1), 16.2 (A/H3N2), and 7.8 (B) folds after vaccination. Geometric mean titers by MNT to all 3 viral strains were of similar magnitude as seen with HAI.

Table 8: Geometric Mean Titer (GMT) response by HAI and MNT for vaccine and placebo recipients

| | | | HAI | | | MNT | |
|----------------|--------|-------|-------|------|-------|-------|-------|
| Vaccine (n=30) | | H1N1 | H3N2 | В | H1N1 | H3N2 | В |
| GMT | Day 1 | 10.0 | 39.5 | 8.8 | 8.7 | 38.6 | 16.2 |
| | Day 22 | 371.9 | 640.0 | 68.1 | 417.4 | 670.3 | 201.6 |
| | Fold | 37.2 | 16.2 | 7.7 | 47.9 | 17.3 | 12.4 |
| Placebo (n=30) | | H1N1 | H3N2 | В | H1N1 | H3N2 | В |
| GMT | Day 1 | 10.6 | 35.6 | 6.9 | 10.8 | 40.0 | 14.6 |
| | Day 22 | 10.7 | 33.6 | 7.0 | 10.5 | 39.1 | 14.3 |
| | Fold | 1.0 | 0.9 | 1.0 | 1.0 | 1.0 | 1.0 |

In summary the data from the phase 1 trial showed the vaccine to be safe and well tolerated. The vaccine was able to induce strong immune response, even among individuals with pre-existing HAI antibodies [7]. Both the safety profile and immunogenicity responses of IVACFLU-S are comparable to licensed inactivated seasonal influenza vaccines (Section 2.2). Furthermore, the immune responses, even at the LB of 95% CI, exceeded the European Medicine Agency and Vietnam Ministry of Health serological criteria for regulatory approval of seasonal influenza vaccines. (8)

Protocol No: IVACFLU-S-0203 529 Dated: 12 March 2018


### 2.2 Data on Clinical Trials from Seasonal Vaccines Similar to IVACFLU-S

### 2.2.1 Flucelvax - Seqirus, Inc

Flucelvax (Influenza Vaccine), a vaccine for intramuscular injection, is a "subunit" influenza vaccine prepared from virus propagated in Madin Darby Canine Kidney (MDCK) cells, a continuous cell line. These cells were adapted to grow freely in suspension in culture medium. The virus is inactivated with \( \mathbb{G}\)-propiolactone, disrupted by the detergent cetyltrimethylammonium bromide and purified through several process steps. Each of the 3 virus strains is produced and purified separately then pooled to formulate the trivalent vaccine. The following safety profile is in the package insert for Flucelvax [9]:

Table 9: Solicited Adverse Reactions in the Safety Population<sup>1</sup> Reported Within 7 Days of Vaccination in Study<sup>1</sup>

| | Adults 18 through 49 Years | |
|---|---|---|
| | Percentages (%) | |
| | Flucelvax<br>N=3813 | Placebo (PBS)<br>N=3894 |
| Local adverse reactions | | 1 |
| Injection site pain | 30 | 10 |
| Erythema | 13 | 10 |
| Induration | 6 | 3 |
| Swelling | 6 | 3 |
| Ecchymosis | 4 | 4 |
| Systemic adverse reactions | | |
| Headache | 15 | 15 |
| Fatigue | 10 | 10 |
| Myalgia | 12 | 7 |
| Malaise | 8 | 6 |
| Chills | 6 | 6 |
| Arthralgia | 3 | 3 |
| Sweating | 3 | 3 |
| Fever (≥38 <sup>0</sup> C) | 1 | <1 |

<sup>&</sup>lt;sup>1</sup>Safety population: all participants in the exposed population who provided post vaccination safety data Flucelvax has the following efficacy profile, as stated in its package insert:

Dated: 12 March 2018


Table 10: Percentage (%) of participants with Post-Vaccination HAI Titers ≥ 1:40 and Seroconversion in Adult Flucelvax Recipients 18 through 49 Years and 50 through 64 Years of Age

| | | 18 through 49 Years | | 50 through 64 Years | |
|---|---|---|---|---|---|
| | Vaccine | % | % 1 | % | % 1 |
| Study | strain | HAI Titer≥1:40 | Seroconversion <sup>1</sup> | HAI Titer≥1:40 | Seroconversion ' |
| | ou an i | (95% CI) | (95% CI) | (95% CI) | (95% CI) |
| | | N=228 | N=228 | | |
| Study 1 US, | A/H1N1 | 99 | 78 | | |
| Finland, | | (97-100) | (72-83) | | |
| Poland<br>2007– | A/H3N2 | 99<br>(98-100) | 59<br>(53-66) | | |
| 2008<br>N=228 | В | 78<br>(72-83) | 51<br>(45-58) | | |
| | | N=478 | N=478 | N=340 | N=340 |
| Study 2<br>Poland<br>2004– | A/H1N1 | 94<br>(91-96) | 73<br>(69-77) | 84<br>(79-88) | 57<br>(52-63) |
| | | 18 through 49 Years | | 50 through 64 Years | |
| 2005 | A/H3N2 | 99<br>(98-100) | 63<br>(59-68) | 99<br>(97-100) | 66<br>(61-71) |
| N=818 | В | 93<br>(90-95) | 88<br>(84-90) | 87<br>(83-90) | 77<br>(70-79) |
| | | N=307 | N=307 | | |
| Study 3<br>US<br>2005– | A/H1N1 | 96<br>(94-98) | 62<br>(57-68) | | |
| | A/H3N2 | 91<br>(87-94) | 85<br>(81-89) | | |
| 2006<br>N=307 | В | 94<br>(91-96) | 77<br>(72-81) | | |

<sup>&</sup>lt;sup>1</sup> Rates of seroconversion = percentage of participants with either a pre-vaccination HAI titer < 1:10 and a post-vaccination HAI titer ≥ 1:40 or a pre-vaccination HAI titer ≥ 1:10 and at least a four-fold rise in post-vaccination HAI antibody titer

### 2.2.2 Fluzone®- Sanofi Pasteur

Fluzone (Influenza Vaccine) for intramuscular injection is an inactivated influenza vaccine, prepared from influenza viruses propagated in embryonated chicken eggs. The virus-containing allantoic fluid is harvested and inactivated with formaldehyde. Influenza virus is concentrated and purified in a linear sucrose density gradient solution using a continuous flow centrifuge. The virus is then chemically disrupted using a non-ionic surfactant, octylphenol ethoxylate (Triton® X-100), producing a "split virus". The split virus is further purified and then suspended in sodium phosphate-buffered isotonic sodium chloride solution. Fluzone has the following safety profile as stated in the package insert [10]:

IVACFLU-S, Phase 2/3


Table 11: Frequency of Solicited Injection-Site Reactions and Systemic Adverse Events within 7 Days after Vaccination with Fluzone, Adults 18 Through 64 Years of Age

| | (N <sup>a</sup> =1392-1394)<br>Percentage | | |
|---|---|---|---|
| | Any | Grade 2 <sup>b</sup> | Grade 3 <sup>C</sup> |
| Injection-Site Erythema | 13.2 | 2.1 | 0.9 |
| Injection-Site Induration | 10.0 | 2.3 | 0.5 |
| Injection-Site Swelling | 8.4 | 2.1 | 0.9 |
| Injection-Site Pain | 53.7 | 5.8 | 0.8 |
| Injection-Site Pruritus | 9.3 | 0.4 | 0.0 |
| Injection-Site Ecchymosis | 6.2 | 1.1 | 0.4 |
| Headache | 30.3 | 6.5 | 1.6 |
| Myalgia | 30.8 | 5.5 | 1.4 |
| Malaise | 22.2 | 5.5 | 1.8 |
| Shivering | 6.2 | 1.1 | 0.6 |
| Fever <sup>d</sup> (≥99.5°F) | 2.6 | 0.4 | 0.2 |

<sup>&</sup>lt;sup>a</sup> N is the number of vaccinated participants with available data for the events listed

Myalgia, Malaise, and Shivering: prevents daily activities

Fluzone has the following efficacy profile, as stated in its package insert:

Table 12: Percentage (%) with Pre and Post-Vaccination HAI Titers ≥1:40 and Seroconversion in Adult Fluzone Recipients 18 through 64 Years of Age

| Antigen | Pre-Vaccination Titer ≥1:40<br>% (95% CI) N=1285-1286 | Post-Vaccination <sup>a</sup><br>Titer ≥1:40<br>% (95% CI) N=1283-1285 | Seroconversion <sup>b</sup> % (95% CI) N=1283-1285 |
|---|---|---|---|
| A (H1N1) | 39.1 (36.4; 41.8) | 91.7 (90.0; 93.1) | 60.5 (57.7; 63.2) |
| A (H3N2) | 33.6 (31.0; 36.2) | 91.4 (89.8; 92.9) | 74.8 (72.3; 77.1) |

<sup>&</sup>lt;sup>b</sup> Grade 2 - Injection-site erythema, Injection-site induration, Injection-site swelling, and Injection-site ecchymosis: ≥ 2.5 cm to <5 cm; Injection-site pain and Injection-site pruritus: sufficiently discomforting to interfere with normal behavior or activities; Fever: >100.4°F to ≤102.2°F; Headache, Myalgia, Malaise, and Shivering: interferes with daily activities

<sup>&</sup>lt;sup>c</sup> Grade 3 - Injection-site erythema, Injection-site induration, Injection-site swelling, and Injection-site ecchymosis: ≥5 cm; Injection-site pain: incapacitating, unable to perform usual activities; Injection-site pruritus: incapacitating, unable to perform usual activities, may have/or required medical care or absenteeism; Fever: >102.2°F; Headache,

<sup>&</sup>lt;sup>d</sup> Fever - The percentage of temperature measurements that were taken by oral or axillary routes, or not recorded were 99.6%, 0.0%, and 0.4%, respectively

Protocol No: IVACFLU-S-0203 532 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017


| В | 41.2 (38.5; 44.0) | 89.3 (87.4; 90.9) | 54.2 (51.4; 56.9) |
|---|-------------------|-------------------|-------------------|

<sup>&</sup>lt;sup>a</sup>Post-vaccination HAI titers drawn at 28 days post-dose

#### 2.2.3 Fluarix - GSK

FLUARIX is a vaccine prepared from influenza viruses propagated in embryonated chicken eggs. Each of the influenza viruses is produced and purified separately. After harvesting the virus-containing fluids, each influenza virus is concentrated and purified by zonal centrifugation using a linear sucrose density gradient solution containing detergent to disrupt the viruses. Following dilution, the vaccine is further purified by diafiltration. Each influenza virus solution is inactivated by the consecutive effects of sodium deoxycholate and formaldehyde leading to the production of a "split virus." Each split inactivated virus is then suspended in sodium phosphate-buffered isotonic sodium chloride solution. The vaccine is formulated from the 3 split inactivated virus solutions. The following safety profile is reported in the package insert for Fluarix [11]:

Table 13: Incidence of Solicited Local Adverse Reactions or General Adverse Events within 4 Days of Vaccination in Adults Aged 18 through 64 Years

| | Fluarix N = 760 | Placebo N = 192 |
|-------------------------|-----------------|-----------------|
| | % | % |
| Local Adverse Reactions | | • |
| Pain | 55 | 12 |
| Redness | 18 | 10 |
| Swelling | 9 | 6 |
| General Adverse Events | • | • |
| Muscle aches | 23 | 12 |
| Fatigue | 20 | 18 |
| Headache | 19 | 21 |
| Arthralgia | 6 | 6 |
| Shivering | 3 | 3 |
| Fever ≥100.4°F (38.0°C) | 2 | 2 |

Fluarix has the following efficacy reported in its package insert:

Table 14: Rates with HAI Titers ≥1:40 and Rates of Seroconversion to Each Antigen following Fluarix or Placebo (21 Days after Vaccination) in Adults Aged 18 through 64 Years

<sup>&</sup>lt;sup>b</sup> Seroconversion: Paired samples with pre-vaccination HAI titer <1:10 and post-vaccination (28 days post-dose) titer ≥1:40 or a minimum 4-fold increase for participants with pre-vaccination titer ≥1:10
Protocol No: IVACFLU-S-0203 533 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017


| | FLUARIX <sup>b</sup> N = 745 | | Place bo | |
|---|---|---|---|---|
| | % (95% CI) | | N = 190 | |
| | | | % (95% CI) | |
| | Pre - | Post- | Pre - | Post- |
| | vaccination | vaccination | vaccination | vaccination |
| With HAI Titers ≥1:40 | | | | |
| A/New Caledonia/20/99 (H1N1) | 54.8 | 96.6 | 52.1 | 51.1 |
| | (51.1, 58.4) | (95.1, 97.8) | (44.8, 59.4) | (43.7, 58.4) |
| A/Wyoming/3/2003 (H3N2) | 68.7 | 99.1 | 65.3 | 65.3 |
| | (65.3, 72) | (98.1, 99.6) | (58, 72) | (58, 72) |
| B/Jiangsu/10/2003 | 49.5 | 98.8 | 48.9 | 51.1 |
| | (45.9, 53.2) | (97.7, 99.4) | (41.6, 56.3) | (43.7, 58.4) |
| Se roconve rsion | Post-vaccination | | Post-va | ccination |
| A/New Caledonia/20/99 (H1N1) | 59.6 | | 0 | |
| | (56, 63.1) | | (0, | 1.9) |
| A/Wyoming/3/2003 (H3N2) | 61.9 | | 1.1 | |
| | (58.3, 65.4) | | (0.1 | , 3.8) |
| B/Jiangsu/10/2003 | 77.6 | | | 1.1 |
| | (74.4, 80.5) | | (0.1 | , 3.8) |

### 2.3 Rationale of Current Study

Vaccination is currently the most effective means of preventing influenza infection. However global influenza vaccine coverage is low and vaccine production capacity is concentrated mostly in industrialized countries. In the event of antigenic shift in the hemagglutinin (HA) of influenza leading to pandemic influenza, it is probable that global supply of a pandemic influenza will be limited due to insufficient vaccine production capacity. It is also recognized that pandemic vaccine production capacity is dependent on seasonal vaccine capacity and demand, and the dependence of this demand on evidence and policies supporting the use of influenza vaccines.

WHO GAP with financial support from Biomedical Advanced Research and Development Authority (BARDA) - the US Department of Health and Human Services and technical assistance from PATH have provided technical and financial support to Institute of Vaccine and Medical Biologics (IVAC) for improving technology, scaling-up, production of clinical lots and carrying out pre-clinical studies and clinical trials. The goal is to have a licensed, Vietnamese-made seasonal influenza vaccine and through that expertise to eventually develop and gain approval of a pandemic influenza vaccine.

The phase 1 trial of the IVAC seasonal trivalent inactivated split virion influenza vaccine

Protocol No: IVACFLU-S-0203 534 Dated: 12 March 2018


completed in Mar, 2016 identified no safety concerns and demonstrated the vaccine to be highly immunogenic [7]. Given the promising findings, the current study proposes to expand on the safety data of the vaccine and to confirm the immunological findings, including individuals up to age 60 with the goal of seeking regulatory approval for indication in non-elderly adults based on the Vietnam Ministry of Health Guidance on Clinical Trial of Influenza Vaccine serological criteria for assessing seasonal influenza [8]. The immediate benefit of licensure of a seasonal influenza vaccine in this age group will be among health care workers (HCW) who are at higher risk of influenza infection as compared to healthy adults who work in non-health care settings [12]. Furthermore vaccinating health care workers against influenza reduces the transmission of the virus in health care settings, decreases staff illness and absenteeism, and indirectly benefits patients by decreasing their chance of being infected [13]. In particular patients who are too young to receive the vaccine (<6 months of age) and those who have poor immunological responses (elderly and immune-compromised). Recent epidemiological data also suggest that vaccinating non-elderly (<65 years old) adults may also protect higher risk individuals in their community, with the potential to prevent up to 5.9% of influenza diagnosis in elderly individuals [14]. Seasonal vaccine is also recommended by WHO to be administrated to pregnant women in order to protect the fetus and mother during the pregnancy. Finally, licensure initially in this age group will also help facilitate future bridging licensure studies in other populations that are vulnerable to influenza infection and its complications.

#### 2.4 Dose Rationale

The rationale for dose selection of seasonal influenza vaccines is widely accepted in the scientific community. This study uses the WHO-recommended dose of 15 mcg of HA per strain as measured by single radiation immunodiffusion (SRID) assay.

### 2.5 Potential Risks and Benefits of Inactivated, split Influenza Vaccine

### 2.5.1 Potential Risks

We expect this study vaccine to cause side effects similar to those seen in the Phase 1 study and in other inactivated, trivalent influenza vaccines particularly other split virion influenza vaccines. From worldwide use, we know that administering seasonal influenza vaccine may cause the participant immediate mild pain in the arm. Other side effects include pain and inflammation (redness/swelling) at the injection site or systemic symptoms such as headache, fever, tiredness, and body aches. It is very rare, but serious or allergic reactions may also happen.

These potential risks are addressed by several measures:

• The study is supervised by a physician and the study staff are trained and equipped to handle any vaccine reaction. To manage immediate reactions, participants remain at the study site at least 30 minutes after injection.

Protocol No: IVACFLU-S-0203 535 Dated: 12 March 2018


- The safety of the study is overseen by a Protocol Safety Review Team (PSRT) that meets regularly (generally weekly) to review safety information up to Day 22.
- The study staff check in with the participants at 1 day following vaccination to check on their health status.

#### 2.5.2 Potential Benefits

It is possible that a participant may not benefit from trial participation as some will receive placebo. Even though the IVACFLU-S vaccine contains virus strains recommended by the WHO in February 2016 for use in the 2016-2017 Northern hemisphere influenza season [6], there is the possibility that these may not match the circulating strains in the community. Furthermore, the IVACFLU-S vaccine is not licensed and its efficacy is being evaluated in the current trial.

### 3 Study Objectives and Endpoints

### 3.1 Study Objectives

### 3.1.1 Primary Objectives, Phase 2

**Safety:** To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults, 18 to 60 years of age.

### 3.1.2 Primary Objectives, Phase 3

**Safety:** To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent split virion, inactivated influenza vaccine in adults, 18 to 60 years of age.

**Immunogenicity:** To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single intramuscular dose of IVACFLU-S seasonal trivalent split virion, inactivated influenza vaccine in adults, 18 to 45 and 46 to 60 years of age.

# 3.1.3 Secondary Objective, Phase 3

**Immunogenicity:** To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single dose of IVACFLU-S seasonal trivalent split virion, inactivated influenza vaccine in adults with and without pre-existing Hemagglutination Inhibition (HAI) antibody

#### 3.2 Study Outcome Measures (Endpoints)

### 3.2.1 Primary Endpoints

#### A. Primary Safety Endpoints, Phase 2 and 3

The number and proportion of participants reporting the following events:

Protocol No: IVACFLU-S-0203 536 Dated: 12 March 2018


- A. Solicited local adverse events, including redness / erythema, swelling / induration, pain within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- B. Solicited systemic adverse events, including fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- C. Unsolicited Adverse Events (AEs) occurring within 21 days post vaccination.
- D. Serious Adverse Events (SAE) occurring during the entire study period (Days 1-91).

### B. Primary Immunogenicity Endpoint, Phase 3

- A. Number and percentage of participants by age groups (18-45, 46-60) with seroconversion against each of the 3 vaccine antigens post-vaccination. Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
  - pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or
  - pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 22
- B. Number and percentage of participants by age groups (18-45, 46-60) with a HAI antibody titer ≥1:40 to each of the 3 vaccine antigens measured on Day 22 post vaccination
- C. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens
- D. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/prevaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens

# 3.2.2 Secondary Immunogenicity Endpoints, Phase 3

- A. Number and percentage of participants by age groups (18-45, 46-60) who develop at least a four-fold increase in HAI antibody titer to each of the vaccine antigen post vaccination measured on Day 22 by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.
- B. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.

Protocol No: IVACFLU-S-0203 537 Dated: 12 March 2018


C. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/pre-vaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.

# 4 Study Design

IVACFLU-S, Phase 2/3

# 4.1 Study Design

This is a phase 2/3, double-blind, randomized, placebo-controlled trial to evaluate the safety and immunogenicity of a single dose the IVACFLU-S seasonal trivalent inactivated influenza vaccine in male and female, ages 18 to 60 years old. Phase 2 will be conducted at 1 site of Long An and will involve 252 participants randomized to receive either IVACFLU-S or placebo at a ratio of 5:1. Following determination of safe to proceed based on PSRT review of Day 8 safety data from all Phase 2 participants and with approval from Vietnam Ministry of Health (MOH), Phase 3 enrollment will commence at 2 sites of Long An and Dong Nai. The Phase 3 components will include 636 participants randomized to receive either IVACFLU-S or placebo at a ratio of 5:1. Randomization of both Phase 2 and 3 volunteers will be stratified by age group as per schema below (Table 15). The sample size takes into account a dropout rate of 5% in the vaccine group to have at least 200 participants in phase 2 and 500 participants in phase 3 at the end of the study.

Table 15: Schema for randomization

| Age<br>group | IVACFLU-S | Placebo | Total |
|--------------|-----------|---------|-------|
| Phase 2 | | | |
| 18 - 45 | 105 | 21 | 126 |
| 46 - 60 | 105 | 21 | 126 |
| Phase 3 | | | |
| 18 - 45 | 265 | 53 | 318 |
| 46 - 60 | 265 | 53 | 318 |

Figure 1: Enrollment and schedule of trial activities

1110.1V1101E0-5-0203 530 Euled. 12 Millen 20




Total study participation duration for one participant: about 91 days

IVACFLU-S, Phase 2/3

Figure 2: Summary of study design

<sup>\*</sup>At Ben Luc site in phase 3, sera samples will be collected prior to vaccination on S1/D1 and D22

IVACFLU-S, Phase 2/3


Date: 09/02/2017




Phase 3:



Protocol No: IVACFLU-S-0203 540 Dated: 12 March 2018


Safety will be assessed in all Phase 2 and 3 participants through Day 91. Immunogenicity will be assessed only in Phase 3 participants. Blood samples will be collected at Day 1 before vaccination in a subset of 252 individuals randomized at one of the study sites to get evaluable samples from at least 200 vaccine recipients (100 each from both age groups) and 40 placebo recipients (20 each from both age groups) and 21 days after vaccination.

# 4.2 Design Rational

Inactivated influenza vaccine has a well established safety profile having been prescribed to millions of individuals globally, including children, the elderly, pregnant women, individuals with chronic disease and immune suppression. Inactivated influenza vaccine also has well established international guidance including quantification of antigen, manufacturing, testing specifications for final bulk and final products, and requirements for national control authorities [15,16]. Because of predictable immunogenicity, dose finding studies of traditional, non-adjuvanted inactivated influenza are often not required. In agreement with National Regulatory Authorities (NRAs), several manufacturers have initiated pivotal licensure Phase 3 inactivated influenza vaccine trials after encouraging safety and immunogenicity data from Phase 1 without conducting Phase 2 studies. Subsequent to NRA approval, these vaccines received or were submitted for WHO prequalification. This approach towards clinical development and licensure of influenza vaccine was presented by the WHO at the IVAC-Vietnam MOH (representatives from Administration of Science, Technology and Training (ASTT)) consultative meeting conducted on 1 March 2016. A follow-up consultative meeting with the ASTT representatives, MOH held on 20 April 2016 included presentation of the IVACFLU-S Phase 1 safety and immunogenicity data; and feedback by MOH of a preliminary P2/3 study design. Based on the Phase 1 results and experience of licensure procedures from other manufacturers and countries that did not include Phase 2 trial, the ASTT representatives, MOH endorsed this current Phase 2/3 design and that the immunogenicity data will be based on HAI only and that evaluation of efficacy will be based on HAI immunogenicity results instead of protective efficacy.

With this seamless phase 2/3 design, the transition procedure from the phase 2 to the phase 3 will be as follows:

- Investigator will prepare the interim study report with information on trial performance, participant dispositions, demographic and key baseline characteristics, blinded data on solicited AEs and unsolicited AEs (please see the interim study report template in the appendix C) until day 8 of the last participants of the phase 2.
- This report will be submitted to the IRB of PI HCM and then to MOH IEC for expedited review and approval in order to check if there is any concern on the safety or trial performance before moving to the phase 3.
- The tentative break for the review by both committees is about 8 weeks since the last participants in the phase 2 complete the D8 visit.

# 4.3 Study sites

The Phase 2 of this study will be conducted in District Health Center (DHC) of Ben Luc, Long An


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 541 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Province. The Phase 3 of the study will be conducted at 2 sites: District Health Center (DHC) of Ben Luc, Long An Province and District Health Center (DHC) of Long Thanh, Dong Nai Province. In both phases of the study, most of study activities will be conducted in the District Health Centers (DHC) of Ben Luc and Long Thanh. Study subjects will be transported by car to DHCs for study visits. District Health Centers and District Hospitals of Ben Luc and Long Thanh are very close to each other which makes the referral convenient in case of any medical emergency.

The Preventive Medicine Center (PMC) of Long An province and District Health Center (DHC) of Ben Luc district have been satellite sites for several vaccine clinical trials (including phase 1 of H1N1 and A/H5N1 influenza vaccines by IVAC) conducted in collaboration with Pasteur Institute in Ho Chi Minh city (PI HCMC). The staff of the DHC, as well as the staff of PMC, have experience in implementing vaccine trials. They also have experience in working with contract research organizations (CROs). The Preventive Medicine Center (PMC) of Dong Nai province and District Health Center (DHC) of Long Thanh district have some experience in conducting epidemiological studies and surveillance such as Dengue and diabetes. The DHCs of both districts manage and control the Expanded Program for Immunization (EPI) program and have pre-qualified WHO cold chain equipment for vaccine storage.

# 5 Study Enrollment and Withdrawal

### 5.1 Description of Participants, Source of Participants

This trial will enroll approximately 888 male and female adults age 18 to 60 years from the Long An and Dong Nai Provinces in Vietnam. Pregnant women, breast feeding women and children are excluded from the study.

The study staff will work through the appropriate health district and commune health workers to recruit potential participants, using IRB-approved methods. For recruitment, each village keeps population/household register books that contain information on the composition of each family in the village. The commune staff will work with population collaborators/village health workers to make a list of potential study participants from these register books to identify which families to approach. They will go household to household and use information from the protocol (specifically the "Information Sheet" from the consent document) to highlight the broad concepts of the study and eligibility criteria. They will assess interest of potentially eligible people and create a list from their household visits. These people will be invited to an information meeting to learn more about the study. After the information session, each person will have a 1:1 meeting with the study Pls to further discuss the trial and ask any questions they have. The investigator will assess the potential participant's understanding of key aspects of the study, such as the voluntary nature of study participation and potential risks and benefits, using an assessment of understanding. The investigator will review with the particiant any answers they did not understand in order to clarify any misunderstandings. Only after that will the participant sign the ICF, if they are interested.

Protocol No: IVACFLU-S-0203 542 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017


The study staff will follow inclusion/exclusion criteria to determine eligibility. Screening will be conducted on all people interested in joining the study who have signed the study consent, and their results will be reviewed with them, regardless of eligibility.

### 5.2 Participant Inclusion Criteria

All participants must meet all of the following criteria to be considered eligible to participate in the study:

- Aged 18 through 60 years on the day of screening/enrollment.
- Literate (by self-report) and willing to provide written informed consent.
- Able to attend all scheduled visits and to comply with all trial procedures.
- Healthy or medically stable, as established by medical history and physical examination. For
  individuals with medical conditions, symptoms/signs, if present must be stable under
  controlled or unchanged for the past 3 months. If medication is used to treat the condition, the
  medication dose must have been stable for at least 1 month preceding vaccination.

### For female participants:

Not breastfeeding or pregnant (based on negative urine pregnancy test) or plan to become
pregnant up to Day 22. Women who are not surgically sterile (hysterectomy or tubal
ligation) or post-menopausal for more than 1 year must have negative pregnancy test and,
be willing to utilize reliable birth control measures (intrauterine device, hormonal
contraception, condom or diaphragm with spermicide) through the Day 22 visit.

## 5.3 Participant Exclusion Criteria

Participants meeting any of the following criteria will be excluded from participation:

- Current or recent (within two weeks of enrollment) acute severe illness with or without fever.
- Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
- Receipt of any non-study vaccine within 4 weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 22 visit.
- Received seasonal influenza vaccine in last 6 months
- Receipt of immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 22 visit.
- Known or suspected congenital or acquired immunodeficiency.
- Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, ≥ 0.5 mg per kg per day; topical steroids are allowed.)

Protocol No: IVACFLU-S-0203 543 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


- Unstable illness by history or physical examination, that in the opinion of the investigator, might interfere with the conduct or results of the study or pose additional risk to the participant.
- Hypersensitivity after previous administration of any vaccine.
- Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein, and rubber (from the vaccine vial stoppers).
- Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion.
- Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
- Current alcohol or drug addiction that in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
- · History of Guillain-Barré Syndrome
- Neoplastic disease or any hematologic malignancy.
- Any condition that, in the opinion of the investigator, would increase the health risk to the
  participant if he/she participates in the study, or would interfere with the evaluation of the study
  objectives.

### 5.4 Treatment Assignment Procedures

### 5.4.1 Randomization Procedures

This is a double-blind, randomized, controlled trial with 2 groups: vaccine and placebo. The ratio of vaccine to placebo recipients will be 5:1. Each participant will be assigned a unique screening number assigned by the investigator after signing the informed consent. After an individual is determined to be eligible for study participation, the participant will be randomized according to age group by assigning a unique participant identification number sequentially in ascending order from the randomization schedule.

The complete randomization schedule that contains the participant identification number and the corresponding randomization assignment will be produced using computer software prior to the initiation of the study.

The Investigator will maintain a screening/enrollment log. The log will contain essential information including participant name, date of screening, gender, date of birth, whether or not the participant meets eligibility criteria, whether participant is enrolled and date, and if not enrolled, reason why the participant is not enrolled or not randomized.

Once a participant identification number has been assigned to a participant, it will not be used again. Additional participants may be randomized into the study at the discretion of the sponsor in the case of any participant who is randomized but does not receive any study vaccine.

Protocol No: IVACFLU-S-0203 544 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### 5.4.2 Blinding and Unblinding Procedures

The randomization will be conducted by an organization or individual not involved in the conduct of the study.

The randomization lists for participants will be used by IVAC to label study vaccine and placebo vials and then will be immediately sealed. It will be opened only after the clinical trial database is declared complete and locked. In the case of any unblinding, researchers must report this in writing to the overseeing Ethics Committee.

The vaccine and placebo vials will be packaged and labeled in such a way that they have similar appearance. The labeling will be done at IVAC before study vaccine and placebo are shipped. Study product injected into each participant will be recorded on the Case Report Form (CRF) using the exact allocation code for each product received by each participant.

The allocation codes link treatment identification with each participant via participant identification numbers. These will be maintained in a secure location, by an individual not involved in the conduct of the study. If any participant experiences an SAE possibly related to receipt of study treatment and the investigator determines it is necessary to unblind, treatment allocation to the participant may be communicated to the investigator.

### 5.4.3 Reasons for Withdrawal

Participants in this study receive only one dose of study product, administered at time enrollment, Day 1. Furthermore, the safety follow-up is minimally intrusive and of short duration. Given these factors and the importance of collecting full safety data from all participants, the reasons for terminating from the study should be minimal but may include the following:

- Participant withdraws consent.
- PI decides that termination is in the best interest of the participant.
- The sponsor terminates the study.

# 5.4.4 Handling of Withdrawals

If a participant withdraws from the study for any reason prior to the planned study duration, every attempt is made to document the participant's health status and follow procedures outlined in section 8.3

### 5.4.5 Strategies to Maintain and Recruit Additional Participants

This is a relatively short trial with only one injection and 3 planned in-clinic study visits and one final study visit via telephone per participant. Strategies to maintain retention in the trial include treating them respectfully, making sure they understand the study and potential side effects, and close communication with each participant about how the study unfolds. Given the short duration

Protocol No: IVACFLU-S-0203 545 Dated: 12 March 2018


of the trial and anticipated side effects of the study vaccine, participant withdrawal and loss of follow-up is expected to be low. Participants who discontinue after the trial is closed to enrollment will not be replaced.

### 6 Termination of the Trial

### 6.1 Termination According to the Protocol

Termination of the trial is the date of the last visit (Day 91) of the last participant participating in the trial, according to the trial scheme.

# 6.2 Suspension and/or Premature Termination of the Trial

The trial might be suspended at any time by IVAC, the Vietnam MOH, any ethical review committee overseeing this study, or by the investigator for any safety concern. This includes, for example, and without limitation, an SAE resulting in death or an unusually high rate of SAEs. IVAC may suspend the study in the event that study conduct is found to be below GCP standards.

In the event of new data that indicate an increased level of risk to participating participants, the clinical trial will be suspended until IVAC, the Vietnam MOH, and all ethical review committees have reviewed relevant data and agreed that the trial may continue.

# 7 Study Products

## 7.1 Study Product Descriptions

### 7.1.1 Acquisition

IVAC will provide both the study vaccine and placebo for this trial.

IVACFLU-S is seasonal inactivated, split virion, trivalent influenza vaccine (A/H3N2, A/H1N1, and B), produced in GCP facility by IVAC uses embryonated chicken eggs. This vaccine is purified by sucrose gradient ultracentrifugation (Alfa Wassermann, West Caldwell, NJ), and inactivated with formaldehyde. The following vaccine strains are recommende by WHO for the influenza season of 2016-2017 in northern hemisphere:

- NYMC X-179A (A/California/07/2009) (H1N1)
- NYMC X-263B (A/HongKong/4801/2014) (H3N2)
- NYMC BX-35 (B/Brisbane/60/2008) (B)

The investigator or qualified designated staff member will be personally responsible for vaccine receipt and management. IVAC will determine with the investigator or the designated staff

Protocol No: IVACFLU-S-0203 546 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


member, the date(s) and time(s) of delivery of vaccine to the study clinic. Study vaccine and placebo, manufactured by IVAC, will be supplied to the study clinic by IVAC under controlled temperature conditions.

# 7.1.2 Formulation, Packaging and Labeling (Seasonal influenza vaccine, IVACFLU-S)

IVACFLU-S is formulated to contain 15 mcg hemagglutinin (HA) from each of the three vaccine strains per 0.5 mL dose, and filled in single dose vials. Each 0.5 mL dose may contain residual amounts of formaldehyde (not more than 0.02%).

IVACFLU-S is a transparent, colorless or opaque white solution, sterile. Antibiotics are not used in the manufacture of IVACFLU-S. IVACFLU-S does not contain latex. The future package insert will describe the vaccine as follows:

| Product name: | Seasonal Influenza Vaccine |
|---|---|
| Trademark: | IVACFLU-S |
| Active substance: | Surface antigen containing hemagglutinin (HA) |
| Formulation: | 15 $\mu$ g (mcg) HA of each of the three strains in 0.5* mL PBS pH 7.2 |
| | *Volume is slightly higher to allow 0.5mL to be extracted |
| Product form: | Trivalent, purified split virion, inactivated |
| Pharmaceutical form: | Injectable biologic |
| Administration route: | Intramuscular (IM) |
| Dosage: | 0.5 mL per dose |
| Storage: | From + 2°C to+ 8°C, avoid freezing |

## <u>Placebo</u>

Placebo is the Phosphate Buffered Saline (PBS) manufactured by IVAC with pH 7.2, will also be in 0.5 mL single-dose vials. The formulation is as follows:

| NaCI: | 4.500 mg |
|------------------------------------------------------|----------|
| Na <sub>2</sub> HPO <sub>4</sub> .2H <sub>2</sub> O: | 0.685 mg |
| NaH <sub>2</sub> PO <sub>4</sub> .2H <sub>2</sub> O: | 0.186 mg |
| Water For Injection (qs): | 0.5 mL |

# **Packaging**

Protocol No: IVACFLU-S-0203 547 Dated: 12 March 2018


Date: 09/02/2017

IVACFLU-S, Phase 2/3


IVACFLU-S vaccine and placebo will be filled in glass vials at a dose volume of 0.5 ml, and covered with a pharmaceutically acceptable rubber stopper, sealing aluminum cap and single-use flip-off plastic lid. Packaging will be done to assure that the vials are intact and vaccine of high quality. A continuous temperature data logger will be placed inside each carton box to monitor product temperature during the process of transportation, storage, and delivery of the product. The carton boxes will also be labeled with "product to be used for clinical trial purposes only" and information on the product storage temperature (from +2°C to +8°C).

The study product must not be used if the package or labeling appears to be tampered with, the label is illegible or the physical properties (color and transparency) are altered.

Picture of vaccine vial and box:



Picture of placebo vial and box:



Sample of blinding label:

548 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018


Date: 09/02/2017




# 7.1.3 Stability and Storage

IVACFLU-S, Phase 2/3

Study product must be stored at a temperature between +2 degrees Celsius (°C) to +8°C. The shelf-life is 12 months in that condition. Storage temperature must be monitored daily and documented on an appropriate form. Back-up power or storage must be available in case of primary power failure. Study vaccine and placebo must never be frozen. Their temperature will be monitored at the manufacturer, during transport, and at the clinical trial site.

In certain instances during transportation and storage for e.g. at some point during movement of IP from the IVAC cold store to the refrigerated truck, from refrigerated truck/fridge to cold boxes or vaccine carriers etc., study product may be exposed to temperatures outside recommended storage temperature range. If the study product is exposed to the temperature not exceeding 22°C for less than 10 minutes and the number of such temperature excursions are no more than 5 times, then the study product can be used. In case of other accidental disruptions of the cold chain, the products may not be administered and the investigator or the responsible person should contact IVAC to receive further instructions. In such cases, the investigator must receive written consent (through facsimile or emailed, scanned copy) of IVAC before any study product may be used.

### 7.1.4 Lot number, Expiry date, Quality control results of study vaccine lots

In 2016, IVAC had produced 3 lots of study vaccine which are 004-01-16, 005-01-16, 006-01-These vaccine lots were tested by National Institute for Control of Vaccines and Biologocals (NICVB) and met the quality requirement with corresponding certification numbers 00416/VXVR-NC, 00516/VXVR-NC and 00616/VXVR-NC dated 22/12/2016; and one lot of placebo 007P-01-16 was also tested by NICBV with certification number 00716/VXVR-NC dated 29/12/2016.

The vaccine lot number IVACFLU-S 004-01-16 (manufacturing date 29/11/2016, expiration date 05/12/2017) and placebo lot number VACFLU-S 007P-01-16 (manufacturing date 02/12/2016, expiration date 05/12/2017) were used as study materials in this phase 2/3 clinical trial. Details on the test results of these lots are in the appendix E "Quality certification by NICBV" for the study product lots.

Other detailed information on the 2 study product lots can be found in the Investigator Brochure (IB).


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 549 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### 7.2 Dosage, Preparation and Administration of Study Products

# 7.2.1 Dosage and Schedule

A single dose level of IVACFLU-S will be evaluated in this study. The dose will be a total of 0.5 mL containing 15 mcg HA for each component. The vaccine is to be delivered intramuscularly preferably into the deltoid of the non-dominant arm.

# 7.2.2 Precautions and Warnings

- IVACFLU-S is only to be used for adults 18 to 60 years of age participating in this study who meet the inclusion/exclusion criteria. It is forbidden to use the vaccine for any other purpose.
- 2. Strict compliance with the regulations of the MOH on the use of vaccines and biologicals is required.
- 3. Vaccination must be intramuscularly preferably into the deltoid of the non-dominant arm.
- Study product vials that have had any temperature excursions outside the allowable time/temperature enumerated in section 7.1.3, may not be used. Contact IVAC for further instructions.
- 5. IVACFLU-S or placebo solution is a homogenous preparation, colorless or opaque white. Do not inject if the study product vial appears to have unusual content or if the liquid in the vials has changed color.
- 6. Only health workers who have been trained and have valid certificate of safe immunization for this research study may administer study product to enrolled participants, assuring proper intramuscular injection technique and sterile injection.
- 7. Only one person may be injected with one needle and syringe.
- 8. Study participants must remain in the clinic and be monitored for 30 minutes after vaccination.
- 9. The study vaccination clinic should have adequate facilities for monitoring and treating any reactions. Drugs to treat anaphylaxis must be available, as must specialist doctors for such an emergency. Prompt referral to additional needed facilities must be available.

# 7.2.3 Preparation and Administration

To prepare and administer study product, vaccination facilities and investigators must comply with current Minsitry of Health regulations on vaccination. The step-by-step instructions for the investigator (or delegated staff) are as follows:

- Wash hands or clean hands with hand sanitizer. Prepare the study vaccine/placebo, needles, syringes, and sharps safety box ahead of time.
- Specific study procedures will be developed and include selecting the appropriate vial for each participant, gently shaking the vaccine vial, withdraw the 0.5-mL dose of study vaccine/placebo from the vial using a sterile needle and syringe. Careful records must be maintained to ensure and document that each participant receives the correct dose. Once the dose vial has been penetrated, the withdrawn study vaccine/placebo should be used

Protocol No: IVACFLU-S-0203 550 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


promptly.

- Make sure you have sufficient equipment to provide every participant with a safe injection and to dispose of injection materials safely.
- Make sure you have emergency drug and equipment kits in both the vaccination area and the observation area.
- Greet the participant in a friendly manner. Ask whether he/she has any questions or concerns about injection and respond to his/her questions and concerns in a truthful and pleasant manner.
- Confirm the participant identity.
- Ensure the participant is seated.
- Inform the participant that for consistency in the study, all participants will be vaccinated preferably in the deltoid of the non-dominant arm.
- Use the cotton swab with 70° alcohol to clean and disinfect the site for injection
- Inject intramuscularly the entire contents of the syringe into the deltoid region of the upper arm.
- While the plunger is still depressed, remove the needle from the participant's arm.
- Apply a dry cotton swab with pressure to the injection site.
- <u>Do not recap the needle</u>. Dispose of the needle and syringe in a sharps container. Store the empty vial in a safe place (not the refrigerator) until the end of the study. The vial must not be disposed of until monitors have verified that it is allowed.
- Record the date of vaccination and vaccine vial number on the participant's vaccination CRF.
- Ask the participant to rest for 30 Minutes.
- While the participant is resting, provide the Diary Card, ruler and thermometer and explain how to use them for recording symptoms. Remind them of upcoming phone calls/visits.
- For 30 Minutes following vaccination, observe the participant and ask about the participant's well-being.
- Before the participant leaves, instruct the participant to seek medical assistance if adverse
  events occur that require medical evaluation and treatment.

### 7.3 Modification of Study Product for a Participant

There is no dose adjustment for the product in the study.

# 7.4 Accountability Procedures for Study Product

The study vaccine and placebo will be kept in a secure place in cold storage (with backup power and/or storage) at the District Health Centers segregated from other products. During the study, the investigator or the person in charge of research product management will record information related to the delivery of vaccine and placebo to the trial site, conduct inventory at the trial site, check the number of doses given to the participants, check the number of unused doses. At the end of the study, the site will receive instruction from the Sponsor regarding the final disposition of any remaining study products.

### At the vaccination site

Protocol No: IVACFLU-S-0203 551 Dated: 12 March 2018


On scheduled vaccination days, study vaccine and placebo will be kept in the cold boxes with proper temperature control and monitoring.

Standard procedures will be followed at the trial site to maintain proper transport, receipt, storage and return of study products.

In the case of interruptions of the cold chain other than that described in the section 7.1.3 above, the investigator or qualified designated staff member must contact IVAC to get further instructions. The investigator must receive the written consent from IVAC before clinical trial products can be used.

### 7.5 Assessment of Compliance with Use of the Study Products

Compliance with use of the study products will be closely monitored during the trial by the research team, IVAC and trial monitors.

#### 7.6 Concomitant Medications/Treatment

Concomitant medications for the treatment of pre-existing medical condition, and per AEs / SAEs reporting period outlined in Table 1 and Section 10.3 will be documented throughout the course of the study. Treatment of conditions that are not exclusionary should continue, if needed by the participant. Subsequent changes in concomitant treatment during the trial must also be reflected in the CRF. Women included in the trial who are using hormonal contraception for pregnancy prevention should using these products through Day 22. Use of such products must also be documented in the CRF.

### 7.7 Unauthorized Products

The following products are not authorized to be used during the study:

- 1. Any concomitant medicine or biologic specifically prescribed for the treatment of a condition which is an exclusion criterion for participation in the trial.
- All non-study vaccines or biologics (including blood products). (Can be used after Day 22.)

Other concomitant products are allowed.

Participants will be requested not to take analgesic or antipyretic drugs in a preventive way (before or soon after injection), as such medications might change the reactogenicity profiles of study vaccine and placebo. Participants may take antipyretic drugs after injection, however, to treat a high fever.

Protocol No: IVACFLU-S-0203 552 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


If during the trial a situation arises where there is an adverse reaction or AE requiring treatment and prescription of unauthorized products or products not stipulated by the protocol, then such products may be prescribed. However, IVAC must be informed of such an occurrence within 48 hours. Information on the products (trade name, dosing or change in dosing, indications, start date, and termination date) must be recorded in the CRF.

# 8 Study Schedule; Description of Visits

The total duration for this study is approximately 22 months; with approximately 12 months (Sep 2016 to Sep 2017) for preparation and implementation of both phases of the study; and approximately 10 months for data analysis, CSR completion and review, approval by local IRBs and Ministry of Health. The recruitment and screening is expected to take no more than 3 weeks for phase 2 and 5 weeks for phase 3 study. In both the studies there are 3 scheduled in-clinic visits and one final study visit via telephone.

# The total expected duration of the study:

| First participant enrolled in study | D1 of first participant |
|---|---|
| The last participant enrolled in study | For phase 2: Day 1 of last subject is estimated approximately 3 weeks from Day 1 of first subject |
| | For Phase 3: Day 1 of last subject is estimated approximately 4-5 months from Day 1 of first subject from phase 2 |
| The last participant completes the trial | D91 of last participant |
| Lock database | approximately 4 weeks after D91 of last participant |
| Clinical trial report | Approximately 5 months from database lock |

# 8.1 Screening

Prior to inclusion into the vaccine study, each participant will be screened through medical history interview and general physical examination. Because screening procedures are required to assess eligibility, they will be performed only after a study consent form has been signed. The investigator or designee will record the screening IDs of all participants who enter screening; whether they entered the trial or failed screening, and the reason for screen failure on the screening/enrollment log.


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 553 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### 8.1.1 Screening and Enrollment/Vaccination (S1/D1)

After assessing understanding and obtaining consent for the study, participants will be screened for eligibility through medical history review and general physical examination. Women of child bearing potential will have a urine pregnancy test. Screening and enrollment/vaccination will occur on the same day (S1/Day 1), although there is a 4-day window allowed, if the participant has second thoughts and needs more time to consider trial participation. If S1 and D1 are conducted separately, a targeted (symptom-based) physical exam with vital signs (heart rate, temperature, blood pressure), urine pregnancy test (for women of child bearing potential only), and brief medical history update will be performed on the day of vaccination (Day 1) to ensure continued eligibility

After participants are consented, the following activities will occur:

- 1. The participant will be interviewed to collect baseline demographic data
- 2. A study clinician will interview the participant to collect a detailed medical history.
- 3. For women with child bearing potential, a urine pregnancy test will be done.
- 4. A study clinician will perform a general physical examination. Results will be reviewed by study staff and with the participant to confirm eligibility prior to conduct of further procedures. If a person is considered ineligible based on medical history and physical examination, the study clinician will tell the person that he or she is not eligible.
- 5. For participants at one site in the phase 3 only: Prior to administration of study product to 252participants at the Ben Luc site in the Phase 3, a blood specimen for HAI test will be collected. Specimen collection information must be documented on the CRF. About 5 mLs of blood will be collected. There will be no blood collection in the Phase 2 study.
- 6. The person performing the injection will confirm that the study product about to be injected is the correct one for this participant.
- 7. The participant will be administered one injection of study product in the deltoid muscle, preferably the non-dominant arm. (This may be switched to the dominant arm if the participant desires).
- 8. The participant will be observed for 30 minutes after administration. If the participant experiences an immediate adverse reaction, he/she will be treated and the event will be recorded on the appropriate CRF.
- 9. The participant will be given a Diary Card, thermometer and ruler in which the participant will be asked to record any local and/or systemic reactions that might appear starting from the evening of Day 1 to Day 7. Concomitant medications and other AEs may be recorded on the Dairy Card, too. The participant will be instructed how to use the Diary Card, thermometer and ruler. All relevant explanations should be included in the Diary Card. The Diary Card will also have contact information for the investigators, should the

Protocol No: IVACFLU-S-0203 554 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


participant have any questions. The participant will be informed that a member of the investigator's team will visit the participant the next 24 hours (Day 2) in phase 2 and visit/call in phase 3 and also call her/him 4 days (Day 5) after vaccination to check on the participant's completion of the Dairy Card and participant's well-being.

10. The participant will be instructed that if the participant experiences an AE requiring medical care, the participant should inform the investigator as soon as possible and seek medical care as appropriate. If the participant visits a health care provider, the participant should be sure to inform the health care provider of participation in this study and provide the health care provider with the investigator's contact information.

# 8.2 Follow-up Periods

# 8.2.1 First Week after Injection (Days 1 to 7)

- 1. The participant will complete the Diary Card daily, starting on the evening reporting any local or systemic reactions experienced and medications taken.
- 2. The participant will have been instructed that if he/she experiences an AE requiring medical care, the participant should inform the investigator as soon as possible and seek medical care as appropriate. If the participant visits a health care provider, the participant should be sure to inform the health care provider of participation in this study and provide the health care provider with the investigator's contact information. The participant should obtain in writing the names of medications prescribed by the health care provider.
- 3. One day after vaccination (Day 2) a member of the investigator's clinical team will visit the participant in phase 2 and visit/call in phase 3 and also call on 4 days (Day 5) to check that the participant is correctly completing the Diary Card and to check on the participant's well-being. If local and systemic reactions suspected to be Grade 3 or higher are reported, the participant will be requested to return to the study clinic for evaluation.

# 8.2.2 Seventh Day after Injection (Day 8 ± 1)

- 1. Study staff will confirm participant identity.
- Study staff will review the participant Diary Card and interim history with the participant and inquire about any new medical events since medical histories were last updated. Any AEs that have occurred and meet reporting requirements, will be recorded in the appropriate section(s) of the CRF. Diary Card information will be entered into the database.
- 3. The participant will have temperature, pulse rate, and blood pressure recorded. A study clinician will perform a targeted (symptom based) physical examination and record the information Results will be reviewed by study staff and with the participant.
- 4. The participant will be instructed to inform the investigator as soon as possible if he/she experiences an AE requiring medical care and to seek medical care as appropriate. If the participant visits a health care provider, the participant should be sure to inform the

Protocol No: IVACFLU-S-0203 555 Dated: 12 March 2018

IVACFLU-S, Phase 2/3

NTIAL Date: 09/02/2017


health care provider of participation in this study and give the health care provider the contact information for the investigator.

### 8.2.3 Second and Third weeks after Injection (Days 9-21)

There are no scheduled visits during this period. Participants may be asked to come to the study clinic if the investigator follows up on any laboratory or clinical issue. The participant will inform the study clinic of any medical events and seek medical care as needed. The participant will be instructed to give the contact information of the study investigator in case they consult any health care provider outside the study.

# 8.2.4 Final Visit (Day 22; ± 1)

Day 22 is the last scheduled in-clinic visit for the participants for closing out AEs and reported medications (Phase 2 & Phase 3) and collection of immunogenicity samples for the Phase 3 portion of the study.

- 1. Study staff will confirm participant identity.
- 2. Phase 2 & 3: Study staff will review interim medical histories and concomitant medications with the participant since these were last updated. Results will be recorded in the appropriate section of the CRFs.
- Phase 3 only: Blood specimens from participants who underwent blood collection at enrollment (S1/D1) will be collected for anti-influenza serologic assays. Specimen collection information must be documented on the CRF and in specimen collection logs. About 5 mL of blood will be collected.

#### 8.2.5 Final Study Visit (Day 91; ± 7)

- 1. The participant will be contacted via telephone and identity confirmed.
- Study staff will review interim medical histories and concomitant medications with the participant since these were last updated. No new concomitant medication will be recorded unless it relates to a newly identified SAE.
- 3. Study staff will ask about any medical event that would constitute an SAE since the last visit. No new AE information will be recorded unless it qualifies as an SAE.
- 4. If an SAE is reported, the clinician should record the SAE on the appropriate form, notify the entities who require notification, and refer the participant for treatment of the SAE, if warranted.

After recording the information, the participant will be discharged from the study.


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 556 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### 8.3 Early Termination Visit

If a participant withdraws from the study for any reason prior to the planned study duration, every attempt is made to complete the following:

- Report of local and systemic reactogenicity and AEs are reviewed by PI (or designee).
- For participants (from one site in the phase 3) who withdraw from the study prior to scheduled immunogenicity laboratory testing, specimens are obtained for immunogenicity analysis if the participants agree to do so.
- Diary Card information is reviewed with the volunteer in detail by site staff, if in use since the last visit.
- Injection site(s) examination and a full physical examination are performed (if indicated).

IVAC must be informed within 48 hours of all instances of the premature termination of a participant's participation in the trial.

If the participant develops a reaction to study vaccine which the investigator believes threatens the participant's well-being, the withdrawn participant must be treated or transferred to a treatment facility.

#### 8.4 Unscheduled Visits

Participants may present to the study center during operating hours for an unscheduled visit should they experience any AE or if the participant's condition requires medical intervention. Data for any examinations or other procedures performed on the participant at an unscheduled visit must be recorded on the appropriate CRFs.

### 9 Study Evaluations

## 9.1 Clinical Evaluations

## 9.1.1 Vital Signs

- Temperature in degrees Celsius (recorded to the nearest 0.1 degree) will be measured by oral thermometer.
- Blood pressure in mm of mercury and pulse rates in beats per minute will be measured by automated device or manually

### 9.1.2 Medical History

At enrollment, medical histories must be thoroughly reviewed with the participant. The following medical conditions, in particular, will be assessed:

Protocol No: IVACFLU-S-0203 557 Dated: 12 March 2018


- Current or recent (within two weeks of enrollment) acute illness with or without fever.
- Recent vaccination history.

IVACFLU-S, Phase 2/3

- Recent receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy within 3 months before enrollment.
- Hypersensitivity of any kind, but particularly to vaccines.
- Clinically relevant history of renal, gastrointestinal, hepatic, cardiovascular, hematological, dermatological, endocrine, neurological, pulmonary or immunological diseases.
- Seizures, including history of febrile seizures, or any other neurologic disorder.
- Known or suspected immunologic impairment of any kind.
- Known HIV infection.
- Known active TB disease.
- Alcohol or drug use.
- Concomitant medications that are ongoing (including trade name, dosing, indications, start date).
- For women, pregnancy, menstrual and contraceptive history and/or history of surgical sterility.

# 9.1.3 Physical Examination

### **General Physical Examinations**

Qualified study clinicians will conduct a physical examination of all participants at S1/D1. This physical examination will include the following:

- · Recording of general appearance
- Physical examination of all organ systems. This includes the following:
  - o neurologic examination, including cranial nerve examination
  - chest auscultation
  - examination of lymph nodes (axillary and cervical)
  - o heart auscultation
  - o abdomen palpation (to check for liver size)
- Measurement of the following vital signs:
  - body temperature
  - o blood pressure
  - o pulse/heart rate
- \* Grade 1 elevated blood pressure (140 to < 160 mmHg systolic OR 90 to < 100 mmHg diastolic) will not be considered to be exclusionary at screening, unless judged to be clinically significant by the PI.

#### **Targeted Physical Examination**

The targeted Physical examination focuses on symptoms reported by the participant and the presence or absence of local and systemic reactogenicity. If no symptoms are reported by the participant, the Targeted PE does not need to be performed. The exam will be made by a clinician on Day 1(only if D1 is on a different day from S1) and Day 8. Evaluation must be made prior to administration of injection of study product if done on Day 1.

Protocol No: IVACFLU-S-0203 558 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017


#### 9.1.4 Injection Site Examination

Assessment of local Injection site reaction 30 minutes after vaccination will be done by trained study personnel and graded for severity according to the toxicity grading table in Appendix A

- Erythema /redness will be examined under proper lighting conditions and measured with a ruler if present.
- Swelling/induration will be examined by palpation and visual inspection under proper lighting conditions. The examiner may temporarily mark skin at margins of visible swelling/induration, then measure with a ruler the maximum diameter
- Pain will be assessed by (a) inquiring as to whether there is significant discomfort at rest and/or (b) whether movement of the injection site causes discomfort, impacts limb movement or daily activity.

### 9.2 Laboratory Evaluations

### 9.2.1 Clinical Laboratory Evaluations

### **Pregnancy Test**

In order to confirm pregnancy status of females with potential to become pregnant, a qualitative human chorionic gonadotropin (hCG) test will be done on a urine sample. Pregnancy testing will be done on Day S1/D1, before vaccination. If Day S1 and D1 are conducted separately, the urine pregnancy test most be done on both visits. No injection of study product may be given to a woman without a pregnancy test being done and to any woman with a positive pregnancy test.

There are no safety laboratory tests in the study.

### 9.2.2 Special Assays

The HAI is the most frequently used serologic test for determining immunologic response to influenza vaccination. Serum specimens will be tested for the presence and titer of HAI antibodies to each one of the influenza strains represented in the vaccine. This testing will be performed by VisMederi srl laboratory, Siena, Italy, by using a validated assay. For these assays, serum specimen collection will occur on Days 1 and 22. Sample collection on Day 1 must occur prior to administration of study product.

## 9.2.3 Preparation, Processing, and Transport Specimens

#### **Blood Specimens**

Blood (serum) will be collected for HAI antibody serology.

### Collection of Blood

Following universal precautions, blood will be collected from the forearm into tubes appropriate for collection of serum for HAI assay. Volumes of blood required for HAI assays at different timepoints are shown in the table below.


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 559 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | Collection<br>Tube | Volume of blood | S1/D1<br>(pre-vac) | D22<br>(Last study<br>visit) |
|---|---|---|---|---|
| Serum for anti-<br>influenza<br>serologic assays | Serum<br>separator | 5 mL tube | <b>√</b> | <b>✓</b> |

(The total volume of blood planned to be collected from each participant during the course of the study will be less than 15 milliliters.)

#### Processing of Sera

Immediately after collection, the blood specimen tube will be made to stand upright to clot at room temperature before transport to the laboratory at Pasteur Institute. At the laboratory, specimens will be centrifuged before division.

#### Division of Sera

Serum specimens for anti-influenza serologic assays will be divided. Specimen division should be performed for only one participant at a time to avoid mixing blood tubes. Each serum specimen will be divided into 4 aliquots as follows:

- 1st aliquot: 0.6 mL for HAI assay
- 2<sup>nd</sup> aliquot: 0.6 mL for back up 1 for HAI assay
- 3<sup>rd</sup> aliquot: 0.6 mL for back up 2 for HAI assay
- 4<sup>th</sup> aliquot: the remaining serum sample for back up and archive
- The study participant number, date of collection, blood specimen number, number of divisions obtained, and the date and time of division will be specified on a serologic specimen log form.
   On this form, comments may be made on the quality of specimens (e.g., hemolyzed, contaminated, etc.).

## Conditions for Transport and Storage of Sera

Serum specimens for anti-influenza serologic assays will be immediately put in the freezer equal or lower than -20°C after division and stored at this temperature until use. All handling will be done to prevent unnecessary freeze-thaw cycles (i.e., back-up samples should not be thawed unless required for testing). Temperature monitoring will be done to assure maintenance of cold chain and specimen quality.

#### **Urine Specimens**

Urine will be collected for pregnancy testing on visit S1/D1 (prior to vaccination). If D1 is conducted separately from S1, a urine pregnancy test should be done at each visit and prior to vaccination on D1.

No urine specimens will be stored after testing.


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 560 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# 10 Assessment of Safety and Adverse Events

#### 10.1 Adverse Events

An Adverse Event is any unfavorable and unintended sign (including a designated out-of-range laboratory finding), symptom, or disease temporally associated with the use of a study product, whether or not considered related to the product. The occurrence of an AE might come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care. Information to be collected on AEs includes event description, time of onset, clinician's assessment of severity, relationship to study product, and time of resolution/stabilization of the event. AE assessment should be made only by those with the training and authority to make a diagnosis.

Any medical condition that was present at the time that the participant was enrolled should not be reported as an AE, but should be reported as a pre-existing condition on the Medical History Form. However, if this condition occurs with greater frequency or severity during the study, it should be recorded as an AE

## 10.1.1 Solicited Local and Systemic Adverse Events

- Solicited adverse events are pre-specific local and systemic adverse events that are common
  or known to be associated with vaccination that are actively monitored as indicators of vaccine
  reactogenicity. Investigators will not be required to assess causality of solicited adverse
  events if the onset is during the solicitation periods. If a solicited adverse event progresses
  beyond the solicited period, it will continue to be reported as a solicited adverse event. If the
  solicited adverse event occurs after the solicitation period it will be reported as an unsolicited
  AE.
- For this trial, solicited local and systemic AEs will be assessed by study staff 30 minutes after vaccination then daily for 7 days by the participants. Participants will be provided a thermometer, ruler and a diary to record the presence or absence of solicited AEs, severity of the solicited AE and use of concomitant medication. The severity of the solicited local and systemic adverse events will be graded using the Toxicity Table for Grading Adverse Events (Appendix A). The specific solicited local and systemic adverse events that will be reported for this trial are:

## • Solicited local adverse event (at site of injection):

- Erythema / redness based on size in cm
- Swelling / induration (hardness at site of injection ) based on size in cm
- Pain

Protocol No: IVACFLU-S-0203 561 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### Systemic Reactions:

- Fever--Body temperature
- Fatigue/malaise
- Generalized muscle aches
- Joint aches
- Chills
- Nausea
- Vomiting
- Headache

### 10.1.2 Unsolicited Adverse Events

Unsolicited adverse events are any AEs that occur any time after the vaccine/placebo is given (temporally related to study product), whether or not deemed "related" to the product, and are not solicited (specifically asked of the participant). Unsolicited AEs can be observed by study staff while the participant is at a clinic for a study visit or reported by the participant at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination will be recorded as an unsolicited AE.

# 10.2 Serious Adverse Events

An SAE is defined as an AE that meets one of the following conditions:

- Death.
- Life-threatening (participant at immediate risk of death.) (The term "life-threatening" in the
  definition of "serious" refers to an event in which the patient was at risk of death at the time of
  the event; it does not refer to an event that hypothetically might have caused death if it were
  more severe).
- Requires inpatient hospitalization or prolongation of existing hospitalization.
- Results in congenital anomaly/birth defect. (Only in the case of a woman becoming pregnant during the study period after administration of at least one injection of study product. All pregnancies must be followed to term and outcome reported to IVAC and regulatory agencies.)

Protocol No: IVACFLU-S-0203 562 Dated: 12 March 2018


- Results in a persistent or significant disability or incapacity.
- Important medical events that might not result in death, be life-threatening, or require
  hospitalization might be considered SAEs when, based upon appropriate medical judgment,
  the event might jeopardize the well-being of the participant and require medical or surgical
  intervention to prevent one of the outcomes listed above. (Medical and scientific judgment
  should be exercised in deciding whether reporting these events is appropriate.)

All SAEs must be reviewed and evaluated by a study clinician to determine relationship to study vaccine as outlined in Section 10.5 and recorded on an SAE form and reported, as specified in Section 10.9. All such SAEs should also be followed until satisfactory resolution or until the investigator deems the event to be chronic or the participant to be stable.

## 10.3 AE/SAE Reporting Period and Parameter

Safety events are reported from the time of study injection (Day 1) through completion of the study at Day 91. Specifically, solicited AEs to assess local and systemic reactogenicities will be collected at 30 minutes and then daily for 7 days thereafter. If a solicited AE starts during the 7 days post vaccination period and continues beyond the 7 days it will continue to be reported as a solicited AE. SAEs will be reported from Day 1 through the end of the study at Day 91. Unsolicited AEs will be reported from Day 1 to Day 22 inclusive.

### 10.4 Severity of Event

IVACFLU-S, Phase 2/3

This study will use the Toxicity Table for Grading Adverse Events (see appendix A). For events not included in the table, the following guidelines will be used to quantify intensity <u>not included</u> on the table, the following guidelines will be used to quantify intensity:

| Grade | Description for grading when an event is not on Toxicity Table |
|---|---|
| 1 (Mild) | Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated. |
| 2 (Moderate) | Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated. |
| 3 (Severe) | Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated. |
| 4 (Life threatening) | Potentially life-threatening symptoms causing inability to perform basic self-<br>care functions with intervention indicated to prevent permanent impairment,<br>persistent disability, or death. |

Protocol No: IVACFLU-S-0203 563 Dated: 12 March 2018


Date: 09/02/2017

IVACFLU-S, Phase 2/3


**Basic Self-care Functions – Adult**: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

**Usual Social & Functional Activities – Adult:** Activities which adults perform on a routine basis and those which are part of regular activities of daily living, for example going to work, shopping, cooking, use of transportation or pursuing a hobby.

### Changes in Severity of an Event

Changes in the severity of an AE should be documented to allow an assessment of the duration of the event at each level of intensity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

### 10.5 Relationship to Study Vaccines

The clinician's assessment of an AE's relationship to study product is part of the documentation process. The clinician must determine whether there is a reasonable possibility that the investigational product(s) caused or contributed to an AE. It is essential to have the best assessment possible as to whether adverse events are related to investigational products.

The relationship assessment, based on clinical judgment, should rely on the following:

- A temporal (time-based) relationship between the event and administration of the investigational product
- A plausible biological mechanism for the investigational product to cause the AE
- A possible alternative etiology for the AE
- Previous reports of similar AEs associated with the investigational product or other vaccines in the same class

To help assess, the following guidelines will be used:

<u>Related</u> – There is a reasonable possibility that the study vaccine caused the AE. "Reasonable possibility" means that there is evidence to suggest a causal relationship between the study product and the AE.

<u>Not Related</u> – There is not a reasonable possibility that the administration of the study product caused the event.

Any solicited local or systemic reactogenicity that occurs during the 5-day period post-injection is automatically regarded as related.

Protocol No: IVACFLU-S-0203 564 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


### 10.6 Follow up of AE

All reported AEs should be followed until resolution or stabilization, or until the participant's participation in the study ends. Participants who have an ongoing study product-related SAE at study completion or at discontinuation from the study will be followed by the PI or his designee until the event is resolved or determined to be irreversible, chronic, or stable by the PI.

## 10.7 General Guidelines for Recording AEs

To improve the quality and precision of acquired AE data, the PI should observe the following guidelines:

- Whenever possible, use recognized medical terms when recording AEs on the AE CRF. Do not use colloquialisms and/or abbreviations.
- If known, record the diagnosis (i.e., disease or syndrome) rather than component signs, symptoms and laboratory values on the AE CRF (e.g., record congestive heart failure rather than dyspnea, rales, and cyanosis). However, signs and symptoms that are considered unrelated to an encountered syndrome or disease should be recorded as individual AEs on the CRF (e.g., if congestive heart failure and severe headache are observed at the same time, each event should be recorded as an individual AE).
- AEs occurring secondary to other events (e.g., sequelae) should be identified by the
  primary cause. A "primary" AE, if clearly identifiable, generally represents the most
  accurate clinical term to record on the AE CRF. If a primary serious AE (SAE) is recorded
  on an SAE CRF, events occurring secondary to the primary event should be described in
  the narrative description of the case.

For example:

Orthostatic  $\rightarrow$  Fainting and  $\rightarrow$  Head  $\rightarrow$  Neck pain hypotension fall to floor trauma

The primary AE is orthostatic hypotension.

- Death is an outcome of an event. The event that resulted in the death should be recorded and reported on the SAE CRF.
- For hospitalizations for surgical or diagnostic procedures, the illness leading to the surgical
  or diagnostic procedure should be recorded as the SAE, not the procedure itself. The
  procedure should be captured in the case narrative as part of the action taken in response
  to the illness.
- Pregnancies are not considered AEs. Participants will be instructed to notify the study team if they become pregnant during the course of the study. They will be recorded on a separate Pregnancy CRF. Pregnancy outcomes that include stillbirth and any congenital anomalies must be reported as SAEs.

Protocol No: IVACFLU-S-0203 565 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 10.8 Unexpected Allergic Reaction

# Immediate Reactions (within 30 minutes)

All participants will be observed for 30 minutes after administration of study product, with appropriate medical treatment readily available in case of an anaphylactic reaction following the administration of study product. Immediate reactions will be assessed by a study physician or appropriately trained medical staff. All reactions that occur during this time will be recorded on the CRF. Any immediate reaction which meets the criteria for an SAE must also be documented on an SAE form.

Emergency medicines will be available at the study clinic to be ready to give first aid if any adverse reactions or events should occur among any participant participating in this research. If anaphylaxis occurs after vaccination, it must be treated in accordance with current MOH regulations on handling anaphylaxis. Treatment for mild reactions after vaccination will be per "Guidance on the treatment of post injection reactions" issued under the Decision No 2535 by Ministry of Health, Vietnam (17). The applied treatment methods must be recorded and kept in the participant file.

# 10.9 Reporting Procedures

#### 10.9.1 Serious Adverse Events

All SAEs must be documented and reported to IVAC or its designate, even if the investigator considers that the SAE is not related to treatment. The study clinician will complete a **Serious Adverse Event Form** within the following timelines of such events:

- All deaths and immediately life-threatening events, whether related or unrelated, will be recorded on the Serious Adverse Event Form and sent by fax or email within 24 hours of site awareness.
- SAEs other than death and immediately life-threatening events (i.e., events resulting in
  hospitalization or prolongation of hospitalization; persistent or significant disability or
  incapacity, or other significant events determined by the investigator to be SAEs), regardless
  of relationship, will be reported via email or fax by the site within 24 hours of becoming aware
  of the event.

IVAC will be primarily responsible for medical monitoring of serious adverse events documented by the investigator. Investigator and PI HCM City will be responsible for reporting the SAEs to local regulatory authorities in accordance with local regulatory safety reporting guidelines. Medical Officers from PATH serving as technical consultants will review all serious adverse events and provide guidance regarding SAE management including classification and reporting. Details for review of serious adverse events and other unanticipated problems will be in an SOP drafted prior to study initiation.

Protocol No: IVACFLU-S-0203 566 Dated: 12 March 2018


#### 10.9.2 Reporting of AEs

Collected SAEs and AEs will be reported to responsible ethical review committees according to their requested timelines. An SOP for reporting to the responsible committees will be developed with reporting requirements and timelines prior to study initiation. It will be the investigator's responsibility to assure that all reportable events are reported to the proper authority or to IVAC and/or its designate in a timely manner and according to the SOP. PATH technical consultants may assist the investigator with regulatory reporting, per the finalized SOP.

### 10.9.3 Other Unexpected Issues/Unanticipated Problems

During study process, if there are any problems related to the trial (unanticipated problems), the Principal Investigator is responsible for reporting to IVAC and PATH to discuss reasonable ways of handling the problem. The Principal Investigator is responsible for reporting any unanticipated problems that affect the health, welfare or rights of study participants or that may impact the integrity of the study data to the ethics committees involved in the review of the research. The Principal Investigator should maintain written documentation of all unanticipated problems and their reporting and resolution.

# 10.9.4 Reporting of Pregnancy

Although women are not tested for pregnancy after vaccination and women are supposed to use effective birth control until Day 22, it is possible that a woman could report a pregnancy during the study. All pregnancies detected among women enrolled in the trial who receive study product must be reported on a Pregnancy Report CRF. All pregnancies must be followed to term and outcome reported to IVAC and regulatory agencies. Unblinding of allocation of treatment of female participants who become pregnant will not occur until after study completion, unless medically indicated.

# 11 Safety Oversight

### 11.1 Protocol Safety Review Team

Routine safety monitoring will be conducted by the Protocol Safety Review Team (PSRT). The PSRT will comprised of at least 4 members: the sponsor Medical Monitor, PATH Medical Officer/s, Contract Research Organization (CRO) Pharmacovigilance Medical Monitor and protocol Principal Investigator (or designate). PSRT members are selected based of their experience and expertise in the conduct and safety oversight of vaccine clinical trials.

During the vaccination phase of the trial, the PSRT reviews blinded cumulative solicited local and systemic reactions and AEs on a weekly basis. Frequencies of review post the vaccination phase will be at the discretion of the PSRT but no less than once a month.

Protocol No: IVACFLU-S-0203 567 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 11.1.1 Expedited Safety Review

Safety events listed in table 1 require expedited PSRT review within 36 hours of submission of the safety information to data management and or SAE reporting system. Members of the PSRT will be notified of these events through the CRO pharmacovigilance system.

| Event and relationship to study agent as assessed | Severity Grade |
|---------------------------------------------------|----------------|
| by investigator or CRO Pharmacovigilance | |
| Medical Monitor | |
| SAE, related | All grades |
| Unsolicited AE, related | 4 |
| Local reactions – erythema or induration | 4 |

### 11.1.2 Study Safety Pauses

This study has no formal pause rules. However if during the weekly or expedited safety reviews the PSRT identifies safety concerns that warrant a safety pause, the PSRT will notify the sponsor. If a decision is made to pause the study, all enrollment will be held pending wider consultation with the PATH, funders and sponsor on whether to lift the pause or discontinued the study prematurely.

IVAC retains the right to temporarily suspend or prematurely discontinue this study at any time for matters related to safety. If the study is stopped or suspended prematurely, IVAC will inform the local principal investigator as well as regulatory authorities about the decision and the reasons for termination or suspension. If such action is taken, all efforts must be made to ensure the safety of the participants enrolled in the study. The principal investigator will assist IVAC in informing the responsible IEC and provide the reason for the suspension or termination. In case of premature study or study clinic closure, the monitor will conduct all activities as indicated in the close out monitoring visit.

# 11.2 Data Safety Monitoring Board

Given the wide global experience with seasonal influenza vaccines and the safety profile observed in the Phase 1 study, there will not be any Data Safety Monitoring Board (DSMB) for this study. The PSRT will be responsible for close safety oversight of the study.

### 12 Monitoring and Auditing

### 12.1 Monitoring Plan

Individuals qualified by education, training and experience will carefully monitor the study. The study monitors (from QuintilesIMS) will periodically contact the site and perform on-site visits. The extent, nature, and frequency of site visits will be based on such considerations as study

Protocol No: IVACFLU-S-0203 568 Dated: 12 March 2018


objectives, study design and complexity, and enrollment rate; periodicity and nature of monitoring activities will be described in the Monitoring Plan. The Monitoring Plan will detail reporting requirements to IVAC to keep it apprised of study progress. Representatives of IVAC or its designees may participate in monitoring visits or visit the study clinic on its own to provide proper oversight.

# 12.2 Set-up Visit (Site Initiation)

The study monitor will contact the site prior to the start of the study to discuss the protocol and data collection procedures with site personnel. Prior to enrollment of participants at the study clinic, specific regulatory documents must be available, including approvals from the Vietnam Ministry of Health and from institutional review boards of the participating institutions. Curriculum vitae for key investigators must also be available. IVAC or CRO will inform the investigator of any additional documents that need to be provided.

### 12.3 Routine Monitoring Visits

Monitoring will be conducted according to an agreed upon Monitoring Plan. The study may use a Risk Based Monitoring approach that will be targeted to issues most critical to the rights and welfare of study participants and the veracity and integrity of study data. The individuals responsible for monitoring the study will periodically review the progress of the study and should have access to all records necessary to ensure the ethical and safe conduct of the study and the integrity/validity of the recorded data.

During site visits and contacts, the monitor will:

- Assess if consent was properly obtained
- 2. Assess adherence to the protocol eligibility criteria
- 3. Look for evidence that randomization was followed
- 4. Look for evidence that blinding was maintained
- 5. Check on study conduct and documentation of procedures/assessments related to the study endpoints:
  - Specimens obtained correctly
  - Specimens labeled correctly
- Check on study conduct and documentation of protocol-required safety assessments, including SAEs
- 7. Ensure that there is documentation of withdrawals and deaths and reasons provided.

As part of study conduct, the Principal Investigator agrees to allow the monitor direct access to all relevant documents and to allocate his/her time and the time of his/her staff to the monitor to
Protocol No: IVACFLU-S-0203 569 Dated: 12 March 2018


discuss findings and any relevant issues. The study consent also makes participants aware that medical records relevant to events in the study may be accessed and viewed by people conducting and overseeing the study.

The Principal Investigator also agrees to allow representatives of IVAC or its designees to occasionally accompany the monitor during site visits.

#### 12.4 Close-out Visit

Upon completion of the study, the study monitor and the investigator will conduct the following activities:

- Data clarification and/or resolution.
- Accounting, reconciliation and disposition of used and unused study products according to the instructions of the sponsor.
- Review of site study records for completeness.
- Ensure study data is handled according to instructions by IVAC.

#### 12.5 Audits and Inspections

For the purpose of compliance with applicable regulatory guidelines IVAC or its designees or national regulatory authorities may conduct a site audit. This could occur at any time from site initiation to after conclusion of the study. If the national regulatory authority requests an inspection, the Principal Investigator must inform IVAC immediately about this request.

The Principal Investigator will allow the auditor direct access to all relevant documents and to allocate his/her time and the time of his/her staff to the auditor to discuss findings and any relevant issues.

# 13 Statistical Considerations

# 13.1 Study Hypothesis

#### Safety:

A single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) will be safe and well tolerated in adults 18 to 60 years of age.

#### Immunogenicity:

A single dose of IVACFLU-S seasonal trivalent split, inactivated influenza vaccine will induce immune responses to each of the three vaccine antigens to meet one or both age group specific Vietnam Ministry of Health licensure requirements.

Protocol No: IVACFLU-S-0203 570 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 13.2 Sample Size Considerations

This is a Phase 2/3 trial with primary objective to evaluate the safety and immunogenicity of one dose of IVACFLU-S. The sample size for this study was selected in response to MOH's requirement for additional safety data from Phase 2 before proceeding to Phase 3 and for primary safety and immunogenicity analysis to satisfy the MOH licensure requirement for influenza vaccine in adults from age 18 through 60. Total sample size for the Phase 2 is approximately 250 participants (at least 200 randomized to vaccine and 40 randomized to placebo). Phase 3 sample size is approximately 650 participants (at least 500 randomized to vaccine and 100 randomized to placebo). The two age groups (18 to 45, 46 to 60) will be equally distributed in both phases of the study. Block randomization will be stratified by site and age group. To account for potential drop-outs (expected to be low) and to address the challenge of stopping enrollment at a precise number due to the large sample size, sample size allows for an overage of approximately 5%. The sample size of this trial reflects guidance and endorsement by MOH at the MOH-IVAC Consultation Meeting held on 20 April 2016.

## 13.3 Safety

There will be 740 subjects randomized to IVACFLU-S arm in the phase 2/3 study; with account of 5% drout-out rate; there would be at least 700 evaluable participants for safety analysis. If no vaccine-related serious adverse events are observed in 700 vaccine recipients, study would able to exclude events occurring at approximately 0.43% based on the upper bound of the one sided 95% Confidence Interval (CI)) using the Clopper-Pearson method. The probability of observing at least one vaccine-related serious adverse event in 700 subjects is 90 % and >95% if the true rate of such events is 0.33 % and 0.43% respectively. The precision of the estimate of AEs judged to be related to IVACFLU-S as bounded by 95% CI is presented in Table 16.

However, the full analysis population will be used for safety analysis, not the assumed number of 700 valuable subject.

Table 16: Exact 95% Confidence Intervals around Potential Number of Study Related Adverse Events

| Sample size | Number of events | 2-sided exact 95% CI |
|-------------|------------------|----------------------|
| 700 | 0 | [0, 0.52*] |
| | 1 | [<0.01, 0.79] |
| | 2 | [0.03, 1.02] |
| | 3 | [0.08, 1.24] |
| | 5 | [0.23, 1.65] |

<sup>\*</sup>one sided,97.5% CI

IVACFLU-S, Phase 2/3


Date: 09/02/2017


#### 13.4 Immunogenicity

The Vietnam MOH guidance on serological immune response requirements [11] for influenza vaccine as summarized in Table 17 is a modification of the EMEA/CPMP serological criteria for assessing seasonal influenza for licensure [18].

Table 17: Vietnam MOH Criteria for Evaluation of Influenza Vaccine Immune Responses

| | Age Group | |
|---|---|---|
| | 18 – 45 | 46 |
| Proportion achieving a HAI titer ≥ 1:40 (seroprotection) | ≥70% | ≥60% |
| Proportion achieving at least 4 fold rise in HAI titer (seroconversion) | ≥40% | ≥30% |
| GMT rise in HAI titer | ≥2.5 times | ≥2.0 times |

Of the three criteria, seroconversion has been the most frequent criteria not meeting licensure threshold [19]. Though the study assumption is based on Phase 1 immunogenicity data for adults 18-45 years of age, we anticipate the immune response in those 46 - 60 will be comparable since significant decline in antibody response is most associated with those who are  $\geq 65$  years of age [20]. Taken together with the immunogenicity results of the IVACFLU-S phase 1 study (section 2.1.6), the sample size consideration for immunogenicity for the study was based on the precision of the estimate of percent of vaccine recipients with HAI seroconversion and seroprotection responses. With a sample size of 100 evaluable vaccine recipients from each age group, the study provides the precision of immunogenicity response as estimated by width of 95% CI of  $\leq \pm 10.2\%$  around the range of estimated response rate (Table 18). An increase in sample size by 50% to 150 provides very limited statistical benefit as it only reduces the maximal width of 95% CI by 1.9% to  $\leq \pm 8.3\%$ . All power calculations were made using 10000 simulations of binomial responses to each strain, based on assumed true response rates and pass/fail criteria. All calculations were made using SAS version 9.3.

Table 18: Observed Response Rate in 100 participants receiving study vaccine and Corresponding 95% CI

| Number of responder (%) | 2-sided exact 95% CI |
|-------------------------|----------------------|
| 90 (90%) | [82.4%, 95.1%] |
| 80 (80%) | [70.8%, 87.3%] |
| 70 (70%) | [60.0%, 78.8%] |
| 60 (60%) | [49.7%, 69.7%] |

Protocol No: IVACFLU-S-0203 572 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017

50 (50%) [39.8%, 60.2%] 40 (40%) [30.3%, 50.3%] 30 (30%) [21.2%, 39.9%]

## 13.4.1 Probability for demonstrating seroconversion criteria for licensure

For the 18-45 year old cohort, if the true seroconversion response to each strain is  $\geq$ 49%, then there is 91% probability that the point estimate for seroconversion to all three strains will be  $\geq$ 40%. Likewise, if the true seroconversion response to each strain is  $\geq$ 60%, then there is 92% probability that the lower bound of the exact 95% CI for seroconversion to all strains will be  $\geq$ 40%. For the older age cohort (46-60 year old), if the true seroconversion response to each strain is  $\geq$ 39%, then there is 93% probability that the point estimate for seroconversion to all three strains will be  $\geq$ 30%. Given that the lowest seroconversion response in the IVAC Phase 1 trial was to B viral strain at 76.7% (95% CI, 57.7 90.1), there is high probability (Table 19) of demonstrating age group specific seroconversion requirement with a sample size of 100 evaluable participants per age group who received the study vaccine.

Table 19: Probability of demonstrating seroconversion response to all 3 viral strains by age groups and assumed true response to each viral strain

| | True response | | |
|---|---|---|---|
| Age group (point estimate response) | Probability > 90% | Probability > 95% | Probability > 99% |
| 18-45 (≥40%) | ≥49% | ≥51% | ≥54% |
| 46- 60 (≥30%) | ≥39% | ≥40% | ≥43% |

# 13.4.2 Probability for demonstrating seroprotection criteria for licensure

For the 18-45 year old cohort there is 92% probability that the point estimate for seroprotection to all three strains will be  $\geq$  70% if the true response to each strain is  $\geq$ 78%. Likewise if the true response to each strain is  $\geq$ 87%, then there is 95% probability that the lower bound of the exact 95% CI for seroprotection to all strains will be  $\geq$ 70%. In the older age cohort (46-60 year old), if the true seroprotection response to each strain is  $\geq$ 69%, then there is 93% probability that the point estimate for seroprotection to all three strains will be  $\geq$ 60%. Given that the lowest seroprotection response in the IVAC Phase 1 trial was to B viral strain at 93.3% (95% CI 77.9; 99.2), there is high probability (Table 20) of demonstrating age group specific seroprotection requirement with a sample size of 100 evaluable participants per age group who received the study vaccine.

IVACFLU-S, Phase 2/3

ENTIAL Date: 09/02/2017


Table 20: Probability of demonstrating seroprotection response to all 3 viral strains by age groups and assumed true response to each viral strain

| | True response | | |
|---|---|---|---|
| Age group (point estimate response) | Probability > 90% | Probability > 95% | Probability > 99% |
| 18-45 (≥70%) | ≥ 78% | ≥ 79% | ≥ 81% |
| 46- 60 (≥60%) | ≥ 69% | ≥ 70% | ≥ 72% |

# 13.5 Data Analysis

A detailed Statistical Analysis Plan (SAP) for preparation of the final study report will be prepared by the CRO statistican. The SAP will be submitted to PATH and IVAC for approval prior to database lock and unblinding. Analysis will be conducted only after all related data have been cleaned and locked. Given the short duration of clinical follow-up and potential delays in generating immunogenicity results, analysis of safety and immunogenicity data can be conducted independently. All statistical analyses will be performed using recent version of data management software.

# 13.6 Definition of Analysis Sets

# Definitions of populations to be analyzed are:

# **Enrolled Population**

All screened participants who are randomized, regardless of the participant's randomization and treatment status in the trial.

#### Full Analysis (FA) Population

All participants in the enrolled population who were randomized and received a study vaccination. This population will serve as the primary analysis population for all safety objectives. The analysis based on this population will serve as the supportive results for all safety objectives. Participants will be analyzed as randomized.

#### Per Protocol (PP) population

All participants in the Full Analysis population who have valid post vaccination immunogenicity measures with no major protocol violations that are determined to potentially interfere with the

Protocol No: IVACFLU-S-0203 574 Dated: 12 March 2018


immunogenicity assessment of the study vaccine. This population will serve as the primary analysis population for all immunogenicity objectives.

The criteria for exclusion of participants from the Per Protocol Population will be established before breaking the blind and will be based on the blinded review of protocol violations.

# 13.7 Analysis of Safety Endpoints

The safety profile of IVACFLU-S will be evaluated by the number and proportion of participants experiencing AEs by severity, relatedness to vaccination of the following four categories for all participants and by age group (solicited AEs will be considered related to study product):

- A. Solicited local adverse events, including redness / erythema, swelling / induration vital, pain within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- B. Solicited systemic adverse events, including fever, fatigue, malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- C. Unsolicited AEs occurring within 21 days post vaccination.
- D. Serious Adverse Events occurring during the entire study period (Days 1-91). .

Counts of all events will be reported and summarized according to event severity, as "any local AE", or "any systemic AE", and by relationship to administration of study product, as deemed by a blinded study clinician. Percentages of participants experiencing each reaction or event, or at least one reaction or event will be calculated along with two-sided exact 95% CIs. For solicited AEs, Fisher's exact test or Cochran-Mantel-Haenszel test will be used to compare the proportion of participants between the two treatment groups. In addition, no formal hypothesis testing with multiplicity adjustment will be performed. No statistical testing will be performed for unsolicited AEs; including SAEs.

#### 13.8 Analysis of Immunogenicity Endpoints

#### **Primary Endpoint:**

A. Number and percentage of participants with seroconversion against each of the 3 vaccine antigens post-vaccination. Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:

- pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or</li>
- pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 22
- B. Number and percentage of participants with a HAI antibody titer ≥1:40 to each of the 3 vaccine antigens measured on Day 22 post vaccination

Protocol No: IVACFLU-S-0203 575 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


- C. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) for each of the 3 vaccine antigens
- D. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/pre-vaccination) for each of the 3 vaccine antigens

Titers below the lowest limit of quantitation (i.e. below the starting dilution of assay reported as "< 10") will be set to half that limit (i.e. 10/ 2 = 5). If a titer is reported as greater or equal to the upper limit of the assay, it will be set to that limit.

# **Secondary Immunogenicity Endpoints:**

The secondary immunogenicity endpoints will be analyzed by the following:

- A. Number and percentage of participants who develop at least a four-fold increase in HAI antibody titer to each of the vaccine antigen post vaccination measured on Day 22 by prevaccination HAI antibody titer of <1:10 or ≥1:10.
- B. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) for each of the 3 vaccine antigens by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.
- C. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/pre-vaccination) for each of the 3 vaccine antigens by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.

The licenture requirements are based on on the point estimate of response in the vaccine group and are not based on comparison to a control. So there will be no formal statistical testing to compare immune response between vaccine and placebo. There are two types of immunogenicity measurements against each of the 3 vaccine antigens, percentages of subjects with immune response and Geometric Mean Titers (GMT) that will be used to evaluate this study objective. For each percentage of subjects with the defined immune responses, the percentage and its corresponding 2-sided exact (Clopper-Pearson) binomial 95% confidence interval (95% CI) around the percentage will be computed for each treatment group and by age group. GMT along with the corresponding two-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs, will be summarized by treatment group on Day1 and Day 22. The same approach will be used to summarize GMFR of Day 22/Day1 separately by treatment group and age group.

#### 13.9 Interim Analysis

All the safety data till day 8 from participants in the phase 2 will be analyzed and reviewed by the PSRT team. In addition all grade 3 and above unsolicited AEs and SAEs till the data cutoff date will also be part of interim report. The same data will be presented to IRBs and MOH for review and approval before initiating phase 3 study.

Protocol No: IVACFLU-S-0203 576 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 14 Data Management

The PI is responsible for ensuring the accuracy, completeness, and timeliness of the data reported. Data collection is the responsibility of the clinical trial staff at the study site under the supervision of the site PIs or designee. Data collection must be completed as soon as possible to allow for timely review of safety information. A CRO with data management expertise will be contracted to be responsible for data management activities, including quality review, analysis, and reporting of the study data according to SOPs.

# 14.1 Case Report Form (CRF)

CRFs will be developed and data will be managed to the extent possible in accordance with internationally agreed-upon standards, such as the Clinical Data Acquisition Standards Harmonization, which defines basic standards for the collection of clinical trial data, and/or The Society for Clinical Data Management's Good Clinical Data Management Guidelines (21). The study will use paper CRFs and transfer the data into an electronic CRF provided by the Data Management CRO.

All the information required by the study protocol must be recorded on the paper CRF provided by the sponsor. All data must be entered legibly. An explanation must be provided for any missing data. Data entered onto the paper CRFs must be accurate, legible, contemporaneous, original (or traceable to the original source) and attributable.

All source documents and CRFs should be completed in a neat, legible manner to ensure accurate interpretation of data. Black or blue ink is required to ensure clarity of reproduced copies. When making changes or corrections, study staff are to cross out the original entry with a single line, and initial and date the change. Do not erase, overwrite, or use correction fluid or tape on the original. All clinical source documents and laboratory reports must be reviewed by the Principal Investigator or designated qualified experts, who will ensure that they are accurate and complete.

The investigator must sign and date each CRF or a set of CRFs for each participant, attesting to his/her responsibility for the quality of all data recorded and that the data represent a complete and accurate record of each participant's participation in the study.

All participants will be assigned a unique screening number and participant identification number at study enrollment – one or both of these numbers will be included on all forms and in the trial database and will serve to link study data to specific individuals. CRFs will be entered, verified for accuracy, linked by study participant number, and managed using database management software, with proper security and controls and the ability to identify who is entering or making changes to the data in the system. Immunologic data will be sent separately to the data management center from the testing laboratory via secured electronic transmission.

Protocol No: IVACFLU-S-0203 577 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 14.2 Source Documents and Source Document Access

Prior to the start of the trial, the sponsor will determine which documents or data fields completed by the investigative team will be considered source documents and documented on a Source Documentation Table. Source documents for this study may be outpatient charts, inpatient charts, laboratory analysis forms, questionnaires, and specimen collection logs. For many data fields, the paper CRF will be the source document.

Only authorized study staff and representatives of IVAC, study monitors authorized by IVAC, PATH, members of ethics review committees, and regulatory agencies may have direct access to source documents containing participant data. Participant identification will be revealed to authorized representatives of these organizations only when necessary.

## 14.3 Database Management and Analysis Software

A CRO will be hired to perform data management for this study. The software used for data management will depend on what is suggested by the CRO, however, it will be validated and will meet widely accepted criteria for maintaining an electronic study database.

All statistical analyses will be performed using a recent version of standard data management software.

Medical history and AEs will be coded using a recent version of the MedDRA dictionary. The frequency count and percentage of participants will be summarized according to the coded terms of system organ class and preferred term. Participant-wise data listings will be provided.

#### 14.4 Entering, Cleaning and Management of Database

A CRO will develop a procedure for entering, cleaning and managing the database. The CRO will perform data management, data analysis and report writing. A Data Management Plan will be drafted by the CRO and submitted to IVAC or its designees to approve before implementation.

#### 14.5 Source Data Verification

For source data verification (SDV), the monitor (on behalf of the study Sponsor) must have direct access to source documents that support the data recorded, e.g., medical records, original laboratory records and ICFs. If source data are electronic, these data must be printed, signed and dated by the site PI and stored in the participant's study file. Essential documents, including ICFs, must be filed and kept in the study files.

Protocol No: IVACFLU-S-0203 578 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 14.6 Database Locking Procedures

A final database lock for the primary safety analysis will occur after all participants have completed all follow-up visits, including the Day 91 safety contact, review of the severity of any AEs has been performed and finalized, all data queries have been resolved to the satisfaction of the sponsor and monitoring is complete.

Immunology data will be maintained in a separate immunology database. These data will also be locked.

#### 14.7 Study Record Retention

Study data will be kept for 15 years after completion of the study. No records will be destroyed without the written consent of IVAC. It is the responsibility of IVAC to inform the PI when these documents no longer need to be retained.

## 15 Quality Control and Quality Assurance

#### 15.1 General Considerations

The study will be conducted in accordance with the procedures specified in the protocol and staff will be guided by written procedures that further explain important protocol implementation activities. Study data collection forms will be designed to guide staff on study conduct; forms also will include areas for documenting that activities did, in fact, occur (even if these activities did not require recording of data) and in the appropriate sequence. All study staff must attend mandatory protocol implementation training prior to participant enrollment.

Written procedures will be developed for key study procedures and refined/revised as necessary.

Study data are recorded on CRFs and then entered into the database throughout the study. After data have been entered in the study database, they are checked systematically by data management staff according to a pre-specified data validation plan. Queries are generated for site staff to clarify or correct throughout the study. An audit trail will be kept of all changes to the data. All listings of the database will be reviewed and discussed for assessment of consistency and medical plausibility. After resolution of all issues the database will be locked.

#### 15.2 Trainings

Each member of the research team will have documentation of his or her qualifications and experience to conduct his or her study responsibilities. In addition, the research team will be trained on all aspects of conducting the protocol. The study monitor is authorized to conduct retraining, if it is identified as a need from monitoring findings.

Protocol No: IVACFLU-S-0203 579 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# 16 Ethics/Protection of Human Subjects

#### 16.1 Ethical Standard

This study will be conducted in full conformity with the Vietnam GCP guidelines of MOH, and with the Declaration of Helsinki, in addition to all other Vietnam MOH regulatory requirements and current laws in order to ensure the best protection for study participants.

Study participants may not forego vaccination with a licensed, seasonal influenza vaccine while participating in this study. The vaccination with a licensed influenza vaccine will not be provided as part of the study. However the participants will not be stopped from receiving a licensed influenza vaccine after day 22, from outside the study. The participants should inform the study team if and when they receive a licensed influenza vaccine. Currently, imported seasonal influenza vaccines have been used in fee-based immunization services, mostly in big cities in Vietnam and the prices are not affordable for population in lower income groups especially at rural areas. Vietnam government has not introduced seasonal flu vaccine in national immunization program yet. Therefore, the availability of seasonal flu vaccines is limited or vaccines are not undertaken widely in Vietnam, even among high risk groups (health care workers, pregnant women, chronic respiratory disease group)

#### 16.2 Financing and Insurance

PATH will fund this trial. Any financial engagement with the clinical study clinic will be regulated by a separate agreement.

IVAC will maintain insurance to cover treatment for study related injuries and other insurance as necessary to meet its obligations under Vietnam law. This product liability insurance will cover product related injuries that cause death, illness leading to hospitalization, and disability. In addition, IVAC and PI HCMC will have an agreement letters with Ben Luc and Long Thanh district hospitals involved in the trial to provide treatment for any injuries for trial participants, whether or not the injuries are serious or caused by the vaccine.

#### 16.3 Assurance of Emergency Medical Care and Care for other Adverse Events

Study participants will be observed by qualified clinicians after each vaccination, and emergency care will be immediately available to participants who need it. If additional urgent care or resources are needed, depending on each case, the participant will be provided urgent care and transported to a hospital at higher level if needed.

Most adverse events that are expected and non-emergent can be handled at the study clinic by the clinical staff as they occur at no cost to the participant. These could be events such as fainting or feeling lightheaded, or swelling from the injection of the study products or blood draws.

Protocol No: IVACFLU-S-0203 580 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 16.4 Institutional Review Boards and Independent Ethics Committee

No human subject research activities will be conducted without the review and approval of all relevant ethics committees of the entities involved in the study. The protocol and all amendments will have initial and continuing review and approval by an independent ethics committee (IEC) responsible for clinical trials in Vietnam. This IEC is the Vietnam MOH Ethics Committee, which is the ultimate authority for decisions related to this trial. The MOH will acknowledge the review by participating institutions' IRBs which are designed to ensure that their staff meet their responsibilities in conducting this human subjects research. In Vietnam, the investigator is responsible for completing and submitting to the MOH the complete set of documents on the clinical trial for their review of the clinical trial application.

The study clinic's institution maintains an institutional review board. This study will be reviewed and approved by the institution's IRB prior to submission of Vietnam MOH IEC. All amendments will be approved by Vietnam MOH IEC before implementation, as appropriate.

The PI or designee shall maintain copies of all application documents and forward copies of all IRB and IEC documents and approvals to IVAC or its designee prior to the start of the study. The approval letters must identify all documents approved and list the study clinic, the study investigator, protocol title, version number, and date and, ICF version number and date, and the date of IRB or IEC approval. The PI will sign all approved versions of the protocol.

The PI is responsible for notifying the IEC and all IRBs of problems related to risks for participants, according to the requirements of the IEC and each IRB.

The PI may not change or deviate from the protocol without prior written IRB/ IEC approval of appropriate amendments, except when necessary to eliminate immediate hazards to the participants or when the changes involve only logistical or administrative aspects of the study (e.g., change of telephone number, etc.).

IVAC will report to the MOH and the IEC/IRBs any new information related to the study vaccine which possibly affect the safety of participants or their risk/benefit ratio for participating in this trial. Reports on the implementation of projects are to be periodically submitted to the Ethics Committee of the MOH.

The PI will be responsible for reporting to the MOH and the IEC/IRBs when the clinical study has been completed. This must occur within 90 days after the last involvement of participants in any study procedure. If the clinical study is terminated earlier than planned, the notice must be submitted to the MOH and the IEC/IRBs within 15 days and the reasons must be clearly explained.

## 16.5 Media Planning for Participant and Community Engagement

To establish trust and support from the community, the study team, along with the representatives of the provincial preventive medicine centers and district health centers will hold meetings in the

Protocol No: IVACFLU-S-0203 581 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


commune of the study site location to provide information on the seasonal influenza, risks to people with underlining diseases, mortality, prevention methods, common adverse reactions after vaccination and research efforts of Vietnam in developing this vaccine to the whole population of participating communes.

Before conducting the study, a risk media plan will be developed between WHO, IVAC, and NIHE in case there is media interest in the study. This plan will address issues such as who are appropriate contacts for each of the trial partners in case of contact by the media; identification of appropriate spokesperson for each entity; and an Internal Q&A on the vaccine candidate, trial, partner(s), project, and other issues as necessary.

#### 16.6 Informed Consent Process

The potential participants who agree to participate will then be invited to attend meetings to hear additional information and, if interested, sign the ICF to allow screening to begin. During implementation, the participants will be made aware of any new information relating to products or the clinical trial that may affect their decision to remain in the study.

The following issues must be included in discussions with potential participants prior to obtaining their informed consent to participate in the study:

- Discussion with the participants of the purpose of research, the time duration that the
  participants need to participate, the procedures involved in the study, the scientific
  evidence that justifies conducting this experimental trial in humans, and the potential risks
  and known benefits of participating in the research.
- Randomization and the chance of receiving either the study vaccine or the placebo.
- That the study staff will not know which study product (vaccine or placebo) the participant will receive and that the study staff and participant will have no way to choose which product is received by the participant.
- That the participant's participation is voluntary, and the participant's refusal to participate
  will not result in any fine or in any loss of rights or access to medical care that the
  participant is normally already entitled receive.
- That in the event of unforeseen circumstances or needs, the investigator may decide to withdraw the participant from continued participation in the research even without the consent of the participant.
- That the participant will be provided with the results of any new important findings related
  to the trial or the study vaccine which may influence the participant's decision on whether
  to continue to participate in the research.
- That the participant will be told the number of other participants participating in the research.
- That the participant will be told who to notify as the point of contact with the investigator
  and IRBs in case the research participant would like to know more information regarding
  the trial and his/her rights as a research participant.
- That the investigator is responsible for collecting from the participant signed and dated

Protocol No: IVACFLU-S-0203 582 Dated: 12 March 2018


written informed consent forms regarding participation in the study before the participant may participate in the research; that the participant will be given a signed and dated copy of the form to keep; and that the investigator must keep the original signed and dated informed consent form in the investigator's research files.

At the first meeting, participants will be told information about the purpose of the study and the procedures involved, as well as the possible risks, benefits and alternatives to joining the study. The participant will be informed of the voluntary nature of participation in the trial and that the volunteer has the right to refuse to join or to withdraw from the trial at any time, and that this refusal will not affect the quality of the participant's care.

Written informed consent of the participant must be obtained before performing any trial procedures. Participants will be made aware that authorized representatives of health agencies and IVAC will have access to their confidential medical information for the purposes of monitoring trial conduct or performing audits.

Written informed consent will be obtained from each participant before screening in duplicate on Day S1. On Day 1, after a participant is fully screened and eligibility is confirmed for entry the participant will be randomized to receive either vaccine or placebo. If Day 1 is conducted on a different day from S1 (there is 4-day window), eligibility must be confirmed again on Day of Injection (D1) including Targeted physical examination (PE) and urine pregnancy test.

ICFs will embody the elements of consent as described in the Declaration of Helsinki and the ICH Harmonized Tripartite Guidelines for Good Clinical Practice. Original ICFs must be kept on file by the investigator for possible inspection by regulatory authorities or IVAC. The participant must receive a copy (or second original) of the signed and dated ICF(s), and any subsequent updates or amendments to the ICF. The study monitor shall check the documentation of the individual ICFs during each monitoring visit.

Participants will be informed that they will be compensated for 450.000 VND (~20 USD) per site visit for their time and effort for participation in this trial and for travel to and meals during study visits.

#### 16.7 Inclusion of Women, Minorities, and Children

Enrollment in this study is open to healthy adults of any gender and race or ethnicity who are able to read the study consent and complete the Diary Cards. Pregnant women and children are excluded from the study because safety has not been determined in these populations. No person may be denied enrollment based on gender or race or ethnicity. The investigator may enroll different races and ethnicities in proportion to their presence in the local population; however, no special recruitment methods will be used to ensure certain levels of participation by any specific minorities residing in the source population. The trial is open to adults 18 through 60 years of age only.

Protocol No: IVACFLU-S-0203 583 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 16.8 Participant Confidentiality:

#### 16.8.1 Confidentiality of Data

By signing the protocol, the Principal Investigator agrees that the study protocol, documentation, data, and all other information generated regarding the vaccines will be held in strict confidence. The investigator may divulge such information within regulatory restrictions and ethical considerations only to ethical review committees or similar expert boards or committees, and their affiliated institutions and employees, only under an appropriate understanding of confidentiality with such board or committee, and their affiliated institutions and employees. No information concerning the study or the data may be released to any unauthorized third party without prior written approval of IVAC. Any regulatory agency deemed appropriate, may consult study documents in order to verify CRF data. Investigators will ensure that all employees involved in the study respect confidentiality.

Medical information about individual participants obtained during the course of this study is confidential and may not be disclosed to third parties, except authorized monitors, auditors or inspectors or as a requirement by law. Confidentiality will be ensured by the use of study participant numbers for the identification of each participant; these study participant numbers will also be used for participant data in the participant files at the site and for the CRFs.

## 16.8.2 Confidentiality of Participant Records

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and their agents. This confidentiality is extended to cover testing of biological specimens in addition to the clinical information relating to participating participants.

Study participants will not be identified by name on any data collection form or on any other documentation sent to IVAC and will not be reported by name in any report or publication resulting from data collected in this study.

Documents and data pertaining to the study will be kept in a locked room or in locked files under the responsibility of the Principal Investigator. IVAC will conduct periodic monitoring visits to ensure that the data are stored securely. Only study clinicians, study staff, monitors or the sponsor or its designee will be granted access to the study data and records. Study data will be kept for 15 years after completion of the study, in compliance with Vietnam law.

The PI will keep individual data confidential to the extent permitted by law. Information will not be released to anyone other than the participant unless required to do so by law or directed by the participant (e.g., to release information to his or her health care provider).

Protocol No: IVACFLU-S-0203 584 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### 16.9 Sharing of Study Results

#### 16.9.1 Sharing of Study Results with the Participant

When the clinical study report is completed, the investigator will share summary results (without any identifiers) with participants via printed materials. These will be submitted for approval by all applicable ethics committees before distribution to study participants.

## 16.9.2 Incidental Health Findings

The investigator may release participant physical examination results data to the participant's primary care physician only if the participant agrees in writing. The clinical staff will share and discuss any incidental health findings with the participant and help the participant seek proper medical follow-up.

#### 16.9.3 Sharing of Study Results with the Community

After the study results are approved by the Independent Ethic Committee, Ministry of Health, a workshop will be organized to report the results to national and local level with the participation of sponsor, study group representatives, representatives of Ministry of Health, the authorities and health officials of the provincial, district and commune levels. The results of this study will later be published in peer-review international and national scientific journals to share information for the international community.

#### 16.10 Study Discontinuation

Study discontinuation is not expected to occur. However, if the study is discontinued for safety reasons, participants will be informed of the reasons for discontinuation and of the implications/potential consequences for the participant.

#### 16.11 Future Use of Stored Specimens

Blood specimens will be maintained to allow re-testing either in Vietnam or outside Vietnam, if needed and for characterizing assays in the development of seasonal influenza vaccine. The specimens will be maintained at IVAC or a storage place designated by IVAC. Specimens will not be labeled with any personally-identifying information. The use of the specimens will be for laboratory quality control only and do not constitute human subjects research as the purpose is not generalizable knowledge, however, if a participant does not consent to their samples being used in this way, the samples will be destroyed when they are no longer needed for the study results.

Protocol No: IVACFLU-S-0203 585 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Date: 09/02/2017

#### 16.12 Potential Risks and How They are Addressed

**Physical Risks**: The main risks of this study are risks of physical injury. Administration of study product may cause the participant immediate mild pain in the arm. Other side effects include pain and inflammation at the injection site or systemic symptoms such as fever and body aches. These are all explained to participants in the consent form.

Serious or allergic reactions also may be possible. This risk is addressed by trying to screen out people who have had an allergic reaction to vaccines in the past and who may have an allergy to one of the components of the vaccine. Should an allergic reaction occur with vaccination, the study clinic will follow its SOP for handling medical emergencies and have supportive medicines in place, in addition to trained staff.

Besides administration of study product, collection of blood specimens may cause some discomfort to participants. Venipuncture is sometimes associated with fainting, discomfort or pain, bleeding, bruising, redness, swelling, local hardness, and/or infection at the puncture site. This risk is addressed by having trained staff draw the blood.

Study participants will be observed closely by qualified clinicians and care will be immediately available to participants after vaccination, including emergency care, if needed. If additional urgent care or resources are needed, the participant will be transported to a local hospital. This hospital will be identified by the investigator prior to study initiation. The study will provide this care to the participant at no cost to the participant.

In the case of expected and unexpected reactions after the use of vaccines, study participants will receive appropriate medical care and treatment. IVAC will pay the entire cost of medical treatment and resolve these cases according to current regulations in Vietnam.

Medical care will be provided for participants in this study. This includes the following:

- monitoring of participants closely for 30 minutes after vaccination and providing emergency care for any immediate reactions.
- monitoring of participants for adverse events which are not life-threatening and providing care for these at nearby local hospitals and treatment centers.
- monitoring of participants for severe adverse events and providing care for these at local hospitals and treatment centers.

During the study period if serious adverse event occurs that is related to the participant's participation in the trial or to the study products, IVAC will ensure coverage for the full cost of treatment according to the laws of Vietnam for research participants. The study clinic will establish an agreement with nearby treatment centers to provide treatment at no cost to the participant for abnormal reactions that are not life-threatening, but nonetheless warrant medical observation or care.

Protocol No: IVACFLU-S-0203 586 Dated: 12 March 2018

IVACFLU-S, Phase 2/3 Version: 4.0 CONFIDENTIAL Date: 09/02/2017


**Risks to Privacy:** Anyone participating in research using their real name and medical information can face a loss of privacy. These risks are mitigated by using unique IDs in place of a participant's name, restricting access to study information, and not naming or identifying a participant in any publication.

# 16.13 Benefits to Study Participants

Study participants may not benefit from being in the study, however, there is potential for some benefit:

• People may benefit from the physical exams that is done in the study, as it may reveal information about their health that they did not know before.

#### 17 Noncompliance and Unanticipated Problems

Noncompliance includes protocol deviations and violations, as stated below.

**Protocol deviations:** Any departure from the approved protocol, trial documents or any other information relating to the conduct of the trial that does not result in harm to the trial participants and does not significantly affect the study outcomes or data integrity or ethical conduct. Examples of deviations may include, but are not limited to:

- A missed protocol visit or a protocol visit date deviation outside the study visit window
- Isolated incident of a missed or incomplete study evaluation (e.g. exam)

**Protocol Violation**: Any departure from the approved protocol, trial documents or any other information relating to the conduct of the study which may affect the safety of trial participants or the study outcome. Examples of violations may include, but are not limited to:

- Failure to obtain informed consent (i.e. no documentary evidence);
- Enrolment of participants that do not meet the inclusion/exclusion criteria;
- Undertaking a procedure not approved by the IRB or Licensing Authority (unless for immediate safety reasons);
- Failure to report adverse events, serious adverse events in accordance with the legislation and sponsor and protocol requirements, such that trial participants, or the public, are put at significant risk;
- Investigational Product(s) dispensing, labeling or dosing error.

Protocol No: IVACFLU-S-0203 587 Dated: 12 March 2018


**Unanticipated Problems:** Problems that may or may not be adverse events but that, when they occur, are unexpected in terms of the frequency or severity (for AEs); related to the research; and put the participants or others at a greater risk of physical, psychological, economical, or social harm than what was previously known or recognized.

It is the responsibility of the site to use continuous vigilance to identify and report deviations and unanticipated problems to IVAC in a timely manner after identification. If required, reports of protocol deviations/violations must be sent to the research ethics committees overseeing the research. The PI and his/her staff are responsible for knowing and adhering to their research ethics committee's/IRB's requirements for reporting noncompliance and unanticipated problems.

# 18 Human Resource for the Study

# 18.1 Human Resource for the Study

The study research team will be qualified by experience, education, and training to conduct their responsibilities on this study.

The study clinic will make arrangements with local health centers to adequately care for participants who experience side effects/illnesses that need care beyond what the study clinic can provide.

The research team may use Commune Health Centers to prepare a list for potential participants, keep contact with study participants, and conduct home visits (if needed).

# 18.2 Training Plan

All key personnel (those responsible for the design and conduct of this study) will have completed Human Subjects Protection and/or GCP Training, as appropriate to their role, prior to interaction with any participants or to having access to their confidential study data. In addition, staff will be trained on any written procedures that pertain to their role in the study.

# 19 Clinical Study Report and Publication Policy

#### 19.1 Clinical Study Report

A Clinical Study Report (CSR) comprised of text and results tables reflecting all safety and immunogenicity data will be generated by IVAC or its designates. The CSR will be compliant with ICH E: 3 guidelines.

Protocol No: IVACFLU-S-0203 588 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


All data, documents, any recordings and information transferred to any contractor or obtained or prepared by any contractor, his/her consultants or persons associated by contractual relationships with any contractor during the trials, belong to IVAC.

Following completion of the clinical study report, the investigators, working with IVAC and representatives, are expected to publish the results, negative or positive, of this research in peer-reviewed scientific journal(s). IVAC may not prohibit the public dissemination of the results of this trial.

## 19.2 Publication Policy

The International Committee of Medical Journal Editors (ICMJE) member journals have adopted a trials-registration policy as a condition for publication. This policy requires that all clinical trials be registered in a public trials registry. It will be the responsibility of IVAC/PATH to register this trial in an acceptable registry. ICMJE authorship criteria will be strictly followed for publication of any manuscript(s) arising from this trial.

Ho Chi Minh City, date month year 20....

**Director of the Institution** 

**Principal Investigator** 


Date: 09/02/2017

Phan Cong Hung, MD

Hanoi, date month year 20.....

Director of the Administration of Science Technology and Training

Protocol No: IVACFLU-S-0203 589 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


#### REFERENCES

- 1. Fineberg HV. Pandemic preparedness and response–lessons from the H1N1 influenza of 2009. N Engl J Med 2014;370:1335–42.
- 2. Lafond KE, Nair H, Rasooly MH, Valente F, Booy R, Rahman M, et al. Global role and burden of influenza in pediatric respiratory hospitalizations, 1982–2012: a systematic analysis. PLoS Med 2016;13:e1001977.
- 3. Friede M, Palkonyay L, Alfonso C, Pervikov Y, Torelli G, Wood D, et al. WHO initiative to increase global and equitable access to influenza vaccine in the event of a pandemic: supporting developing country production capacity through technology transfer. Vaccine 2011;29(Suppl 1):A2–7.
- 4. Saha S, Chadha M, Al MA, Rahman M, Sturm-Ramirez K, Chittaganpitch M, et al.Influenza seasonality and vaccination timing in tropical and subtropical areas of southern and south-eastern Asia. Bull World Health Organ 2014;92:318–30.
- 5. WHO FluNet, Influenza Laboratory Suveillance Information by the Global Influenza Surveillance and Response System (GISRS) (<a href="www.who.int/flunet">www.who.int/flunet</a>) <a href="http://gamapserver.who.int/gareports/Default.aspx?ReportNo=1">http://gamapserver.who.int/gareports/Default.aspx?ReportNo=1</a>, [accessed on 17 October 2016].
- 6. <a href="http://www.who.int/influenza/vaccines/virus/candidates\_reagents/2016\_17\_north">http://www.who.int/influenza/vaccines/virus/candidates\_reagents/2016\_17\_north</a> [accessed on 17 October 2016].
- 7. Anh DD, Thiem VD, Anh NT, Huong VM, Nga NT, Thang TC, Thai DH, Chien VC, Holt R, Wahid R, Flores J, Berlanda Scorza F, Taylor DN.Randomized safety and immunogenicity trial of a seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) in healthy young Vietnamese adults. Vaccine. 2016 Oct 26;34(45):5457-5462.
- 8. Guidance on Clinical Trial of Influenza Vaccine. Ministry Of Health (Administration of Science Technology And Training), Hanoi, Vietnam, 2013.
- http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UC M329134.pdf [accessed on 17 October 2016].
- http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UC M305089.pdf [accessed on 17 October 2016].
- 11. <a href="http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM335392.pdf">http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM335392.pdf</a> [accessed on 17 October 2016].
- 12. Stefan P. Kuster, Prakesh S. Shah, Brenda L. Coleman, Po-Po Lam, Agnes Tong, Anne Wormsbecker, Allison McGeer. Incidence of Influenza in Healthy Adults and Healthcare Workers: A Systematic Review and Meta-Analysis PLOS Published: October 18, 2011
- 13. Pearson ML, Bridges CB, Harper SA. Influenza vaccination of health-care personnel [published correction appears in MMWR Recomm Rep. 2006;55(9):252]. MMWR Recomm Rep 2006;55(RR-2):1–16
- 14. Taksler GB, Rothberg MB, Cutler DM. Association of Influenza Vaccination Coverage in Younger Adults With Influenza-Related Illness in the Elderly. Clin Infect Dis. 2015 Nov 15;61(10):1495-503. doi: 10.1093/cid/civ630
- 15. World Health Organization WHO Technical Report Series, No. 927, 2005 Annex 3 Recommendations for the production and control of influenza vaccine (inactivated) [accessed on 17 October 2016].
- 16. <a href="http://www.ema.europa.eu/docs/en">http://www.ema.europa.eu/docs/en</a> GB/document library/Scientific guideline/2013/03/ WC500139747.pdf [accessed on 17 October 2016].
- · The Guidance on the treatment of post injection reactions issued under the decision No

Protocol No: IVACFLU-S-0203 590 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


2535/QD-BYT by Ministry of Health, Vietnam; <a href="http://vncdc.gov.vn/vi/huong-dan-giam-sat-phong-chong-dich-benh/329/quyet-dinh-ve-viec-ban-hanh-huong-dan-theo-doi-cham-soc-xu-tri-phan-ung-sau-tiem-chung">http://vncdc.gov.vn/vi/huong-dan-giam-sat-phong-chong-dich-benh/329/quyet-dinh-ve-viec-ban-hanh-huong-dan-theo-doi-cham-soc-xu-tri-phan-ung-sau-tiem-chung</a>

- 17. Committee for Proprietary Medicinal Products (CPMP). Note for guidance on harmonization of requirements for influenza vaccines. CPMP/BWP/214/96. The European Agency for the Evaluation of Medicinal Products (EMEA), March 1997
- 18. Voordouw AC, Beyer WE, Smith DJ, Sturkenboom MC, Stricker BH. Evaluation of serological trials submitted for annual re-licensure of influenza vaccines to regulatory authorities between 1992 and 2002. Vaccine. 2009 Dec 11;28(2):392-7.
- 19. Goodwin K, Viboud C, Simonsen L .Antibody response to influenza vaccination in the elderly: a quantitative review.. Vaccine. 2006 Feb 20;24(8):1159-69.
- 20. <a href="https://www.cdisc.org/sites/default/files/members/standard/foundational/cdash/cdash\_std">https://www.cdisc.org/sites/default/files/members/standard/foundational/cdash/cdash\_std</a>
  <a href="https://www.cdisc.org/sites/default/files/members/standard/foundational/cdash/cdash\_std">https://www.cdisc.org/sites/default/files/members/standard/foundational/cdash/cdash\_std</a>
  <a href="https://www.cdisc.org/sites/default/files/members/sites/def

Protocol No: IVACFLU-S-0203 591 Dated: 12 March 2018


Date: 09/02/2017


**APPENDIX A: Table of Grading Severity** 

# IVACFLU-S TABLE OF GRADING SEVERITY FOR CERTAIN EVENTS<sup>1</sup>

# I. <u>Instructions and Clarifications</u>

IVACFLU-S, Phase 2/3

#### Estimating Severity Grade for Parameters Not Identified in the Table

In order to grade a clinical AE that is not identified in the DAIDS AE grading table, refer to the protocol.

## Determining Severity Grade for Parameters "Between Grades"

If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE. If a laboratory value that is graded as a multiple of the ULN or LLN falls between two grades, select the higher of the two grades for the AE. For example, Grade 1 is 2.5 x ULN and Grade 2 is 2.6 x ULN for a parameter. If the lab value is 2.53 x ULN (which is between the two grades), the severity of this AE would be Grade 2, the higher of the two grades.

#### Values Below Grade 1

Any laboratory value that is between either the LLN or ULN and Grade 1 should not be graded.

# <u>Determining Severity Grade when Local Laboratory Normal Values Overlap with Grade 1</u> Ranges

In these situations, the severity grading is based on the ranges in the DAIDS AE Grading Table, even when there is a reference to the local lab LLN.

For example: Phosphate, Serum, Low, Adult and Pediatric > 14 years Grade 1 range is 2.50 mg/dL - < LLN. A particular laboratory's normal range for Phosphate is 2.1 – 3.8 mg/dL. A participant's actual lab value is 2.5. In this case, the value of 2.5 exceeds the LLN for the local lab, but will be graded as Grade 1 per DAIDS AE Grading Table.

\_

<sup>&</sup>lt;sup>1</sup> Based On The DAIDS Table For Grading the Severity of Adult And Pediatric Adverse Events, Version 2.0, November 2014; and Guidance For Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials; FDA, 2007.

Protocol No: IVACFLU-S-0203 592 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# II. Definitions of terms used in the Table:

Basic Self-care Functions Adult

Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

LLN Lower limit of normal

Medical Intervention Use of pharmacologic or biologic agent(s) for

treatment of an AE

NA Not Applicable

Operative Intervention Surgical OR other invasive mechanical

procedures.

ULN Upper limit of normal

Usual Social & Functional Activities Adult

Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc.

Version 1.0 593 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203

IVACFLU-S, Phase 2/3


| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE-THREATENING |
|---|---|---|---|---|
| ESTIMATING SEVER | RITY GRADE | | | |
| Blood Pressure<br>Abnormalities<br>Hypertension | 140 to < 160 mmHg<br>systolic OR 90 to <<br>100 mmHg diastolic | ≥ 160 to < 180 mmHg<br>systolic OR ≥ 100 to <<br>110 mmHg diastolic | ≥ 180 mmHg systolic<br>OR ≥ 110 mmHg<br>diastolic | Life-threatening<br>consequences in a<br>participant not<br>previously diagnosed<br>with hypertension (e.g.,<br>malignant hypertension)<br>OR Hospitalization<br>indicated |
| SYSTEMIC | | | | |
| Acute Allergic<br>Reaction | Localized urticaria<br>(wheals) with no<br>medical intervention<br>indicated | Localized urticaria with intervention indicated OR Mild angioedema with no intervention indicated | Generalized urticaria OR Angioedema with intervention indicated OR Symptoms of mild bronchospasm | Acute anaphylaxis OR<br>Life-threatening<br>bronchospasm OR<br>Laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue or Malaise<br>Report only one | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating<br>symptoms of fatigue or<br>malaise causing inability<br>to perform basic self-<br>care functions |
| Arthralgia (Joint<br>Pain) | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Incapacitating joint pain causing inability to perform basic self-care functions |
| Fever (non-axillary temperatures only) | 38.0 to < 38.6°C | ≥ 38.6 to < 39.3°C | ≥ 39.3 to < 40.0°C | ≥ 40.0°C |
| Fever (axillary) | 37.7 – 38.1°C | 38.2 – 38.8°C | 38.9 – 40.0°C | > 40.0°C |
| Nausea | Transient (< 24 hours)<br>or intermittent AND<br>No or minimal<br>interference with oral<br>intake | Persistent nausea<br>resulting in decreased<br>oral intake for 24 to 48<br>hours | Persistent nausea<br>resulting in minimal oral<br>intake for > 48 hours<br>OR Rehydration<br>indicated (e.g., IV fluids) | Life-threatening<br>consequences (e.g.,<br>hypotensive shock) |
| Vomiting | Transient or intermittent AND No or minimal interference with oral intake | Frequent episodes with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated (e.g., IV fluids) | Life-threatening<br>consequences (e.g.,<br>hypotensive shock |

Protocol No: IVACFLU-S-0203 594 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE-THREATENING |
|---|---|---|---|---|
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated OR Headache with significant impairment of alertness or other neurologic function |
| INJECTION SITE RE | ACTIONS | | | |
| Injection Site Pain or<br>Tenderness<br>Report only one | Pain or tenderness<br>causing no or minimal<br>limitation of use of<br>limb | Pain or tenderness<br>causing greater than<br>minimal limitation of<br>use of limb | Pain or tenderness causing inability to perform usual social & functional activities | Pain or tenderness<br>causing inability to<br>perform basic self-care<br>function OR<br>Hospitalization indicated |
| Injection Site Erythema or Redness Report only one > 15 years of age | 2.5 to < 5 cm in<br>diameter OR 6.25 to <<br>25 cm² surface area<br>AND Symptoms<br>causing no or minimal<br>interference with<br>usual social &<br>functional activities | ≥ 5 to < 10 cm in diameter OR ≥ 25 to < 100 cm² surface area OR Symptoms causing greater than minimal interference with usual social & functional activities | ≥ 10 cm in diameter OR ≥ 100 cm² surface area OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage OR Symptoms causing inability to perform usual social & functional activities | Potentially life-<br>threatening<br>consequences (e.g.,<br>abscess, exfoliative<br>dermatitis, necrosis<br>involving dermis or<br>deeper tissue) |
| Injection Site Induration or Swelling Report only one > 15 years of age | Same as for Injection<br>Site Erythema or<br>Redness, > 15 years<br>of age | Same as for Injection<br>Site Erythema or<br>Redness, > 15 years<br>of age | Same as for Injection<br>Site Erythema or<br>Redness, > 15 years of<br>age | Same as for Injection<br>Site Erythema or<br>Redness, > 15 years of<br>age |

Protocol No: IVACFLU-S-0203 595 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# **APPENDIX B: Roles and responsibilities matrix**

| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Objective 1: Phase 2/3 S | tudy Developed | | | | |
| 1 | Develop protocol | tudy Beveloped | PATH | WHO | IVAC | CRO |
| | Draft protocol synopsis prepared | С | R/A | С | С | ı |
| | Protocol drafted | С | R/A | С | С | I |
| | Protocol finalized and ready for submission | А | R/A | С | Α | I |
| 2 | Prepare investigational p | product and | PATH | WHO | IVAC | CRO |
| | Prepare summary batch record for production and QC testing for 3 lots | I | I | I | R/A | |
| | Send samples of 3 lots to NICVB for release testing | I | I | I | R/A | |
| | Filling, packaging,<br>labelling investigational<br>product and placebo | ı | С | I | R/A | |
| | QC testing for placebo | I | I | I | R/A | |
| | Coding investigational products | I | Α | I | Α | R |
| | Labeling of investigational products | 1 | I | I | R/A | I |
| 3 | Select CTU and site | | PATH | WHO | IVAC | CRO |
| | Clinical site(s) initially assessed/proposed | С | R | I | C/A | |
| | Clinical site agreed upon | R | ı | ı | Α | |
| | Specialty (serology) lab(s) initially assessed/proposed | С | R | I | C/A | |
| | Specialty (serology) lab(s) agreed upon | С | R | I | Α | |
| 4 | Register Phase 2/3 study | | PATH | WHO | IVAC | CRO |

IVACFLU-S Version 1.0 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Petition to conduct<br>clinical trial submitted<br>(including proposed site,<br>PI and Protocol<br>Synopsis) | I | С | I | R/A | |
| | Investigator's Brochure updated for submission | I | С | I | R/A | |
| | - Summary information on investigational product updated | I | С | I | R/A | |
| | -Summary information on MSV/WSV updated | I | С | I | R/A | |
| | - Lot release certificates<br>from NICVB for 3<br>consecutive lots<br>obtained | I | С | I | R/A | I |
| | Receives MOH approval<br>or address MOH<br>feedback on<br>"registration" | I | С | I | R/A | I |
| 5 | Develop<br>investigational dossier | | PATH | WHO | IVAC | CRO |
| | Investigator's Brochure provided to site | I | I | I | R/A | I |
| | Informed consent forms (ICFs) developed according the protocol and translated | С | R | I | C/A | I |
| | Clinical Trial Agreement (CTA) drafted | С | R/A | I | С | I |
| | CTU/site budget preparation | С | R/A | I | I | |
| | Additional specialty lab budget preparation | С | R/A | I | I | |
| | Contract for Clinical trial and MOU prepared and signed | А | R/A | I | Α | I |

IVACFLU-S Version 1.0 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Insurances for subjects | I | I | I | R/A | I |
| | Clinical Trial Agreement<br>signed by parties after<br>MOH approval | R | R/A | I | R | I |
| 6 | "Investigational dossier" approved | | PATH | WHO | IVAC | CRO |
| | "Application" form submitted to PI HCMC's IRB | R | С | I | С | I |
| | Obtain approval letter<br>and meeting minutes of<br>the IRB of PI HCMC<br>Review Meeting | R | С | I | С | _ |
| | Obtain supporting letter from Provincial Level and People's Committee | R | С | I | С | I |
| | Submission packages to MOH's IRB | R | С | I | С | I |
| | Present/Defend the dossier to MOH | R | С | I | С | I |
| | Receives approval or feedback from MOH on investigational dossier | R | I | I | I | I |
| | Addresses any issues raised by MOH | R | R/A | I | R | I |
| | Submit package and obtain approval from WIRB (PATH REC) | I | R/A | I | I | I |
| | Objective 2: Phase 2/3 S | tudy Implemented | | | | |
| 7 | Pre- trial preparation | | PATH | WHO | IVAC | CRO |
| | Pre-study progress reporting | R/A | R/A | I | I | I |
| | Randomization plan developed | I | R/A | I | С | R |
| | Clinical monitoring plan developed | I | C/A | I | Α | R |

IVACFLU-S Version 1.0 598 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|
| Safety monitoring plan developed | I | C/A | I | Α | R |
| Interim SAP and immunogenicity analysis plans | I | C/A | I | А | R |
| Study registered with international trial registry (e.g. clinicaltrials.gov) | I | R | I | А | I |
| Lab reagents/materials<br>for taking blood<br>purchased | R | R/A | I | I | |
| Preparation meeting with field site staff and community | R/A | С | I | С | I |
| The list of eligible subjects constructed | R/A | С | I | С | I |
| 8 Develop study materials | | | | | |
| Investigator's File established (including all logs) | R | R/A | I | С | R |
| Protocol issued to investigative staff | С | R/A | I | R/A | I |
| Site SOP's developed | R/A | R/A | I | А | I |
| eCRFs and completion guidelines developed | С | С | I | I | R/A |
| SOPs relating to cold chain maintenance developed | А | R/A | I | R/A | I |
| Manual of Operations Developed | С | R/A | I | С | I |
| Pharmacy and Lab Manuals Developed | С | R/A | I | С | I |
| ICF printed | R | С | ı | I | Α |
| CRFs printed and transported to site | С | С | I | I | R/A |
| 9 Pre-trial training | | PATH | WHO | IVAC | CRO |

IVACFLU-S Version 1.0 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Training Plan Developed | R | R/A | I | С | С |
| | RE/GCP training for required personnel provided | R | С | I | С | I |
| | Protocol training for sub-<br>investigators and staff<br>provided | R | R/A | I | С | I |
| | Data management training | С | С | I | I | R/A |
| | Trial practice run training conducted | R | R/A | I | С | I |
| 10 | Vaccine transportation a | ind management | PATH | WHO | IVAC | CRO |
| | Pre-trial cold-chain assessment | С | R/A | I | R/A | I |
| | Provide Product Certificate of Analysis to site | I | I | I | R/A | I |
| | Provide shipment information to site and/or handling agent | I | С | I | R/A | I |
| | Shipment of vaccine to site | I | I | I | R/A | ı |
| | Receipt of vaccine at site | R/A | I | I | С | I |
| | Return of unused vaccine to manufacturer | R/A | I | I | С | А |
| 11 | Overall study<br>responsibilities<br>fulfilled | | PATH | WHO | IVAC | CRO |
| | Investigative staff identified, recruited and/or hired | R | C/A | I | C/A | I |
| | Implementation Plan<br>Developed | R | C/A | I | С | С |
| | Financial management | R/A | R/A | ı | l | |
| | Study teleconference organization | I | С | I | А | R/A |

IVACFLU-S Version 1.0 600 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Study teleconference | R | R | | R | R/A |
| | participation | | | | | |
| | Study implementation | R/A | C/A | I | C/A | С |
| | Progress reports to WHO, PATH and IVAC | R | Α | I | А | R/A |
| | Reports to Safety Monitoring Groups | С | R/A | I | С | R/A |
| 40 | Conduct transport and to | PATH | \\/\!\ | | 000 | |
| 12 | specimens | | | WHO | IVAC | CRO |
| | Specialty Laboratory(s) (serology) | | | | | |
| | Coordination of transport of samples from site to specialty lab(s) | R/A | С | I | С | I |
| | Laboratory sample testing | 1 | C/A | I | С | I |
| 13 | Clinical/Medical Monitoring | | PATH | WHO | IVAC | CRO |
| | CRO identified for site monitoring | I | С | R/A | I | |
| | CRO appoints medical monitor | I | R/A | I | С | R/A |
| | Conduct/participate prestudy site visits | С | R | I | C/A | I |
| | Conduct site initiation/activation | С | С | I | С | R/A |
| | Conduct interim monitoring | С | С | I | I | R/A |
| 14 | <u>Develop Statistical</u><br><u>Analysis Plan (SAP)</u> | | PATH | WHO | IVAC | CRO |
| | Develop SAP | l | С | I | I | R/A |
| | Approve SAP | I | R/A | I | Α | С |
| 15 | Clinical Study Report | | PATH | WHO | IVAC | CRO |
| | Write Clinical Study<br>Report | 1 | С | I | С | R/A |
| | Write Clinical Study<br>Report MOH template | С | R/A | I | С | I |

Protocol No: IVACFLU-S-0203 601 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


| | ACTIVITY | PI HCMC<br>(Investigator,<br>Clinical Trial Unit,<br>Clinical Site,<br>Laboratories) | PATH | WHO | IVAC<br>(Sponsor) | CRO |
|---|---|---|---|---|---|---|
| | Review Drafts of CSR;<br>Approve of Final CSR | I | R/A | I | R/A | С |
| 16 | Trial Master File (TMF) | | PATH | WHO | IVAC | CRO |
| | Develop and Manage<br>Trial Master File | С | I | I | С | R/A |
| | Ensure completeness of TMF | R | C/A | I | С | С |
| | Submit TMF to Sponsor | I | I | I | С | R/A |

# Note:

R = Responsibility

C = Consulted

I = Informed

A = Approved


Date: 09/02/2017

Protocol No: IVACFLU-S-0203 602 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


# APPENDIX C: Template of interim study report of the phase 2/3

- 1. Cover pages (according to the CSR template by MOH VN)
- Study title, protocol number
- Key individuals and institution involving the study.
- Timeline of study implementation of the phase 2
- 2. Protocol synopsis
- 3. Study plan
- 4. Overall phase 2 status until D8
- Enrollment/screening counts: total participants screened/enrolled/failured
- Screening failure summary: illegibility, withdraw consent, study no longer for enrollment, others
- Study progress: total S1/D1 visit, total D8 visit
- Early termination
- Protocol violation/deviation
- Demographic and key baseline characteristics
- 5. Overall Reactogencicity report until D8 (blinded data and not presented by treatment group)
- Local solicited AEs
- Systemic solicited AEs
- 6. Demographic and baseline characteristics
- 7. Unsolicited AEs until D8 and grade 3 and above unsolicited AEs till data cutoff date (blinded data and not presented by treatment group)
- 8. SAEs till data cut-off date
- 9. Conclusion

Protocol No: IVACFLU-S-0203 603 Dated: 12 March 2018


# **APPENDIX D: Assessment of Understanding**

IVACFLU-S, Phase 2/3

# List of questions to evaluate the understanding of consent process by participants

**Directions:** After providing and explaining information about the study in the information sheet, and answering questions asked by participant. It is necessary to evaluate the understanding of participant in order to see if they correctly understand about the study before asking she/he to sign in the consent form. Investigator should ask all questions below, if the participant answers well those questions, she/he will be asked to sign the ICF. If she/he cannot or wrongly answer any question, investigator has to explain again to her/him and asks some more questions to make sure the correct understanding by participant before signing the ICF.

**Read this to the participant:** We have talked about the study together. Now I want to ask you some questions to see how well I explained the study to you.

- 1. Can you tell me which vaccine is tested in this study and what disease is this vaccine trying to prevent?
- 2. Is your participation in this study voluntary or are you forced to join it?
- 3. If you join the study do you have to stay in it, even if you want to leave it early?
- 4. Will everyone in the study get the study vaccine?
- 5. According to you, does your participation bring any benefit for yourself and for the community (other people)?
- 6. According to you, what reactions/risks may you have if you participate in this study (receive the study product)?

Protocol No: IVACFLU-S-0203 604 Dated: 12 March 2018


Date: 09/02/2017


# APPENDIX E: Quality Certification by NICBV for study product lots

Product name: IVACFLU-S (Trivalent, inactivated, split virion seasonal influenza vaccine)

**Lot number:** 004-01-16 **Packaging unit:** 0.5ml/dose/vial

Manufacture date: 29 November, 2016 Expired date: 05 December, 2017

Manufacturer: Institute of Vaccine and Medical Biologicals (IVAC)

# **RESULTS:**

IVACFLU-S, Phase 2/3

| # | Indicator/Testi | Acceptance criteria of the | Result | Evaluation |
|---|---|---|---|---|
| | ng | manufacturer | | |
| 1. | Filling volume | ≥ volume in label (0.5 | 0,596; 0,604; 0,596; | Pass |
| | | ml/vial) | 0,596; 0,599 | |
| 2. | Visual | The solution is clear, | Pass | Pass |
| | | colorless or opaque white, | | |
| | G | no sediment, no particle | 0 | |
| 3. | Sterility | No growth of bacteria and | Pass | Pass |
| | | fungi in culture medium after | | |
| | | 14 days | | |
| 4. | pН | 6.5 – 7.5 | 7.04 | Pass |
| 5. | Identity | Positive reaction with | Positive | Pass |
| 0. | 13.0.11.0 | specific antiserum of each | | |
| | | strain | | |
| 6. | HA content | ≥ 15µg for each strain | Type B: 17,92 μg/dose | |
| | (potency) | | Type H1N1:19,71 μg/ dose | |
| | | | Type 111101:19,71 μg/ dose | |
| | | | Type H3N2: 20,03 μg/ dose | |
| 7. | Endotoxin | ≤ 100 EU | 8 EU/dose | Pass |
| | | | <u> </u> | |
| 8. | | | Pass | Pass |
| | | are in good health and gain weight after 7 monitoring | | |
| | | days | | |
| 9. | Protein content | ≤ 300 μg/ml | μg/ml 288.47 | |
| J . | (μg/dose) | | | Pass |
| 10. | Formaldehyde | ≤ 0.02 % | 0.00055 % | Pass |
| | content (%) | · ··· | | |
Protocol No: IVACFLU-S-0203 605 Dated: 12 March 2018

IVACFLU-S, Phase 2/3


Product name: PLACEBO

**Lot number:** 007P-01-16 **Packaging:** 0.5ml/dose/vial

Manufacture date: 02 December 2016 Expired date: 05 December 2017

Manufacturer: Institute of Vaccine and Medical Biologicals (IVAC)

## **RESULTS:**

| # | Indicator/Testing | Acceptance criteria of the | Result | Evaluation |
|---|---|---|---|---|
| | | manufacturer | | |
| 1 | Visual | The solution is clear, colorless or | Pass | Pass |
| | | opaque white, no sediment, no | | |
| | | particle | | |
| 2 | Filling volume | ≥ volume in label (0.5 ml/vial) | 0,598; 0,594; | Pass |
| | | | 0,595; 0,594; | |
| | | | 0,592 | |
| 3 | Sterility | No growth of bacteria and fungi in | Pass | Pass |
| | | culture medium after 14 days | | |
| 4 | рН | 6.5 - 7.5 | 7.21 | Pass |
| 5 | Endotoxin | ≤ 1.25 EU | 0.625 EU/dose | Pass |
| 6 | General safety | All the mice and guinea pigs are in | Pass | Pass |
| | | good health and gain weight after | | |
| | | 7 monitoring days | | |
| 7 | NaCl content (%) | ≤ 1% | 0.90% | Pass |

Protocol No: IVACFLU-S-0203 606 Dated: 12 March 2018

## 16.1.2 Sample case report form

| Document | Date |
|---------------------------------------|------------------|
| Annotated Case Report Form, Version 4 | 02 May 2017 |
| Blank Subject Diary Card, Version 1 | 14 December 2016 |
| eCRF Design Approval Form, Version 4 | 02 May 2017 |

Protocol No: IVACFLU-S-0203 607 Dated: 12 March 2018

Annotated Study Book for Study Design: IVACFLU-S-0203

Study Design Version: 1.0

Sponsor: Institute of Vaccines and Medical Biologicals (IVAC)

Protocol: IVACFLU-S-0203 eCRF Version 04.00 IYA06804

Generated by Central Designer <sup>™</sup> May 2, 2017 8:49PM Protocol No: IVACFLU-S-0203 608 Dated: 12 March 2018

| | Element | | Sys | stem | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Assessment | CRF | System<br>Screening<br>(SCRVIS)<br>[S] | System<br>Enrollment<br>(ENRVIS)<br>[S] | Screening<br>(SCR)<br>[S] | Day<br>1<br>(DAY<br>1)<br>[U] | Day<br>2<br>(Day<br>2)<br>[S] | Day<br>5<br>(Day<br>5)<br>[S] | Day<br>8<br>(DAY<br>8)<br>[S] | Day<br>22<br>(DAY<br>22)<br>[S] | Day<br>91<br>(Day<br>91)<br>[S] | Unscheduled<br>Visit<br>(UNS VIS)<br>[U/R] | Log<br>(LOG<br>VIS)<br>[U] | Common<br>(Common)<br>[U] | End<br>of<br>Study<br>(EOS)<br>[U] |
| | Visit Start Hours | | 0 | 0 | 0 | 1 | 25 | 121 | 193 | 529 | 2185 | 2186 | 2187 | 2188 | 2189 |
| 1 | SYSTEM SCREENING | SYSSCR | 1 | | | | | | | | | | | | |
| 2 | SYSTEM ENROLLMENT | ENROL | | 1 | | | | | | | | | | | |
| 3 | DATE OF VISIT | DOV | | | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | | |
| 4 | SUBJECT IDENTIFICATION FORM | SUBID | | | 2 | | | | | | | | | | |
| 5 | DEMOGRAPHICS | DEMOG | | | 3 | | | | | | | | | | |
| 6 | CURRENT MEDICAL CONDITION | MHX | | | 4 | 2-DF | | | | | | | | | |
| 7 | SCREENING PHYSICAL EXAM | PE | | | 5 | | | | | | | | | | |
| 8 | URINE PREGNANCY TEST | UPREG | | | 6-DF | 4-DF | | | | | | 5-DF | | | |
| 9 | RANDOMIZATION | ELIG | | | 7 | 5-DF | | | | | | | | | |
| 10 | TARGETED PE | TPE | | | | 3-DF | | | 2 | 3 | | 3-DF | | | |
| 11 | ANTI-INFLUENZA SEROLOGIC ASSAY | ANTI INF<br>SER | | | | 6-DF | | | | 2-DF | | 4-DF | | | |
| 12 | VACCINATION | VAC | | | | 7 | | | | | | | | | |
| 13 | 30-MINUTE REACTOGENICITY | ROG | | | | 8 | | | | | | | | | |
| 14 | CONTACT | TELECONT | | | | | 2 | 2 | | | 2 | | | | |
| 15 | SOLICITED LOCAL REACTOGENICITY | LOCAL | | | | | | | 3 | | | | | | |
| 16 | SOLICITED SYSTEMIC REACTOGENICITY | SYSTEMIC | | | | | | | 4 | | | | | | |
| 17 | UNSCHEDULED ASSESSMENT FORMS | UNSFM | | | | | | | | | | 2 | | | |
| 18 | LOG | LOGFM | | | | | | | | | | | 1 | | |
| 19 | UNSOLICITED ADVERSE EVENT | AEUNSOL | | | | | | | | | | | 2-DF-<br>RF | | |
| 20 | SERIOUS ADVERSE EVENT | SAE | | | | | | | | | | | 3-DF-<br>RF | | |
| 21 | CONCOMITANT MEDICATIONS | СМ | | | | | | | | | | | 4-DF-<br>RF | | |
| 22 | MISSED VISIT FORM | MISSED<br>VISIT FORM | | | | | | | | | | | | 1 | |
| 23 | REPORT OF PREGNANCY | REPORT OF PREGNANCY | | | | | | | | | | | | 2-DF | |
| 24 | END OF STUDY | EOSFM | | | | | | | | | | | | | 1 |
| 25 | INVESTIGATOR SIGNATURE | SIGN | | | | | | | | | | | | | 2 |

Protocol No: IVACFLU-S-0203 609 Dated: 12 March 2018

| IVACFLU-S-0203: SYSTEM SCREENING (SYSSCR) [SYSSCR] | | |
|---|---|---|
| Sys | stem Screening [SYSSCRSC] | |
| 1. | Subject Initials [hidden] [Initials] | [SUBINI] |
| | Date of birth<br>[Date of birth] | [SCRDOBDT] |

| RDE Analytics: RD_SYSSCR | | |
|--------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| SUBINI | SUBINI | VARCHAR2 |
| | SUBINI_ND | VARCHAR2 |
| SCRDOBDT | SCRDOBDT | DATE |
| | SCRDOBDT_DTS | VARCHAR2 |
| | SCRDOBDT_DTR | VARCHAR2 |
| | SCRDOBDT_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 610 Dated: 12 March 2018

| Sys | stem Enrollment [SYSENRSC] | |
|----------|------------------------------------------------|----------------|
| 1.*<br>• | Screening ID [Screening ID] | [SCRNUMZ] A5* |
| 2. | InForm Subject ID [hidden] [InForm Subject ID] | [INSUBJID] A20 |

| RDE Analytics: RD_SYSENR | | |
|--------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| SCRNUMZ | SCRNUMZ | VARCHAR2 |
| | SCRNUMZ_ND | VARCHAR2 |
| INSUBJID | INSUBJID | VARCHAR2 |
| | INSUBJID_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 611 Dated: 12 March 2018

| IVACFLU-S-0203: DATE OF VISIT (DOV) [DOV1] | | |
|---|---|---|
| Date of Visit [DOVSC] | | |
| 1.* | Date of Visit [Date of Visit] | [DOVDT]<br> Req |
| Key: [*] = Item is required [✓] = Source verification required Note: Source verification critical settinos made in Inform will override any settinos made in Central Designer. | | |

| RDE Analytics: RD_DOV1 | | |
|------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| DOVDT | DOVDT | DATE |
| | DOVDT_DTS | VARCHAR2 |
| | DOVDT_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 612 Dated: 12 March 2018

| [VACFLU-S-0203: Subject identification form (SUBID) [SUBID] |
|---|
| SUBIDSC [SUBIDSC] |
| ] |
| [InForm Subject ID] A20 Jupdate Subject Randomization Number [Update Subject Randomization Number] [InJudate Subject Randomization Number] |

| Study Object Descriptions: Subject identification for | | |
|---|---|---|
| Туре | RefName | Description |
| Form | SUBID | SUBJECT IDENTIFICATION FORM |

| RDE Analytics: RD_SUBID | | |
|-------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| SCRNUMZ | SCRNUMZ | VARCHAR2 |
| | SCRNUMZ_ND | VARCHAR2 |
| INSUBJID | INSUBJID | VARCHAR2 |
| | INSUBJID_ND | VARCHAR2 |
| SUBRAND | SUBRAND_C | VARCHAR2 |
| | SUBRAND | VARCHAR2 |
| | SUBRAND_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 613 Dated: 12 March 2018

| ΙV | IVACFLU-S-0203: DEMOGRAPHICS (DEMOG) [DM] | |
|---|---|---|
| Sul | Subject Information [DM1SC] | |
| 1.* | Informed Consent Signed [ Informed Consent for Screening 1] | [ICFA] [A:1] \( \text{ [ICFADT]} \\ Yes \\ Date of signing \\ Req \( \sqrt{ / Req } \sqrt{ / Req } \( \text{ (2017-2018)} \) [A:2] \( \text{ No} \) |
| Dei | mographic Details [DM2SC] | |
| 2.* | Date of birth<br>[Date of birth] | [DOBDT] |
| 3.* | Ethnicity<br>[Ethnicity] | [DMETH] [A:1] □ Kinh [A:2] □ Khmer [A:3] □ Hoa [A:4] □ Other |
| 4.* Sex [Sex] [GENDR] [A:1] | | |
| | Key: [*] = Item is required [ ✓ ] = Source verification required Note: Source verification critical settings made in Inform will override any settings made in Central Designer. | |

| RDE Analytics: RD_DM | | |
|-----------------------|------------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| ICFA | ICFA_C | VARCHAR2 |
| | ICFA | VARCHAR2 |
| | ICFA_ND | VARCHAR2 |
| ICFA - ICFADT | ICFADT | DATE |
| | ICFADT_DTS | VARCHAR2 |
| DOBDT | DOBDT | DATE |
| | DOBDT_DTS | VARCHAR2 |
| | DOBDT_DTR | VARCHAR2 |
| | DOBDT_ND | VARCHAR2 |
| DMETH | DMETH_ND | VARCHAR2 |
| DMETH - Kinh | DMETH_CITMETH1_C | VARCHAR2 |
| | DMETH_CITMETH1 | VARCHAR2 |
| DMETH - Khmer | DMETH_CITMETH2_C | VARCHAR2 |
| | DMETH_CITMETH2 | VARCHAR2 |
| DMETH - Hoa | DMETH_CITMETH3_C | VARCHAR2 |
| | DMETH_CITMETH3 | VARCHAR2 |
| DMETH - Other | DMETH_CITMETH4_C | VARCHAR2 |
| | DMETH_CITMETH4 | VARCHAR2 |
| GENDER | GENDER_C | VARCHAR2 |
| | GENDER | VARCHAR2 |
| | GENDER_ND | VARCHAR2 |
| GENDER - BEARING | BEARING_C | VARCHAR2 |
| | BEARING | VARCHAR2 |

Protocol No: IVACFLU-S-0203 614 Dated: 12 March 2018

| IV | IVACFLU-S-0203: CURRENT MEDICAL CONDITION (MHX) [MHX] | | | | | |
|---|---|---|---|---|---|---|
| Current Medical Condition [MHXSC] | | | | | | |
| Plea | Please record all current medical conditions on Current Medical Condition form in Screening visit; Please ONLY record concurrent medical conditions if any updates on Day 1. | | | | | |
| 1.* | Does the subject have any current medical conditions/ updates of [Any current medical conditions/ updates on Day 1? ] | tes on Day 1? [MHYN] [A:1] | | | dates on Day 1? | Yes |
| | Current Medical Condition Number | System | Conditi | on | Taking Medication for this current condition? | |
| 2. | | | | | | |
| CUE | RRENT MEDICAL CONDITION Entry [MHX1SC] | | | | | |
| 2.1 | Current Medical Condition Number [read-only] [Current Medical Condition Number] | [MHNUM]<br>N3 | | | | |
| 2.2 | • System<br>[System] | M3 [MHSYS] (A:1] | | | | |
| 2.3 | Condition [Condition] | [MHTERM]<br>A200* | | | | |
| 2.4 | Taking Medication for this current condition? [Taking Medication for this current condition?] | [MHMED] [A:1] ①Yes, Please complete Concomitant Medications form [A:2] ②No | | | | |
| | Key: [*] = Item is required [ ✓ ] = Source verification required [★] = ASCII Only Note: Source verification critical settings made in InForm will override any settings made in Central Designer | | | | | |

| RDE Analytics: RD_MHX | | |
|-----------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| MHYN | MHYN_C | VARCHAR2 |
| | MHYN | VARCHAR2 |
| | MHYN_ND | VARCHAR2 |
| RD_MHX_MHX1SC | | |
| MHNUM | MHNUM | NUMBER |
| | MHNUM_ND | VARCHAR2 |
| MHSYS | MHSYS_C | VARCHAR2 |
| | MHSYS | VARCHAR2 |
| | MHSYS_ND | VARCHAR2 |
| MHSYS - MHSYSSP | MHSYSSP | VARCHAR2 |
| MHTERM | MHTERM | VARCHAR2 |
| | MHTERM_ND | VARCHAR2 |
| MHMED | MHMED_C | VARCHAR2 |
| | MHMED | VARCHAR2 |
| | MHMED_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 615 Dated: 12 March 2018

| IV | IVACFLU-S-0203: SCREENING PHYSICAL EXAM (PE) [PE] | | |
|---|---|---|---|
| | Screening Examination Details [PESC] | | |
| | Examination Date<br>[Examination Date] | [PEVSDT]<br> Req ♥ / Req ♥ / Req ♥ (2017-2018) | |
| Vita | ital Signs [PE1SC] | | |
| | Body temperature (oral)<br>(Body temperature) | [VSTENCMP] [VSTEMP] Body temperature (oral) XX.X °C(b) [VSTRE] Finding [A:1] Normal [A:2] Abnormal - NCS | |
| | | [A:3] | |
| | Blood Pressure [Blood Pressure] | [VSBPCMP] [VSBPCM] [SYSBP] N3 mmHg <sup>[b]</sup> N3 mmHg <sup>[b]</sup> N3 mmHg <sup>[b]</sup> Systolic Diastolic [VSBRE] Finding [A:1] Normal [A:1] Normal - NCS [A:3] NBORMAN - NCS [A:4] NBORMAN - NCS [A:4] NBORM | |
| | Pulse Rate<br> Pulse Rate | [VSHRCMP] [VSHR] Pulse Rate N3 beats/min[b] [VSHRE] Finding [A:1] | |
| Phy | sical Examination [PE2SC] | | |
| 5.*<br>• | Are there any abnormal and clinically significant PE findings?<br>[Any abnormal and clinically significant PE findings?] | [PERES] [A:1] Yes [A:2] No If Yes, please complete Abnormal Findings below. | |
| | PE number | Area/System | Finding |
| 6. | | | |
| _ | ormal Findings Entry [PE3SC] | | 1 |
| 6.1 | PE number [read-only] [PE number] | [PENUM] | |
| 6.2 <sup>*</sup> | Area/System<br>[Area/System] | [PESYSPD] [A:1] [PESYS] [CIPESYS] [A:2] [PEDESOTH] Other, specify: A100 * | |
| 6.3 | Finding<br>[Finding] | [PERES1] [A:1] | |
| Ke | /: [*] = Item is required [ ✓ ] = Source verification required [b] = B | ase Unit [*] = ASCII Only | |

| Codelist Values Tables: SCREENING PHYSICAL EXAM | | | | | |
|---|---|---|---|---|---|
| Codelist RefName | Data Variable RefName | | | | |
| dPESYS | String | General Appearance | 1 | citmPESYS1 | PESYS |
| l l | | ENT | 2 | citmPESYS2 | |
| | | Neurologic | 8 | citmPESYS8 | 1 |
| | | Chest auscultation | 6 | citmPESYS6 | |
| | | Lymph nodes (cervical & axillary) | 4 | citmPESYS4 | |
| | | Abdomen palpation | 7 | citmPESYS7 | |
| | | Musculoskeletal | 9 | citmPESYS9 | |

| RDE Analytics: RD_PE | | |
|-----------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| PEVSDT | PEVSDT | DATE |
| | PEVSDT_DTS | VARCHAR2 |

Version 1.0 Protocol No: IVACFLU-S-0203 616 Dated: 12 March 2018

| | PEVSDT_ND | VARCHAR2 |
|--------------------|-------------|----------|
| VSTEMCMP | VSTEMCMP_ND | VARCHAR2 |
| VSTEMCMP - VSTEMP | VSTEMP | FLOAT |
| | VSTEMP_U | VARCHAR2 |
| VSTEMCMP - VSTRE | VSTRE_C | VARCHAR2 |
| | VSTRE | VARCHAR2 |
| VSTEMCMP - VSTGR | VSTGR_C | VARCHAR2 |
| | VSTGR | VARCHAR2 |
| VSBPCMP | VSBPCMP_ND | VARCHAR2 |
| VSBPCMP - SYSBP | SYSBP | NUMBER |
| | SYSBP_U | VARCHAR2 |
| VSBPCMP - DIABP | DIABP | NUMBER |
| | DIABP_U | VARCHAR2 |
| VSBPCMP - VSBRE | VSBRE_C | VARCHAR2 |
| | VSBRE | VARCHAR2 |
| VSBPCMP - VBSGR | VBSGR_C | VARCHAR2 |
| | VBSGR | VARCHAR2 |
| VSHRCMP | VSHRCMP_ND | VARCHAR2 |
| VSHRCMP - VSHR | VSHR | NUMBER |
| | VSHR_U | VARCHAR2 |
| VSHRCMP - VSHRE | VSHRE_C | VARCHAR2 |
| | VSHRE | VARCHAR2 |
| VSHRCMP - HRSPec | HRSPEC | VARCHAR2 |
| PERES | PERES_C | VARCHAR2 |
| | PERES | VARCHAR2 |
| | PERES_ND | VARCHAR2 |
| RD_PE_PE3SC | | |
| PENUM | PENUM | NUMBER |
| | PENUM_ND | VARCHAR2 |
| PESYSPD | PESYSPD_C | VARCHAR2 |
| | PESYSPD | VARCHAR2 |
| | PESYSPD_ND | VARCHAR2 |
| PESYSPD - PESYS | PESYS_C | VARCHAR2 |
| | PESYS | VARCHAR2 |
| PESYSPD - PEDESOTH | PEDESOTH | VARCHAR2 |
| PERES1 | PERES1_C | VARCHAR2 |
| | PERES1 | VARCHAR2 |
| | PERES1_ND | VARCHAR2 |
| PERES1 - PECM | PECM | VARCHAR2 |

Protocol No: IVACFLU-S-0203 617 Dated: 12 March 2018

| ΤΛ | ACFLU-S-0203: URINE PREGNANCY TEST (UPREG) [UPREG] | |
|---|---|---|
| Uri | ine Pregnancy Test [UPREGSC] | |
| 1.*<br>• | Date of Urine Collection [Date of Urine Collection] | [UPREGDT]<br> Req ☑ / Req ☑ / Req ☑ (2017-2018) |
| 2.* | Result Reading Time<br>[Result Reading Time] | [UPREGTM] Req ☑ : Req ☑ 24-hour clock |
| 3.*<br>• | Result:<br>[Result] | [UPREGRES] [A:1] O Positive [A:2] Negative |

| RDE Analytics: RD_UPREG | | |
|---|---|---|
| Data Variable RefName RD Column Name Column Data T | | |
| UPREGDT | UPREGDT | DATE |
| | UPREGDT_DTS | VARCHAR2 |
| | UPREGDT_ND | VARCHAR2 |
| UPREGTM | UPREGTM | DATE |
| | UPREGTM_TMS | VARCHAR2 |
| | UPREGTM_ND | VARCHAR2 |
| UPREGRES | UPREGRES_C | VARCHAR2 |
| | UPREGRES | VARCHAR2 |
| | UPREGRES_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 618 Dated: 12 March 2018



| RDE Analytics: RD_ELIG | | |
|----------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| ELIGYN | ELIGYN_C | VARCHAR2 |
| | ELIGYN | VARCHAR2 |
| | ELIGYN_ND | VARCHAR2 |
| ELIGYN - ELIGRES | ELIGRES_C | VARCHAR2 |
| | ELIGRES | VARCHAR2 |
| ELIGYN - ELIGNUM | ELIGNUM | VARCHAR2 |
| ELIGYN - ELIGOTHC | ELIGOTHC | VARCHAR2 |
| ELIGRANDYN | ELIGRANDYN_C | VARCHAR2 |
| | ELIGRANDYN | VARCHAR2 |
| | ELIGRANDYN_ND | VARCHAR2 |
| ELIGRANDYN - ELIGSUBID | ELIGSUBID | VARCHAR2 |
| ELIGRANDYN - ELIGSFREAS | ELIGSFREAS_C | VARCHAR2 |
| | ELIGSFREAS | VARCHAR2 |
| ELIGRANDYN - ELIGSFREASOTH | ELIGSFREASOTH | VARCHAR2 |

Protocol No: IVACFLU-S-0203 619 Dated: 12 March 2018

| ΙV | IVACFLU-S-0203: TARGETED PE (TPE) [TPE] | | |
|---|---|---|---|
| Targeted PE [TPESC] | | | |
| 1.* | Was the Targeted PE done? | [PETVSYN] | |
| - | [Was the Targeted PE done?] | [A:1] [PETVSDT] | |
| | | Yes Examination Date | |
| | | Req 🕶 / Req 🕶 / Req 🕶 (2017-2018) | |
| | | [A:2] ONO | |
| Vita | ital Signs [TPE1SC] | | |
| 2. | Body temperature (oral) | [VSTEMPCMP1] | |
| ~ | [Body temperature] | [VSTEMP1] xx.x °C[b] | |
| | | [VSTEMPF] | |
| | | Finding | |
| | | [A:1] Normal | |
| | | [A:2] OAbnormal, NCS [A:3] [VSTEMP1GR] | |
| | | Abnormal, CS<br>Grading Scale | |
| | | [A:0] Oungradable | |
| | | [A:1] (1 (38.0 - <38.6°C) | |
| | | [A:2] (2 (38.6 - <39.3°C) | |
| | | [A:3] | |
| 2 | Plond Braceura | [VSBPCMP2] | |
| 3. | Blood Pressure<br>[Blood Pressure] | [VSBPCMP1] | |
| | | [SYSBP1] [DIABP1] N3 mmHg[b] N3 mmHg[b] | |
| | | Systolic Diastolic | |
| | | [VSBPF] | |
| | | Finding [A:1] Normal | |
| | | [A:2] OAbnormal, NCS | |
| | | [A:3] [VBBPG1] | |
| | | Abnormal, CS<br>Grading Scale | |
| | | [A:0] O Ungradable | |
| | | [A:1] $\bigcirc$ 1 140 to < 160 mmHg systolic OR 90 to < 100 mr<br>[A:2] $\bigcirc$ 2 $\geq$ 160 to < 180 mmHg systolic OR $\geq$ 100 to < 1 | |
| | | [A:3] $\bigcirc$ 3 $\geq$ 180 mmHg systolic OR $\geq$ 110 mmHg diastolic | 10 mmig diastolic |
| | | [A:4] O4 Life Threatening | |
| 4. | Pulse Rate | [VSHRCMP1] | |
| ~ | [Pulse Rate] | [VSHR1] N3 beats/min <sup>[b]</sup> | |
| | | N3 beats/minter [VSHRF] | |
| | | Finding | |
| | | [A:1] ONormal | |
| | | [A:2] OAbnormal, NCS [A:3] O[VSBPSP1] | |
| | | Abnormal, CS | |
| | | Specify: A200* | |
| T- | geted Dhysical Evamination (TDE2CC) | | |
| 5. | geted Physical Examination [TPE2SC] Physical examination is not required unless subject reports | [PETVSYN1] | |
| J. | symptoms. Did the subject have any symptoms that required | [A:1] QYes | |
| | evaluation? [Did the subject have any symptoms that required evaluation?] | [A:2] | |
| Н | | If Yes, please complete Abnormal Findings below. | Eind: |
| 6. | PE number | Area/System | Finding |
| ٠<br>• | | | |
| Abı | normal Findings Entry [TPE3SC] | | |
| 6.1 | PE number [read-only] [PE number] | [TPENUM] | |
| <u> </u> | | N3 | |
| 6.2 | * Area/System<br>[Area/System] | [TPESYSPD] [A:1] [TPESYS] | |
| • | [///cd/system] | [clTPESYS] 🗸 | |
| | | [A:2] Other specify: | |
| | | Other, specify: A200* | |
| - | * Finding | [TPERES] | |
| 6.3 | [Finding] | [A:1] Abnormal, NCS | |
| | | [A:2] [TPEDES] | |
| | | Abnormal, CS<br>Specify current medical condition number if Day 1, AE numl | ber if other visit |
| | | A200* | |
| Ke | Key: [*] = Item is required [▼] = Source verification required [b] = Base Unit [★] = ASCII Only | | |
| No | Note: Source verification critical settings made in Inform will override any settings made in Central Designer. | | |

| Codelist Values Tables: TARGETED PE | | | | | |
|---|---|---|---|---|---|
| Codelist RefName | Codelist Data Type | Label | Code | Codelist Item RefName | Data Variable RefName |
| cITPESYS | String | ENT | 1 | citmTPESYS1 | TPESYS |
| | | Neurological | 2 | citmTPESYS2 | |
| | | Chest auscultation | 3 | citmTPESYS3 | |
| | | Heart auscultation | 4 | citmTPESYS4 | |
| | | Abdomen | 5 | citmTPESYS5 | |
| | | Lymph nodes | 6 | citmTPESYS6 | |

Protocol No: IVACFLU-S-0203 620 Dated: 12 March 2018

| RDE Analytics: RD_TPE | | |
|------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| PETVSYN | PETVSYN_C | VARCHAR2 |
| | PETVSYN | VARCHAR2 |
| | PETVSYN_ND | VARCHAR2 |
| PETVSYN - PETVSDT | PETVSDT | DATE |
| | PETVSDT_DTS | VARCHAR2 |
| VSTEMPCMP1 | VSTEMPCMP1_ND | VARCHAR2 |
| VSTEMPCMP1 - VSTEMP1 | VSTEMP1 | FLOAT |
| | VSTEMP1_U | VARCHAR2 |
| VSTEMPCMP1 - VSTEMPF | VSTEMPF_C | VARCHAR2 |
| | VSTEMPF | VARCHAR2 |
| VSTEMPCMP1 - VSTEMP1GR | VSTEMP1GR_C | VARCHAR2 |
| | VSTEMP1GR | VARCHAR2 |
| VSBPCMP2 | VSBPCMP2_ND | VARCHAR2 |
| VSBPCMP2 - SYSBP1 | SYSBP1 | NUMBER |
| | SYSBP1_U | VARCHAR2 |
| VSBPCMP2 - DIABP1 | DIABP1 | NUMBER |
| | DIABP1_U | VARCHAR2 |
| VSBPCMP2 - VSBPF | VSBPF_C | VARCHAR2 |
| | VSBPF | VARCHAR2 |
| VSBPCMP2 - VBBPG1 | VBBPG1_C | VARCHAR2 |
| | VBBPG1 | VARCHAR2 |
| VSHRCMP1 | VSHRCMP1_ND | VARCHAR2 |
| VSHRCMP1 - VSHR1 | VSHR1 | NUMBER |
| | VSHR1_U | VARCHAR2 |
| VSHRCMP1 - VSHRF | VSHRF_C | VARCHAR2 |
| | VSHRF | VARCHAR2 |
| VSHRCMP1 - VSBPSP1 | VSBPSP1 | VARCHAR2 |
| PETVSYN1 | PETVSYN1_C | VARCHAR2 |
| | PETVSYN1 | VARCHAR2 |
| | PETVSYN1_ND | VARCHAR2 |
| RD_TPE_TPE3SC | | |
| TPENUM | TPENUM | NUMBER |
| | TPENUM_ND | VARCHAR2 |
| TPESYSPD | TPESYSPD_C | VARCHAR2 |
| | TPESYSPD | VARCHAR2 |
| | TPESYSPD_ND | VARCHAR2 |
| TPESYSPD - TPESYS | TPESYS_C | VARCHAR2 |
| | TPESYS | VARCHAR2 |
| TPESYSPD - TPEDESOTH | TPEDESOTH | VARCHAR2 |
| TPERES | TPERES_C | VARCHAR2 |
| | TPERES | VARCHAR2 |
| | TPERES_ND | VARCHAR2 |
| TPERES - TPEDES | TPEDES | VARCHAR2 |

Protocol No: IVACFLU-S-0203 621 Dated: 12 March 2018

| IVACFLU-S-0203: ANTI-INFLUENZA SEROLOGIC ASSAY (ANTI INF SER) [AISA] |
|---|
| Anti-Influenza Serologic Assay [AISASC] |
| 1. * Was the blood sample collected? [AISPERF] [A:1] ○[AISADT] Yes Date and Time of blood collection Req □ / Req □ / Req □ (2017-2018) Req □ : Req □ 24-hour clock [A:2] ○ No |
| Key: [*] = Item is required [✓] = Source verification required Note: Source verification critical settings made in Inform will override any settings made in Central Designer. |

| RDE Analytics: RD_AISA | | |
|------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| AISPERF | AISPERF_C | VARCHAR2 |
| | AISPERF | VARCHAR2 |
| | AISPERF_ND | VARCHAR2 |
| AISPERF - AISADT | AISADT | DATE |
| | AISADT_DTS | VARCHAR2 |

Protocol No: IVACFLU-S-0203 622 Dated: 12 March 2018

| ΙV | VACFLU-S-0203: VACCINATION (VAC) [VAC] | |
|---|---|---|
| Sub | ubject Vaccination [VAC3SC] | |
| 1.* | Was the subject given an injection of the study product at this visit? [Was the subject given an injection of the study product at this visit?] | [VACCYN] [A:1] ○Yes [A:2] ○ [VACOTH] No please specify reason and please complete Day 1 visit. A200 * |
| Rar | Randomization Code [VAC1SC] | |
| 2. | Study product code:<br>[Study product code] | [ELIGPROD] A5* |
| Vac | ccination [VAC2SC] | |
| 3. | Date and Time of Vaccination [Date and Time of Vaccination] | [VACDT] Req ♥ / Req ♥ (2017-2018) Req ♥ : Req ▼ 24-hour clock |
| | In which arm was the injection given? [In which arm was the injection given?] | [VACARM] [A:1] OLeft [A:2] ORight |
| | Key: [ v ] = Source verification required [ *] = ASCII Only Note: Source verification critical settings made in Inform will override any settings made in Central Designer. | |

| RDE Analytics: RD_VAC | | |
|-----------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| VACCYN | VACCYN_C | VARCHAR2 |
| | VACCYN | VARCHAR2 |
| | VACCYN_ND | VARCHAR2 |
| VACCYN - VACOTH | VACOTH | VARCHAR2 |
| ELIGPROD | ELIGPROD | VARCHAR2 |
| | ELIGPROD_ND | VARCHAR2 |
| VACDT | VACDT | DATE |
| | VACDT_DTS | VARCHAR2 |
| | VACDT_ND | VARCHAR2 |
| VACARM | VACARM_C | VARCHAR2 |
| | VACARM | VARCHAR2 |
| | VACARM_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 Dated: 12 March 2018

| - | ACFLU-S-0203: 30-MINUTE REACTOGENICITY (ROG) [ROG] | |
|---|---|---|
| 30 | Minutes [ROG4SC] | T. |
| 1.* | Temperature (Temperature) | [ROGTEMP30] |
| \ \ \ | [Temperature] | Temperature (oral) XX.X °C[b] |
| | | [ROGTEMFD] |
| | | Finding [A:1] Normal |
| | | [A:2] Abnormal, NCS |
| | | [A:3] [ROGYGS30] |
| | | Abnormal, CS |
| | | Grading Scale [A:0] Olngradable |
| | | [A:1] (38.0 - <38.6°C) |
| | | [A:2] O2 (38.6 - <39.3°C) |
| | | [A:3] (39.3 - <40.0°C) |
| | | [A:4] ○4 (≥ 40.0°C) |
| 2.* | Any local / systemic reaction? | [ROGYN30] |
| Z. | [Any local / systemic reaction?] | [A:2] No |
| | | [A:1] OYes |
| | | (If Yes, complete below) |
| 30 | Minutes Local Reactions [ROG5SC] | |
| 3. | Redness (cm) | [ROGREDPD30] |
| ~ | [Redness] | [A:1] None |
| | | [A:2] [ROGRED30C0] |
| | | [ROGRED30] xx.x cm <sup>[b]</sup> |
| | | [ROGRED30GR] Grade [A:0] Oungradable |
| | | [A:1] 1, 2.5 to < 5 cm in diameter |
| | | [A:2] 02, 5 to < 10 cm in diameter |
| | | [A:3] ()3, >= 10 cm in diameter |
| | | [A:4] 04, Necrosis, or exfoliative dermatitis (for redness) |
| 4. | Swelling (cm) | [ROGSWELLPD30] |
| Ü | [Swelling] | [A:1] None |
| | | [A:2] [ROGSWE30CO] |
| | | [ROGSWELL30] |
| | | xx.x cm <sup>[b]</sup> |
| | | [ROGSWE30GR] |
| | | Grade [A:0] ○Ungradable |
| | | [A:1] ①1, 2.5 to < 5 cm in diameter |
| | | [A:2] Q2, 5 to < 10 cm in diameter |
| | | [A:3] 03, >= 10 cm in diameter [A:4] 04, Necrosis, or exfoliative dermatitis (for redness) |
| _ | | _ |
| 5. | Induration (hardness) (cm) | [ROGINDPD30] |
| | [Induration] | [A:1] None<br>[A:2] [ROGIND30CO] |
| | | [ROGIND30] |
| | | xx.x cm <sup>[b]</sup> |
| | | [ROGIND30GR] |
| | | Grade [A:0] Oungradable |
| | | [A:1] 01, 2.5 to < 5 cm in diameter |
| | | [A:2] Q2, 5 to < 10 cm in diameter |
| | | [A:3] (A:3) (A:3) 3, >= 10 cm in diameter |
| | | [A:4] Q4, Necrosis, or exfoliative dermatitis (for redness) |
| 6. | Pain | [ROGPAIN30] |
| ~ | [Pain] | [cIROGRES] |
| 7. | Tenderness | [ROGTEND30] |
| ~ | [Tenderness] | [clROGRES] V |
| 30 | <br>Minutes Systemic Reactions [ROG6SC] | |
| - | | [DOCTION 201 |
| 8. | Fatigue/Malaise<br>[Fatigue/Malaise] | [ROGTIRED30] [CIROGRES] |
| Ŀ | | |
| 9. | Generalized Muscle Aches | [ROGMUSCLE30] |
| Ľ | [Generalized Muscle Aches] | [clROGRES] |
| | Joint Aches | [ROGJOINT30] |
| ~ | [Joint Aches] | [ciROGRES] |
| 11. | Chills | [ROGCHILLS30] |
| ¥. | [Chills] | [cirogres] |
| 12 | Neuron | [DOCNAUSEA20] |
| 12. | Nausea<br>[Nausea] | [ROGNAUSEA30] [ciROGRES] |
| 13. | Vomiting | [ROGVOM30] |
| _ | [Vomiting] | [clROGRES] 🗸 |
| 14. | Headache | [ROGHEAD30] |
| ~ | [Headache] | [cIROGRES] |
| V. | ey: [ ] = Source verification required [b] = Base Unit | |
| | by: $[ \lor ] = Source verification required [b] = Base Unitthe: Source verification critical settings made in InForm will override any settings made in Central Desi$ | gner. |

| Codelist Values Tables: 30-MINUTE REACTOGENICITY | | | | | |
|---|---|---|---|---|---|
| Codelist RefName | Codelist Data Type | Label | Code | Codelist Item RefName | Data Variable RefName |
| dROGRES | String | 0, None | 1 | citmROGRES1 | ROGPAIN30,<br>ROGTEND30, |
| | | 1, Mild | 2 | citmROGRES2 | ROGTIRED30,<br>ROGMUSCLE30, |
| | | 2, Moderate | 3 | citmROGRES3 | ROGJOINT30, |
| | | 3, Severe | 4 | CITMROGRES4 | ROGCHILLS30,<br>ROGNAUSEA30, |
| | | 4, Potentially Life Threatening | 5 | citmRoGERRE5 | ROGVOM30,<br>ROGHEAD30 |

| RDE Analytics: RD_ROG | | |
|-----------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| ROGTEMCO | ROGTEMCO_ND | VARCHAR2 |
| ROGTEMCO - ROGTEMP30 | ROGTEMP30 | FLOAT |

Dated: 12 March 2018

| Protocol No: IVACFLU-S-02 | 03 | | |
|---------------------------|----|---|---|
| I | I | 1 | 1 |

| | ROGTEMP30_U | VARCHAR2 |
|---------------------------|-----------------|----------|
| ROGTEMCO - ROGTEMFD | ROGTEMFD_C | VARCHAR2 |
| | ROGTEMFD | VARCHAR2 |
| ROGTEMCO - ROGYGS30 | ROGYGS30_C | VARCHAR2 |
| | ROGYGS30 | VARCHAR2 |
| ROGYN30 | ROGYN30_C | VARCHAR2 |
| | ROGYN30 | VARCHAR2 |
| | ROGYN30_ND | VARCHAR2 |
| ROGREDPD30 | ROGREDPD30_C | VARCHAR2 |
| NOGINEEN BS0 | ROGREDPD30 | VARCHAR2 |
| | ROGREDPD30_ND | VARCHAR2 |
| ROGREDPD30 - ROGRED30 | ROGRED30_ND | FLOAT |
| ROGREDFD30 - ROGRED30 | ROGRED30_U | VARCHAR2 |
| ROGREDPD30 - ROGRED30GR | | VARCHAR2 |
| RUGREDPD30 - RUGRED30GR | ROGRED30GR_C | |
| | ROGRED30GR | VARCHAR2 |
| ROGSWELLPD30 | ROGSWELLPD30_C | VARCHAR2 |
| | ROGSWELLPD30 | VARCHAR2 |
| | ROGSWELLPD30_ND | |
| ROGSWELLPD30 - ROGSWELL30 | ROGSWELL30 | FLOAT |
| | ROGSWELL30_U | VARCHAR2 |
| ROGSWELLPD30 - ROGSWE30GR | ROGSWE30GR_C | VARCHAR2 |
| | ROGSWE30GR | VARCHAR2 |
| ROGINDPD30 | ROGINDPD30_C | VARCHAR2 |
| | ROGINDPD30 | VARCHAR2 |
| | ROGINDPD30_ND | VARCHAR2 |
| ROGINDPD30 - ROGIND30 | ROGIND30 | FLOAT |
| | ROGIND30_U | VARCHAR2 |
| ROGINDPD30 - ROGIND30GR | ROGIND30GR_C | VARCHAR2 |
| | ROGIND30GR | VARCHAR2 |
| ROGPAIN30 | ROGPAIN30_C | VARCHAR2 |
| | ROGPAIN30 | VARCHAR2 |
| | ROGPAIN30_ND | VARCHAR2 |
| ROGTEND30 | ROGTEND30_C | VARCHAR2 |
| | ROGTEND30 | VARCHAR2 |
| | ROGTEND30_ND | VARCHAR2 |
| ROGTIRED30 | ROGTIRED30_C | VARCHAR2 |
| | ROGTIRED30 | VARCHAR2 |
| | ROGTIRED30_ND | VARCHAR2 |
| ROGMUSCLE30 | ROGMUSCLE30_C | VARCHAR2 |
| NOGI-103CEE30 | ROGMUSCLE30 | VARCHAR2 |
| | ROGMUSCLE30_ND | VARCHAR2 |
| ROGIOINT30 | | VARCHAR2 |
| ROGJOINT30 | ROGJOINT30_C | |
| | ROGJOINT30 | VARCHAR2 |
| | ROGJOINT30_ND | VARCHAR2 |
| ROGCHILLS30 | ROGCHILLS30_C | VARCHAR2 |
| | ROGCHILLS30 | VARCHAR2 |
| | ROGCHILLS30_ND | VARCHAR2 |
| ROGNAUSEA30 | ROGNAUSEA30_C | VARCHAR2 |
| | ROGNAUSEA30 | VARCHAR2 |
| | ROGNAUSEA30_ND | VARCHAR2 |
| ROGVOM30 | ROGVOM30_C | VARCHAR2 |
| | ROGVOM30 | VARCHAR2 |
| | ROGVOM30_ND | VARCHAR2 |
| ROGHEAD30 | ROGHEAD30_C | VARCHAR2 |
| | ROGHEAD30 | VARCHAR2 |
| | ROGHEAD30_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 625 Dated: 12 March 2018

| ΙV | [VACFLU-S-0203: Contact (TELECONT) [TELECONT] | |
|---|---|---|
| Cor | Contact [TELECONT] | |
| 1.* Date of contact [Date of contact] TELEDATE Req V / Req V / Req V (2017-2018) | | |
| | Subject Contacted? [Subject Contacted?] | [TELEYN] [A:1] |
| Key: [*] = Item is required [✓] = Source verification required Note: Source verification critical settinos made in Inform will override any settinos made in Central Designer. | | |

| Study | Study Object Descriptions: Contact | |
|-------|------------------------------------|-------------|
| Туре | RefName | Description |
| Form | TELECONT | CONTACT |

| RDE Analytics: RD_TELECONT | | |
|----------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| TELEDATE | TELEDATE | DATE |
| | TELEDATE_DTS | VARCHAR2 |
| | TELEDATE_ND | VARCHAR2 |
| TELEYN | TELEYN_C | VARCHAR2 |
| | TELEYN | VARCHAR2 |
| | TELEYN_ND | VARCHAR2 |


Dated: 12 March 2018

| 1.* | al Reactogenicity [SLRSC] Did the subject report any local reactogenicity during Days 1 to 7? | [SLRYN] |
|---|---|---|
| • | [Did the subject report any local reactogenicity during Days 1 to 7?] | [A:1] O Yes<br>[A:2] O No |
| ai | n at injection site [SLR2SC] Pain at injection site | [SLRPAINWK] |
| - | [Pain at injection site] | [A:1] None all week |
| 3.<br>• | Evening Day 1 [Day 1 Pain at injection site] | [SLRPAIND1] [cIROGRES] |
| 4.<br>• | Day 2 [Day 2 Pain at injection site] | [SLRPAIND2] [clrOGRES] |
| 5.<br>✔ | Day 3 [Day 3 Pain at injection site] | [SIRPAIND3] [cIROGRES] |
| 5.<br>• | Day 4 [Day 4 Pain at injection site] | [SLRPAIND4]<br>[cirogres] |
| 7.<br>• | Day 5<br>[Day 5 Pain at injection site] | [SLRPAINDS] [cIROGRES] |
| B.<br>✔ | Day 6 [Day 6 Pain at injection site] | [SLRPAIND6] [cIROGRES] |
| 9.<br>• | Day 7 [Day 7 Pain at injection site] | [SLRPAIND7] [cIROGRES] |
| 10. | After Day 7: Ongoing? [Ongoing] | [SLRPAINONG] [A:2] \( \)\ \ |
| Ter | derness at injection site [SLR3SC] | |
| 11.<br>• | derness at injection site [SLRSSU] Tenderness at injection site [Tenderness at injection site] | [SLRTENDWK] [A:1] None all week |
| 12. | Evening Day 1 [Day 1 Tenderness at injection site] | [SLRTENDD1] [CIROGRES] |
| 13.<br>• | Day 2<br>[Day 2 Tenderness at injection site] | [SLRTENDD2] [cIROGRES] |
| 14.<br>• | Day 3<br>[Day 3 Tenderness at injection site] | [SLRTENDD3] [cirogres] |
| 15.<br>• | Day 4 [Day 4 Tenderness at injection site] | [SLRTENDD4] [clROGRES] |
| 16.<br>• | Day 5<br>[Day 5 Tenderness at injection site] | [SLRTENDDS] [cIROGRES] |
| 17.<br>• | Day 6<br>[Day 6 Tenderness at injection site] | [SLRTENDD6] [cIROGRES] |
| 18.<br>• | Day 7<br>[Day 7 Tenderness at injection site] | [SLRTENDD7] [clROGRES] |
| 19. | After Day 7: Ongoing? [Ongoing] | [SLRTENDONG] [A:2] ○ No [A:1] ○ [SLRTENDONGCMP] Yes [SLRTENDSEV] Highest severity until resolution: [cliseV] □ [SLRTENDEDAT] End date Req ○ / Req ○ / Req ○ (2017-2018) |
| Rec | Iness at injection site [SLR4SC] | |
| 20. | Redness at injection site [Redness at injection site] | [SLRREDWK] [A:1] None all week |
| 21. | Evening Day 1 [Day 1 Redness at injection site] | [SLREDD1]<br>[cIROGRES] ✓ |
| 22. | Day 2<br>[Day 2 Redness at injection site] | [SLREDD2] [CIROGRES] |
| 23.<br>• | Day 3<br>[Day 3 Redness at injection site] | [SLREDD3] [cirogres] |
| 24.<br>• | Day 4<br>[Day 4 Redness at injection site] | [SLREDD4] [cIROGRES] ✓ |
| 25.<br>• | Day 5<br>[Day 5 Redness at injection site] | [SLREDD5] [CIROGRES] ✓ |
| 26.<br>• | Day 6<br>[Day 6 Redness at injection site] | [SLREDD6] [CIROGRES] |
| 27.<br>• | Day 7<br>[Day 7 Redness at injection site] | [SLREDD7] [CIROGRES] |
| 28. | After Day 7: Ongoing? [Ongoing] | [SLRREDONG] [A:2] ○ NO [A:1] ○ [SLRREDONGCMP] Yes [SLRREDSEV] Highest severity until resolution: [clSEV] ▼ [SLRREDEDAT] End date Req ▼ / Req ▼ / Req ▼ (2017-2018) |
| | elling at injection site [SLR5SC] Swelling at injection site | [SLRSWELLWK] |

Protocol No: IVACFLU-S-0203 627 Dated: 12 March 2018

| 31. | Day 2<br>[Day 2 Swelling at injection site] | [SLRSWELLD2] [cIROGRES] |
|---|---|---|
| 32.<br>• | Day 3<br>[Day 3 Swelling at injection site] | [SLRSWELLD3] [CIROGRES] |
| 33. | Day 4<br>[Day 4 Swelling at injection site] | [SLRSWELLD4] [CIROGRES] |
| 34. | Day 5<br>[Day 5 Swelling at injection site] | [SLRSWELLD5] [CIROGRES] |
| 35.<br>• | Day 6<br>[Day 6 Swelling at injection site] | [SLRSWELLD6]<br>[CIROGRES] |
| 36.<br>✔ | Day 7<br>[Day 7 Swelling at injection site] | [SLRSWELLD7] [cIROGRES] |
| 37. | After Day 7: Ongoing? [Ongoing] | [SLRSWELLONG] [A:12] No [A:12] SLRSWELLONGCMP] Yes Highest severity until resolution: [cisev] [cisev] [SLRSWELLEDAT] End date Req / Req / Req (2017-2018) |
| Har | dness at injection site [SLR6SC] | |
| 38.<br>✓ | Hardness at injection site<br>[Hardness at injection site] | [SLRINDWK] [A:I] □None all week |
| 39.<br>✔ | Evening Day 1 [Day 1 Hardness at injection site] | [SLRINDD1] [clrogres] |
| 40.<br>• | Day 2<br>[Day 2 Hardness at injection site] | [SLRINDD2] [cIROGRES] |
| 41. | Day 3<br>[Day 3 Hardness at injection site] | [SLRINDD3]<br>[CIROGRES] |
| 42.<br>• | Day 4<br>[Day 4 Hardness at injection site] | [SLRINDD4] [cIROGRES] |
| 43.<br>• | Day 5<br>[Day 5 Hardness at injection site] | [SLRINDD5] [CIROGRES] |
| 44.<br>• | Day 6 [Day 6 Hardness at injection site] | [SLRINDD6]<br>[cIROGRES] |
| 45.<br>• | Day 7<br>[Day 7 Hardness at injection site] | [SLRINDD7] [cirogres] |
| 46. | After Day 7: Ongoing? [Ongoing] | [SLRINDONG] [A:2] No [A:12] SLRINDONGCMP] Yes [SLRINDSEV] Highest severity until resolution: [CISEV] |
| | | [SLRINDEDAT] End date Req / Req / Req (2017-2018) |
| | ey: $[*]$ = Item is required $[\checkmark]$ = Source verification required<br>the: Source verification critical settings made in InForm will override any settings made in Central Desi | gner. |

| Codelist RefName | Codelist Data Type | Label | Code | Codelist Item RefName | Data Variable RefName |
|---|---|---|---|---|---|
| dROGRES | String | 0, None | 1 | citmROGRES1 | SLRPAIND1,<br>SLRPAIND2,<br>SLRPAIND3,<br>SLRPAIND4,<br>SLRPAIND5,<br>SLRPAIND5,<br>SLRPAIND5,<br>SLRPAIND7, |
| | | 1, Mild | 2 | citmROGRES2 | SLRTENDD1,<br>SLRTENDD1,<br>SLRTENDD2,<br>SLRTENDD3,<br>SLRTENDD4,<br>SLRTENDD5,<br>SLRTENDD6,<br>SLRTENDD7. |
| | | 2, Moderate | 3 | citmROGRES3 | SLRREDD1,<br>SLRREDD2,<br>SLRREDD3,<br>SLRREDD4,<br>SLRREDD5,<br>SLRREDD6,<br>SLRREDD7, |
| | | 3, Severe | 4 | CITMROGRES4 | SLRSWELLD1,<br>SLRSWELLD2,<br>SLRSWELLD3,<br>SLRSWELLD4,<br>SLRSWELLD5,<br>SLRSWELLD6,<br>SLRSWELLD7, |
| | | 4, Potentially Life Threatening | 5 | citmRoGERRE5 | SLRINDD1,<br>SLRINDD2,<br>SLRINDD3,<br>SLRINDD4,<br>SLRINDD5,<br>SLRINDD6,<br>SLRINDD7 |
| cISEV | String | Grade 1 | 1 | citmSEV1 | SLRPAINSEV, |
| | | Grade 2 | 2 | citmSEV2 | SLRTENDSEV,<br>SLRREDSEV, |
| | | Grade 3 | 3 | citmSEV3 | SLRSWELLSEV,<br>SLRINDSEV |
| | | Grade 4 | 4 | citmSEV4 | SERTINDSEN |

| RDE Analytics: RD_SLR | |
|-----------------------|------------------------------|
| RD Column Name | Column Data Type |
| SLRYN_C | VARCHAR2 |
| SLRYN | VARCHAR2 |
| SLRYN_ND | VARCHAR2 |
| | RD Column Name SLRYN_C SLRYN |

Dated: 12 March 2018

| SLRPAINWK | SLRPAINWK_C | VARCHAR2 |
|---|---|---|
| | SLRPAINWK | VARCHAR2 |
| | SLRPAINWK_ND | VARCHAR2 |
| SLRPAIND1 | SLRPAIND1_C | VARCHAR2 |
| | SLRPAIND1 | VARCHAR2 |
| | SLRPAIND1_ND | VARCHAR2 |
| SLRPAIND2 | SLRPAIND2_C | VARCHAR2 |
| | SLRPAIND2<br>SLRPAIND2 ND | VARCHAR2<br>VARCHAR2 |
| SLRPAIND3 | SLRPAIND3_C | VARCHAR2<br>VARCHAR2 |
| SERFAINDS | SLRPAIND3_C | VARCHAR2 |
| | SLRPAIND3_ND | VARCHAR2 |
| SLRPAIND4 | SLRPAIND4_C | VARCHAR2 |
| | SLRPAIND4 | VARCHAR2 |
| | SLRPAIND4_ND | VARCHAR2 |
| SLRPAIND5 | SLRPAIND5_C | VARCHAR2 |
| | SLRPAIND5 | VARCHAR2 |
| | SLRPAIND5_ND | VARCHAR2 |
| SLRPAIND6 | SLRPAIND6_C | VARCHAR2 |
| | SLRPAIND6 | VARCHAR2 |
| | SLRPAIND6_ND | VARCHAR2 |
| SLRPAIND7 | SLRPAIND7_C | VARCHAR2<br>VARCHAR2 |
| | SLRPAIND7<br>SLRPAIND7_ND | VARCHAR2 |
| SLRPAINONG | SLRPAINONG_C | VARCHAR2 |
| SERI AINONG | SLRPAINONG | VARCHAR2 |
| | SLRPAINONG_ND | VARCHAR2 |
| SLRPAINONG - SLRPAINSEV | SLRPAINSEV_C | VARCHAR2 |
| | SLRPAINSEV | VARCHAR2 |
| SLRPAINONG - SLRPAINEDAT | SLRPAINEDAT | DATE |
| | SLRPAINEDAT_DTS | VARCHAR2 |
| SLRTENDWK | SLRTENDWK_ND | VARCHAR2 |
| SLRTENDWK - None all week | SLRTENDWK_CITMNONEWEEK1_C | VARCHAR2 |
| | SLRTENDWK_CITMNONEWEEK1 | VARCHAR2 |
| SLRTENDD1 | SLRTENDD1_C | VARCHAR2 |
| | SLRTENDD1 | VARCHAR2 |
| | SLRTENDD1_ND | VARCHAR2 |
| SLRTENDD2 | SLRTENDD2_C | VARCHAR2 |
| | SLRTENDD2<br>SLRTENDD2_ND | VARCHAR2<br>VARCHAR2 |
| SLRTENDD3 | SLRTENDD3_C | VARCHAR2 |
| SERVENDOS | SLRTENDD3 | VARCHAR2 |
| | SLRTENDD3_ND | VARCHAR2 |
| SLRTENDD4 | SLRTENDD4_C | VARCHAR2 |
| | SLRTENDD4 | VARCHAR2 |
| | SLRTENDD4_ND | VARCHAR2 |
| SLRTENDD5 | SLRTENDD5_C | VARCHAR2 |
| | SLRTENDD5 | VARCHAR2 |
| | SLRTENDD5_ND | VARCHAR2 |
| SLRTENDD6 | SLRTENDD6_C | VARCHAR2 |
| | SLRTENDD6 | VARCHAR2 |
| CLRTENDDZ | SLRTENDD6_ND | |
| SLRTENDD7 | SLRTENDD7_C<br>SLRTENDD7 | VARCHAR2<br>VARCHAR2 |
| | SLRTENDD7_ND | VARCHAR2 |
| SLRTENDONG | SLRTENDONG_C | VARCHAR2 |
| | SLRTENDONG | VARCHAR2 |
| | SLRTENDONG_ND | VARCHAR2 |
| SLRTENDONG - SLRTENDSEV | SLRTENDSEV_C | VARCHAR2 |
| | SLRTENDSEV | VARCHAR2 |
| SLRTENDONG - SLRTENDEDAT | SLRTENDEDAT | DATE |
| | SLRTENDEDAT_DTS | VARCHAR2 |
| SLRREDWK | SLRREDWK_ND | VARCHAR2 |
| SLRREDWK - None all week | SLRREDWK_CITMNONEWEEK1_C | VARCHAR2 |
| SLRREDD1 | SLRREDWK_CITMNONEWEEK1 SLRREDD1 C | VARCHAR2<br>VARCHAR2 |
| SERREDDI | | |
| | SLRREDD1<br>SLRREDD1 ND | VARCHAR2<br>VARCHAR2 |
| SLRREDD2 | SLRREDD2_C | VARCHAR2 |
| | SLRREDD2 | VARCHAR2 |
| | SLRREDD2_ND | VARCHAR2 |
| SLRREDD3 | SLRREDD3_C | VARCHAR2 |
| | SLRREDD3 | VARCHAR2 |
| | SLRREDD3_ND | VARCHAR2 |
| SLRREDD4 | SLRREDD4_C | VARCHAR2 |
| | SLRREDD4 | VARCHAR2 |
| | SLRREDD4_ND | VARCHAR2 |
| SLRREDD5 | SLRREDD5_C | VARCHAR2 |
| | SLRREDD5 | VARCHAR2 |

629 Dated: 12 March 2018

| | SLRREDD5_ND | VARCHAR2 |
|---|---|---|
| SLRREDD6 | SLRREDD6 C | VARCHAR2 |
| DEM.EDD0 | SLRREDD6 | VARCHAR2 |
| | SLRREDD6 ND | VARCHAR2 |
| SLRREDD7 | SLRREDD7_C | VARCHAR2 |
| | SLRREDD7 | VARCHAR2 |
| | SLRREDD7_ND | VARCHAR2 |
| SLRREDONG | SLRREDONG_C | VARCHAR2 |
| | SLRREDONG | VARCHAR2 |
| | SLRREDONG_ND | VARCHAR2 |
| SLRREDONG - SLRREDSEV | SLRREDSEV_C | VARCHAR2 |
| | SLRREDSEV | VARCHAR2 |
| SLRREDONG - SLRREDEDAT | SLRREDEDAT | DATE |
| | SLRREDEDAT_DTS | VARCHAR2 |
| SLRSWELLWK | SLRSWELLWK ND | VARCHAR2 |
| SLRSWELLWK - None all week | SLRSWELLWK_CITMNONEWEEK1_C | - |
| | SLRSWELLWK_CITMNONEWEEK1 | VARCHAR2 |
| SLRSWELLD1 | SLRSWELLD1_C | VARCHAR2 |
| | SLRSWELLD1 | VARCHAR2 |
| | SLRSWELLD1_ND | VARCHAR2 |
| SLRSWELLD2 | SLRSWELLD2 C | VARCHAR2 |
| | SLRSWELLD2 | VARCHAR2 |
| | SLRSWELLD2 ND | VARCHAR2 |
| SLRSWELLD3 | SLRSWELLD3_C | VARCHAR2 |
| | SLRSWELLD3 | VARCHAR2 |
| | SLRSWELLD3 ND | VARCHAR2 |
| SLRSWELLD4 | SLRSWELLD3_ND | VARCHAR2 |
| JENOWELLD4 | SLRSWELLD4_C | VARCHAR2 |
| | SLRSWELLD4 ND | VARCHAR2 |
| SLRSWELLD5 | SLRSWELLD5_C | VARCHAR2 |
| SEKSWELLDS | | VARCHAR2 |
| | SLRSWELLD5_ND | |
| SLRSWELLD6 | | VARCHAR2<br>VARCHAR2 |
| SEKSWELLDO | SLRSWELLD6_C | - |
| | SLRSWELLD6 | VARCHAR2 |
| | SLRSWELLD6_ND | VARCHAR2 |
| SLRSWELLD7 | SLRSWELLD7_C | VARCHAR2 |
| | SLRSWELLD7 | VARCHAR2 |
| | SLRSWELLD7_ND | VARCHAR2 |
| SLRSWELLONG | SLRSWELLONG_C | VARCHAR2 |
| | SLRSWELLONG | VARCHAR2 |
| | SLRSWELLONG_ND | VARCHAR2 |
| SLRSWELLONG - SLRSWELLSEV | SLRSWELLSEV_C | VARCHAR2 |
| CLECKELLONG CLECKELLEDAT | SLRSWELLSEV | VARCHAR2 |
| SLRSWELLONG - SLRSWELLEDAT | | DATE |
| CI DINIDUM | SLRSWELLEDAT_DTS | VARCHAR2 |
| SLRINDWK | SLRINDWK_ND | VARCHAR2 |
| SLRINDWK - None all week | SLRINDWK_CITMNONEWEEK1_C | VARCHAR2 |
| CI DINIDD4 | SLRINDWK_CITMNONEWEEK1 | VARCHAR2 |
| SLRINDD1 | SLRINDD1_C | VARCHAR2 |
| | SLRINDD1 | VARCHAR2 |
| CI DINIDDO | SLRINDD1_ND | VARCHAR2 |
| SLRINDD2 | SLRINDD2_C | VARCHAR2 |
| | SLRINDD2 | VARCHAR2 |
| CI DINIDD3 | SLRINDD2_ND | |
| SLRINDD3 | SLRINDD3_C | VARCHAR2 |
| | SLRINDD3 | VARCHAR2 |
| CI DINDD4 | SLRINDD3_ND<br>SLRINDD4 C | VARCHAR2 |
| SLRINDD4 | | VARCHAR2 |
| | SLRINDD4 | VARCHAR2 |
| SI RINDD5 | SLRINDD4_ND | VARCHAR2 |
| SEKTINDO | SLRINDD5_C | VARCHAR2 |
| | SLRINDD5 | VARCHAR2 |
| CLDINDDG | SLRINDD5_ND | VARCHAR2 |
| SLRINDD6 | SLRINDD6_C | VARCHAR2 |
| | SLRINDD6 | VARCHAR2 |
| CI DINIDO 7 | SLRINDD6_ND | VARCHAR2 |
| SLRINDD7 | SLRINDD7_C | VARCHAR2 |
| | SLRINDD7 | VARCHAR2 |
| | SLRINDD7_ND | VARCHAR2 |
| SLRINDONG | SLRINDONG_C | VARCHAR2 |
| | SLRINDONG | VARCHAR2 |
| | SLRINDONG_ND | VARCHAR2 |
| SLRINDONG - SLRINDSEV | SLRINDSEV_C | VARCHAR2 |
| | SLRINDSEV | VARCHAR2 |
| SLRINDONG - SLRINDEDAT | SLRINDEDAT | DATE |
| | SLRINDEDAT_DTS | VARCHAR2 |

Protocol No: IVACFLU-S-0203 630 Dated: 12 March 2018

| 1.* | Did the subject report any systemic reactogenicity during Days 1 to 7? | [SSRYN] |
|---|---|---|
| • | Did the subject report any systemic reactogenicity during Days 1 to 7?] | [A:1] OYES<br>[A:2] ONO |
| | nperature (oral) [SLR1SC_1] Evening Day 1 | [SLRTEMPD1_1] |
| .* | [Day 1 Temperature] | xx.x °C[b] |
| .* | Day 2 [Day 2 Temperature] | [SLRTEMPD2_1] XX.X.X. |
| .* | Day 3 [Day 3 Temperature] | [SLRTEMPD3_1] XX.X.X. |
| .* | Day 4 [Day 4 Temperature] | [SLRTEMPD4_1] XX.X. |
| .* | Day 5<br>[Day 5 Temperature] | [SLRTEMPD5_1] XX.X.X. |
| ,* | Day 6<br>[Day 6 Temperature] | [SLRTEMPD6_1] XX.X. |
| 3.*<br>• | Day 7<br>[Day 7 Temperature] | [SLRTEMPD7_1] XX.X °C[b] |
| •.* | After Day 7: Ongoing? [Ongoing] | [SLRTEMPONG_1] [A:2] |
| | igue/Malaise [SSR1SC] Fatigue/Malaise | [SSRTIREDWK] |
| 10. | ratigue/malaise<br>[Fatigue/Malaise]<br>Evening Day 1 | [A:1] None all week |
| | Day 1 Fatigue/Malaise] | [ciROGRES] V |
| 3. | Day 2 Fatigue/Malaise] | [cirogres] V |
| _ | [Day 3 Fatigue/Malaise] | [clROGRES] |
| .4.<br>• | Day 4 [Day 4 Fatigue/Malaise] | [SSRTIREDD4] [CIROGRES] |
| l5.<br>✓ | Day 5<br>[Day 5 Fatigue/Malaise] | [SSRTIREDD5] [clROGRES] |
| l6.<br>✓ | Day 6 [Day 6 Fatigue/Malaise] | [SSRTIREDG] [clrogers] |
| 7. | Day 7 Fatigue/Malaise] | [SSATIREDO7] [CIROGRES] [SSSATIREDONG] |
| 18. | After Day 7: Ongoing? [Ongoing] | [A:2] No [SSRTIREDCMP] Yes [SSRTIREDSEV] Highest severity until resolution: [clSEV] [SSRTIREDSEV] [SSRTIREDEDAT] End date Req / Req / Req (2017-2018) |
| _ | neralized Muscle Aches [SSR2SC] | |
| ~ | Generalized Muscle Aches<br>[Generalized Muscle Aches] | [SSRNUSWK] [A:1] None all week |
| _ | Evening Day 1 [Day 1 Generalized Muscle Aches] | [SSRMUSD1] [CIROGRES] |
| _ | Day 2 [Day 2 Generalized Muscle Aches] | [SSRMUSD2]<br>[CIROGRES] W |
| 22.<br>•<br>23. | Day 3 [Day 3 Generalized Muscle Aches] Day 4 | [SSRMUSD3] [clROGRES] [SSRMUSD4] |
| 23.<br>✓<br>24. | Day 4 Day 5 Day 5 | [SSRMUSD5] |
| ¥.<br>✓<br>25. | Day 5 Generalized Muscle Aches] | [SSRMUSD6] |
| • | [Day 6 Generalized Muscle Aches] | [SSRMUSD7] |
| 26.<br>• | Day 7 [Day 7 Generalized Muscle Aches] After Day 7: Opening 7 | [SSKMUSDY] [CRIRGORES] W |
| 27.<br>✔ | After Day 7: Ongoing? [Ongoing] | [A:2] ONO [A:2] No [A:2] No [A:3] SERMUSONGCMP] Yes [SSRMUSSEV] Highest severity until resolution: [clsv] |
| | | [SSRMUSEDAT] End date Req ✓ / Req ✓ / Req ✓ (2017-2018) |
| Joir | nt Aches [SSR3SC] | |
| 28. | Joint Aches<br>[Joint Aches] | [SSRJNTWK] [A:1] □None all week |
| | Evening Day 1 | [SSRJNTD1] |

Protocol No: IVACFLU-S-0203 631 Dated: 12 March 2018

| , | [Day 1 Joint Aches] | [clrogres] 🗸 |
|---|---|---|
| 30. | Day 2 | [SSRJNTD2] |
| 31. | [Day 2 Joint Aches] Day 3 | [CIROGRES] [SRJNTD3] |
| 32. | [Day 3 Joint Aches] | [cirogres] [SSRINTD4] |
| • | Day 4<br>[Day 4 Joint Aches] | [cirogres] |
| 33.<br>• | Day 5<br>[Day 5 Joint Aches] | [SSRJNTD5] [cirogres] |
| 34.<br>• | Day 6<br>[Day 6 Joint Aches] | [SSRJNTD6] [CIROGRES] |
| 35.<br>• | Day 7 [Day 7 Joint Aches] | [SSRJNTD7]<br>[cIROGRES] |
| 36. | After Day 7: Ongoing? [Ongoing] | [SSRINTONG] [A:2] ○NO |
| | | [A:1] OSSINTONGCMP] Yes |
| | | [SSRINTSEV] Highest severity until resolution: [clsev] |
| | | [SSRJNTEDAT] End date Req ♥ / Req ♥ / Req ♥ (2017-2018) |
| - | Is [SSR4SC] Chills | [SSRCHILWK] |
| ~ | [Chills] | [A:1] None all week |
| 38.<br><b>✓</b> | Evening Day 1<br>[Day 1 Chills] | [SSRCHILD1] [clROGRES] |
| 39.<br>✔ | Day 2<br>[Day 2 Chills] | [SSRCHILD2] [cirogres] |
| 40.<br>• | Day 3<br>[Day 3 Chills] | [SSRCHILD3] [cIROGRES] |
| 41. | Day 4<br>[Day 4 Chills] | [SSRCHILD4] [cirogres] |
| 42. | Day 5<br>[Day 5 Chills] | [SSRCHILD5] [clrogres] |
| 43. | Day 6<br>[Day 6 Chills] | [SSRCHILD6] [cirogres] |
| 44. | Day 7 [Day 7 Chills] | [SSRCHILD7] [ciRoGRES] V |
| 45. | After Day 7: Ongoing? | [SSRCHILONG] |
| | [Ongoing] | [A:2] No<br>[A:1] SSRCHILONGCMP] Yes |
| | | [SSRCHILSEV] Highest severity until resolution: [clSEV] |
| | | [SSRCHILEDAT] |
| Nau | sea [SSR5SC] | End date Req 💟 / Req 💟 / 2017-2018) |
| 46.<br>• | Nausea<br>[Nausea] | [SSRNAUWK] [A:1] □None all week |
| 47.<br>• | Evening Day 1<br>[Day 1 Nausea] | [SSRNAUD1] [clROGRES] |
| 48. | Day 2<br>[Day 2 Nausea] | [SSRNAUD2] [ciROGRES] |
| 49. | Day 3 | [SSRNAUD3] |
| 50. | [Day 3 Nausea] Day 4 | [cirogres] V |
| 51. | [Day 4 Nausea] Day 5 | [cIROGRES] V |
| • | [Day 5 Nausea] | [clrogres] 🗸 |
| _ | Day 6<br>[Day 6 Nausea] | [SSRNAUD6]<br>[cirogres] |
| 53.<br>✓ | Day 7<br>[Day 7 Nausea] | [SSRNAUD7]<br>[cIROGRES] |
| 54.<br>• | After Day 7: Ongoing? [Ongoing] | [SSRNAUONG] [A:2] NO FESTIVATION COMP. |
| | | [A:1] O[SSRNAUONGCMP] Yes [SSRNAUSEV] |
| | | Highest severity until resolution: [clSEV] |
| 14. | siting (CCDCCC) | End date Req / Req / Req (2017-2018) |
| 55. | iting [SSR6SC] Vomiting [Vomiting] | [SSRYOMWK] |
| 56. | [Vomiting] Evening Day 1 [Day 1 Vomiting] | [A:1] None all week [SSRVMMD] |
| 57. | [Day 1 Vomiting] Day 2 | [cirogres] V |
| 58. | [Day 2 Vomiting] Day 3 | [cirogres] [SRYOMD3] |
| 1.4 | | I-Inconco |
| 59. | [Day 3 Vomiting] Day 4 | [cirogres] [SRYOMD4] |
| 59.<br>• | Day 4<br>[Day 4 Vomiting] | [SSRVOMD4]<br>[cIROGRES] |
| 59. | Day 4 | [SSRVOMD4] |

Protocol No: IVACFLU-S-0203 632

IVACFLU-S Version 1.0 Dated: 12 March 2018

| - | | [cirogres] 🗸 |
|---|---|---|
| 62.<br>• | Day 7<br>[Day 7 Vomiting] | [SSRVOMD7]<br>[ciROGRES] |
| 63. | After Day 7: Ongoing? [Ongoing] | [SSRVOMONG] [A:1] |
| Hea | adache [SSR7SC] | |
| 64.<br>✔ | Headache<br>[Headache] | [SSRHEADWK] [A:1] □None all week |
| 65.<br>• | Evening Day 1<br>[Day 1 Headache] | [SSRHEADD1] [CIROGRES] |
| 66.<br>• | Day 2<br>[Day 2 Headache] | [SSRHEADD2]<br>[cirogres] |
| 67.<br>• | Day 3<br>[Day 3 Headache] | [SSRHEADD3]<br>[cirogres] |
| 68.<br>• | Day 4<br>[Day 4 Headache] | [SSRHEADD4] [cirogres] |
| 69.<br>• | Day 5<br>[Day 5 Headache] | [SSRHEADD5] [cirogres] |
| 70.<br>• | Day 6<br>[Day 6 Headache] | [SSRHEADD6] [cirogres] |
| 71. | Day 7<br>[Day 7 Headache] | [SSRHEADD7] [cirogres] |
| 72. | After Day 7: Ongoing? [Ongoing] | [SSRHEADONG] [A:2] ○ No [A:1] ○ [SSRHEADONGCMP] Yes [SSRHEADSEV] Highest severity until resolution: [cISEV] ▼ [SSRHEADEDAT] End date Req ▼ / Req ▼ / Req ▼ (2017-2018) |
| | ey: $[*] = $ Item is required $[ \checkmark ] = $ Source verification required $[b] = $ Base Unit ote: Source verification critical settings made in InForm will override any settings made in Central Designation. | gner. |

| Codelist RefName | Codelist Data Type | Label | Code | Codelist Item RefName | Data Variable RefName |
|---|---|---|---|---|---|
| dROGRES | String | 0, None | 1 | citmROGRES1 | SSRTIREDD 1,<br>SSRTIREDD 2,<br>SSRTIREDD 3,<br>SSRTIREDD 4,<br>SSRTIREDD 5,<br>SSRTIREDD 6,<br>SSRTIREDD 7,<br>SSRMUSD 1,<br>SSRMUSD 1,<br>SSRMUSD 2, |
| | | 1, Mild | 2 | citmROGRES2 | SSRMUSD3,<br>SSRMUSD4,<br>SSRMUSD5,<br>SSRMUSD6,<br>SSRMUSD7,<br>SSRNITD1,<br>SSRNITD2,<br>SSRNITD2,<br>SSRNITD3,<br>SSRNITD4,<br>SSRNITD5, |
| | | 2, Moderate | 3 | citmROGRES3 | SSRINTD6,<br>SSRINTD7,<br>SSRCHILD1,<br>SSRCHILD2,<br>SSRCHILD3,<br>SSRCHILD4,<br>SSRCHILD5,<br>SSRCHILD6,<br>SSRCHILD7,<br>SSRCHILD7,<br>SSRNAUD1, |
| | | 3, Severe | 4 | CITMROGRES4 | SSRNAUD2,<br>SSRNAUD3,<br>SSRNAUD4,<br>SSRNAUD5,<br>SSRNAUD6,<br>SSRNAUD7,<br>SSRVOMD1,<br>SSRVOMD2,<br>SSRVOMD3,<br>SSRVOMD4, |
| | | 4, Potentially Life Threatening | 5 | citmRoGERRE5 | SSRVOMD5,<br>SSRVOMD6,<br>SSRVOMD7,<br>SSRHEADD1,<br>SSRHEADD2,<br>SSRHEADD3,<br>SSRHEADD4,<br>SSRHEADD5,<br>SSRHEADD5,<br>SSRHEADD6,<br>SSRHEADD7 |
| clSEV | String | Grade 1 | 1 | citmSEV1 | SSRTIREDSEV,<br>SSRMUSSEV, |
| | | Grade 2 | 2 | citmSEV2 | SSRINTSEV,<br>SSRCHILSEV, |
| | | Grade 3 | 3 | citmSEV3 | SSRNAUSEV, |
| | | Grade 4 | 4 | citmSEV4 | SSRVOMSEV,<br>SSRHEADSEV |

| RDE Analytics: RD_SSR | | |
|-----------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| SSRYN | SSRYN_C | VARCHAR2 |
| | SSRYN | VARCHAR2 |
| | SSRYN_ND | VARCHAR2 |

Dated: 12 March 2018

SLRTEMPD1\_1 FLOAT SLRTEMPD1 1 SLRTEMPD1 1 U VARCHAR2 SLRTEMPD1\_1\_ND VARCHAR2 SLRTEMPD2 1 SLRTEMPD2\_1 FLOAT SLRTEMPD2\_1\_U VARCHAR2 SLRTEMPD2\_1\_ND VARCHAR2 SLRTEMPD3\_1 SLRTEMPD3\_1 FLOAT SLRTEMPD3 1 U VARCHAR2 SLRTEMPD3 1 ND VARCHAR2 SLRTEMPD4 1 SLRTEMPD4 1 FLOAT SLRTEMPD4\_1\_U VARCHAR2 SLRTEMPD4\_1\_ND VARCHAR2 SLRTEMPD5\_1 SLRTEMPD5\_1\_U VARCHAR2 SLRTEMPD5\_1\_ND VARCHAR2 SLRTEMPD6 1 SLRTEMPD6 1 FLOAT SLRTEMPD6 1 U VARCHAR2 SLRTEMPD6\_1\_ND VARCHAR2 SLRTEMPD7 1 SLRTEMPD7\_1 FLOAT SLRTEMPD7\_1\_U VARCHAR2 SLRTEMPD7\_1\_ND VARCHAR2 SLRTEMPONG\_1 SLRTEMPONG\_1\_C VARCHAR2 VARCHAR2 SLRTEMPONG\_1 SLRTEMPONG 1 ND VARCHAR2 SLRTEMPONG\_1 - SLRTEMPSEV\_1 SLRTEMPSEV\_1\_C VARCHAR2 SLRTEMPSEV 1 VARCHAR2 SLRTEMPONG\_1 - SLRTEMPEDAT\_1 SLRTEMPEDAT\_1 DATE SLRTEMPEDAT\_1\_DTS VARCHAR2 SSRTIREDWK VARCHAR2 SSRTIREDWK\_ND SSRTIREDWK\_CITMNONEWEEK1\_C VARCHAR2 SSRTIREDWK - None all week SSRTIREDWK CITMNONEWEEK1 VARCHAR2 SSRTIREDD1 SSRTIREDD1 C VARCHAR2 SSRTIREDD1 VARCHAR2 SSRTIREDD1\_ND VARCHAR2 SSRTIREDD2 SSRTIREDD2\_C VARCHAR2 VARCHAR2 SSRTIREDD2 SSRTIREDD2\_ND VARCHAR2 SSRTIREDD3 VARCHAR2 SSRTIREDD3 C SSRTIREDD3 VARCHAR2 SSRTIREDD3 ND VARCHAR2 SSRTIREDD4 SSRTIREDD4\_C VARCHAR2 SSRTIREDD4 VARCHAR2 SSRTIREDD4\_ND VARCHAR2 SSRTIREDD5 SSRTIREDD5\_C VARCHAR2 SSRTIREDD5 VARCHAR2 VARCHAR2 SSRTIREDD5 ND SSRTIREDD6 VARCHAR2 SSRTIREDD6 C SSRTIREDD6 VARCHAR2 SSRTIREDD6 ND VARCHAR2 SSRTIREDD7 SSRTIREDD7\_C VARCHAR2 SSRTIREDD7 VARCHAR2 SSRTIREDD7\_ND VARCHAR2 SSRTIREDONG SSRTIREDONG\_C VARCHAR2 SSRTIREDONG VARCHAR2 SSRTIREDONG ND VARCHAR2 SSRTIREDONG - SSRTIREDSEV SSRTIREDSEV C VARCHAR2 SSRTIREDSEV VARCHAR2 SSRTIREDONG - SSRTIREDEDAT SSRTIREDEDAT DATE SSRTIREDEDAT\_DTS VARCHAR2 SSRMUSWK SSRMUSWK\_ND SSRMUSWK - None all week SSRMUSWK\_CITMNONEWEEK1\_C VARCHAR2 SSRMUSWK CITMNONEWEEK1 VARCHAR2 SSRMUSD1 SSRMUSD1 C VARCHAR2 SSRMUSD1 VARCHAR2 SSRMUSD1\_ND VARCHAR2 SSRMUSD2 SSRMUSD2\_C VARCHAR2 SSRMUSD2\_ND VARCHAR2 SSRMUSD3 VARCHAR2 SSRMUSD3\_C SSRMUSD3 VARCHAR2 SSRMUSD3 ND VARCHAR2 SSRMIISD4 SSRMUSD4\_C VARCHAR2 SSRMUSD4 VARCHAR2 SSRMUSD4\_ND VARCHAR2 SSRMUSD5 SSRMUSD5\_C VARCHAR2 SSRMUSD5 VARCHAR2 SSRMUSD5\_ND VARCHAR2 SSRMUSD6 SSRMUSD6 C VARCHAR2

SSRMUSD6

VARCHAR2

Dated: 12 March 2018

| | SSRMUSD6_ND | VARCHAR2 |
|---|---|---|
| SSRMUSD7 | SSRMUSD7 C | VARCHAR2 |
| | SSRMUSD7 | VARCHAR2 |
| | SSRMUSD7_ND | VARCHAR2 |
| SSRMUSONG | SSRMUSONG_C | VARCHAR2 |
| | SSRMUSONG | VARCHAR2 |
| | SSRMUSONG_ND | VARCHAR2 |
| SSRMUSONG - SSRMUSSEV | SSRMUSSEV_C | VARCHAR2 |
| | SSRMUSSEV | VARCHAR2 |
| SSRMUSONG - SSRMUSEDAT | SSRMUSEDAT | DATE |
| | SSRMUSEDAT_DTS | VARCHAR2 |
| SSRJNTWK - None all week | SSRJNTWK_ND | VARCHAR2 |
| SSRJINI WK - Notice all week | SSRJNTWK_CITMNONEWEEK1_C SSRJNTWK CITMNONEWEEK1 | VARCHAR2 |
| SSRINTD1 | SSRJNTD1_C | VARCHAR2 |
| | SSRJNTD1 | VARCHAR2 |
| | SSRJNTD1_ND | VARCHAR2 |
| SSRJNTD2 | SSRJNTD2_C | VARCHAR2 |
| | SSRJNTD2 | VARCHAR2 |
| | SSRJNTD2_ND | VARCHAR2 |
| SSRJNTD3 | SSRJNTD3_C | VARCHAR2 |
| | SSRJNTD3 | VARCHAR2 |
| | SSRJNTD3_ND | VARCHAR2 |
| SSRJNTD4 | SSRJNTD4_C | VARCHAR2 |
| | SSRJNTD4 | VARCHAR2 |
| SSRJNTD5 | SSRJNTD4_ND | VARCHAR2<br>VARCHAR2 |
| SOLINING | SSRJNTD5_C<br>SSRJNTD5 | VARCHAR2<br>VARCHAR2 |
| | SSRJNTD5_ND | VARCHAR2 |
| SSRJNTD6 | SSRINTD6 C | VARCHAR2 |
| | SSRJNTD6 | VARCHAR2 |
| | SSRJNTD6_ND | VARCHAR2 |
| SSRJNTD7 | SSRJNTD7_C | VARCHAR2 |
| | SSRJNTD7 | VARCHAR2 |
| | SSRJNTD7_ND | VARCHAR2 |
| SSRJNTONG | SSRJNTONG_C | VARCHAR2 |
| | SSRJNTONG | VARCHAR2 |
| | SSRJNTONG_ND | VARCHAR2 |
| SSRJNTONG - SSRJNTSEV | SSRJNTSEV_C | VARCHAR2 |
| | SSRJNTSEV | VARCHAR2 |
| CCDINITONIC CCDINITEDAT | CCDINTEDAT | |
| SSRJNTONG - SSRJNTEDAT | SSRINTEDAT DTS | DATE |
| | SSRJNTEDAT_DTS | VARCHAR2 |
| SSRCHILWK | SSRINTEDAT_DTS SSRCHILWK_ND | VARCHAR2<br>VARCHAR2 |
| | SSRJNTEDAT_DTS | VARCHAR2 |
| SSRCHILWK | SSRJNTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C | VARCHAR2<br>VARCHAR2<br>VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week | SSRJNTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1 | VARCHAR2<br>VARCHAR2<br>VARCHAR2<br>VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week | SSRJNTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1 SSRCHILD1_C | VARCHAR2<br>VARCHAR2<br>VARCHAR2<br>VARCHAR2<br>VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_ND SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C SSRCHILD2_SSRCHILD2_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1 SSRCHILD1_C SSRCHILD1 LO SSRCHILD1 ND SSRCHILD2_C SSRCHILD2 SSRCHILD2 SSRCHILD2 SSRCHILD2_ND SSRCHILD3_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILIWK_CITMNONEWEEK1 SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_NC SSRCHILD3_NC SSRCHILD3_NC | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_D SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_SSRCHILD3_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3 | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_D SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_SSRCHILD3_SSRCHILD3_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3 SSRCHILD3 SSRCHILD3_SSRCHILD3 SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4 | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_DD SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILIWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_D SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4 SSRCHILD4_SSRCHILD4_SSRCHILD4_SSRCHILD4_SSRCHILD4_SSRCHILD5_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_D SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_ND SSRCHILD4_ND SSRCHILD5_C SSRCHILD5 | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 | SSRNNTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITIMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILLD1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_ND SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6 SSRCHILD6 SSRCHILD6 SSRCHILD6_SSRCHILD6_ND SSRCHILD6_SSRCHILD6_ND SSRCHILD6_ND SSRCHILD6_ND SSRCHILD6_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD6_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_C SSRCHILD7_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD6_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_C SSRCHILD7_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD5 | SSRNNTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD6_C SSRCHILD7_C SSRCHILD7_C SSRCHILD7 SSRCHILD7_SSRCHILD7 SSRCHILD7_ND SSRCHILD7_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD5 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILMK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_ND SSRCHILD4_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD6_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7_C SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITIMNONEWEEK1_C SSRCHILLOT_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD4_ND SSRCHILD4_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD4_C SSRCHILD4_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7_ND SSRCHILD5_C SSRCHILD7_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_ND SSRCHILD7_C SSRCHILD7_ND SSRCHILD0_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILUNK_CITMNONEWEEK1 SSRCHILD1_C SSRCHILD1 SSRCHILD1 SSRCHILD2 SSRCHILD2_C SSRCHILD2_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD6_C SSRCHILD7_DD SSRCHILD7_DD SSRCHILDNG_C SSRCHILDNG_C SSRCHILDNG_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILO7 SSRCHILONG - SSRCHILSEV | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_C SSRCHILD3_C SSRCHILD3_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7_C SSRCHILD7_C SSRCHILD7_C SSRCHILD7_SSRCHILD0_SSRCHILD0_SSRCHILD0_SSRCHILD0_SSRCHILD0_SSRCHILD0_ND SSRCHILD0_ND SSRCHILSEV_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILONG SSRCHILONG - SSRCHILSEV SSRCHILONG - SSRCHILEDAT SSRNAUWK | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILLMK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1 SSRCHILD1_ND SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILDNG_C SSRCHILDNG_C SSRCHILDNG_C SSRCHILDNG_ND SSRCHILDNG_ND SSRCHILDNG_ND SSRCHILDNG_ND SSRCHILSEV_C SSRCHILEDAT_DTS SSRCHILEDAT_DTS SSRCHILEDAT_DTS | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILONG - SSRCHILSEV SSRCHILONG - SSRCHILEDAT | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILLD1 SSRCHILD1 SSRCHILD1 SSRCHILD1 SSRCHILD2 SSRCHILD2 SSRCHILD2 SSRCHILD2 SSRCHILD3 SSRCHILD3 SSRCHILD3 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD6 SSRCHILD6 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD6 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILONG SSRCHILONG SSRCHILONG SSRCHILONG SSRCHILONG SSRCHILONG SSRCHILONG SSRCHILDS SSRCHILDS SSRCHILDS SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD7 SSRCHILD8 SSRCHILD8 SSRCHILD9 SSRCHILDD4 SSRCHILDD4 SSRCHILDD4 SSRCHILDD4 SSRCHILDD4 SSRCHILDDAT SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT_DTS SSRNAUWK_ND | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILONG - SSRCHILSEV SSRCHILONG - SSRCHILEDAT SSRCHILONG - SSRCHILEDAT SSRNAUWK - None all week | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2 SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_C SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_C SSRCHILD7 SSRCHILD7_C SSRCHILD7 SSRCHILONG_C SSRCHILONG_C SSRCHILONG_SSRCHILONG_ND SSRCHILONG_ND SSRCHILSEV_C SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRNAUWK_CITMNONEWEEK1_C SSRNAUWK_CITMNONEWEEK1_C | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILONG SSRCHILONG - SSRCHILSEV SSRCHILONG - SSRCHILEDAT SSRNAUWK | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2_C SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD4_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD7 SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILDS_ND SSRCHILDS_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD7_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD7_ND SSRCHILD7_ | VARCHAR2 |
| SSRCHILWK SSRCHILWK - None all week SSRCHILD1 SSRCHILD2 SSRCHILD3 SSRCHILD4 SSRCHILD5 SSRCHILD5 SSRCHILD6 SSRCHILD7 SSRCHILONG - SSRCHILSEV SSRCHILONG - SSRCHILEDAT SSRCHILONG - SSRCHILEDAT SSRNAUWK - None all week | SSRINTEDAT_DTS SSRCHILWK_ND SSRCHILWK_CITMNONEWEEK1_C SSRCHILWK_CITMNONEWEEK1_C SSRCHILD1_C SSRCHILD1_C SSRCHILD2_C SSRCHILD2 SSRCHILD2_ND SSRCHILD2_ND SSRCHILD3_ND SSRCHILD3_C SSRCHILD3_ND SSRCHILD4_C SSRCHILD4_C SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_C SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD5_ND SSRCHILD6_C SSRCHILD6_C SSRCHILD6_C SSRCHILD6_ND SSRCHILD7_C SSRCHILD7 SSRCHILD7_C SSRCHILD7 SSRCHILONG_C SSRCHILONG_C SSRCHILONG_SSRCHILONG_ND SSRCHILONG_ND SSRCHILSEV_C SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRCHILEDAT SSRNAUWK_CITMNONEWEEK1_C SSRNAUWK_CITMNONEWEEK1_C | VARCHAR2 |

635 Dated: 12 March 2018

| SSRNAUD2 | SSRNAUD2_C | VARCHAR2 |
|---|---|---|
| | SSRNAUD2 | VARCHAR2 |
| | SSRNAUD2_ND | VARCHAR2 |
| SSRNAUD3 | SSRNAUD3_C | VARCHAR2 |
| | SSRNAUD3 | VARCHAR2 |
| | SSRNAUD3_ND | VARCHAR2 |
| SSRNAUD4 | SSRNAUD4_C | VARCHAR2 |
| | SSRNAUD4 | VARCHAR2 |
| | SSRNAUD4_ND | VARCHAR2 |
| SSRNAUD5 | SSRNAUD5_C | VARCHAR2 |
| | SSRNAUD5 | VARCHAR2 |
| | SSRNAUD5_ND | VARCHAR2 |
| SSRNAUD6 | SSRNAUD6_C | VARCHAR2 |
| | SSRNAUD6 | VARCHAR2 |
| | SSRNAUD6_ND | VARCHAR2 |
| SSRNAUD7 | SSRNAUD7_C | VARCHAR2 |
| | SSRNAUD7 | VARCHAR2 |
| | SSRNAUD7_ND | VARCHAR2 |
| SSRNAUONG | SSRNAUONG_C | VARCHAR2 |
| | SSRNAUONG | VARCHAR2 |
| | SSRNAUONG_ND | VARCHAR2 |
| SSRNAUONG - SSRNAUSEV | SSRNAUSEV_C | VARCHAR2 |
| | SSRNAUSEV | VARCHAR2 |
| SSRNAUONG - SSRNAUEDAT | SSRNAUEDAT | DATE |
| | SSRNAUEDAT_DTS | VARCHAR2 |
| SSRVOMWK | SSRVOMWK_ND | VARCHAR2 |
| SSRVOMWK - None all week | SSRVOMWK_CITMNONEWEEK1_C | VARCHAR2 |
| | SSRVOMWK_CITMNONEWEEK1 | VARCHAR2 |
| SSRVOMD1 | SSRVOMD1_C | VARCHAR2 |
| • | SSRVOMD1 | VARCHAR2 |
| | SSRVOMD1_ND | VARCHAR2 |
| SSRVOMD2 | SSRVOMD2_C | VARCHAR2 |
| | SSRVOMD2 | VARCHAR2 |
| | SSRVOMD2_ND | VARCHAR2 |
| SSRVOMD3 | SSRVOMD3_C | VARCHAR2 |
| 55114-61-12-5 | SSRVOMD3 | VARCHAR2 |
| | SSRVOMD3_ND | VARCHAR2 |
| SSRVOMD4 | SSRVOMD4_C | VARCHAR2 |
| SSKV611B 1 | SSRVOMD4 | VARCHAR2 |
| | SSRVOMD4_ND | VARCHAR2 |
| SSRVOMD5 | SSRVOMD5_C | VARCHAR2 |
| 55.1.4-61.12-5 | SSRVOMD5 | VARCHAR2 |
| | SSRVOMD5_ND | VARCHAR2 |
| SSRVOMD6 | SSRVOMD6 C | VARCHAR2 |
| 55.1.7.67.1.5.0 | SSRVOMD6 | VARCHAR2 |
| | SSRVOMD6_ND | VARCHAR2 |
| SSRVOMD7 | SSRVOMD7 C | VARCHAR2 |
| 5511157 | SSRVOMD7 | VARCHAR2 |
| | SSRVOMD7_ND | VARCHAR2 |
| SSRVOMONG | SSRVOMONG_C | VARCHAR2 |
| 331(40)101(4 | SSRVOMONG | VARCHAR2 |
| | SSRVOMONG_ND | VARCHAR2 |
| SSRVOMONG - SSRVOMSEV | SSRVOMSEV_C | VARCHAR2 |
| 33KVOHONG - 33KVOH3LV | SSRVOMSEV_C | VARCHAR2 |
| CCDVOMONG CCDVOMEDAT | SSRVOMEDAT | |
| SSRVOMONG - SSRVOMEDAT | SSRVOMEDAT DTS | DATE<br>VARCHAR2 |
| SSRHEADWK | SSRVOMEDAT_DTS SSRHEADWK_ND | VARCHAR2<br>VARCHAR2 |
| SSRHEADWK - None all week | SSRHEADWK_ND SSRHEADWK_CITMNONEWEEK1_C | VARCHAR2 |
| SOMILADIVIN - Notice dil Week | SSRHEADWK_CITMNONEWEEK1_C | VARCHAR2<br>VARCHAR2 |
| SSRHEADD1 | SSRHEADWK_CITMNONEWEEKI | VARCHAR2 |
| JUNIEMDD1 | | VARCHAR2<br>VARCHAR2 |
| | SSRHEADD1 ND | |
| CCDUEADD3 | SSRHEADD1_ND | VARCHAR2 |
| SSRHEADD2 | SSRHEADD2_C | VARCHAR2 |
| | SSRHEADD2 | VARCHAR2 |
| SSRHEADD3 | SSRHEADD2_ND | VARCHAR2 |
| SOUTENDO | SSRHEADD3_C | VARCHAR2 |
| | SSRHEADD3 | VARCHAR2 |
| CODUCADDA | SSRHEADD3_ND | VARCHAR2 |
| | SSRHEADD4_C | VARCHAR2 |
| SSRHEADD4 | | VARCHAR2 |
| 33KIILADD4 | SSRHEADD4 | VARGUETE |
| | SSRHEADD4_ND | VARCHAR2 |
| SSRHEADD5 | SSRHEADD4_ND<br>SSRHEADD5_C | VARCHAR2 |
| | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 | VARCHAR2<br>VARCHAR2 |
| | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 SSRHEADD5_ND | VARCHAR2 |
| | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 | VARCHAR2<br>VARCHAR2 |
| SSRHEADD5 | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 SSRHEADD5_ND | VARCHAR2<br>VARCHAR2<br>VARCHAR2 |
| SSRHEADD5 | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 SSRHEADD5_ND SSRHEADD6_C | VARCHAR2<br>VARCHAR2<br>VARCHAR2 |
| SSRHEADD5 | SSRHEADD4_ND SSRHEADD5_C SSRHEADD5 SSRHEADD5_ND SSRHEADD6_C SSRHEADD6_C | VARCHAR2<br>VARCHAR2<br>VARCHAR2<br>VARCHAR2<br>VARCHAR2 |

Protocol No: IVACFLU-S-0203 636 Dated: 12 March 2018

| | SSRHEADD7_ND | VARCHAR2 |
|--------------------------|-----------------|----------|
| SSRHEADONG | SSRHEADONG_C | VARCHAR2 |
| | SSRHEADONG | VARCHAR2 |
| | SSRHEADONG_ND | VARCHAR2 |
| SSRHEADONG - SSRHEADSEV | SSRHEADSEV_C | VARCHAR2 |
| | SSRHEADSEV | VARCHAR2 |
| SSRHEADONG - SSRHEADEDAT | SSRHEADEDAT | DATE |
| | SSRHEADEDAT DTS | VARCHAR2 |

Protocol No: IVACFLU-S-0203 637 Dated: 12 March 2018

| nscheduled Assessment Forms [UNSFMSC] | |
|---|---|
| Reason for Unscheduled visit [Reason for Unscheduled visit] | [UNSREAS] [A:3] |
| * Unscheduled Assessment Forms<br>[Unscheduled Assessment Forms] | [UNSFORM] [A:1] ☐ Targeted PE [A:4] ☐ Urine Pregnancy Test [A:6] ☐ Anti-Influenza Serologic Assay |

| RDE Analytics: RD_UNSFM | | |
|---|---|---|
| Data Variable RefName | RD Column Name | Column Data Type |
| UNSREAS | UNSREAS_C | VARCHAR2 |
| | UNSREAS | VARCHAR2 |
| | UNSREAS_ND | VARCHAR2 |
| UNSREAS - UNSREASOTH | UNSREASOTH | VARCHAR2 |
| UNSFORM | UNSFORM_ND | VARCHAR2 |
| UNSFORM - Targeted PE | UNSFORM_CITMUNLIST1_C | VARCHAR2 |
| | UNSFORM_CITMUNLIST1 | VARCHAR2 |
| UNSFORM - Urine Pregnancy Test | UNSFORM_CITMUNLIST4_C | VARCHAR2 |
| | UNSFORM_CITMUNLIST4 | VARCHAR2 |
| UNSFORM - Anti-Influenza Serologic Assay | UNSFORM_CITMUNLIST6_C | VARCHAR2 |
| | UNSFORM_CITMUNLIST6 | VARCHAR2 |

Protocol No: IVACFLU-S-0203 638 Dated: 12 March 2018

| .og [LOGFMSC] | |
|---|---|
| * Were any Unsolicited Adverse Events reported? [Were any Unsolicited Adverse Events reported?] | [LOGAE] [A::1] |
| * Were any Serious Adverse Events reported? [Were any Serious Adverse Events reported?] | [LOGSAE] [A::1] ② Yes [A::2] ② No If Yes, please record the details on the SAE form. |
| .* Were any Concomitant Medications reported? [Were any Concomitant Medications reported?] | [LOGCM] [A:1] Yes [A:2] No If Yes, please record the details on the CM form. |

| RDE Analytics: RD | _LOGFM | |
|---|---|---|
| Data Variable RefName | RD Column Name Column Data | |
| LOGAE | LOGAE_C | VARCHAR2 |
| | LOGAE | VARCHAR2 |
| | LOGAE_ND | VARCHAR2 |
| LOGSAE | LOGSAE_C | VARCHAR2 |
| | LOGSAE | VARCHAR2 |
| | LOGSAE_ND | VARCHAR2 |
| LOGCM | LOGCM_C | VARCHAR2 |
| | LOGCM | VARCHAR2 |
| | LOGCM_ND | VARCHAR2 |

Dated: 12 March 2018

| LE Number | Adverse Event | Start Date | Stop Date | Severity | Serious? | Treatment Required | Action Taken | Relationship to Study Product | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| olicited Adv | erse Event [AESC | ] | | | | | | | |
| | | | | 100 | | | | | |
| Start Date | | | | | | | | | |
| [Start Date] | | | | Re | eq 🔽 / Req | / Req (2017-2018) | | | |
| Stop Date<br>[Stop Date] | | | | | | / Req (2017-2018) | | | |
| Severity<br>[Severity] | | | | [A<br>[A | [AEINT] [A:1] Mild (Grade 1) [A:2] Moderate (Grade 2) [A:3] Severe (Grade 3) [A:4] Ulfe threatening (Grade 4) | | | | |
| Serious?<br>[Serious?] | | | | [4 | [AESER] [A:1] ○Yes: Complete the SAE form and report to sponsor, IRB and regulatory authorities. [A:2] ○ No | | | | |
| | | | | [4 | [AETRT] [A:1] | | | | |
| | | | | [A<br>[A | EACN] A:1] None A:2] Disco A:3] [AEA Othe | ntinued<br>CNO]<br>r, please specify | | | |
| | | | | [4 | [AEREL] [A:1] Related [A:2] Not Related | | | | |
| Outcome<br>[Outcome] | | | | [A<br>[A<br>[A<br>[A | (A:1) | | | | |
| | AE Number [AE Number [AE Number [AE Number [AE Number [AE Number Stop Date [Start Date]] Stop Date [Stop Date] Severity [Severity] Treatment [Treatment Action Take [Action Take]] Relationship [Relationship] | Start Date [Start Date [Start Date [Start Date] Stop Date [Stop Date [Stop Date] Seventy [Seventy] Treatment Required [Treatment Required] Action Taken [ Action Taken] Relationship to Study Product [Relationship to Study Product Outcome | AE Number [read-only] [AE Number] Adverse Event [Adverse Event] Adverse Event [Adverse Event] Stap Date [Start Date] Stop Date [Stop Date] Severity [Severity] Treatment Required [Treatment Required] Action Taken [ Action Taken] Relationship to Study Product [Relationship to Study Product] Outcome | AE Number [read-only] [AE Number] Adverse Event [Adverse Event] Adverse Event [Adverse Event] Start Date [Start Date] Stop Date [Stop Date] Severity [Severity] Treatment Required [Treatment Required] Action Taken [ Action Taken] Relationship to Study Product [Relationship to Study Product] Outcome | AE Number [read-only] [AE Number [read-only] [AIEN Unmber] Adverse Event [Adverse Event] Start Date [Start Date] Stop Date [Stop Date] Stop Date [Stop Date] Severity [Severity] [A [ | Action Taken Act | AE Number Fread-only | AENUMP REAL RESTDT Req Req | Activate Activate |

| RDE Analytics: RD | | |
|-----------------------|----------------|----------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| AENUM | AENUM | NUMBER |
| | AENUM_ND | VARCHAR2 |
| AETERM | AETERM | VARCHAR2 |
| | AETERM_ND | VARCHAR2 |
| AESTDT | AESTDT | DATE |
| | AESTDT_DTS | VARCHAR2 |
| | AESTDT_ND | VARCHAR2 |
| AEEDT | AEEDT | DATE |
| | AEEDT_DTS | VARCHAR2 |
| | AEEDT_ND | VARCHAR2 |
| AEINT | AEINT_C | VARCHAR2 |
| | AEINT | VARCHAR2 |
| | AEINT_ND | VARCHAR2 |
| AESER | AESER_C | VARCHAR2 |
| | AESER | VARCHAR2 |
| | AESER_ND | VARCHAR2 |
| AETRT | AETRT_C | VARCHAR2 |
| | AETRT | VARCHAR2 |
| | AETRT_ND | VARCHAR2 |
| AEACN | AEACN_C | VARCHAR2 |
| | AEACN | VARCHAR2 |
| | AEACN_ND | VARCHAR2 |
| AEACN - AEACNO | AEACNO | VARCHAR2 |
| AEREL | AEREL_C | VARCHAR2 |
| | AEREL | VARCHAR2 |
| | ALKEL | |
| | AEREL_ND | VARCHAR2 |
| AEOUT | | VARCHAR2<br>VARCHAR2 |
| AEOUT | AEREL_ND | - |

Protocol No: IVACFLU-S-0203 640 Dated: 12 March 2018

| # | SAE | Type of | | Date of | Serious A | dverse Event | Onset | Re | solved | Serious | | Relationship | | Outcome | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| t | Number | Report | | birth | Na | me(s) | Date | ' | Date | Criteria | | Produ | ıct | 1 | Narrati | ve |
| _ | | | | | n. If multip | le SAEs, com | plete a fo | rm fo | or each S/ | AE. | | | | | | |
| er | _ | rse Event [S<br>ber [read-or | | c] | | | [SAEN | UM] | | | | | | | | |
| | [SAE Number] | | | | | | N3 | | | | | | | | | |
| 2.* | Type of Report [Type of Report] Sex [read-only] [Sex] | | | | | | [SAER | | itial | | | | | | | |
| | | | | | | | | ○Fo | llow-up | | | | | | | |
| 3. | | | | | | | [SAEG | ENDE | R] | | | | | | | |
| | | | | | | | [A:1]<br>[A:2] | | | | | | | | | |
| 1. | Date of b | Date of birth [read-only] | | | | | | OBDT | 1 | | _ | | | | | |
| | [Date of | dverse Even | t Nas | (-) | | | Req/Ui | | / Req/Unk | / Req | (1918-201 | .8) | | | | |
| 5.*<br>• | | Adverse Eve | | | | | A200 | | | | | | | | | |
| 5.* | Onset Da | ite | | | | | [SAES | rDT] | | | | | | | | |
| ~ | [Onset D | ate] | | | | | | | eq 🛂 / Re | (2017- | 2018) | | | | | |
| 7.<br>• | Resolved<br>[Resolve | | | | | | Req V | | eq 🔽 / Re | q 🔽 (2017- | 2018) | | | | | |
| в.* | Serious ( | Criteria (chec | k all | that apply | ) | | [SAECI | RIT] | AEDCMP] | | | | | | | |
| ٠ | [ | | | | | | 2=3 | D€ | eath<br>CAUSE] | | | | | | | |
| | | | | | | | | Pr | | se of Death | | | | | | |
| | | | | | | | | , | 200 | | | | | | | |
| | | | | | | | | L | | | | | | | | |
| | | | | | | | | | DEATHDT]<br>ate of deat | h Req 🛂 / | Req 🗸 / F | eq 🟏 (2017-20 | 18) | | | |
| | | | | | | | | | EATHCERT<br>as a death | r]<br>certificate | obtained? | | | | | |
| | | | | | | | | | 4:1] ( Yes<br>4:2] ( No | 5 | | | | | | |
| | | | | | | | | [4 | 4:3] OPer | nding | | | | | | |
| | | | | | | | | W | utopsy]<br>as Autopsy | performed | ? | | | | | |
| | | | | | | | | [/ | Yes | AEREPORT] | | | | | | |
| | | | | | | | | | [A: | the report a<br>:1] OYes | vallabler | | | | | |
| | | | | | | | (A:2) No (A:2) No (A:3) Pending (A:2) Life-threatening (A:3) [SAEHOSCMP] [ISAEHOSCMP] | | | | | | | | | |
| | | | | | | ΓΔ·21 | | | | | | | | | | |
| | | | | | | [A:3] | | | | | | | | | | |
| | | | | | | | | Initial or prolonged hospitalization [HoSADDT] Admission Date Req / Req / Req (2017-2018) [HOSDDT] Discharge Date Req / Req / Req (2017-2018) [A:3] Persistent or significant disability/incapacity [A:5] Congenital anomaly/inth defect [A:6] SAESOT] Medically significant event Please specify reason | | | | | | | | |
| | | | | | | | [A:4] | | | | | | | | | |
| | | | | | | | [A:5] | | | | | | | | | |
| | | | | | | | [A:6] | | | | | | | | | |
| | | | | | | | | | 200* | y reason | | | | | | |
| 9.* | Severity | | | | | | [SAEII | IT] | | | | | | | | |
| ~ | [Severity | .] | | | | | [A:1]<br>[A:2] | | ld<br>oderate | | | | | | | |
| | | | | | | | [A:3] | OSe | | ina | | | | | | |
| 10. | * Relations | hip to Study | Prod | uct | | | [SAER | - | e uneaten | III 9 | | | | | | |
| <b>v</b> | | ship to Study | | | | | [A:1] | No | t Related<br>AERELSP] | | | | | | | |
| | | | | | | | [A.2] | Re | lated | de investiga | tor rational | e | | | | |
| | | | | | | | | | 200* | | | | | | | |
| 11. | Outcome | | | | | | [SAEO | | | | | | | | | |
| • | [Outcom | ej | | | | | [A:1]<br>[A:2] | | solved<br>ngoing | | | | | | | |
| | | | | | | | | ОВе | come stab | le/chronic | | | | | | |
| | | | | | | | | | eatn<br>iknown | | | | | | | |
| | rative [SA | | | | | | | | | | | | | | | |
| 12.*<br>• | Descripti | | ical p | presentatio | | the event(s), | A2000 | | | | | | | | | |
| | explain t | ne event. | | | er assessme | nts which help | | | | | | | | | | |
| | [Event D | escription/Ca | ise Ni | arrative] | | | | | | | | | | | | |
| | 1 | | | | | | | | | | | | | | | 1 |

IVACFLU-S Version 1.0 641 Dated: 12 March 2018

| SAE Count [hidden] | [SAEC] |
|---|---|
| [SAE Count] | N3 |
| : [ v ] = Source verification required [ *] = ASCII Only | ngs mada in Central Decigner |

| RDE Analytics: RD_SAE | | |
|---|---|---|
| Data Variable RefName | RD Column Name | Column Data Type |
| SAENUM | SAENUM | NUMBER |
| | SAENUM_ND | VARCHAR2 |
| SAERPT | SAERPT_C | VARCHAR2 |
| | SAERPT | VARCHAR2 |
| | SAERPT_ND | VARCHAR2 |
| SAEGENDER | SAEGENDER_C | VARCHAR2 |
| | SAEGENDER | VARCHAR2 |
| | SAEGENDER_ND | VARCHAR2 |
| SAEDOBDT | SAEDOBDT | DATE |
| | SAEDOBDT_DTS | VARCHAR2 |
| | SAEDOBDT_DTR | VARCHAR2 |
| | SAEDOBDT_ND | VARCHAR2 |
| SAETERM | SAETERM | VARCHAR2 |
| | SAETERM_ND | VARCHAR2 |
| SAESTDT | SAESTDT | DATE |
| | SAESTDT_DTS | VARCHAR2 |
| | SAESTDT_ND | VARCHAR2 |
| SAEEDT | SAEEDT | DATE |
| <del> </del> | SAEEDT_DTS | VARCHAR2 |
| | SAEEDT_ND | VARCHAR2 |
| SAECRIT | | VARCHAR2 |
| SAECRIT - Death | SAECRIT_ND<br>SAECRIT_SAEDCMP_C | VARCHAR2 |
| JALCKII - DEdIII | | VARCHAR2 |
| CAFCRYT BOAUGE | SAECRIT_SAEDCMP | |
| SAECRIT - DCAUSE SAECRIT - DEATHDT | DCAUSE | VARCHAR2 |
| SAECRII - DEATHDI | DEATHDT | DATE |
| | DEATHDT_DTS | VARCHAR2 |
| SAECRIT - DEATHCERT | DEATHCERT_C | VARCHAR2 |
| | DEATHCERT | VARCHAR2 |
| SAECRIT - AUTOPSY | AUTOPSY_C | VARCHAR2 |
| | AUTOPSY | VARCHAR2 |
| SAECRIT - SAEREPORT | SAEREPORT_C | VARCHAR2 |
| | SAEREPORT | VARCHAR2 |
| SAECRIT - Life-threatening | SAECRIT_CITMSAECRT2_C | |
| | SAECRIT_CITMSAECRT2 | VARCHAR2 |
| SAECRIT - Initial or prolonged hospitalization | SAECRIT_SAEHOSCMP_C | VARCHAR2 |
| | SAECRIT_SAEHOSCMP | VARCHAR2 |
| SAECRIT - HOSADDT | HOSADDT | DATE |
| | HOSADDT_DTS | VARCHAR2 |
| SAECRIT - HOSDSDT | HOSDSDT | DATE |
| | HOSDSDT_DTS | VARCHAR2 |
| SAECRIT - Persistent or significant disability/incapacity | SAECRIT_CITMSAECRT4_C | VARCHAR2 |
| | SAECRIT_CITMSAECRT4 | VARCHAR2 |
| SAECRIT - Congenital anomaly/birth defect | SAECRIT_CITMSAECRT5_C | VARCHAR2 |
| | SAECRIT_CITMSAECRT5 | VARCHAR2 |
| SAECRIT - Medically significant event | SAECRIT_SAESOT_C | VARCHAR2 |
| | SAECRIT_SAESOT | VARCHAR2 |
| SAECRIT - SAESOT | SAESOT | VARCHAR2 |
| SAEINT | SAEINT_C | VARCHAR2 |
| | SAEINT | VARCHAR2 |
| | SAEINT_ND | VARCHAR2 |
| SAEREL | SAEREL_C | VARCHAR2 |
| | SAEREL | VARCHAR2 |
| | SAEREL_ND | VARCHAR2 |
| SAEREL - SAERELSP | SAERELSP | VARCHAR2 |
| SAEOUT | SAEOUT_C | VARCHAR2 |
| | SAEOUT | VARCHAR2 |
| | SAEOUT_ND | VARCHAR2 |
| CATAGOM | SAENCOM | VARCHAR2 |
| SAENCOM | | |
| SAENCOM | SAENCOM ND | VARCHAR2 |
| SAEC | SAENCOM_ND<br>SAEC | VARCHAR2<br>NUMBER |


| col No: IVACFLU-S-0203 | 642 | Dated: 12 March 2018 |
|-----------------------------|------|----------------------|
| 001 110. 1 V 11C1 EC 5 0205 | 0-12 | Dated. 12 March 2010 |

| Sequence Number (read-only) Total | ACFLU-S-0203: CONCC | | NS (CM) Dose Unit | | | Frequency | Start Date | Stop Date | Indicatio |
|---|---|---|---|---|---|---|---|---|---|
| Sequence Number (read-only) Total | | | | | | | | | |
| 16 Sequence (funder) 17 18 18 18 18 18 18 18 | ncomitant Medications [CMSC] | | | | | | | | |
| Technology A200* A100* A | CM Sequence Number [read-onl<br>[CM Sequence Number] | y]<br> | 1 | 1 | | | | | |
| Colsost Align Colsost Align Colsost Align Colsost Align Colsost Align Colsost Cols | Medication Name | | | IG] | | | | | |
| ALDO CHANNIST CH | | | 1,7200 | | | | | | |
| ALDO CHANNIST CH | | | | | | | | | |
| CHAINT (A.1) CUNTILIST) (CHAINT) (A.2) CUNTILIST) (CHAINT) (A.2) CUNTILIST) (CHAINT) (A.2) CUNTILIST) (CHAINT) (CH | Dose | | | E] | | | | | |
| ALJ CHANNEL | [Dose] | | A100* | | | | | | |
| CHROUTE A 100 * CHRO | Unit | | [CMUNI | T] | | | | | |
| ADD CHARDOT | [Unit] | | [A:1] ( | [CICMUNIT] | | | | | |
| Please specify A100* [CHROUTS] [A10] [CHROUT] [A20] [ROUTOT] [A21] [REST] [CHROUT] [A22] [ROUTOT] [A22] [ROUTOT] [A23] [A24] [A24] [A25] [A24] [A25] [A24] [A25] [A25] [A26] [A26] [A27] [A27] [A28] [A29] [A29] [A29] [A20] [A20] [A20] [A21] [A20] [A21] [A21] [A21] [A22] [A23] [A23] [A24] [A24] [A25] [A26] [A26] [A26] [A27] [A28] [A28] [A28] [A28] [A28] [A28] [A28] [A29] [A29] [A20] [A20] [A20] [A20] [A20] [A21] [A21] [A21] [A22] [A23] [A23] [A24] [A24] [A25] [A26] [A26] [A26] [A27] [A27] [A28] [A28] [A28] [A28] [A28] [A29] [A21] [A21] [A21] [A21] [A22] [A23] [A23] [A23] [A24] [A24] [A25] [A26] [A26] [A26] [A27] [A27] [A27] [A28] [A28] [A28] [A28] [A28] [A29] [A21] [A21] [A21] [A21] [A22] [A22] [A23] [A23] [A23] [A24] [A24] [A25] [A24] [A25] [A26] [A26] [A26] [A27] [A27] [A28] [A28] [A28] [A28] [A28] [A28] [A28] [A29] [A21] [A21] [A21] [A21] [A22] [A23] [A23] [A23] [A24] [A24] [A25] [A26] [A26] [A26] [A27] [A27] [A27] [A28] | | | [A:2] ( | [UNITOT] | | | | | |
| CMNOVES (ALS) CRUSTO (ALS) ( | | | | Please specify | | | | | |
| equency equency (A2) (REAST) | | | | A100* | | | | | |
| CCHRROUT | Route of Administration | | | | | | | | |
| A2 ORAPICO | [Route of Administration] | | [A:1] ( | [RLIST] | | | | | |
| Continue Condition Condi | | | [A:2] ( | [ROUTOT] | | | | | |
| equency COMPREC) C | | | | Other | | | | | |
| A.2 | | | | | | | | | |
| A.2 | Frequency | | CMERE | 01 | | | | | |
| A-22 CHANDO | [Frequency] | | | [FREQLIST] | | | | | |
| art Date tart Date tart Date COMPTO A100 * RegUnk / RegUn | | | ΓΔ·21 <b>(</b> | [CICMFREQ] | | | | | |
| art Date tart D | | | [/2] | other | | | | | |
| Reguluk Regu | | | | | | | | | |
| Reg/Unk Peq Reg/Unk P | | | | | | | | | |
| Condition Cond | Start Date<br>[Start Date] | | | | Req (1956-201 | 8) | | | |
| RegUNk RegUnk RegUnk RegUnk Regund Re | Stop Date<br>[Stop Date] | | [CMEND | ]<br>TCMENDT1 | | | | | |
| CMIND (A:3) CMMH (A:3) CMMHNO_1 CMMHNO_2 CMMHNO_3 CMMHNO_4 CMMHNO_5 CUrrent Medical Current Medical | [ | | | Req/Unk V / Req/ | Unk 🗸 / Req 🛂 | (2017-2018) | | | |
| A:3] CMMH) Current Medical Condition Current Medical C | To disease: | | | | | | | | |
| Condition 1 CMMHNO_1 CMMHNO_2 CMMHNO_3 CMMHNO_5 CUrrent Medical Current Medical Cur | [Indication] | | [A:3] | [СММН] | | | | | |
| Condition 1 Condition 2 Condition 3 Condition 4 Condition 5 N2 N2 N2 N2 N2 N2 N2 | | | | [CMMHNO_1] [ | CMMHNO_2] [C | ммнио_з] [см | IMHNO_4] [CM | MHNO_5] | |
| N2 | | | | Current Medical C | urrent Medical Cu | ırrent Medical Cur | rent Medical Curr | ent Medical | |
| [A:1] | | | | | | | | dition 5 | |
| Unsolicited AE 1 Unsolicited AE 2 Unsolicited AE 3 Unsolicited AE 3 Unsolicited AE 5 Unsol | | | [A:1] | CMAE] | VZ IV | 2 102 | IVZ | | |
| Unsolicited AE 1 Unsolicited AE 3 Unsolicited AE 3 Unsolicited AE 4 Unsolicited AE 5 N2 | | | | Unsolicited AE | CMAENO_2] [ | CMAENO_3] [C | MAENO_4] [C | MAENO_5] | |
| [A:2] | | | | Unsolicited AE 1 L | Insolicited AE 2 U | nsolicited AE 3 Ur | | | |
| Solicites (CHSDACH) AE [A:1] | | | [A:2] | CMINDSAECM1 | | VZ IV | 2 14. | 2 | |
| [A:2] CMLOCI (A:2] CMLOCI (A:2] CMLOCI (A:2] CMLOCI (A:3] Temperature (oral) (A:3] | | | | Solicited [CMSAI | 30-Min [A:2] | Follow-Up | | | |
| [A:1] | | | | [Syster | nLocal] | _ | | | |
| System [A:1] emperature (oral) A:2] Fatigue/Malaise A:3] Fatigue/Malaise A:3] Generalized Muscle A:4] Fatigue/Malaise A:5] | | | | [A:1] | [CMSYS] | | [A:2] [ | CMLOC] | |
| [A:3] Generalized Muscle Aches [A:4] Joint Aches Injection site Aches [A:5] Chills [A:5] Chills [A:7] Wornting [A:7] Wornting [A:7] Wornting [A:8] Headache [A:9] ○[CMINDOTH] Other, Please specify: A200 ★ [*] = Item is required [✔] = Source verification required [★] = ASCII Only Associated form = UNSOLICITED ADVENSE EVENT. | | | | | System [A:1] | | orai) L | ocai [A:1] Pa<br>sit | e |
| [A:3] _ Joint Aches | | | | | [A:3] | Generalized Mu | uscle | ini | ection site |
| [A:5] Chills [A:4] Swelling at injection site [A:5] | | | | | | Joint Aches | | | |
| [A:37] Vomiting [A:5] | | | | | | | | [A:4] Sw | elling at |
| [A:89] CIMINDOTH] Other, Please specify: A200 * [*] = Item is required [*] = Source verification required [*] = ASCII Only Associated form = UNSOLICITED ADVENSE EVENT. | | | | | [A:7] | Vomiting | | [A:5] Ha | rdness at |
| Other, Please specify: A200 ★ [*] = Item is required [ ✓ ] = Source verification required [ ★ ] = ASCII Only Associated form = UNSOLICITED ADVERSE EVENT. | | | [A+002 | CCMINDOTH1 | | | | "", | |
| [*] = Item is required [ ✓ ] = Source verification required [★] = ASCII Only Associated form = UNSOLICITED ADVENSE EVENT. | | | [A:99] | Other, Please spe | cify: | | | | |
| Associated form = UNSOLICITED ADVERSE EVENT. | | | | A200* | | | | | |
| Associated form = UNSOLICITED ADVERSE EVENT. | | | | | | | | | |
| Associated form = UNSOLICITED ADVERSE EVENT. | ev: [*] = Item is required [.4.3] C | ource verification required [+1 | ASCII Colu | | | | | | |
| Source verification critical settings made in InForm will override any settings made in Central Designer. | ote: Associated form = UNSOLICITED | ADVERSE EVENT. | | e in Central Designer | | | | | |

| Codelist Values Tables: CONCOMITANT MEDICATIONS | | | | | |
|---|---|---|---|---|---|
| Codelist RefName | Codelist Data Type | Label | Code | Codelist Item RefName | Data Variable RefName |
| dCMUNIT | String | amp = ampules | 1 | citmCMUNIT1 | UNITLIST |
| | | cap = capsules | 2 | citmCMUNIT2 | |
| | | g = gram | 3 | citmCMUNIT3 | |
| | | mg = milligram | 4 | citmCMUNIT4 | |
| | | mcg = microgram | 5 | citmCMUNIT5 | |
| | | gtts = drops | 6 | citmCMUNIT6 | |
| | | mL = milliliters | 7 | citmCMUNIT7 | |
| | | puffs = puffs | 8 | citmCMUNIT8 | |
| | | tab = tablets | 9 | citmCMUNIT9 | |
| | | sup = suppository | 10 | citmCMUNIT10 | |
| | | vial = vials | 11 | citmCMUNIT11 | |
| | | oint = ointment | 12 | citmCMUNIT12 | |

Protocol No: IVACFLU-S-0203 643 Dated: 12 March 2018

| | | pas = paste | 13 | citmCMUNIT13 | |
|---------|--------|-------------------|----|--------------|----------|
| dCMROUT | String | 1 = oral | 1 | citmCMROUT1 | RLIST |
| | | 2 = intramuscular | 2 | citmCMROUT2 | |
| | | 3 = subcutaneous | 3 | citmCMROUT3 | |
| | | 4 = intravenous | 4 | citmCMROUT4 | |
| | | 5 = aerosol | 5 | citmCMROUT5 | |
| | | 6 = apply on skin | 6 | citmCMROUT6 | |
| | | 7 = Other | 7 | citmCMROUT7 | |
| dCMFREQ | String | 1 = QD | 1 | citmCMFREQ1 | FREQLIST |
| | | 2 = BID | 2 | citmCMFREQ2 | |
| | | 3 = TID | 3 | citmCMFREQ3 | |
| | | 4 = QID | 4 | citmCMFREQ4 | |
| | | 5 = as needed | 5 | citmCMFREQ5 | |
| | | 6 = one time | 6 | citmCMFREQ6 | |
| | | 7 = at bed time | 7 | citmCMFREQ7 | |

| Data Variable RefName | RD Column Name | Column Data Type |
|---|---|---|
| CMSEQ | CMSEQ | NUMBER |
| | CMSEQ_ND | VARCHAR2 |
| CMDRUG | CMDRUG | VARCHAR2 |
| | CMDRUG_ND | VARCHAR2 |
| CMDOSE | CMDOSE | VARCHAR2 |
| | CMDOSE_ND | VARCHAR2 |
| CMUNIT | CMUNIT_C | VARCHAR2 |
| | CMUNIT | VARCHAR2 |
| | CMUNIT_ND | VARCHAR2 |
| CMUNIT - UNITLIST | UNITLIST C | VARCHAR2 |
| | UNITLIST | VARCHAR2 |
| CMUNIT - UNITOT | UNITOT | VARCHAR2 |
| CMROUTE | CMROUTE_C | VARCHAR2 |
| CHROOTE | CMROUTE | VARCHAR2 |
| | | VARCHAR2 |
| CMBOUTE BLICT | CMROUTE_ND | |
| CMROUTE - RLIST | RLIST_C | VARCHAR2 |
| | RLIST | VARCHAR2 |
| CMROUTE - ROUTOT | ROUTOT | VARCHAR2 |
| CMFREQ | CMFREQ_C | VARCHAR2 |
| | CMFREQ | VARCHAR2 |
| | CMFREQ_ND | VARCHAR2 |
| CMFREQ - FREQLIST | FREQLIST_C | VARCHAR2 |
| | FREQLIST | VARCHAR2 |
| CMFREQ - FREQOT | FREQOT | VARCHAR2 |
| CMSTDT | CMSTDT | DATE |
| | CMSTDT_DTS | VARCHAR2 |
| | CMSTDT_DTR | VARCHAR2 |
| | CMSTDT_ND | VARCHAR2 |
| CMEND | CMEND_C | VARCHAR2 |
| | CMEND | VARCHAR2 |
| | CMEND_ND | VARCHAR2 |
| CMEND - CMENDT | CMENDT | DATE |
| CHEND | CMENDT_DTS | VARCHAR2 |
| | CMENDT_DTS CMENDT_DTR | VARCHAR2 |
| CMIND | | VARCHAR2 |
| CMIND | CMIND_C | |
| | CMIND | VARCHAR2 |
| | CMIND_ND | VARCHAR2 |
| CMIND - CMMHNO_1 | CMMHNO_1 | NUMBER |
| CMIND - CMMHNO_2 | CMMHNO_2 | NUMBER |
| CMIND - CMMHNO_3 | CMMHNO_3 | NUMBER |
| CMIND - CMMHNO_4 | CMMHNO_4 | NUMBER |
| CMIND - CMMHNO_5 | CMMHNO_5 | NUMBER |
| CMIND - CMAENO_1 | CMAENO_1 | NUMBER |
| CMIND - CMAENO_2 | CMAENO_2 | NUMBER |
| CMIND - CMAENO_3 | CMAENO_3 | NUMBER |
| CMIND - CMAENO_4 | CMAENO_4 | NUMBER |
| CMIND - CMAENO_5 | CMAENO_5 | NUMBER |
| CMIND - 30-Min | CMSAECAT_CLIT30MIN_C | VARCHAR2 |
| | CMSAECAT_CLIT30MIN | VARCHAR2 |
| CMIND - Follow-Up | CMSAECAT CLITFOLLOWUP C | VARCHAR2 |
| * | CMSAECAT_CLITFOLLOWUP | VARCHAR2 |
| CMIND - System | SYSTEMLOCAL_CMSYS_C | VARCHAR2 |
| | SYSTEMLOCAL_CMSYS | VARCHAR2 |
| CMIND - Temperature (oral) | | |
| CHIND - remperature (oral) | CMSYS_CLITTEMPERATURE_C | VARCHAR2 |
| | CMSYS_CLITTEMPERATURE | VARCHAR2 |
| CMIND - Fatigue/Malaise | CMSYS_CLITFATIGUEMALAISE_C | VARCHAR2 |
| | CMSYS_CLITFATIGUEMALAISE | VARCHAR2 |
| CMIND - Generalized Muscle Aches | | VARCHAR2 |
| | *CMSYS_CLITGENERALIZEDMUSCLEACHES | VARCHAR2 |
| | CHOTO_CELTGENERGICEEDTTOOCEETCHES | |
| CMIND - Joint Aches | CMSYS_CLITJOINTACHES_C | VARCHAR2 |

Protocol No: IVACFLU-S-0203 644 Dated: 12 March 2018

| CMIND - Chills | CMSYS_CLITCHILLS_C | VARCHAR2 |
|---|---|---|
| | CMSYS_CLITCHILLS | VARCHAR2 |
| CMIND - Nausea | CMSYS_CLITNAUSEA_C | VARCHAR2 |
| | CMSYS_CLITNAUSEA | VARCHAR2 |
| CMIND - Vomiting | CMSYS_CLITVOMITING_C | VARCHAR2 |
| | CMSYS_CLITVOMITING | VARCHAR2 |
| CMIND - Headache | CMSYS_CLITHEADACHE_C | VARCHAR2 |
| | CMSYS_CLITHEADACHE | VARCHAR2 |
| CMIND - Local | SYSTEMLOCAL_CMLOC_C | VARCHAR2 |
| | SYSTEMLOCAL_CMLOC | VARCHAR2 |
| CMIND - Pain at injection site | CMLOC_CLITPAIN_C | VARCHAR2 |
| | CMLOC_CLITPAIN | VARCHAR2 |
| CMIND - Tenderness at injection site | CMLOC_CLITTENDERNESS_C | VARCHAR2 |
| | CMLOC_CLITTENDERNESS | VARCHAR2 |
| CMIND - Redness at injection site | CMLOC_CLITREDNESS_C | VARCHAR2 |
| | CMLOC_CLITREDNESS | VARCHAR2 |
| CMIND - Swelling at injection site | CMLOC_CLITSWELLING_C | VARCHAR2 |
| | CMLOC_CLITSWELLING | VARCHAR2 |
| CMIND - Hardness at injection site | CMLOC_CLITHARDNESS_C | VARCHAR2 |
| | CMLOC_CLITHARDNESS | VARCHAR2 |
| CMIND - CMINDOTH | CMINDOTH | VARCHAR2 |
| Key: [*] = The column and/or table na | me in the actual RDE extract may be different. | |

Protocol No: IVACFLU-S-0203 645 Dated: 12 March 2018

| I۷ | ACFLU-S-0203: MISSED VISIT FORM (MISSED | VISIT F | ORM) [I | MISSFORM] | |
|---|---|---|---|---|---|
| Mis | sing Visit [ScMissingVisit] | | | | |
| 1.* | Were any study visits missed?<br>[Any Missing Visit?] | | | [MISSYN] [A:1] | |
| | Study day that was missed | | | Reason visit was missed | Comment |
| 2. | | | | | |
| MIS | SED VISIT FORM Entry [ScMISSEDVISITFORM] | | | | |
| 2.1 | Study day that was missed [Study day that was missed] | [MISSDAY] [A:1] | ay 2<br>ay 5<br>ay 8<br>ay 22 | | |
| 2.2 | Reason visit was missed [Reason visit was missed] | [A:2] QU<br>[A:3] QS<br>[A:4] QS<br>[A:5] QS<br>[A:6] QI | Inable to co | eceased | |
| 2.3 | Comment [Comment] | [MISSCOM<br>A200* | 1 | | |
| | y: [ ▼ ] = Source verification required [★] = ASCII Only te: Source verification critical settings made in InForm will override any setti | ngs made in | Central Desi | gner. | |

| Study ( | Study Object Descriptions: MISSED VISIT FORM | |
|---|---|---|
| Туре | RefName | Description |
| Form | MISSFORM | MISSED VISIT FORM |
| Section | ScMISSEDVISITFORM | MISSED VISIT FORM |

| Data Variable RefName | RD Column Name | Column Data Type |
|-----------------------|----------------|------------------|
| MISSYN | MISSYN_C | VARCHAR2 |
| | MISSYN | VARCHAR2 |
| | MISSYN_ND | VARCHAR2 |
| *RD_MISSFORM_SCMISSI | EDVISITFORM | |
| MISSDAY | MISSDAY_C | VARCHAR2 |
| | MISSDAY | VARCHAR2 |
| | MISSDAY_ND | VARCHAR2 |
| MISSREA | MISSREA_C | VARCHAR2 |
| | MISSREA | VARCHAR2 |
| | MISSREA_ND | VARCHAR2 |
| MISSREA - MISSSPEC | MISSSPEC | VARCHAR2 |
| MISSCOM | MISSCOM | VARCHAR2 |
| | MISSCOM_ND | VARCHAR2 |


Protocol No: IVACFLU-S-0203 646 Dated: 12 March 2018

| RE | PORT OF PREGNANCY [scPREGRPT] | |
|---|---|---|
| 1.* | Pregnancy test date<br>[Pregnancy test date] | [PREGDATE] Req / Req / Req (2017-2018) |
| 2.* | Date of last menstrual period [Date of last menstrual period] | [MENSDATE] Req |
| 3.* | Estimated date of delivery<br>[Estimated date of delivery] | [DELIDATE] Req |
| 1.* | 1, Pregnancy History: [Pregnancy History:] | [NewCompound] [PREGREFO] 1.1, Has the woman been pregnant before? [A:1] ○[RAMMALY] Yes 1.2, Any history of fetal anomalies? [A:1] ○[Yes [A:2] ○[No [PREMATUR] 1.3, Any history of premature births? [A:1] ○[Yes [A:2] ○[No [DEATH] 1.4, Any history of fetal deaths? [A:1] ○[Yes [A:2] ○[No [STILLBRT] 1.5, Any history of still births? [A:1] ○[Yes [A:2] ○[No [MISCARRY] 1.6, Any history of miscarriage? [A:1] ○[Yes [A:2] ○[No [PREGOTH] 1.7 Other problem? [A:1] ○[PREGSPEC] Yes, Specify: A200 ★ |
| 5.*<br>• | 2, Were there any medications taken during the time of conception or during the pregnancy? [Medications taken] | [PREGMED] [A:1] ○Yes, Please complete Concomitant Medications form [A:2] ○No |
| 5.*<br><b>✓</b> | 3, Any additional information? [Any additional information?] | [ADDINFO] [A:1] ○ [PREGDESC] Yes Describe: A200 * [A:2] ○ No |
| 7.*<br>• | Is subject willing to be contacted after delivery? [ Is subject willing to be contacted after delivery? ] | [PREGCONT] [IA:1] |

| Study Object Descriptions: REPORT OF PREGNANCY | | |
|---|---|---|
| Туре | RefName | Description |
| Form | PREGRPT | REPORT OF PREGNANCY |
| Section | scPREGRPT | REPORT OF PREGNANCY |

| RDE Analytics: RD_ | | |
|------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| PREGDATE | PREGDATE | DATE |
| | PREGDATE_DTS | VARCHAR2 |
| | PREGDATE_ND | VARCHAR2 |
| MENSDATE | MENSDATE | DATE |
| | MENSDATE_DTS | VARCHAR2 |
| | MENSDATE_DTR | VARCHAR2 |
| | MENSDATE_ND | VARCHAR2 |
| DELIDATE | DELIDATE | DATE |
| | DELIDATE_DTS | VARCHAR2 |
| | DELIDATE_DTR | VARCHAR2 |
| | DELIDATE_ND | VARCHAR2 |
| NewCompound | NEWCOMPOUND_ND | VARCHAR2 |
| NewCompound - PREGBEFO | PREGBEFO_C | VARCHAR2 |
| | PREGBEFO | VARCHAR2 |
| NewCompound - ANOMALY | ANOMALY_C | VARCHAR2 |
| | ANOMALY | VARCHAR2 |
| NewCompound - PREMATUR | PREMATUR_C | VARCHAR2 |
| | PREMATUR | VARCHAR2 |
| NewCompound - DEATH | DEATH_C | VARCHAR2 |
| | DEATH | VARCHAR2 |
| NewCompound - STILLBRT | STILLBRT_C | VARCHAR2 |
| | STILLBRT | VARCHAR2 |
| NewCompound - MISCARRY | MISCARRY_C | VARCHAR2 |
| | MISCARRY | VARCHAR2 |
| NewCompound - PREGOTH | PREGOTH_C | VARCHAR2 |
| | PREGOTH | VARCHAR2 |
| NewCompound - PREGSPEC | PREGSPEC | VARCHAR2 |
| PREGMED | PREGMED_C | VARCHAR2 |

Protocol No: IVACFLU-S-0203 647 Dated: 12 March 2018

| | PREGMED | VARCHAR2 |
|--------------------|-------------|----------|
| | PREGMED_ND | VARCHAR2 |
| ADDINFO | ADDINFO_C | VARCHAR2 |
| | ADDINFO | VARCHAR2 |
| | ADDINFO_ND | VARCHAR2 |
| ADDINFO - PREGDESC | PREGDESC | VARCHAR2 |
| PREGCONT | PREGCONT_C | VARCHAR2 |
| | PREGCONT | VARCHAR2 |
| | PREGCONT_ND | VARCHAR2 |

Protocol No: IVACFLU-S-0203 648 Dated: 12 March 2018



| RDE Analytics: RD_EOSFM | | |
|-------------------------|----------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| EOSYN | EOSYN_C | VARCHAR2 |
| | EOSYN | VARCHAR2 |
| | EOSYN_ND | VARCHAR2 |
| EOSYN - EOSDT | EOSDT | DATE |
| | EOSDT_DTS | VARCHAR2 |
| EOSYN - EOSRES | EOSRES_C | VARCHAR2 |
| | EOSRES | VARCHAR2 |
| EOSYN - EOSAENUM | EOSAENUM | VARCHAR2 |
| EOSYN - EOSRSNOT | EOSRSNOT | VARCHAR2 |
| EOSYN - EOSVISDT | EOSVISDT | DATE |
| | EOSVISDT_DTS | VARCHAR2 |

Protocol No: IVACFLU-S-0203 649 Dated: 12 March 2018

| IVACFLU-S-0203: INVESTIGATOR SIGNATURE (SIGN) [PISIGN] Signature [SIGNSC] | | |
|---|---|---|
| | (ey: [*] = Item is required [ ✓ ] = Source verification required lote: Source verification critical settings made in InForm will override any settings made in Central Des | gner. |

| RDE Analytics: RD_PISIGN | | |
|--------------------------|--------------------|------------------|
| Data Variable RefName | RD Column Name | Column Data Type |
| SIGNY | SIGNY_ND | VARCHAR2 |
| SIGNY - Yes | SIGNY_CITMSIGNY1_C | VARCHAR2 |
| | SIGNY_CITMSIGNY1 | VARCHAR2 |

Protocol No: IVACFLU-S-0203 650 Dated: 12 March 2018

| InForm Special Property | Property Type | Data Object RefName | Data Object Path RefName |
|---|---|---|---|
| Screening | Visit | SCRVIS | SCRVIS |
| Enrollment | Visit | ENRVIS | ENRVIS |
| Screening | Form | SYSSCR | SCRVIS.SYSSCR |
| Enrollment | Form | SYSENR | ENRVIS.SYSENR |
| Patient Identification | Form | SUBID | SCR.SUBID |
| Study Completion | Form | EOSFM | EOS.EOSFM |
| Reg Docs | Form | Unassigned | Unassigned |
| Visit Report | Form | Unassigned | Unassigned |
| Initials (Screening) | Item | SUBINI | SCRVIS.SYSSCR.SYSSCRSC.SUBINI |
| DOB (Screening) | Item | SCRDOBDT | SCRVIS.SYSSCR.SYSSCRSC.SCRDOBD |
| Screening date (Screening) | Item | Unassigned | Unassigned |
| Patient No. (Enrollment) | Item | INSUBJID | SCR.SUBID.SUBIDSC.INSUBJID<br>ENRVIS.SYSENR.SYSENRSC.INSUBJID |
| Initials (Patient Identification) | Item | Unassigned | Unassigned |
| Completion status (Study Completion) | Item | EOSYN | EOS.EOSFM.EOSSC.EOSYN |
| Drop out reason (Study Completion) | Item | EOSRES | EOS.EOSFM.EOSSC.EOSCMP.EOSRES |
| DOV (Date of Visit) | Item | DOVDT | UNSVIS.DOVI.DOVSC.DOVDT DI.DOVI.DOVSC.DOVDT SCR.DOVI.DOVSC.DOVDT Day2.DOVI.DOVSC.DOVDT Day5.DOVI.DOVSC.DOVDT D8.DOVI.DOVSC.DOVDT D8.DOVI.DOVSC.DOVDT D91.DOVI.DOVSC.DOVDT D91.DOVI.DOVSC.DOVDT VISS.DOVI.DOVSC.DOVDT |
| Randomization field (Randomization) | Item | ELIGSUBID | D1.ELIG.IE2SC.ELIGYCMP.ELIGSUBID<br>SCR.ELIG.IE2SC.ELIGYCMP.ELIGSUBID |

Protocol No: IVACFLU-S-0203 651 Dated: 12 March 2018

| Personal/Protected Health Information Table: IVACFLU-S-0203 |
|---|
| Item RefName Section RefName Form RefName |
| No items have been defined as "Personal/Protected Health Information". |
| Please note: emails sent from the trial server by the InForm application are not encrypted. If you are subject to HIPAA requirements, you should identify and block all Personal/Protected Health Information items that may be included in email notifications. |

Protocol No: IVACFLU-S-0203 652 Dated: 12 March 2018

Unit Conversions For Study Design: IVACFLU-S-0203

No unit conversion data

Protocol No: IVACFLU-S-0203 653 Dated: 12 March 2018

Review States for Study: IVACFLU-S-0203

No Review States have been defined.

IVACFLU-S

Version 1.0 Protocol No: IVACFLU-S-0203 654 Dated: 12 March 2018

| Participant ID | |
|-----------------|-----|
| r articipant iD | l 1 |

## TAKE-HOME DIARY CARD

| (This part is completed by INVESTIGATOR) |
|---|
| FULL NAME of participant: |
| Date of vaccination://2017 |
| Vaccinated arm: |
| Date of the next visit://2017 |
| Date of diary card collection://2017 |
| After reviewing the diary card completed by the participant, the investigator needs to answer the following question: |
| Does the participant have any signs and symptoms which are continuing on day 7? |
| $\square$ No |
| $\square$ Yes $\rightarrow$ Investigator to complete the form titled "Post-vaccination monitoring after day 7" and instruct the participant to monitor ongoing signs and symptoms |
| FULL NAME of investigator: Signature: |

IVACFLU-S-0203 Page 1 of 9

Participant ID

Dated: 12 March 2018

#### TAKE-HOME DIARY CARD

655

#### INSTRUCTIONS

- 1. Take your temperature by mouth each day using the thermometer we gave you.
  - Start taking your temperature later today.
  - Take it around the same time each day.
  - Wait 15 minutes if you had a hot or cold drink.



- Wait for the beep or other indication that the temperature is ready.
- Write the temperature in the space on the Diary Card. If you take your temperature more than once during the day, write the highest temperature for the day on the Diary Card.
- 2. Each day, look at your arm where you received the injection.



- Check for redness and swelling. Touch your arm and feel for hardness at the injection site.
- If you do not find anything, check "None" on the diary card for the day.
- If you see or feel something, place a mark with a pen on either side of the area. Measure the widest part of it with the ruler we have given you.
- Record your measurement on the Diary Card. If you do more than one measurement during the day, record the largest measurement for each day on the Diary Card.
- Example: This person had redness at the injection site. They put
  dots with a pen at the widest points of the redness and measured
  it. It measured 2.4 cm. They wrote 2.4 cm on the Diary Card for
  that day.
- 3. Severity of symptoms:

None: I did not have any discomfort

Mild: I only had minor discomfort. I did my usual activities

Moderate: I noticed the symptom. It bothered me enough that I did not do as much as I

usually do

Severe: I really noticed the symptom. It kept me from doing many of the things I

wanted or needed to do

4. Please contact the study site using the number below if you have any questions:

| l |
|---|
| l |
| l |
| l |
| l |
| l |
| l |

IVACFLU-S-0203 Page 2 of 9

IVACFLU-S Version 1.0 656 Dated: 12 March 2018

| Participant ID |
|----------------|
|----------------|

## TAKE-HOME DIARY CARD **LOCAL REACTIONS** within 7 days post-vaccination

| | Evening Day 1 (Day of vaccination)//2017 | Day 2<br>//2017 | Day 3<br>//2017 | <b>Day 4</b> //2017 | Day 5<br>//2017 | <b>Day 6</b> //2017 | <b>Day 7</b> //2017 |
|---|---|---|---|---|---|---|---|
| Oral<br>temperature | ,_°C | ,_°C | ,_°C | ,_°C | ,_°C | ,_°C | ,°C |
| Pain at injection site | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe |
| Tenderness<br>at injection<br>site | □ None □ Yes, grading: □ Mild □ Moderate □ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe | ☐ None ☐ Yes, grading: ☐ Mild ☐ Moderate ☐ Severe |

IVACFLU-S Version 1.0 657 Dated: 12 March 2018

| Participant ID |
|----------------|
|----------------|

## TAKE-HOME DIARY CARD **LOCAL REACTIONS** within 7 days post-vaccination

| | Evening Day 1 (Day of vaccination)//2017 | Day 2//2017 | Day 3//2017 | Day 4//2017 | Day 5//2017 | Day 6//2017 | Day 7//2017 |
|---|---|---|---|---|---|---|---|
| Redness at injection site | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | ☐ None ☐ Yes, measurement:mm |
| Swelling at injection site | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm |
| Hardness at injection site | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm | □ None □ Yes, measurement:mm |

Version 1.0 Protocol No: IVACFLU-S-0203 658 Dated: 12 March 2018

| Participant ID | | |
|----------------|---|------|
| <b>.</b> | · | <br> |

## TAKE-HOME DIARY CARD **SYSTEMIC REACTIONS** within 7 days post-vaccination

| | Evening Day 1 (Day of vaccination)//2017 | Day 2<br>//2017 | Day 3<br>//2017 | <b>Day 4</b> //2017 | Day 5<br>//2017 | <b>Day 6</b> //2017 | <b>Day 7</b> //2017 |
|---|---|---|---|---|---|---|---|
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| Tiredness/ | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | $\square$ Yes, grading: |
| discomfor | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| t | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Muscle<br>Aches | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Joint<br>Aches | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| Titles | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 659 Dated: 12 March 2018

| Participant ID |
|----------------|
|----------------|

## TAKE-HOME DIARY CARD **SYSTEMIC REACTIONS** within 7 days post-vaccination

| | Evening Day 1 (Day of vaccination)//2017 | Day 2<br>//2017 | Day 3//2017 | <b>Day 4</b> //2017 | Day 5<br>//2017 | <b>Day 6</b> //2017 | <b>Day 7</b> //2017 |
|---|---|---|---|---|---|---|---|
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Headache | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Chills | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Nausea | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |

Version 1.0 Protocol No: IVACFLU-S-0203 660 Dated: 12 March 2018

| Participant ID |
|----------------|
|----------------|

## TAKE-HOME DIARY CARD **SYSTEMIC REACTIONS** within 7 days post-vaccination

| | Evening Day 1 (Day of vaccination)//2017 | Day 2<br>//2017 | <b>Day 3</b> //2017 | <b>Day 4</b> //2017 | Day 5//2017 | <b>Day 6</b> //2017 | <b>Day 7</b> //2017 |
|---|---|---|---|---|---|---|---|
| | □ None | □ None | □ None | □ None | □ None | □ None | □ None |
| | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: | ☐ Yes, grading: |
| Vomiting | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild | ☐ Mild |
| | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate | ☐ Moderate |
| | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe | ☐ Severe |


Dated: 12 March 2018

Participant ID | \_\_\_|

## TAKE-HOME DIARY CARD

| Other COMPLAINT or ILLNESS: Did you have any other things that bothered you? Yes No Record any other complaints or illness which developed or worsened during the 7-day follow-up period after receiving the study injection. List each illness or complaint separately. You may call study doctor for any other complaints or illness. | | | | | |
|---|---|---|---|---|---|
| Complaint or illness | | Start | date | | ast day the illness or<br>emplaint presents <sup>(*)</sup> |
| Example: Cough | | 21/07/ | 2017 | | 23/07/2017 |
| 1. | | | | | |
| 2. | | | | | |
| 3. | | | | | |
| 4. | | | | | |
| 5. | | | | | |
| (*) Write "continuing" if the illness is still going on day 7. | | | | | |
| MEDICATIONS: | | | | | |
| Did you take any medications durin | _ | days after you | r injection? | | |
| | No | | | | |
| If you took medication, list the med medications or the used packaging l | | | | | ir prescription or |
| Medication you took | Why y | you took the | Start dat | | Last day you took medication (*) |
| Example: Paracetamol | | Fever | 21/07/201 | 7 | 22/07/2017 |
| 1. | | | | | |
| 2. | | | | | |
| 3. | | | | | |
| 4. | | | | | |
| 5. | | | | | |

IVACFLU-S-0203 Version 1.0, dated 14/12/2016

<sup>(\*)</sup> Write "continuing" if you still took medication on day 7.

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 662 Dated: 12 March 2018

| Participant ID |
|----------------|

# TAKE-HOME DIARY CARD Other notes (if any)

| <br> |
|------|

Protocol No: IVACFLU-S-0203 Dated: 12 March 2018

Quintiles/MS

eCRF Design Approval Form

Sponsor Name: Institute of Vaccines and Medical Biologicals (IVAC) Protocol Number: IVACFLU-S-

0203 Page 1 of 2

Institute of Vaccines and

Sponsor: Medical Biologicals Project Database ID: IYA06804

(IVAC)

Protocol: IVACFLU-S-0203 Date: 11May2017 (ddmmmyyyy)

Protocol Version: 4.0 Protocol Date: 9Feb2017 (ddmmmyyyy)

Annotated Trial Design (ATD) / Annotated Study Book (ASB) / CRF Design Specification / Study Blank CRF and Study Unique CRF (aCRF):

and Study Unique CRF (aCRF):

Version Number: V4.0

Version Date:

2May2017 (ddmmmyyyy)

Reference: CS\_WI\_DM0404

Authorization confirms review and approval of the eCRF design. QuintilesIMS authorization is obtained using electronic signatures in ELVIS. Signature line and Date are used only if the corresponding Role is with the Sponsor.

| Name: | Tushar Tewari/ Tran Thang | Signature: |
|---|---|---|
| Title:<br>Role: | Sponsor Representative Senior Medical Officer | Signature: Than Date: (ddmmmyyyy) 12 May, 2017 |
| Name: | Shirley Xiong | |
| Title: | Data Team Lead | |
| Name: | Lianying Zhao | |
| Title: | Technical Designer | |
| Name: | Suman Kapoor | Signature: |
| Title: | Statistical Team Lead | Date: (ddmmmyyyy) |
| Name: | Hong Anh Nguyen | |
| Title: | Clinical Lead | |
| Name: | Niamh Page | Signature: |
| Title: | Lifecycle Safety | Date: (ddmmmyyyy) |
| Name: | Flora Amos | Signature: |
| Title: | Therapeutic Medical Advisor (TMA) | Date:<br>(ddmmmyyyy) |

Form No: CS\_FM\_DM118 Revision 8

Effective Date: 01Mar2017

Copyright © 2008, 2009, 2011-2013, 2015, 2017 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 664 Dated: 12 March 2018



eCRF Design Approval Form

Sponsor Name: Institute of Vaccines and Medical Biologicals (IVAC) Protocol Number: IVACFLU-S-0203

Reference: CS\_WI\_DM0404

Page 2 of 2

| Name: | | Signature: |
|---|---|---|
| Title: | Clinical Event Validation and Adjudication (CEVA) | Date: (ddmmmyyyy) |
| Name: | | |
| Title: | Epidemiologist | |
| Additional Information: | | |

| Document Version History | | |
|---|---|---|
| Version | Version Date<br>(dd-mmm-yyyy) | Significant Changes |
| V1.0 | 28-Feb-2017 | Initial version |
| V2.0 | 10-Mar-2017 | <ol> <li>Add two new visits. Day 2 and Day 5.</li> <li>Update Day 91 telephone contact form to Contact form</li> <li>Add 'Result Reading Time' item on Urine pregnancy test from.</li> <li>Update 'Indication' field Current Medical Condition and Unsolicited AE from free text to variable box</li> </ol> |
| V3.0 | 21-Mar-2017 | Add 'Day 2' and 'Day 5' in the 'study day that was missed field' on 'Missed visit' form. |
| V4.0 | 2-May-2017 | <ol> <li>Year range for CM start date, change from 2017-2018 to 1956-2018</li> <li>Add item 3 "Update Subject Randomization Number" onto subject identification form</li> </ol> |

Form No: CS\_FM\_DM118 Revision 8

Effective Date: 01Mar2017

Copyright © 2008, 2009, 2011-2013, 2015, 2017 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 665 Dated: 12 March 2018



## Document Approval Signature(s)

This document has been signed electronically in compliance with Quintiles electronic signature policies and procedures. This page is a manifestation of the electronic signatures, which may be confirmed within the Quintiles source system in accordance with Quintiles records retention policies.

Note: the Title field in the signature block has been intentionally left blank.

UserName: Zhao, Lianying (q820274)

Title:

Date: Thursday, 11 May 2017, 06:34 AM Eastern Time

Meaning: I Approve the Document

\_\_\_\_\_

UserName: Page, Niamh (q601811)

Title:

Date: Thursday, 11 May 2017, 07:27 AM Eastern Time

Meaning: I Approve the Document

\_\_\_\_\_

UserName: Nguyen, Hong Anh (q813460)

Title:

Date: Thursday, 11 May 2017, 08:30 AM Eastern Time

Meaning: I Approve the Document

UserName: Xiong, Shirley (q832662)

Title:

Date: Thursday, 11 May 2017, 09:42 PM Eastern Time

Meaning: I Approve the Document

UserName: Kapoor, Suman (q805805)

Title:

Date: Thursday, 11 May 2017, 10:20 PM Eastern Time

Meaning: I Approve the Document

\_\_\_\_\_

Protocol No: IVACFLU-S-0203 666 Dated: 12 March 2018



## Document Approval Signature(s)

This document has been signed electronically in compliance with Quintiles electronic signature policies and procedures. This page is a manifestation of the electronic signatures, which may be confirmed within the Quintiles source system in accordance with Quintiles records retention policies.

Note: the Title field in the signature block has been intentionally left blank.

UserName: Amos, Flora (q828871)

Title:

Date: Thursday, 11 May 2017, 11:38 PM Eastern Time

Meaning: I Approve the Document

Protocol No: IVACFLU-S-0203 667 Dated: 12 March 2018

# 16.1.3 List of IECs or IRBs and Representative Written Information for Subject and Sample Consent Forms

## 16.1.3.1. List of IRBS and/or IECs by Investigator

| Study Center | IRB/EC Name/Address |
|---|---|
| | The World Health Organization Research Ethics Review Committee 20, Avenue Appia –CH-1211 Geneva 27, Switzerland |
| 201 and 203 | Pasteur Institute Ethics Committee in Biomedical Research Pasteur Institute in Ho Chi Minh City 167 Pasteur, Ward 8, District 3 Ho Chi Minh City, Vietnam |
| | Ethics Committee in Biomedical Research - Ministry of Health<br>138 Giang Vo Street, Ba Dinh Street<br>Hanoi, Vietnam |

Protocol No: IVACFLU-S-0203 668 Dated: 12 March 2018

16.1.3.2. Sample of Written Subject Information and Consent Form

| Document | Date |
|---|---|
| Site Specific Information Sheet and Informed Consent Forms (Phase 2), Site 201, Version 4 | 09 February 2017 |
| Site Specific Information Sheet and Informed Consent Forms (Phase 3), Site 201, Version 4 | 09 February 2017 |
| Site Specific Information Sheet and Informed Consent Forms (Phase 3), Site 203, Version 4 | 09 February 2017 |

Protocol No: IVACFLU-S-0203 669 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### INFORMATION SHEET and INFORMED CONSENT FORMS

for "screening" and "participation in the research study" entitled:

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

| Sponsor: | Institute of Vaccines and Medical Biologicals (IVAC) |
|---|---|
| Funder: | PATH |
| Study implementer: | Pasteur Institute in Ho Chi Minh City (PIHCMC) |
| Full name of volunteer: | |
| Participant screening code: | |
| Participant identification code (if recruited): | |

#### **CONSENT FOR PHASE 2**

#### Introduction

You are invited to participate in a research study. This is a study of an experimental seasonal influenza vaccine called IVACFLU-S. We will call it the "study vaccine." The study vaccine has not been approved for sale in Vietnam. It can only be used in research. This vaccine was made in Vietnam by the Institute of Vaccines and Biologicals (IVAC), Ministry of Health.

The vaccine was used in a Phase 1 study of 60 people in the Hung Ha district health center. In the Phase 1 study, the vaccine did not cause any serious health problems. Most of the side effects were mild and did not last long. Now we will test the study vaccine in a larger study of about 888 people. If the study shows good results, IVAC will apply to license the vaccine in Vietnam. The study is a combination of a Phase 2 study and a Phase 3 study. **You are being asked to join the Phase 2 part of the study with 252 participants.** For this study, we want to see if the study vaccine continues to be safe for people to use. You will not have any blood drawn in this study.

The following groups are involved in the study: Institute of Vaccines and Biologicals, the Pasteur Institute, Ho Chi Minh City, Long An Preventive Medicine Centers and the Ben Luc district health centers. The study is funded through the US Biomedical Advanced Research and Development Authority (BARDA), PATH, an international nonprofit organization, and the World Health Organization (WHO).

This information sheet explains the study and your part in the study. Please take as much time as you need to read this information. Talk with friends, relatives and your doctor if you wish. You can ask us any questions you want.

#### What you should know about this study:

1. Being in this study is voluntary. You can refuse to join or leave any time after you have joined without penalty or loss of any rights you normally have.

---

Protocol No: IVACFLU-S-0203 670 Dated: 12 March 2018

## IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

- 2. You may or may not benefit from being in the study. If you join, you may help other people in your community and Vietnam.
- 3. You will receive 1 injection of the study vaccine or a placebo. The placebo is sterile salt water. It will not prepare your body to fight influenza infections. You and the researcher will not know if you were given study vaccine or placebo until the end of the study. This is decided by chance. However, each person in the study has a greater chance of getting the study vaccine. For every person who gets the placebo, 5 people will get the study vaccine.
- 4. You will have physical examinations by a clinician. If you are a woman, you will have a urine test for pregnancy. You must agree to use birth control until 3 weeks (21 days) after your injection. We will counsel you on reliable birth control methods (intrauterine devices, hormonal contraception, condoms or diaphragm with spermicide) and help you get it for free.
- 5. In research of vaccines, there is a risk of harm. Please take your time to understand the risks. Ask any questions you have.
- 6. During the study, we will tell you of any new information about the vaccine. This new information might affect your decision to stay in the study. You may leave the study at any time.

#### What is a seasonal influenza vaccine?

The influenza virus is a very small germ that can be passed from person to person through the fluids in your nose, throat, mouth and lungs. Influenza virus can cause an illness in a person's airways that lasts about one week. Usually, the illness comes with a high fever, cough, headache and tiredness. Some influenza illnesses can be severe, especially among the young, old, and people with chronic diseases.

Most healthy people do not think of the flu as a serious illness. They may feel bad and miss some work. They are not aware that the flu causes many hospitalizations and early deaths for the young, old, and persons with chronic diseases. The flu has been linked with increases in miscarriage and heart attacks. In this study, we will teach you how to prevent getting the flu and giving it to others.

A vaccine is one of the best protections against influenza. There are different types of influenza and even those types may change slightly from one year to the next. Every year, the World Health Organization (WHO) receives information from countries all over the world about what types of influenza they are seeing in their country. The WHO uses this information to predict which types of influenza may be causing problems in the coming year. It tells the vaccine manufactures what type of vaccine they should make each year to help fight influenza infection. Companies can put together several types of influenza vaccines into one injection. This is called seasonal influenza vaccine.

#### What should I know about the study vaccine manufactured by IVAC?

IVAC made the influenza vaccine that will be used in this study. The WHO and PATH (an international nonprofit organization) have supported IVAC to make influenza vaccine. They helped IVAC meet the standards necessary to make a good product. The vaccine has had testing done to show that it was made correctly. The tests showed that study vaccine can be used in humans in vaccine studies. The vaccine cannot give you influenza.

#### What is the goal of this study?

This study's goal is to describe the safety and the body's responses to 1 injection of the study vaccine.

#### How is the vaccine given?

We will give the vaccine by injecting it into the muscle of your upper arm. We will give it only once.

Protocol No: IVACFLU-S-0203 671 Dated: 12 March 2018

### IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

We divide the people in the study into 2 groups. One group (210 people) will get an injection of the study vaccine and the other group (42 people) will get an injection of a liquid that does not have the vaccine in it (the placebo). The placebo is sterile salt water. A computer decides which group you are in. Neither you nor the study doctor can decide or will know. In this study, people have a much greater chance of getting the study vaccine than getting the placebo. For every person who gets the placebo in the study, 5 will get the study vaccine.

#### How long will I be in this study?

If you join, you will be in the study for about 3 months after your injection. However, you will only need to come to the study site during the first 3 weeks.

#### What will happen during screening for this study?

If you agree to be in this study, we will do some things to see if you can join; this is called "screening". You will be provided information about the study and you need to sign this consent before we do any screening.

- 1. For screening:
  - A clinician will ask about your health history.
  - The clinician will do a physical exam. We will take your temperature, pulse, and blood pressure.
  - If you are a woman who is able to get pregnant, we will do a urine pregnancy test see if you are pregnant.
     Pregnant women cannot get the study products.
- 2. Women who could become pregnant must have already been using reliable birth control (intrauterine device, hormonal contraception, or condoms) to be in the study.

We will go over the results of screening with you. If we find you have a health issue, we will advise you on how to get proper treatment. Because we cannot tell ahead of time how many people who enter screening will qualify and want to join the study, we may have to exclude some people from the study, even if they qualify and want to join.

#### What will happen in this study?

If the questions and the physical exam show that you can be in the study, we will ask if you still would like to join. If you agree, you can have the study injection the same day as your screening visit. You can take a few more days to think about it, if you want. You can always change your mind if you do not want to be in the study. Nothing bad will happen if you decide not to join or leave after you have joined.

#### 1. Product injection:

- If the injection is given to you on a different day from the screening visit, we will again take your temperature, pulse and blood pressure and do a urine pregnancy test on women who can become pregnant. Pregnant women will not receive the injection.
- We will give you your injection of study vaccine or placebo. The injection will be into a muscle in your upper arm.
- You will be asked to stay in the study clinic for at least 30 minutes. During this time, the study staff will
  check to see if you have any reactions to the injection.
- The study staff will show you how to complete a Diary Card. We want you to record any reaction or
  medical event and any medications you take on this form. Record each day for 7 days since the day of
  your injection.
- 2. The study staff will visit your home one day after your injection and call you 4 days after your injection to check on your well-being and see if you are completing the Diary Card.
- 3. Seven (7) days after you are given the injection, you will return to the study clinic.
  - We will take your oral temperature, pulse, and blood pressure. A clinician will do a physical exam only if
    you report symptoms.

IVACFLU-S-0203\_ICF\_ Phase 2\_Ben Luc Version 4.0, dated 09/02/2017

Protocol No: IVACFLU-S-0203 672 Dated: 12 March 2018

IVAC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

- We will go over the Diary Card with you to make sure we understand what you wrote.
- 4. Over the next 2 weeks (14 days) you will have no clinic visits, but we want you to tell us if you have any health concerns. If needed, we will examine you or refer you to care.
- 5. Twenty-one (21) days after you are given the injection, you will return to the study clinic.
  - We will take your temperature, pulse, and blood pressure. The clinician will do a physical exam only
    if you report symptoms.
  - If you are a women who could become pregnant, we will tell you that you no longer need to use birth
    control for the study.
- 6. Three months after your injection a member of the study staff will call you.
  - We will ask about health problems you told us were continuing at your last visit.
  - We will ask you about medications you told us you were still using at your last visit.
  - We will ask about any new, serious health problems that may have happened since we saw you last.
  - We will thank you for being in the study. This will end your study participation.
- 7. After the Phase 2 part of the study, we will do a Phase 3 part. It will take many months to finish the study and know the results. When we know the results, we will send you a letter so that you know the study results, too.

#### In summary, if you join the study:

- You will visit the Study Clinic 3 times over about 3 weeks and one time for consent meeting.
- Women will provide a urine sample before their injection. We will use it for a pregnancy test. Women should be using reliable birth control for at least 3 weeks after their injection.
- You will receive only 1 injection of study vaccine or placebo.
- You will be completing a Diary Card for 7 days since the date of the injection
- We will visit your home one day after the injection and call you 4 days after the injection to check on your well-being.
- We will contact you about 3 months after the injection to find out about your health
- During the study, we will tell you about new information or changes in the study that may affect your health or your willingness to continue.
- You will be informed about the study results and all exams related to your health.
- We will send you a letter with the study results, including what study product you received.

Almost all of the procedures we do in this study are like what happens when you have regular health care. The part of this study that is not standard treatment is when we give you the study vaccine or placebo.

#### What are my responsibilities?

- Tell us if you have ever had a bad reaction to a vaccine or allergy to eggs, chicken or rubber.
- Inform us if you are pregnant or breast feeding.
- Come to the study visits and do your best to follow directions.
- Tell us if you have moved.
- Tell us if you do not like something about the study.
- Tell us if you want to leave the study.
- Tell your study doctor about any changes in your health that occur during the study as well as any changes in your medications during the study.
- While participating in this study, you may not take part in any other research project.

IVACFLU-S-0203\_ICF\_ Phase 2\_Ben Luc Version 4.0, dated 09/02/2017 Protocol No: IVACFLU-S-0203 673 Dated: 12 March 2018

IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### What harm could happen?

Sometimes bad things can happen in a study of a vaccine. Think about these when deciding if you want to join. Here is what we know that could happen during the study:

- Receiving the injection of vaccine or placebo can cause pain, redness, swelling, hardness or infection where
  the needle was put in. Also the whole body may feel feverish or have muscle aches or nausea (feeling like you
  may throw up). In the earlier study of the vaccine, people report pain and tenderness the most. Most of the
  side effects were mild, meaning that people did not limit their activities because of the injection.
- It is very rare, but sometimes people have a serious allergic reaction to a vaccine. This can be life-threatening.
   We can provide emergency care, if needed.
- There may be harm, even serious harm that we do not know about yet.
- We do not know if the study vaccine is safe for use in pregnancy. That is why we ask women to agree to use reliable birth control during the study.
- We do our best to keep your study records and private information confidential. However, there is always a
  risk that someone who is not supposed to may see your information by accident. If this happens, we will tell
  you.
- To be in the study, you must not have had a flu vaccine in the past 6 months and you must wait until 3 weeks
  after your injection to have any licensed vaccines. Because of this, it is possible that you could get exposed to
  seasonal influenza and get the flu during the study. We will teach you ways to protect yourself and others
  from the flu.

#### What if I am injured?

If you have an injury and need help, contact Dr. Phan Cong Hung or Dr. Hoang Anh Thang to let him know what is happening. Their numbers are at the end of this form. Dr. Phan Cong Hung or Dr. Hoang Anh Thang can consult and help you get the care you need. The IVAC has arranged for the Ben Luc district hospital to provide you with free treatment for any injuries that happen during the study. The IVAC does not plan to pay any additional money to you unless directed by the Ministry of Health, which reviews research injuries.

#### What if I become pregnant?

We will test for pregnancy before you receive your injection. If you become pregnant and have received an injection on the study, we will ask you to stay in the study. Because you received a study product, we want to watch after your health. If the study ends and you are still pregnant, we will stay in touch with you to report on the outcome of the pregnancy and health of the baby.

#### What are the known benefits of participating in this research study?

There may not be any benefit to you personally. However, you may benefit from the physical exams. If you receive the study vaccine, we do not know if it will protect you against an infection with seasonal influenza. People in the study will contribute information about a vaccine against influenza. This may eventually help Vietnam have access to a new influenza vaccine that is made locally.

#### What are my alternatives to participating in this research study?

You can choose not to join the study. You can get an approved seasonal influenza vaccine from a public or private health care center, however, you will have to pay for the vaccine.

#### What if I want to leave the study?

If you want to leave the study, please tell us. We will ask you to come for at least one more study visit just to check on your health.

Protocol No: IVACFLU-S-0203 674 Dated: 12 March 2018

IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

### Can I be taken off the study without my consent?

The researcher can take you off the study for the following reasons:

- You have trouble following the directions of the study staff
- We find out you have been enrolled in the study, but you should not have been enrolled.

In most cases, we will ask you to stay in the study and continue to be assessed by the study staff. If you are asked (or choose) to leave the study altogether, we will ask about your health before you leave.

#### Who will see my personal information in this research study?

We will keep all of your personal information confidential unless the law requires us to release it.

We keep your study forms locked. The following people/groups will be allowed to see your confidential information:

- People involved in doing the research
- People paying for the study
- People from groups that make sure the study is being done well
- People from health agencies that keep track of an illness you may have

We will take great care with information that can identify you, such as your name. Your name will be seen only by people who need to see it for their work on the study. For example, the study staff need to know your name. Also, study monitors will come to the site to check your consent form, which has your name. You will not be identified by name in publications of this study.

#### Will I be paid for my participation in the study?

- There are no costs to you for participation in this study.
- All physical exams will be free of cost to you.
- You will receive payment for your time and effort to be in this study. You will receive VND 450,000 for each
  study visit to the Health Center. Therefore, if you participate in all activities until the end of the study, you
  will receive a total amount of VND 1.800,000 for 3 site visits and a consent meeting.

#### How will I know the study results?

The researchers will provide a written summary of the study results to you. This could take a year or longer from when you started the study. Also, information about the study will be posted on a public website called clinicaltrials.gov. You can go to www.clinicaltrials.gov to view this or other studies. Your personal information is kept out of any study reports.

We will review any individual safety results with you as they are available during the study.

#### Who may I contact if I have additional questions?

The study staff can answer anything you do not understand.

You should immediately report to Dr. Phan Cong Hung or Dr. Hoang Anh Thang or other study staff if:

- You are having any injuries that you think may be caused by being in the study.
- You are in need of urgent medical care.

Protocol No: IVACFLU-S-0203 675 Dated: 12 March 2018

IVAC **PIHCMC** 

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

Dr. Phan Cong Hung (PI) Dr. Hoang Anh Thang Pasteur Institute in Ho Chi Minh City Pasteur Institute in Ho Chi Minh City 168 Pasteur Street, Ward 8, District 3, 168 Pasteur street, Ward 8, District 3, HCM City. HCM City. Cell phone: 093 528 8287 Cell phone: 090 322 4407

You may also contact the administrator of the research ethics committee with any questions or concerns about how you are being treated on this study or your rights as a study volunteer:

IRB of Pasteur Institute in Ho Chi Minh City

Phone: 08 3820 4013

Protocol No: IVACFLU-S-0203 676 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

| INFORMED CONSENT FORM FOR PHASE 2 | |
|---|---|
| I, | |
| attest that: | _ |
| • I have read and understand the information about the clinical study. | |
| • I was informed by the researchers about this study and enrollment procedures. | |
| <ul> <li>I have had a chance to ask questions about this study. My questions have been answere<br/>satisfaction.</li> </ul> | ed to my |
| • I have had enough time to think about my participation in this study. | |
| • I have been given this information sheet, which describes this study. | |
| <ul> <li>I understand that I have the right to refuse to join or withdraw from this study. I may w time and for any reason.</li> </ul> | vithdraw at any |
| <ul> <li>I am aware that study information could be published in medical journals or put on a p I am aware that this may be done to help medical science. I am aware that my identity masked.</li> </ul> | |
| • I know that if I request it, you will share my screening physical exam results with my r | regular doctor. |
| • I agree to participate in the Phase 2 part of the study. | |
| Full name of volunteer (PRINTED NAME): | |
| Signature of volunteer | |
| Time:: Date:/ | |
| Part to be completed by researcher I provided information to the volunteer on nature and purpose of this study and potential risks of participation in this study. | and benefits |
| Name and Signature of researcher:Date:/ | / |

(Dr. Phan Cong Hung or designee)
Protocol No: IVACFLU-S-0203 677 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### INFORMATION SHEET and INFORMED CONSENT FORMS

for "screening" and "participation in the research study" entitled:

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

| Sponsor: | Institute of Vaccines and Medical Biologicals (IVAC) |
|---|---|
| Funder: | PATH |
| Study implementer: | Pasteur Institute in Ho Chi Minh City (PIHCMC) |
| Full name of volunteer: | |
| Address: | |
| Participant screening code: | |
| Participant identification code (if recruited): | |

## CONSENT FOR PHASE 3 - BEN LUC DISTRICT HEALTH CENTER, LONG AN PROVICE

#### Introduction

You are invited to participate in a research study. This is a study of an experimental seasonal influenza vaccine called IVACFLU-S. We will call it the "study vaccine." The study vaccine has not been approved for sale in Vietnam. It can only be used in research. This vaccine was made in Vietnam by the Institute of Vaccines and Biologicals (IVAC), Ministry of Health.

The vaccine was used in a Phase 1 study of 60 people in the Hung Ha district health center. In the Phase 1 study, the vaccine did not cause any serious health problems. Most of the side effects were mild and did not last long. Now we will test the study vaccine in a larger study of about 888 people. If the study shows good results, IVAC will apply to license the vaccine in Vietnam. The study is a combination of a Phase 2 study and a Phase 3 study.

You are being asked to join the Phase 3 part of the study. About 252 people participated in the Phase 2 study in Ben Luc, Long An. Among them, 210 received the study vaccine. The vaccine was considered acceptable to be used in this Phase 3 part of the study with 636 people. We want to see if the study vaccine continues to be safe for people to use and if it is likely to protect people from the influenza virus.

The following groups are involved in the study: Institute of Vaccines and Biologicals, the Pasteur Institute, Ho Chi Minh City, Long An and Dong Nai Preventive Medicine Centers and the Ben Luc and Long Thanh district health centers. The study is funded through the US Biomedical Advanced Research and Development Authority (BARDA), PATH, an international nonprofit organization, and the World Health Organization (WHO).

This information sheet explains the study and your part in the study. Please take as much time as you need to read this information. Talk with friends, relatives and your doctor if you wish. You can ask us any questions you want.

----

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### What you should know about this study:

- 1. Being in this study is voluntary. You can refuse to join or leave any time after you have joined without penalty or loss of any rights you normally have.
- You may or may not benefit from being in the study. If you join, you may help other people in your community and Vietnam.
- 3. You will receive 1 injection of the study vaccine or a placebo. The placebo is sterile salt water. It will not prepare your body to fight influenza infections. You and the researcher will not know if you were given study vaccine or placebo until the end of the study. This is decided by chance. However, each person in the study has a greater chance of getting the study vaccine. For every person who gets the placebo, 5 people will get the study vaccine.
- 4. You will have physical examinations and 2 blood draws by a clinician.
- 5. If you are a woman, you will have a urine test for pregnancy. You must agree to use birth control until 3 weeks (21 days) after your injection. We will counsel you on reliable birth control methods (intrauterine devices, hormonal contraception, condoms or diaphragm with spermicide) and help you get it for free.
- In research of vaccines, there is a risk of harm. Please take your time to understand the risks. Ask any questions you have.
- 7. During the study, we will tell you of any new information about the vaccine. This new information might affect your decision to stay in the study. You may leave the study at any time.

#### What is a seasonal influenza vaccine?

The influenza virus is a very small germ that can be passed from person to person through the fluids in your nose, throat, mouth and lungs. Influenza virus can cause an illness in a person's airways that lasts about one week. Usually, the illness comes with a high fever, cough, headache and tiredness. Some influenza illnesses can be severe, especially among the young, old, and people with chronic diseases.

Most healthy people do not think of the flu as a serious illness. They may feel bad and miss some work. They are not aware that the flu causes many hospitalizations and early deaths for the young, old, and persons with chronic diseases. The flu has been linked with increases in miscarriage and heart attacks. In this study, we will teach you how to prevent getting the flu and giving it to others.

A vaccine is one of the best protections against influenza. There are different types of influenza and even those types may change slightly from one year to the next. Every year, the World Health Organization (WHO) receives information from countries all over the world about what types of influenza they are seeing in their country. The WHO uses this information to predict which types of influenza may be causing problems in the coming year. It tells the vaccine manufactures what type of vaccine they should make each year to help fight influenza infection. Companies can put together several types of influenza vaccines into one injection. This is called seasonal influenza vaccine.

#### What should I know about the study vaccine manufactured by IVAC?

IVAC made the influenza vaccine that will be used in this study. The WHO and PATH (an international nonprofit organization) have supported IVAC to make influenza vaccine. They helped IVAC meet the standards necessary to make a good product. The vaccine has had testing done to show that it was made correctly. The tests showed that study vaccine can be used in humans in vaccine studies. The vaccine cannot give you influenza.

#### What is the goal of this study?

This study's goal is to describe the safety and the body's responses to 1 injection of the study vaccine.

Protocol No: IVACFLU-S-0203 679 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### How is the vaccine given?

We will give the vaccine by injecting it into the muscle of your upper arm.

We will give it only once.

We divide the people in the study into 2 groups. One group (530 people) will get an injection of the study vaccine and the other group (106 people) will get an injection of a liquid that does not have the vaccine in it (the placebo). The placebo is sterile salt water. A computer decides which group you are in. Neither you nor the study doctor can decide or will know. In this study, people have a much greater chance of getting the study vaccine than getting the placebo. For every person who gets the placebo in the study, 5 will get the study vaccine.

#### How long will I be in this study?

If you join, you will be in the study for about 3 months after your injection. However, you will only need to come to the study site during the first 3 weeks.

#### What will happen during screening for this study?

If you agree to be in this study, we will do some things to see if you can join; this is called "screening". You will be provided information about the study and you need to sign this consent before we do any screening.

- 1. For screening:
  - A clinician will ask about your health history.
  - The clinician will do a physical exam. We will take your temperature, pulse, and blood pressure.
  - If you are a woman who is able to get pregnant, we will do a urine pregnancy test see if you are pregnant.
     Pregnant women cannot get the study products.
- 2. Women who could become pregnant must have already been using reliable birth control (intrauterine device, hormonal contraception, or condoms) to be in the study.

We will go over the results of screening with you. If we find you have a health issue, we will advise you on how to get proper treatment. Because we cannot tell ahead of time how many people who enter screening will qualify and want to join the study, we may have to exclude some people from the study, even if they qualify and want to join.

#### What will happen in this study?

If the questions and the physical exam show that you can be in the study, we will ask if you still would like to join. If you agree, you can have the study injection the same day as your screening visit. You can take a few more days to think about it, if you want. You can always change your mind if you do not want to be in the study. Nothing bad will happen if you decide not to join or leave after you have joined.

#### 1. Product injection:

- If the injection is given to you on a different day from the screening visit, we will again take your temperature, pulse and blood pressure and do a urine pregnancy test on women who can become pregnant. Pregnant women will not receive the injection.
- Before your first injection: The clinician will collect 5 mL (a teaspoon) of blood from a vein in your arm. This blood sample will be used to check to see if your body has reacted to the influenza virus in the past.
- We will give you your injection of study vaccine or placebo. The injection will be into a muscle in your upper arm.
- You will be asked to stay in the study clinic for at least 30 minutes. During this time, the study staff will check to see if you have any reactions to the injection.
- The study staff will show you how to complete a Diary Card. We want you to record any reaction or
  medical event and any medications you take on this form. Record each day for 7 days since the day of
  your injection.

IVACFLU-S-0203\_ICF\_Phase 3\_Ben Luc Version 4.0, dated 09/02/2017

Protocol No: IVACFLU-S-0203 680 Dated: 12 March 2018

IVAC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

- 2. The study staff will visit your home or call you one day after your injection and call you 4 days after your injection to check on your well-being and see if you are completing the Diary Card.
- 3. Seven (7) days after you are given the injection, you will return to the study clinic.
  - We will take your oral temperature, pulse, and blood pressure. A clinician will do a physical exam only if
    you report symptoms.
  - We will go over the Diary Card with you to make sure we understand what you wrote.
- 4. Over the next 2 weeks (14 days) you will have no clinic visits, but we want you to tell us if you have any health concerns. If needed, we will examine you or refer you to care.
- 5. Twenty-one (21) days after you are given the injection, you will return to the study clinic.
  - We will take your temperature, pulse, and blood pressure. The clinician will do a physical exam only
    if you report symptoms.
  - We will take 5 mL (a teaspoon) of blood from a vein in your arm to see how your body is reacting to the influenza vaccine or placebo.
  - If you are a women who could become pregnant, we will tell you that you no longer need to use birth
    control for the study.
- 6. Three months after your injection a member of the study staff will call you.
  - We will ask about health problems you told us were continuing at your last visit.
  - We will ask you about medications you told us you were still using at your last visit.
  - We will ask about any new, serious health problems that may have happened since we saw you last.
  - We will thank you for being in the study. This will end your study participation.
- 7. After the last person finishes the Phase 3 study, it will take about 6 months to know the results. When we know the results, we will send you a letter so that you know the study results, too.

#### In summary, if you join the study:

- You will visit the Study Clinic 3 times over about 3 weeks and one time for consent meeting.
- Women will provide a urine sample before their injection. We will use it for a pregnancy test. Women should be using reliable birth control for at least 3 weeks after their injection.
- You will receive only 1 injection of study vaccine or placebo.
- You will have 2 blood draws from a vein in your arm.
- You will be completing a Diary Card for 7 days since the date of the injection.
- We will visit your home or call you one day after the injection and call you 4 days after the injection to check on your well-being.
- We will contact you about 3 months after the injection to find out about your health
- During the study, we will tell you about new information or changes in the study that may affect your health or your willingness to continue.
- You will be informed about the study results and all exams related to your health.
- We will send you a letter with the study results, including what study product you received.

Almost all of the procedures we do in this study are like what happens when you have regular health care. The part of this study that is not standard treatment is when we give you the study vaccine or placebo.

What will happen to my blood samples?

IVACFLU-S-0203\_ICF\_Phase 3\_Ben Luc Version 4.0, dated 09/02/2017 IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

**Testing in the Study:** We will test blood samples to see if there is an immune response to the vaccine. Those who get the placebo will not have this immune response. Your samples will be sent to a laboratory in Italy for this testing. We will compare the responses of those who got the vaccine to those who got the placebo.

Quality Control by Pasteur Institute Laboratory during the Study: Also, we will use blood samples to help staff at Pasteur Institute Laboratories learn to conduct testing for influenza viruses. We will use a number in place of your name on the labels of the blood samples. The Pasteur Institute Lab will check its results against the results from the laboratory in Italy.

**Using Left-over Samples:** There may be blood samples left over after the study ends. If you agree, we want to continue to use these samples to help improve the quality of testing for influenza or influenza vaccines by Vietnam laboratories. The samples will have a number in place of your name. After 5 years, we will destroy any samples that remain. At the end of this form, we will ask you if you will allow this use of your left-over samples. You can say "no" and still be in this study. You can also say "yes" and change your mind later.

#### What are my responsibilities?

- Tell us if you have ever had a bad reaction to a vaccine or allergy to eggs, chicken or rubber.
- Inform us if you are pregnant or breast feeding.
- Come to the study visits and do your best to follow directions.
- Tell us if you have moved.
- Tell us if you do not like something about the study.
- Tell us if you want to leave the study.
- Tell your study doctor about any changes in your health that occur during the study as well as any changes in your medications during the study.
- While participating in this study, you may not take part in any other research project.

#### What harm could happen?

Sometimes bad things can happen in a study of a vaccine. Think about these when deciding if you want to join. Here is what we know that could happen during the study:

- Drawing blood can cause pain, redness, bruising, swelling, or infection. It is rare, but sometimes people faint
  when having blood taken.
- Receiving the injection of vaccine or placebo can cause pain, redness, swelling, hardness or infection where
  the needle was put in. Also the whole body may feel feverish or have muscle aches or nausea (feeling like you
  may throw up). In the earlier study of the vaccine, people report pain and tenderness the most. Most of the
  side effects were mild, meaning that people did not limit their activities because of the injection.
- It is very rare, but sometimes people have a serious allergic reaction to a vaccine. This can be life-threatening.
   We can provide emergency care, if needed.
- There may be harm, even serious harm that we do not know about yet.
- We do not know if the study vaccine is safe for use in pregnancy. That is why we ask women to agree to use reliable birth control during the study.
- We do our best to keep your study records and private information confidential. However, there is always a
  risk that someone who is not supposed to may see your information by accident. If this happens, we will tell
  you.
- To be in the study, you must not have had a flu vaccine in the past 6 months and you must wait until 3 weeks
  after your injection to have any licensed vaccines. Because of this, it is possible that you could get exposed to
  seasonal influenza and get the flu during the study. We will teach you ways to protect yourself and others
  from the flu.

Protocol No: IVACFLU-S-0203 682 Dated: 12 March 2018

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### What if I am injured?

If you have an injury and need help, contact Dr. Phan Cong Hung or Dr. Hoang Anh Thang to let him know what is happening. Their numbers are at the end of this form. Dr. Phan Cong Hung or Dr. Hoang Anh Thang can consult and help you get the care you need. The IVAC has arranged for the Ben Luc district hospital to provide you with free treatment for any injuries that happen during the study. The IVAC does not plan to pay any additional money to you unless directed by the Ministry of Health, which reviews research injuries.

#### What if I become pregnant?

We will test for pregnancy before you receive your injection. If you become pregnant and have received an injection on the study, we will ask you to stay in the study. Because you received a study product, we want to watch after your health. If the study ends and you are still pregnant, we will stay in touch with you to report on the outcome of the pregnancy and health of the baby.

#### What are the known benefits of participating in this research study?

There may not be any benefit to you personally. However, you may benefit from the physical exams. If you receive the study vaccine, we do not know if it will protect you against an infection with seasonal influenza. People in the study will contribute information about a vaccine against influenza. This may eventually help Vietnam have access to a new influenza vaccine that is made locally.

#### What are my alternatives to participating in this research study?

You can choose not to join the study. You can get an approved seasonal influenza vaccine from a public or private health care center, however, you will have to pay for the vaccine.

#### What if I want to leave the study?

If you want to leave the study, please tell us. We will ask you to come for at least one more study visit just to check on your health.

#### Can I be taken off the study without my consent?

The researcher can take you off the study for the following reasons:

- You have trouble following the directions of the study staff
  - We find out you have been enrolled in the study, but you should not have been enrolled.

In most cases, we will ask you to stay in the study and continue to be assessed by the study staff. If you are asked (or choose) to leave the study altogether, we will ask about your health before you leave.

#### Who will see my personal information in this research study?

We will keep all of your personal information confidential unless the law requires us to release it.

We keep your study forms locked. The following people/groups will be allowed to see your confidential information:

- People involved in doing the research
- People paying for the study
- People from groups that make sure the study is being done well
- People from health agencies that keep track of an illness you may have

We will take great care with information that can identify you, such as your name. Your name will be seen only by people who need to see it for their work on the study. For example, the study staff need to know your name. Also,

IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

study monitors will come to the site to check your consent form, which has your name. You will not be identified by name in publications of this study.

#### Will I be paid for my participation in the study?

- There are no costs to you for participation in this study.
- All physical exams will be free of cost to you.
- You will receive payment for your time and effort to be in this study. You will receive VND 450,000 for each study visit to the Health Center. Therefore, if you participate in all activities until the end of the study, you will receive a total amount of VND 1,800,000 for 3 site visits and a consent meeting.

#### How will I know the study results?

The researchers will provide a written summary of the study results to you. This could take a year or longer from when you started the study. Also, information about the study will be posted on a public website called clinicaltrials.gov. You can go to www.clinicaltrials.gov to view this or other studies. Your personal information is kept out of any study reports.

We will review any individual safety results with you as they are available during the study.

#### Who may I contact if I have additional questions?

The study staff can answer anything you do not understand.

You should immediately report to Dr. Phan Cong Hung or Dr. Hoang Anh Thang or other study staff if:

- You are having any injuries that you think may be caused by being in the study.
- You are in need of urgent medical care.

Dr. Phan Cong Hung (PI)
Pasteur Institute in Ho Chi Minh City
168 Pasteur Street, Ward 8, District 3,
HCM City.
Cell phone: 093 528 8287

Dr. Hoang Anh Thang
Pasteur Institute in Ho Chi Minh City
168 Pasteur Street, Ward 8, District 3,
HCM City.
Cell phone: 090 322 4407

You may also contact the administrator of the research ethics committee with any questions or concerns about how you are being treated on this study or your rights as a study volunteer:

IRB of Pasteur Institute - Ho Chi Minh City

Phone: 08 3820 4013

Protocol No: IVACFLU-S-0203 684 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

### INFORMED CONSENT FORM FOR PHASE 3 - BEN LUC DISTRICT HEALTH CENTER, LONG AN PROVINCE

| I, |
|--------------|
| attest that: |

- I have read and understand the information about the clinical study.
- I was informed by the researchers about this study and enrollment procedures.
- I have had a chance to ask questions about this study. My questions have been answered to my satisfaction.
- I have had enough time to think about my participation in this study.
- I have been given this information sheet, which describes this study.
- I understand that I have the right to refuse to join or withdraw from this study. I may withdraw at any time and for any reason.
- I am aware that study information could be published in medical journals or put on a public website.
   I am aware that this may be done to help medical science. I am aware that my identity will be masked.
- I know that if I request it, you will share my screening physical exam results with my regular doctor.
- I agree to participate in the Phase 3 part of the study.
- Using left-over samples: Will you allow the use of any left over blood samples for 5 years to help laboratories in Vietnam improve their ability to test for influenza or influenza vaccines? (You can say "no" and still be in this vaccine study.) Please sign either box below.

| Yes | Signature: |
|-----|------------|
| No | Signature: |

| Full name of volunteer | (PRINTED NAME): |
|------------------------|-----------------|
| Signature of volunteer | |
| Time:: | Date:// |

#### Part to be completed by researcher

I provided information to the volunteer on nature and purpose of this study and potential risks and benefits of participation in this study.

Protocol No: IVACFLU-S-0203 685 Dated: 12 March 2018

| IVAC | PIHCMC |
|------------------------------------------------|---------|
| Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06 | |
| Name and Signature of researcher: | Date:// |
| (Dr. Phan Cong Hung or designee) | |

Protocol No: IVACFLU-S-0203 686 Dated: 12 March 2018

IVAC PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### INFORMATION SHEET and INFORMED CONSENT FORMS

for "screening" and "participation in the research study" entitled:

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

| Sponsor: | Institute of Vaccines and Medical Biologicals (IVAC) |
|---|---|
| Funder: | PATH |
| Study implementer: | Pasteur Institute in Ho Chi Minh City (PIHCMC) |
| Full name of volunteer: | |
| Address: | |
| Participant screening code: | |
| Participant identification code (if recruited): | |

## CONSENT FOR PHASE 3 - LONG THANH DISTRICT HEALTH CENTER, DONG NAI PROVINCE

#### Introduction

You are invited to participate in a research study. This is a study of an experimental seasonal influenza vaccine called IVACFLU-S. We will call it the "study vaccine." The study vaccine has not been approved for sale in Vietnam. It can only be used in research. This vaccine was made in Vietnam by the Institute of Vaccines and Biologicals (IVAC), Ministry of Health.

The vaccine was used in a Phase 1 study of 60 people in the Hung Ha district health center. In the Phase 1 study, the vaccine did not cause any serious health problems. Most of the side effects were mild and did not last long. Now we will test the study vaccine in a larger study of about 888 people. If the study shows good results, IVAC will apply to license the vaccine in Vietnam. The study is a combination of a Phase 2 study and a Phase 3 study.

You are being asked to join the Phase 3 part of the study. About 252 people participated in the Phase 2 study in Ben Luc, Long An. Among them, 210 received the study vaccine. The vaccine was considered acceptable to be used in this Phase 3 part of the study with 636 people. We want to see if the study vaccine continues to be safe for people to use and if it is likely to protect people from the influenza virus. You will not have any blood drawn in this study.

The following groups are involved in the study: Institute of Vaccines and Biologicals, the Pasteur Institute, Ho Chi Minh City, Long An and Dong Nai Preventive Medicine Centers and the Ben Luc and Long Thanh district health centers. The study is funded through the US Biomedical Advanced Research and Development Authority (BARDA), PATH, an international nonprofit organization, and the World Health Organization (WHO).

This information sheet explains the study and your part in the study. Please take as much time as you need to read this information. Talk with friends, relatives and your doctor if you wish. You can ask us any questions you want.

----

Protocol No: IVACFLU-S-0203 687 Dated: 12 March 2018

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### What you should know about this study:

- 1. Being in this study is voluntary. You can refuse to join or leave any time after you have joined without penalty or loss of any rights you normally have.
- You may or may not benefit from being in the study. If you join, you may help other people in your community and Vietnam.
- 3. You will receive 1 injection of the study vaccine or a placebo. The placebo is sterile salt water. It will not prepare your body to fight influenza infections. You and the researcher will not know if you were given study vaccine or placebo until the end of the study. This is decided by chance. However, each person in the study has a greater chance of getting the study vaccine. For every person who gets the placebo, 5 people will get the study vaccine.
- 4. You will have physical examinations.
- 5. If you are a woman, you will have a urine test for pregnancy. You must agree to use birth control until 3 weeks (21 days) after your injection. We will counsel you on reliable birth control methods (intrauterine devices, hormonal contraception, condoms or diaphragm with spermicide) and help you get it for free.
- In research of vaccines, there is a risk of harm. Please take your time to understand the risks. Ask any questions you have.
- 7. During the study, we will tell you of any new information about the vaccine. This new information might affect your decision to stay in the study. You may leave the study at any time.

#### What is a seasonal influenza vaccine?

The influenza virus is a very small germ that can be passed from person to person through the fluids in your nose, throat, mouth and lungs. Influenza virus can cause an illness in a person's airways that lasts about one week. Usually, the illness comes with a high fever, cough, headache and tiredness. Some influenza illnesses can be severe, especially among the young, old, and people with chronic diseases.

Most healthy people do not think of the flu as a serious illness. They may feel bad and miss some work. They are not aware that the flu causes many hospitalizations and early deaths for the young, old, and persons with chronic diseases. The flu has been linked with increases in miscarriage and heart attacks. In this study, we will teach you how to prevent getting the flu and giving it to others.

A vaccine is one of the best protections against influenza. There are different types of influenza and even those types may change slightly from one year to the next. Every year, the World Health Organization (WHO) receives information from countries all over the world about what types of influenza they are seeing in their country. The WHO uses this information to predict which types of influenza may be causing problems in the coming year. It tells the vaccine manufactures what type of vaccine they should make each year to help fight influenza infection. Companies can put together several types of influenza vaccines into one injection. This is called seasonal influenza vaccine.

#### What should I know about the study vaccine manufactured by IVAC?

IVAC made the influenza vaccine that will be used in this study. The WHO and PATH (an international nonprofit organization) have supported IVAC to make influenza vaccine. They helped IVAC meet the standards necessary to make a good product. The vaccine has had testing done to show that it was made correctly. The tests showed that study vaccine can be used in humans in vaccine studies. The vaccine cannot give you influenza.

#### What is the goal of this study?

This study's goal is to describe the safety and the body's responses to 1 injection of the study vaccine.

Protocol No: IVACFLU-S-0203 688 Dated: 12 March 2018

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### How is the vaccine given?

We will give the vaccine by injecting it into the muscle of your upper arm.

We will give it only once.

We divide the people in the study into 2 groups. One group (530 people) will get an injection of the study vaccine and the other group (106 people) will get an injection of a liquid that does not have the vaccine in it (the placebo). The placebo is sterile salt water. A computer decides which group you are in. Neither you nor the study doctor can decide or will know. In this study, people have a much greater chance of getting the study vaccine than getting the placebo. For every person who gets the placebo in the study, 5 will get the study vaccine.

#### How long will I be in this study?

If you join, you will be in the study for about 3 months after your injection. However, you will only need to come to the study site during the first 3 weeks.

#### What will happen during screening for this study?

If you agree to be in this study, we will do some things to see if you can join; this is called "screening". You will be provided information about the study and you need to sign this consent before we do any screening.

- 1. For screening:
  - A clinician will ask about your health history.
  - The clinician will do a physical exam. We will take your temperature, pulse, and blood pressure.
  - If you are a woman who is able to get pregnant, we will do a urine pregnancy test see if you are pregnant. Pregnant women cannot get the study products.
- 2. Women who could become pregnant must have already been using reliable birth control (intrauterine device, hormonal contraception, or condoms) to be in the study.

We will go over the results of screening with you. If we find you have a health issue, we will advise you on how to get proper treatment. Because we cannot tell ahead of time how many people who enter screening will qualify and want to join the study, we may have to exclude some people from the study, even if they qualify and want to join.

#### What will happen in this study?

If the questions and the physical exam show that you can be in the study, we will ask if you still would like to join. If you agree, you can have the study injection the same day as your screening visit. You can take a few more days to think about it, if you want. You can always change your mind if you do not want to be in the study. Nothing bad will happen if you decide not to join or leave after you have joined.

#### 1. Product injection:

- If the injection is given to you on a different day from the screening visit, we will again take your temperature, pulse and blood pressure and do a urine pregnancy test on women who can become pregnant. Pregnant women will not receive the injection.
- We will give you your injection of study vaccine or placebo. The injection will be into a muscle in your upper arm.
- You will be asked to stay in the study clinic for at least 30 minutes. During this time, the study staff will
  check to see if you have any reactions to the injection.
- The study staff will show you how to complete a Diary Card. We want you to record any reaction or
  medical event and any medications you take on this form. Record each day for 7 days since the day of
  your injection.

Protocol No: IVACFLU-S-0203 689 Dated: 12 March 2018

#### IVAC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

- 2. The study staff will visit your home or call you one day after your injection and call you 4 days after your injection to check on your well-being and see if you are completing the Diary Card.
- 3. Seven (7) days after you are given the injection, you will return to the study clinic.
  - We will take your oral temperature, pulse, and blood pressure. A clinician will do a physical exam only if
    you report symptoms.
  - We will go over the Diary Card with you to make sure we understand what you wrote.
- 4. Over the next 2 weeks (14 days) you will have no clinic visits, but we want you to tell us if you have any health concerns. If needed, we will examine you or refer you to care.
- 5. Twenty-one (21) days after you are given the injection, you will return to the study clinic.
  - We will take your temperature, pulse, and blood pressure. The clinician will do a physical exam only
    if you report symptoms.
  - If you are a women who could become pregnant, we will tell you that you no longer need to use birth
    control for the study.
- 6. Three months after your injection a member of the study staff will call you.
  - We will ask about health problems you told us were continuing at your last visit.
  - We will ask you about medications you told us you were still using at your last visit.
  - We will ask about any new, serious health problems that may have happened since we saw you last.
  - We will thank you for being in the study. This will end your study participation.
- 7. After the last person finishes the Phase 3 study, it will take about 6 months to know the results. When we know the results, we will send you a letter so that you know the study results, too.

#### In summary, if you join the study:

- You will visit the Study Clinic 3 times over about 3 weeks and one time for consent meeting.
- Women will provide a urine sample before their injection. We will use it for a pregnancy test. Women should
  be using reliable birth control for at least 3 weeks after their injection.
- You will receive only 1 injection of study vaccine or placebo.
- You will be completing a Diary Card for 7 days since the date of the injection.
- We will visit your home or call you one day after the injection and call you 4 days after the injection to check on your well-being.
- We will contact you about 3 months after the injection to find out about your health
- During the study, we will tell you about new information or changes in the study that may affect your health or your willingness to continue.
- You will be informed about the study results and all exams related to your health.
- We will send you a letter with the study results, including what study product you received.

Almost all of the procedures we do in this study are like what happens when you have regular health care. The part of this study that is not standard treatment is when we give you the study vaccine or placebo.

#### What are my responsibilities?

- Tell us if you have ever had a bad reaction to a vaccine or allergy to eggs, chicken or rubber.
- Inform us if you are pregnant or breast feeding.
- Come to the study visits and do your best to follow directions.

Protocol No: IVACFLU-S-0203 690 Dated: 12 March 2018

IVAC PIHCMC

#### Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

- Tell us if you have moved.
- Tell us if you do not like something about the study.
- Tell us if you want to leave the study.
- Tell your study doctor about any changes in your health that occur during the study as well as any changes in your medications during the study.
- While participating in this study, you may not take part in any other research project.

#### What harm could happen?

Sometimes bad things can happen in a study of a vaccine. Think about these when deciding if you want to join. Here is what we know that could happen during the study:

- Receiving the injection of vaccine or placebo can cause pain, redness, swelling, hardness or infection where
  the needle was put in. Also the whole body may feel feverish or have muscle aches or nausea (feeling like you
  may throw up). In the earlier study of the vaccine, people report pain and tenderness the most. Most of the
  side effects were mild, meaning that people did not limit their activities because of the injection.
- It is very rare, but sometimes people have a serious allergic reaction to a vaccine. This can be life-threatening.
   We can provide emergency care, if needed.
- There may be harm, even serious harm that we do not know about yet.
- We do not know if the study vaccine is safe for use in pregnancy. That is why we ask women to agree to use reliable birth control during the study.
- We do our best to keep your study records and private information confidential. However, there is always a
  risk that someone who is not supposed to may see your information by accident. If this happens, we will tell
  you.
- To be in the study, you must not have had a flu vaccine in the past 6 months and you must wait until 3 weeks
  after your injection to have any licensed vaccines. Because of this, it is possible that you could get exposed to
  seasonal influenza and get the flu during the study. We will teach you ways to protect yourself and others
  from the flu.

#### What if I am injured?

If you have an injury and need help, contact Dr. Phan Cong Hung or Dr. Hoang Anh Thang to let him know what is happening. Their numbers are at the end of this form. Dr. Phan Cong Hung or Dr. Hoang Anh Thang can consult and help you get the care you need. The IVAC has arranged for the Long Thanh district hospital to provide you with free treatment for any injuries that happen during the study. The IVAC does not plan to pay any additional money to you unless directed by the Ministry of Health, which reviews research injuries.

#### What if I become pregnant?

We will test for pregnancy before you receive your injection. If you become pregnant and have received an injection on the study, we will ask you to stay in the study. Because you received a study product, we want to watch after your health. If the study ends and you are still pregnant, we will stay in touch with you to report on the outcome of the pregnancy and health of the baby.

#### What are the known benefits of participating in this research study?

There may not be any benefit to you personally. However, you may benefit from the physical exams. If you receive the study vaccine, we do not know if it will protect you against an infection with seasonal influenza. People in the study will contribute information about a vaccine against influenza. This may eventually help Vietnam have access to a new influenza vaccine that is made locally.

Protocol No: IVACFLU-S-0203 691 Dated: 12 March 2018

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

#### What are my alternatives to participating in this research study?

You can choose not to join the study. You can get an approved seasonal influenza vaccine from a public or private health care center, however, you will have to pay for the vaccine.

#### What if I want to leave the study?

If you want to leave the study, please tell us. We will ask you to come for at least one more study visit just to check on your health.

#### Can I be taken off the study without my consent?

The researcher can take you off the study for the following reasons:

- You have trouble following the directions of the study staff
- We find out you have been enrolled in the study, but you should not have been enrolled.

In most cases, we will ask you to stay in the study and continue to be assessed by the study staff. If you are asked (or choose) to leave the study altogether, we will ask about your health before you leave.

#### Who will see my personal information in this research study?

We will keep all of your personal information confidential unless the law requires us to release it.

We keep your study forms locked. The following people/groups will be allowed to see your confidential information:

- People involved in doing the research
- People paying for the study
- People from groups that make sure the study is being done well
- People from health agencies that keep track of an illness you may have

We will take great care with information that can identify you, such as your name. Your name will be seen only by people who need to see it for their work on the study. For example, the study staff need to know your name. Also, study monitors will come to the site to check your consent form, which has your name. You will not be identified by name in publications of this study.

#### Will I be paid for my participation in the study?

- There are no costs to you for participation in this study.
- All physical exams will be free of cost to you.
- You will receive payment for your time and effort to be in this study. You will receive VND 450,000 for each study visit to the Health Center. Therefore, if you participate in all activities until the end of the study, you will receive a total amount of VND 1,800,000 for 3 site visits and a consent meeting.

#### How will I know the study results?

The researchers will provide a written summary of the study results to you. This could take a year or longer from when you started the study. Also, information about the study will be posted on a public website called clinicaltrials.gov. You can go to www.clinicaltrials.gov to view this or other studies. Your personal information is kept out of any study reports.

We will review any individual safety results with you as they are available during the study.

#### Who may I contact if I have additional questions?

The study staff can answer anything you do not understand.

----

Protocol No: IVACFLU-S-0203 692 Dated: 12 March 2018

<u>IVAC</u> PIHCMC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

You should immediately report to Dr. Phan Cong Hung or Dr. Hoang Anh Thang or other study staff if:

- You are having any injuries that you think may be caused by being in the study.
- You are in need of urgent medical care.

Dr. Phan Cong Hung (PI)
Pasteur Institute in Ho Chi Minh City
168 Pasteur Street, Ward 8, District 3,
HCM City.
Cell phone: 093 528 8287

Dr. Hoang Anh Thang
Pasteur Institute in Ho Chi Minh City
168 Pasteur Street, Ward 8, District 3,
HCM City.
Cell phone: 093 528 8287

Cell phone: 090 322 4407

You may also contact the administrator of the research ethics committee with any questions or concerns about how you are being treated on this study or your rights as a study volunteer:

IRB of Pasteur Institute - Ho Chi Minh City

Phone: 08 3820 4013

Protocol No: IVACFLU-S-0203 693 Dated: 12 March 2018

IVAC

Protocol: IVACFLU-S-0203. MOH Code: VX.2016.06

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

## INFORMED CONSENT FORM FOR PHASE 3 - LONG THANH DISTRICT HEALTH CENTER, DONG NAI PROVINCE

| I, |
|--------------|
| attest that: |

- I have read and understand the information about the clinical study.
- I was informed by the researchers about this study and enrollment procedures.
- I have had a chance to ask questions about this study. My questions have been answered to my satisfaction.
- I have had enough time to think about my participation in this study.
- I have been given this information sheet, which describes this study.
- I understand that I have the right to refuse to join or withdraw from this study. I may withdraw at any time and for any reason.
- I am aware that study information could be published in medical journals or put on a public website.
   I am aware that this may be done to help medical science. I am aware that my identity will be masked.
- I know that if I request it, you will share my screening physical exam results with my regular doctor.
- I agree to participate in the Phase 3 part of the study.

| | <del></del> |
|---|---|
| Signature of volunteer | |
| Time: : Date:// | |
| Part to be completed by researcher I provided information to the volunteer on nature and purpose of this study and p of participation in this study. | potential risks and benefits |
| Name and Signature of researcher: | Date:// |

Protocol No: IVACFLU-S-0203 694 Dated: 12 March 2018

## 16.1.4 List and description of Investigators and other important participants in the study

Principal Investigators at study centers that consented at least 1 subject are listed below. Curriculum vitae for the Principal Investigators are available upon request.

| Study Center | Principal Investigator | Investigator Address |
|---|---|---|
| 201<br>(District Health<br>Center of Ben Luc<br>district, Long An<br>Province) | PI: Dr. Phan Cong Hung<br>Co-PI: Dr. Nguyen Trong Toan | Pasteur Institute in Ho Chi Minh City<br>167 Pasteur, Ward 8, District 3 |
| 203<br>(District Health<br>Center of Long<br>Thanh district, Dong<br>Nai Province) | PI: Dr. Phan Cong Hung<br>Co-PI: Dr. Nguyen Trong Toan | Ho Chi Minh City<br>Vietnam |

Protocol No: IVACFLU-S-0203 695 Dated: 12 March 2018

## 16.1.5 Signatures of principal investigator(s) and sponsor's responsible medical officer

The signatures of Sponsor's representative and Principal Investigator are available on Title Page (Page 2) of this CSR.

Protocol No: IVACFLU-S-0203 696 Dated: 12 March 2018

# 16.1.6 Listing of subjects receiving test drug(s)/investigational product(s) from specific batches

| Products | Lot | Manufacturing<br>Date | Expiry<br>Date | Manufacturer |
|---|---|---|---|---|
| IVACFLU-S | 004-01-16 | 29/11/16 | 05/12/17 | IVAC |
| 15 mcg | | | | |
| PLACEBO | 007P-01-16 | 02/12/16 | 05/12/17 | IVAC |

IVACELU-S Version 1.0

Protocol No. IVACELU S 0202 607

Protocol No: IVACFLU-S-0203 697 Dated: 12 March 2018

#### 16.1.7 Randomization scheme and codes

#### **Document**

IVACFLU-S-0203 Subject Randomization

IVACFLU-S-0203 Randomization Specification Document Version 2, Dated 31 March 2017

Protocol No: IVACFLU-S-0203 698 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA001 (A001) | IVACFLU-S | IVACFLU-S | 20Mar2017:08:53:00 | A001 | Y |
| IVACFLU-S-0203-201-SA002 (A003) | PLACEBO | PLACEBO | 20Mar2017:08:43:00 | A003 | Y |
| IVACFLU-S-0203-201-SA003 (A004) | IVACFLU-S | IVACFLU-S | 20Mar2017:08:47:00 | A004 | Y |
| IVACFLU-S-0203-201-SA004 (A005) | IVACFLU-S | IVACFLU-S | 20Mar2017:08:59:00 | A005 | Y |
| IVACFLU-S-0203-201-SA005 (A002) | IVACFLU-S | IVACFLU-S | 20Mar2017:08:39:00 | A002 | Y |
| IVACFLU-S-0203-201-SA006() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA007() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA008 (A006) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:05:00 | A006 | Y |
| IVACFLU-S-0203-201-SA009 (A007) | PLACEBO | PLACEBO | 20Mar2017:09:07:00 | A007 | Y |
| IVACFLU-S-0203-201-SA010 (A010) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:20:00 | A010 | Y |
| IVACFLU-S-0203-201-SA011 (A011) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:24:00 | A011 | Y |
| IVACFLU-S-0203-201-SA012 (A009) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:15:00 | A009 | Y |
| IVACFLU-S-0203-201-SA013 (A012) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:36:00 | A012 | Y |
| IVACFLU-S-0203-201-SA014 (A013) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:41:00 | A013 | Y |
| IVACFLU-S-0203-201-SA015 (A019) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:18:00 | A019 | Y |
| IVACFLU-S-0203-201-SA016 (A008) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:11:00 | A008 | Y |
| IVACFLU-S-0203-201-SA017 (A015) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:50:00 | A015 | Y |
| IVACFLU-S-0203-201-SA018 (A018) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:16:00 | A018 | Y |
| IVACFLU-S-0203-201-SA019 (A017) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:55:00 | A017 | Y |
| IVACFLU-S-0203-201-SA020 (A016) | PLACEBO | PLACEBO | 20Mar2017:09:53:00 | A016 | Y |
| IVACFLU-S-0203-201-SA021 (A014) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:45:00 | A014 | Y |
| IVACFLU-S-0203-201-SA022 (A020) | IVACFLU-S | IVACFLU-S | 20Mar2017:11:51:00 | A020 | Y |
| IVACFLU-S-0203-201-SA023 (A021) | PLACEBO | PLACEBO | 22Mar2017:08:32:00 | A021 | Y |
| IVACFLU-S-0203-201-SA024 (A022) | IVACFLU-S | IVACFLU-S | 22Mar2017:08:46:00 | A022 | Y |
| IVACFLU-S-0203-201-SA025 (A023) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:07:00 | A023 | Y |
| IVACFLU-S-0203-201-SA026 (A024) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:10:00 | A024 | Y |
| IVACFLU-S-0203-201-SA027 (A026) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:00:00 | A026 | Y |
| IVACFLU-S-0203-201-SA028 (A025) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:55:00 | A025 | Y |
| IVACFLU-S-0203-201-SA029 (A029) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:18:00 | A029 | Y |
| IVACFLU-S-0203-201-SA030 (A027) | PLACEBO | PLACEBO | 22Mar2017:11:06:00 | A027 | Y |
| IVACFLU-S-0203-201-SA031 (A030) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:20:00 | A030 | Y |
| IVACFLU-S-0203-201-SA032 (A031) | PLACEBO | PLACEBO | 22Mar2017:11:22:00 | A031 | Y |
| IVACFLU-S-0203-201-SA033 (A032) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:24:00 | A032 | Y |
| IVACFLU-S-0203-201-SA034 (A033) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:26:00 | A033 | Y |

Protocol No: IVACFLU-S-0203 699 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA035 (A038) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:36:00 | A038 | Y |
| IVACFLU-S-0203-201-SA036 (A037) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:34:00 | A037 | Y |
| IVACFLU-S-0203-201-SA037 (A036) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:32:00 | A036 | Y |
| IVACFLU-S-0203-201-SA038 (A035) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:29:00 | A035 | Y |
| IVACFLU-S-0203-201-SA039() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA040 (A034) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:27:00 | A034 | Y |
| IVACFLU-S-0203-201-SA041 (A028) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:16:00 | A028 | Y |
| IVACFLU-S-0203-201-SA042 (A040) | PLACEBO | PLACEBO | 22Mar2017:12:00:00 | A040 | Y |
| IVACFLU-S-0203-201-SA043 (A039) | IVACFLU-S | IVACFLU-S | 22Mar2017:11:38:00 | A039 | Y |
| IVACFLU-S-0203-201-SA044 (A041) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:19:00 | A041 | Y |
| IVACFLU-S-0203-201-SA045 (A042) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:21:00 | A042 | Y |
| IVACFLU-S-0203-201-SA046 (A044) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:40:00 | A044 | Y |
| IVACFLU-S-0203-201-SA047 (A043) | PLACEBO | PLACEBO | 23Mar2017:08:38:00 | A043 | Y |
| IVACFLU-S-0203-201-SA048 (A045) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:42:00 | A045 | Y |
| IVACFLU-S-0203-201-SA049() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA050 (A047) | IVACFLU-S | IVACFLU-S | 23Mar2017:09:57:00 | A047 | Y |
| IVACFLU-S-0203-201-SA051 (A046) | IVACFLU-S | IVACFLU-S | 23Mar2017:09:53:00 | A046 | Y |
| IVACFLU-S-0203-201-SA052 (A050) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:53:00 | A050 | Y |
| IVACFLU-S-0203-201-SA053 (A053) | PLACEBO | PLACEBO | 23Mar2017:11:02:00 | A053 | Y |
| IVACFLU-S-0203-201-SA054 (A048) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:42:00 | A048 | Y |
| IVACFLU-S-0203-201-SA055 (A056) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:16:00 | A056 | Y |
| IVACFLU-S-0203-201-SA056 (A051) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:55:00 | A051 | Y |
| IVACFLU-S-0203-201-SA057 (A049) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:44:00 | A049 | Y |
| IVACFLU-S-0203-201-SA058 (A057) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:19:00 | A057 | Y |
| IVACFLU-S-0203-201-SA059 (A052) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:00:00 | A052 | Y |
| IVACFLU-S-0203-201-SA060() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA061 (A055) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:06:00 | A055 | Y |
| IVACFLU-S-0203-201-SA062 (A058) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:32:00 | A058 | Y |
| IVACFLU-S-0203-201-SA063() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA064() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA065 (A054) | IVACFLU-S | IVACFLU-S | 23Mar2017:11:04:00 | A054 | Y |
| IVACFLU-S-0203-201-SA066 (A061) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:01:00 | A061 | Y |
| IVACFLU-S-0203-201-SA067 (A062) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:05:00 | A062 | Y |
| IVACFLU-S-0203-201-SA068 (A060) | PLACEBO | PLACEBO | 23Mar2017:13:57:00 | A060 | Y |
| IVACFLU-S-0203-201-SA069 (A059) | IVACFLU-S | IVACFLU-S | 23Mar2017:13:55:00 | A059 | Y |
| IVACFLU-S-0203-201-SA070 (A066) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:15:00 | A066 | Y |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 700 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA071 (A072) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:39:00 | A072 | Y |
| IVACFLU-S-0203-201-SA072 (A076) | PLACEBO | PLACEBO | 23Mar2017:15:36:00 | A076 | Y |
| IVACFLU-S-0203-201-SA073 (A077) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:41:00 | A077 | Y |
| IVACFLU-S-0203-201-SA074 (A063) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:08:00 | A063 | Y |
| IVACFLU-S-0203-201-SA075 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA076 (A064) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:10:00 | A064 | Y |
| IVACFLU-S-0203-201-SA077 (A068) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:21:00 | A068 | Y |
| IVACFLU-S-0203-201-SA078 (A069) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:26:00 | A069 | Y |
| IVACFLU-S-0203-201-SA079 (A065) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:13:00 | A065 | Y |
| IVACFLU-S-0203-201-SA080 (A071) | PLACEBO | PLACEBO | 23Mar2017:14:37:00 | A071 | Y |
| IVACFLU-S-0203-201-SA081 (A070) | PLACEBO | PLACEBO | 23Mar2017:14:30:00 | A070 | Y |
| IVACFLU-S-0203-201-SA082 (A067) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:17:00 | A067 | Y |
| IVACFLU-S-0203-201-SA083 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA084 (A073) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:43:00 | A073 | Y |
| IVACFLU-S-0203-201-SA085 (A075) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:01:00 | A075 | Y |
| IVACFLU-S-0203-201-SA086 (A074) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:45:00 | A074 | Y |
| IVACFLU-S-0203-201-SA087() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA088 (A079) | PLACEBO | PLACEBO | 24Mar2017:08:12:00 | A079 | Y |
| IVACFLU-S-0203-201-SA089 (A080) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:19:00 | A080 | Y |
| IVACFLU-S-0203-201-SA090 (A078) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:04:00 | A078 | Y |
| IVACFLU-S-0203-201-SA091 (A081) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:58:00 | A081 | Y |
| IVACFLU-S-0203-201-SA092() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA093 (A082) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:59:00 | A082 | Y |
| IVACFLU-S-0203-201-SA094 (A083) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:14:00 | A083 | Y |
| IVACFLU-S-0203-201-SA095 (A092) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:25:00 | A092 | Y |
| IVACFLU-S-0203-201-SA096 (A085) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:29:00 | A085 | Y |
| IVACFLU-S-0203-201-SA097 (A086) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:32:00 | A086 | Y |
| IVACFLU-S-0203-201-SA098 (A084) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:27:00 | A084 | Y |
| IVACFLU-S-0203-201-SA099 (A089) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:08:00 | A089 | Y |
| IVACFLU-S-0203-201-SA100 (A088) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:42:00 | A088 | Y |
| IVACFLU-S-0203-201-SA101() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA102 (A090) | PLACEBO | PLACEBO | 24Mar2017:10:12:00 | A090 | Y |
| IVACFLU-S-0203-201-SA103 (A091) | PLACEBO | PLACEBO | 24Mar2017:10:16:00 | A091 | Y |
| IVACFLU-S-0203-201-SA104 (A087) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:36:00 | A087 | Y |
| IVACFLU-S-0203-201-SA105() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA106 (A094) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:52:00 | A094 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA107 (A093) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:37:00 | A093 | Y |
| IVACFLU-S-0203-201-SA108 (A095) | IVACFLU-S | IVACFLU-S | 24Mar2017:11:05:00 | A095 | Y |
| IVACFLU-S-0203-201-SA109 (A098) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:02:00 | A098 | Y |
| IVACFLU-S-0203-201-SA110 (A097) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:00:00 | A097 | Y |
| IVACFLU-S-0203-201-SA111 (A096) | IVACFLU-S | IVACFLU-S | 24Mar2017:13:54:00 | A096 | Y |
| IVACFLU-S-0203-201-SA112() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA113 (A105) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:34:00 | A105 | Y |
| IVACFLU-S-0203-201-SA114 (A104) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:31:00 | A104 | Y |
| IVACFLU-S-0203-201-SA115 (A103) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:27:00 | A103 | Y |
| IVACFLU-S-0203-201-SA116 (A114) | PLACEBO | PLACEBO | 24Mar2017:14:59:00 | A114 | Y |
| IVACFLU-S-0203-201-SA117 (A102) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:25:00 | A102 | Y |
| IVACFLU-S-0203-201-SA118 (A099) | PLACEBO | PLACEBO | 24Mar2017:14:12:00 | A099 | Y |
| IVACFLU-S-0203-201-SA119 (A100) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:15:00 | A100 | Y |
| IVACFLU-S-0203-201-SA120 (A101) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:23:00 | A101 | Y |
| IVACFLU-S-0203-201-SA121 (A108) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:44:00 | A108 | Y |
| IVACFLU-S-0203-201-SA122 (A115) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:03:00 | A115 | Y |
| IVACFLU-S-0203-201-SA123 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA124 (A107) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:42:00 | A107 | Y |
| IVACFLU-S-0203-201-SA125 (A106) | PLACEBO | PLACEBO | 24Mar2017:14:40:00 | A106 | Y |
| IVACFLU-S-0203-201-SA126 (A109) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:46:00 | A109 | Y |
| IVACFLU-S-0203-201-SA127 (A110) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:50:00 | A110 | Y |
| IVACFLU-S-0203-201-SA128() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA129 (A111) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:52:00 | A111 | Y |
| IVACFLU-S-0203-201-SA130 (A113) | PLACEBO | PLACEBO | 24Mar2017:14:56:00 | A113 | Y |
| IVACFLU-S-0203-201-SA131 (A112) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:54:00 | A112 | Y |
| IVACFLU-S-0203-201-SA132 (A116) | IVACFLU-S | IVACFLU-S | 24Mar2017:16:40:00 | A116 | Y |
| IVACFLU-S-0203-201-SA133 (A122) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:08:00 | A122 | Y |
| IVACFLU-S-0203-201-SA134 (A117) | IVACFLU-S | IVACFLU-S | 26Mar2017:13:53:00 | A117 | Y |
| IVACFLU-S-0203-201-SA135 (A118) | IVACFLU-S | IVACFLU-S | 26Mar2017:13:55:00 | A118 | Y |
| IVACFLU-S-0203-201-SA136 (A120) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:02:00 | A120 | Y |
| IVACFLU-S-0203-201-SA137 (A119) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:00:00 | A119 | Y |
| IVACFLU-S-0203-201-SA138 (A121) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:04:00 | A121 | Y |
| IVACFLU-S-0203-201-SA139 (A123) | PLACEBO | PLACEBO | 26Mar2017:14:12:00 | A123 | Y |
| IVACFLU-S-0203-201-SA140 (A124) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:14:00 | A124 | Y |
| IVACFLU-S-0203-201-SA141 (A125) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:18:00 | A125 | Y |
| IVACFLU-S-0203-201-SA142 (A126) | IVACFLU-S | IVACFLU-S | 26Mar2017:14:40:00 | A126 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA143() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA144() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA145() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA146() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA147() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA148() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA149() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA150() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA151() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA152() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA153() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA154() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA155() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA156() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA157() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA158() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA159() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA160() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA161() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA162() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA163() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA164() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA165() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA166() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA167() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA168() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA169() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA170() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA171() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA172() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA173() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA174() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA175() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA176() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA177() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA178() | SCREEN FAILURE | SCREEN FAILURE | | | |

Version 1.0 Protocol No: IVACFLU-S-0203 703 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SA179() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA180() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA181() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA182() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA183() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA184() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA185() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA186() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA187() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA188() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA189() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA190() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA191() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA192() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA193() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA194() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA195() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA196() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA197() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA198() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA199() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA200() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA201() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA202() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA203() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA204() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA205() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SA206() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB001 (B001) | IVACFLU-S | IVACFLU-S | 20Mar2017:09:29:00 | B001 | Y |
| IVACFLU-S-0203-201-SB002 (B003) | PLACEBO | PLACEBO | 20Mar2017:10:24:00 | B003 | Y |
| IVACFLU-S-0203-201-SB003() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB004 (B007) | PLACEBO | PLACEBO | 20Mar2017:10:42:00 | B007 | Y |
| IVACFLU-S-0203-201-SB005 (B002) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:21:00 | B002 | Y |
| IVACFLU-S-0203-201-SB006 (B008) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:45:00 | B008 | Y |
| IVACFLU-S-0203-201-SB007() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB008() | SCREEN FAILURE | SCREEN FAILURE | | | |

IVACFLU-S-0203-201-SB039 (B032)

IVACFLU-S-0203-201-SB040 (B030)

IVACFLU-S-0203-201-SB041 (B033)

IVACFLU-S-0203-201-SB042 (B034)

IVACFLU-S-0203-201-SB043 (B027)

IVACFLU-S-0203-201-SB044 (B031)

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB009() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB010 (B010) | IVACFLU-S | IVACFLU-S | 20Mar2017:11:11:00 | B010 | Y |
| IVACFLU-S-0203-201-SB011 (B005) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:33:00 | B005 | Y |
| IVACFLU-S-0203-201-SB012() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB013 (B004) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:29:00 | B004 | Y |
| IVACFLU-S-0203-201-SB014 (B006) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:37:00 | B006 | Y |
| IVACFLU-S-0203-201-SB015() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB016() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB017 (B009) | IVACFLU-S | IVACFLU-S | 20Mar2017:10:52:00 | B009 | Y |
| IVACFLU-S-0203-201-SB018 (B011) | IVACFLU-S | IVACFLU-S | 20Mar2017:11:20:00 | B011 | Y |
| IVACFLU-S-0203-201-SB019() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB020 (B013) | IVACFLU-S | IVACFLU-S | 20Mar2017:11:29:00 | B013 | Y |
| IVACFLU-S-0203-201-SB021 (B012) | IVACFLU-S | IVACFLU-S | 20Mar2017:11:26:00 | B012 | Y |
| IVACFLU-S-0203-201-SB022 (B015) | IVACFLU-S | IVACFLU-S | 22Mar2017:08:55:00 | B015 | Y |
| IVACFLU-S-0203-201-SB023 (B014) | IVACFLU-S | IVACFLU-S | 22Mar2017:08:43:00 | B014 | Y |
| IVACFLU-S-0203-201-SB024 (B026) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:29:00 | B026 | Y |
| IVACFLU-S-0203-201-SB025 (B016) | PLACEBO | PLACEBO | 22Mar2017:09:00:00 | B016 | Y |
| IVACFLU-S-0203-201-SB026() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB027() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB028 (B018) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:21:00 | B018 | Y |
| IVACFLU-S-0203-201-SB029 (B028) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:38:00 | B028 | Y |
| IVACFLU-S-0203-201-SB030 (B029) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:53:00 | B029 | Y |
| IVACFLU-S-0203-201-SB031 (B019) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:49:00 | B019 | Y |
| IVACFLU-S-0203-201-SB032 (B017) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:13:00 | B017 | Y |
| IVACFLU-S-0203-201-SB033 (B021) | PLACEBO | PLACEBO | 22Mar2017:10:03:00 | B021 | Y |
| IVACFLU-S-0203-201-SB034() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB035 (B022) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:05:00 | B022 | Y |
| IVACFLU-S-0203-201-SB036 (B020) | IVACFLU-S | IVACFLU-S | 22Mar2017:09:58:00 | B020 | Y |
| IVACFLU-S-0203-201-SB037 (B024) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:15:00 | B024 | Y |
| IVACFLU-S-0203-201-SB038 (B023) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:13:00 | B023 | Y |

IVACFLU-S

**IVACFLU-S** 

IVACFLU-S

**IVACFLU-S** 

PLACEBO

**PLACEBO** 

22Mar2017:11:00:00

22Mar2017:10:57:00

22Mar2017:11:12:00

22Mar2017:11:11:00

22Mar2017:10:35:00

22Mar2017:11:04:00

IVACFLU-S

**IVACFLU-S** 

IVACFLU-S

IVACFLU-S

PLACEBO

PLACEBO

Y

Y Y

Y

Y

Y

B032

B030

B033

B034

B027

B031

Version 1.0 Protocol No: IVACFLU-S-0203 705 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB045 (B025) | IVACFLU-S | IVACFLU-S | 22Mar2017:10:22:00 | B025 | Y |
| IVACFLU-S-0203-201-SB046 (B035) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:29:00 | B035 | Y |
| IVACFLU-S-0203-201-SB047() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB048 (B036) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:45:00 | B036 | Y |
| IVACFLU-S-0203-201-SB049() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB050 (B037) | IVACFLU-S | IVACFLU-S | 23Mar2017:08:59:00 | B037 | Y |
| IVACFLU-S-0203-201-SB051() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB052() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB053 (B044) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:21:00 | B044 | Y |
| IVACFLU-S-0203-201-SB054 (B039) | IVACFLU-S | IVACFLU-S | 23Mar2017:09:48:00 | B039 | Y |
| IVACFLU-S-0203-201-SB055() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB056 (B038) | IVACFLU-S | IVACFLU-S | 23Mar2017:09:20:00 | B038 | Y |
| IVACFLU-S-0203-201-SB057() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB058 (B040) | PLACEBO | PLACEBO | 23Mar2017:09:59:00 | B040 | Y |
| IVACFLU-S-0203-201-SB059 (B041) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:04:00 | B041 | Y |
| IVACFLU-S-0203-201-SB060() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB061() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB062 (B042) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:06:00 | B042 | Y |
| IVACFLU-S-0203-201-SB063 (B046) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:32:00 | B046 | Y |
| IVACFLU-S-0203-201-SB064() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB065 (B045) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:29:00 | B045 | Y |
| IVACFLU-S-0203-201-SB066() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB067 (B043) | PLACEBO | PLACEBO | 23Mar2017:10:11:00 | B043 | Y |
| IVACFLU-S-0203-201-SB068() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB069 (B047) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:35:00 | B047 | Y |
| IVACFLU-S-0203-201-SB070 (B048) | IVACFLU-S | IVACFLU-S | 23Mar2017:10:50:00 | B048 | Y |
| IVACFLU-S-0203-201-SB071() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB072 (B049) | IVACFLU-S | IVACFLU-S | 23Mar2017:14:58:00 | B049 | Y |
| IVACFLU-S-0203-201-SB073() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB074 (B051) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:17:00 | B051 | Y |
| IVACFLU-S-0203-201-SB075() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB076 (B050) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:03:00 | B050 | Y |
| IVACFLU-S-0203-201-SB077 (B053) | PLACEBO | PLACEBO | 23Mar2017:15:29:00 | B053 | Y |
| IVACFLU-S-0203-201-SB078() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB079 (B055) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:50:00 | B055 | Y |
| IVACFLU-S-0203-201-SB080 (B056) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:54:00 | B056 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB081() | SCREEN FAILURE | SCREEN FAILURE | | | Ü |
| IVACFLU-S-0203-201-SB082() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB083 (B052) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:26:00 | B052 | Y |
| IVACFLU-S-0203-201-SB084() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB085() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB086() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB087 (B054) | IVACFLU-S | IVACFLU-S | 23Mar2017:15:38:00 | B054 | Y |
| IVACFLU-S-0203-201-SB088() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB089() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB090() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB091 (B057) | IVACFLU-S | IVACFLU-S | 23Mar2017:16:18:00 | B057 | Y |
| IVACFLU-S-0203-201-SB092 (B058) | IVACFLU-S | IVACFLU-S | 23Mar2017:16:20:00 | B058 | Y |
| IVACFLU-S-0203-201-SB093 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB094() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB095() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB096 (B061) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:21:00 | B061 | Y |
| IVACFLU-S-0203-201-SB097() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB098 (B060) | PLACEBO | PLACEBO | 24Mar2017:08:14:00 | B060 | Y |
| IVACFLU-S-0203-201-SB099 (B064) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:40:00 | B064 | Y |
| IVACFLU-S-0203-201-SB100 (B059) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:10:00 | B059 | Y |
| IVACFLU-S-0203-201-SB101 (B062) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:34:00 | B062 | Y |
| IVACFLU-S-0203-201-SB102() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB103 (B063) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:37:00 | B063 | Y |
| IVACFLU-S-0203-201-SB104 (B065) | IVACFLU-S | IVACFLU-S | 24Mar2017:08:47:00 | B065 | Y |
| IVACFLU-S-0203-201-SB105() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB106 (B069) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:20:00 | B069 | Y |
| IVACFLU-S-0203-201-SB107() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB108() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB109() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB110 (B067) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:08:00 | B067 | Y |
| IVACFLU-S-0203-201-SB111 (B066) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:01:00 | B066 | Y |
| IVACFLU-S-0203-201-SB112 (B068) | IVACFLU-S | IVACFLU-S | 24Mar2017:09:10:00 | B068 | Y |
| IVACFLU-S-0203-201-SB113 (B070) | PLACEBO | PLACEBO | 24Mar2017:10:18:00 | B070 | Y |
| IVACFLU-S-0203-201-SB114 (B075) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:33:00 | B075 | Y |
| IVACFLU-S-0203-201-SB115 (B071) | PLACEBO | PLACEBO | 24Mar2017:10:20:00 | B071 | Y |
| IVACFLU-S-0203-201-SB116 (B072) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:22:00 | B072 | Y |

Version 1.0 Protocol No: IVACFLU-S-0203 707 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB117 (B074) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:30:00 | B074 | Y |
| IVACFLU-S-0203-201-SB118 (B073) | IVACFLU-S | IVACFLU-S | 24Mar2017:10:28:00 | B073 | Y |
| IVACFLU-S-0203-201-SB119 (B076) | PLACEBO | PLACEBO | 24Mar2017:10:39:00 | B076 | Y |
| IVACFLU-S-0203-201-SB120 (B077) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:18:00 | B077 | Y |
| IVACFLU-S-0203-201-SB121 (B078) | IVACFLU-S | IVACFLU-S | 24Mar2017:14:37:00 | B078 | Y |
| IVACFLU-S-0203-201-SB122 (B079) | PLACEBO | PLACEBO | 24Mar2017:15:06:00 | B079 | Y |
| IVACFLU-S-0203-201-SB123() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB124 (B081) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:12:00 | B081 | Y |
| IVACFLU-S-0203-201-SB125() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB126 (B080) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:08:00 | B080 | Y |
| IVACFLU-S-0203-201-SB127() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB128 (B083) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:21:00 | B083 | Y |
| IVACFLU-S-0203-201-SB129 (B085) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:32:00 | B085 | Y |
| IVACFLU-S-0203-201-SB130() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB131 (B082) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:14:00 | B082 | Y |
| IVACFLU-S-0203-201-SB132() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB133 (B086) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:43:00 | B086 | Y |
| IVACFLU-S-0203-201-SB134 (B084) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:28:00 | B084 | Y |
| IVACFLU-S-0203-201-SB135 (B087) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:49:00 | B087 | Y |
| IVACFLU-S-0203-201-SB136() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB137 (B093) | IVACFLU-S | IVACFLU-S | 24Mar2017:16:14:00 | B093 | Y |
| IVACFLU-S-0203-201-SB138() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB139() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB140 (B088) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:51:00 | B088 | Y |
| IVACFLU-S-0203-201-SB141 (B090) | PLACEBO | PLACEBO | 24Mar2017:16:01:00 | B090 | Y |
| IVACFLU-S-0203-201-SB142 (B091) | PLACEBO | PLACEBO | 24Mar2017:16:05:00 | B091 | Y |
| IVACFLU-S-0203-201-SB143 (B092) | IVACFLU-S | IVACFLU-S | 24Mar2017:16:11:00 | B092 | Y |
| IVACFLU-S-0203-201-SB144 (B089) | IVACFLU-S | IVACFLU-S | 24Mar2017:15:54:00 | B089 | Y |
| IVACFLU-S-0203-201-SB145() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB146 (B095) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:21:00 | B095 | Y |
| IVACFLU-S-0203-201-SB147() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB148 (B101) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:50:00 | B101 | Y |
| IVACFLU-S-0203-201-SB149 (B094) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:17:00 | B094 | Y |
| IVACFLU-S-0203-201-SB150 (B097) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:26:00 | B097 | Y |
| IVACFLU-S-0203-201-SB151() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB152 (B096) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:23:00 | B096 | Y |

| Protocol No: IVACFLU-S-0203 | 708 | Dated: 12 March 2018 |
|-----------------------------|-----|----------------------|
|-----------------------------|-----|----------------------|

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB153 (B098) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:29:00 | B098 | Y |
| IVACFLU-S-0203-201-SB154() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB155 (B099) | PLACEBO | PLACEBO | 26Mar2017:08:31:00 | B099 | Y |
| IVACFLU-S-0203-201-SB156 (B102) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:52:00 | B102 | Y |
| IVACFLU-S-0203-201-SB157 (B106) | PLACEBO | PLACEBO | 26Mar2017:09:13:00 | B106 | Y |
| IVACFLU-S-0203-201-SB158 (B103) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:55:00 | B103 | Y |
| IVACFLU-S-0203-201-SB159 (B104) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:59:00 | B104 | Y |
| IVACFLU-S-0203-201-SB160 (B100) | IVACFLU-S | IVACFLU-S | 26Mar2017:08:43:00 | B100 | Y |
| IVACFLU-S-0203-201-SB161 (B107) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:07:00 | B107 | Y |
| IVACFLU-S-0203-201-SB162 (B119) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:49:00 | B119 | Y |
| IVACFLU-S-0203-201-SB163 (B113) | PLACEBO | PLACEBO | 26Mar2017:09:28:00 | B113 | Y |
| IVACFLU-S-0203-201-SB164 (B111) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:23:00 | B111 | Y |
| IVACFLU-S-0203-201-SB165() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB166 (B108) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:09:00 | B108 | Y |
| IVACFLU-S-0203-201-SB167 (B109) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:16:00 | B109 | Y |
| IVACFLU-S-0203-201-SB168 (B105) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:01:00 | B105 | Y |
| IVACFLU-S-0203-201-SB169 (B110) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:20:00 | B110 | Y |
| IVACFLU-S-0203-201-SB170 (B117) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:45:00 | B117 | Y |
| IVACFLU-S-0203-201-SB171 (B115) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:41:00 | B115 | Y |
| IVACFLU-S-0203-201-SB172 (B118) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:47:00 | B118 | Y |
| IVACFLU-S-0203-201-SB173 (B114) | PLACEBO | PLACEBO | 26Mar2017:09:39:00 | B114 | Y |
| IVACFLU-S-0203-201-SB174 (B116) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:43:00 | B116 | Y |
| IVACFLU-S-0203-201-SB175 (B122) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:54:00 | B122 | Y |
| IVACFLU-S-0203-201-SB176 (B112) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:26:00 | B112 | Y |
| IVACFLU-S-0203-201-SB177 (B121) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:53:00 | B121 | Y |
| IVACFLU-S-0203-201-SB178 (B120) | IVACFLU-S | IVACFLU-S | 26Mar2017:09:51:00 | B120 | Y |
| IVACFLU-S-0203-201-SB179() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB180 (B123) | PLACEBO | PLACEBO | 26Mar2017:10:00:00 | B123 | Y |
| IVACFLU-S-0203-201-SB181 (B124) | IVACFLU-S | IVACFLU-S | 26Mar2017:10:07:00 | B124 | Y |
| IVACFLU-S-0203-201-SB182 (B125) | IVACFLU-S | IVACFLU-S | 26Mar2017:10:35:00 | B125 | Y |
| IVACFLU-S-0203-201-SB183 (B126) | IVACFLU-S | IVACFLU-S | 26Mar2017:10:57:00 | B126 | Y |
| IVACFLU-S-0203-201-SB184() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB185() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB186() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB187() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB188 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |


Protocol No: IVACFLU-S-0203 709 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SB189() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB190() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB191() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB192 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB193 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB194() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB195() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB196() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB197() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB198() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB199() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB200() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB201() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB202() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB203() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB204() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB205() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB206() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB207() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB208() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB209() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB210() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB211() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB212() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB213 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB214() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB215() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB216() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB217() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB218() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB219() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB220() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB221() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB222() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SB223 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC001 (C018) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:42:00 | C018 | Y |

IVACFLU-S
Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SC002 (C072) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:23:00 | C072 | Y |
| IVACFLU-S-0203-201-SC002 (C072) | IVACFLU-S | IVACELU-S | 11Jun2017:09:25:00 | C069 | Y |
| IVACFLU-S-0203-201-SC004 (C068) | IVACFLU-S | IVACELU-S | 11Jun2017:08:46:00 | C068 | Y |
| IVACFLU-S-0203-201-SC005 (C081) | PLACEBO | PLACEBO | 11Jun2017:11:10:00 | C081 | Y |
| IVACFLU-S-0203-201-SC006 (C001) | IVACFLU-S | IVACFLU-S | 08Jun2017:11:10:00 | C001 | Y |
| IVACFLU-S-0203-201-SC007 ( ) | SCREEN FAILURE | SCREEN FAILURE | 0034112017.00.21.00 | C001 | 1 |
| IVACFLU-S-0203-201-SC008 (C070) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:59:00 | C070 | Y |
| IVACFLU-S-0203-201-SC009 (C082) | IVACFLU-S | IVACFLU-S | 11Jun2017:11:31:00 | C082 | Y |
| IVACFLU-S-0203-201-SC010 (C008) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:29:00 | C008 | Y |
| IVACFLU-S-0203-201-SC011 (C005) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:12:00 | C005 | Y |
| IVACFLU-S-0203-201-SC012 (C011) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:50:00 | C011 | Y |
| IVACFLU-S-0203-201-SC013 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC014 (C006) | PLACEBO | PLACEBO | 08Jun2017:09:18:00 | C006 | Y |
| IVACFLU-S-0203-201-SC015 (C004) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:00:00 | C004 | Y |
| IVACFLU-S-0203-201-SC016 (C014) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:15:00 | C014 | Y |
| IVACFLU-S-0203-201-SC017 (C015) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:20:00 | C015 | Y |
| IVACFLU-S-0203-201-SC018 (C013) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:05:00 | C013 | Y |
| IVACFLU-S-0203-201-SC019 (C002) | IVACFLU-S | IVACFLU-S | 08Jun2017:08:42:00 | C002 | Y |
| IVACFLU-S-0203-201-SC020 (C016) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:26:00 | C016 | Y |
| IVACFLU-S-0203-201-SC021() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC022 (C009) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:36:00 | C009 | Y |
| IVACFLU-S-0203-201-SC023() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC024 (C012) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:01:00 | C012 | Y |
| IVACFLU-S-0203-201-SC025 (C073) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:35:00 | C073 | Y |
| IVACFLU-S-0203-201-SC026 (C017) | PLACEBO | PLACEBO | 08Jun2017:10:40:00 | C017 | Y |
| IVACFLU-S-0203-201-SC027 (C095) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:11:00 | C095 | Y |
| IVACFLU-S-0203-201-SC028 (C094) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:08:00 | C094 | Y |
| IVACFLU-S-0203-201-SC029 (C097) | PLACEBO | PLACEBO | 11Jun2017:15:18:00 | C097 | Y |
| IVACFLU-S-0203-201-SC030 (C086) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:12:00 | C086 | Y |
| IVACFLU-S-0203-201-SC031 (C090) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:31:00 | C090 | Y |
| IVACFLU-S-0203-201-SC032 (C085) | PLACEBO | PLACEBO | 11Jun2017:14:09:00 | C085 | Y |
| IVACFLU-S-0203-201-SC033 (C091) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:35:00 | C091 | Y |
| IVACFLU-S-0203-201-SC034 (C084) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:05:00 | C084 | Y |
| IVACFLU-S-0203-201-SC035 (C020) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:27:00 | C020 | Y |
| IVACFLU-S-0203-201-SC036 (C023) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:09:00 | C023 | Y |
| IVACFLU-S-0203-201-SC037 (C019) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:10:00 | C019 | Y |


| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SC038 (C123) | IVACFLU-S | IVACFLU-S | 12Jun2017:14:21:00 | C123 | Y |
| IVACFLU-S-0203-201-SC039 (C089) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:24:00 | C089 | Y |
| IVACFLU-S-0203-201-SC040 (C024) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:20:00 | C024 | Y |
| IVACFLU-S-0203-201-SC041 ( ) | SCREEN FAILURE | SCREEN FAILURE | 0034112017.13.20.00 | C02+ | 1 |
| IVACFLU-S-0203-201-SC042 (C096) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:15:00 | C096 | Y |
| IVACFLU-S-0203-201-SC043 (C021) | PLACEBO | PLACEBO | 08Jun2017:14:37:00 | C021 | Y |
| IVACFLU-S-0203-201-SC044 ( ) | SCREEN FAILURE | SCREEN FAILURE | 0004112017.11.37.00 | 0021 | 1 |
| IVACFLU-S-0203-201-SC045 (C092) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:50:00 | C092 | Y |
| IVACFLU-S-0203-201-SC046 ( ) | SCREEN FAILURE | SCREEN FAILURE | 1104112017.10.000 | 2072 | 1 |
| IVACFLU-S-0203-201-SC047 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC048 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC049 (C022) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:44:00 | C022 | Y |
| IVACFLU-S-0203-201-SC050() | SCREEN FAILURE | SCREEN FAILURE | - | | |
| IVACFLU-S-0203-201-SC051 (C088) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:27:00 | C088 | Y |
| IVACFLU-S-0203-201-SC052 (C083) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:00:00 | C083 | Y |
| IVACFLU-S-0203-201-SC053() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC054 (C064) | PLACEBO | PLACEBO | 11Jun2017:08:21:00 | C064 | Y |
| IVACFLU-S-0203-201-SC055() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC056 (C063) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:07:00 | C063 | Y |
| IVACFLU-S-0203-201-SC057 (C062) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:04:00 | C062 | Y |
| IVACFLU-S-0203-201-SC058 (C071) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:05:00 | C071 | Y |
| IVACFLU-S-0203-201-SC059 (C087) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:14:00 | C087 | Y |
| IVACFLU-S-0203-201-SC060 (C061) | IVACFLU-S | IVACFLU-S | 11Jun2017:07:56:00 | C061 | Y |
| IVACFLU-S-0203-201-SC061 (C065) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:26:00 | C065 | Y |
| IVACFLU-S-0203-201-SC062 (C067) | PLACEBO | PLACEBO | 11Jun2017:08:40:00 | C067 | Y |
| IVACFLU-S-0203-201-SC063 (C066) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:29:00 | C066 | Y |
| IVACFLU-S-0203-201-SC064() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC065 (C029) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:03:00 | C029 | Y |
| IVACFLU-S-0203-201-SC066 (C034) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:03:00 | C034 | Y |
| IVACFLU-S-0203-201-SC067 (C025) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:26:00 | C025 | Y |
| IVACFLU-S-0203-201-SC068 (C028) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:58:00 | C028 | Y |
| IVACFLU-S-0203-201-SC069() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC070 (C031) | PLACEBO | PLACEBO | 10Jun2017:09:18:00 | C031 | Y |
| IVACFLU-S-0203-201-SC071 (C111) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:22:00 | C111 | Y |
| IVACFLU-S-0203-201-SC072() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC073 (C027) | PLACEBO | PLACEBO | 10Jun2017:08:43:00 | C027 | Y |

711

Protocol No: IVACFLU-S-0203 712 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SC074 (C116) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:49:00 | C116 | Y |
| IVACFLU-S-0203-201-SC074 (C110) | IVACFLU-S | IVACELU-S IVACELU-S | 10Jun2017:09:12:00 | C030 | Y |
| IVACFLU-S-0203-201-SC075 (C030) | IVACFLU-S | IVACELU-S IVACELU-S | 10Jun2017:09:52:00 | C032 | Y |
| IVACFLU-S-0203-201-SC076 (C032) | IVACFLU-S | IVACELU-S IVACELU-S | 10Jun2017:09:32:00 | C026 | Y |
| IVACFLU-S-0203-201-SC077 (C020) | IVACELU-S IVACELU-S | IVACELU-S IVACELU-S | 10Jun2017:10:49:00 | C039 | Y |
| IVACFLU-S-0203-201-SC078 (C039) | SCREEN FAILURE | SCREEN FAILURE | 103u112017.10.49.00 | C039 | 1 |
| IVACFLU-S-0203-201-SC079 () IVACFLU-S-0203-201-SC080 (C108) | PLACEBO | PLACEBO | 11Jun2017:16:27:00 | C108 | Y |
| IVACFLU-S-0203-201-SC080 (C108) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:53:00 | C040 | Y |
| IVACFLU-S-0203-201-SC081 (C040) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:54:00 | C102 | Y |
| IVACFLU-S-0203-201-SC082 (C102) | IVACELU-S IVACELU-S | IVACELU-S IVACELU-S | 11Jun2017:16:20:00 | C102 | Y |
| IVACFLU-S-0203-201-SC083 (C100) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:20:00 | C100 | Y |
| IVACFLU-S-0203-201-SC084 (C033) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:57:00 | C103 | Y |
| IVACFLU-S-0203-201-SC085 (C103) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:22:00 | C103 | Y |
| | IVACFLU-S | IVACFLU-S | 11Jun2017:15:22:00<br>11Jun2017:15:41:00 | C107 | Y |
| IVACFLU-S-0203-201-SC087 (C100) | IVACFLU-S<br>IVACFLU-S | | | C100<br>C098 | Y |
| IVACFLU-S-0203-201-SC088 (C098) | | IVACELUS | 11Jun2017:15:23:00 | | Y |
| IVACFLU-S-0203-201-SC089 (C105) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:04:00 | C105 | Y |
| IVACFLU-S-0203-201-SC090 (C093) | PLACEBO | PLACEBO | 11Jun2017:15:03:00 | C093 | Y |
| IVACFLU-S-0203-201-SC091 () | SCREEN FAILURE | SCREEN FAILURE | 111 2017 15 20 00 | G000 | *** |
| IVACFLU-S-0203-201-SC092 (C099) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:38:00 | C099 | Y |
| IVACFLU-S-0203-201-SC093 () | SCREEN FAILURE | SCREEN FAILURE | 101 2017 10 47 00 | G020 | *** |
| IVACFLU-S-0203-201-SC094 (C038) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:47:00 | C038 | Y |
| IVACFLU-S-0203-201-SC095 (C036) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:36:00 | C036 | Y |
| IVACFLU-S-0203-201-SC096 () | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC097 () | SCREEN FAILURE | SCREEN FAILURE | | ~~ | |
| IVACFLU-S-0203-201-SC098 (C041) | PLACEBO | PLACEBO | 10Jun2017:10:57:00 | C041 | Y |
| IVACFLU-S-0203-201-SC099 (C010) | PLACEBO | PLACEBO | 08Jun2017:09:45:00 | C010 | Y |
| IVACFLU-S-0203-201-SC100 (C037) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:43:00 | C037 | Y |
| IVACFLU-S-0203-201-SC101 (C101) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:44:00 | C101 | Y |
| IVACFLU-S-0203-201-SC102 (C035) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:26:00 | C035 | Y |
| IVACFLU-S-0203-201-SC103 (C042) | PLACEBO | PLACEBO | 10Jun2017:13:45:00 | C042 | Y |
| IVACFLU-S-0203-201-SC104 (C007) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:24:00 | C007 | Y |
| IVACFLU-S-0203-201-SC105 (C125) | IVACFLU-S | IVACFLU-S | 12Jun2017:15:19:00 | C125 | Y |
| IVACFLU-S-0203-201-SC106 (C124) | IVACFLU-S | IVACFLU-S | 12Jun2017:14:54:00 | C124 | Y |
| IVACFLU-S-0203-201-SC107 (C060) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:38:00 | C060 | Y |
| IVACFLU-S-0203-201-SC108 (C054) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:56:00 | C054 | Y |
| IVACFLU-S-0203-201-SC109 (C056) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:03:00 | C056 | Y |
| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SC110() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC111 (C058) | PLACEBO | PLACEBO | 10Jun2017:15:21:00 | C058 | Y |
| IVACFLU-S-0203-201-SC112 (C051) | PLACEBO | PLACEBO | 10Jun2017:14:46:00 | C051 | Y |
| IVACFLU-S-0203-201-SC113 (C003) | IVACFLU-S | IVACFLU-S | 08Jun2017:08:54:00 | C003 | Y |
| IVACFLU-S-0203-201-SC114 (C126) | IVACFLU-S | IVACFLU-S | 12Jun2017:15:25:00 | C126 | Y |
| IVACFLU-S-0203-201-SC115 (C059) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:28:00 | C059 | Y |
| IVACFLU-S-0203-201-SC116 (C044) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:02:00 | C044 | Y |
| IVACFLU-S-0203-201-SC117 (C045) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:09:00 | C045 | Y |
| IVACFLU-S-0203-201-SC118 (C043) | IVACFLU-S | IVACFLU-S | 10Jun2017:13:50:00 | C043 | Y |
| IVACFLU-S-0203-201-SC119() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC120 (C047) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:17:00 | C047 | Y |
| IVACFLU-S-0203-201-SC121 (C050) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:27:00 | C050 | Y |
| IVACFLU-S-0203-201-SC122 (C055) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:58:00 | C055 | Y |
| IVACFLU-S-0203-201-SC123 (C048) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:20:00 | C048 | Y |
| IVACFLU-S-0203-201-SC124 (C052) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:49:00 | C052 | Y |
| IVACFLU-S-0203-201-SC125 (C053) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:44:00 | C053 | Y |
| IVACFLU-S-0203-201-SC126 (C046) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:14:00 | C046 | Y |
| IVACFLU-S-0203-201-SC127 (C057) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:15:00 | C057 | Y |
| IVACFLU-S-0203-201-SC128 (C049) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:24:00 | C049 | Y |
| IVACFLU-S-0203-201-SC129() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC130 (C119) | PLACEBO | PLACEBO | 12Jun2017:09:09:00 | C119 | Y |
| IVACFLU-S-0203-201-SC131 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC132 (C078) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:55:00 | C078 | Y |
| IVACFLU-S-0203-201-SC133 (C077) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:45:00 | C077 | Y |
| IVACFLU-S-0203-201-SC134 (C120) | IVACFLU-S | IVACFLU-S | 12Jun2017:09:05:00 | C120 | Y |
| IVACFLU-S-0203-201-SC135 (C122) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:18:00 | C122 | Y |
| IVACFLU-S-0203-201-SC136 (C075) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:11:00 | C075 | Y |
| IVACFLU-S-0203-201-SC137 (C076) | PLACEBO | PLACEBO | 11Jun2017:10:15:00 | C076 | Y |
| IVACFLU-S-0203-201-SC138 (C079) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:59:00 | C079 | Y |
| IVACFLU-S-0203-201-SC139() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC140 (C080) | IVACFLU-S | IVACFLU-S | 11Jun2017:11:14:00 | C080 | Y |
| IVACFLU-S-0203-201-SC141() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC142 (C118) | PLACEBO | PLACEBO | 12Jun2017:08:57:00 | C118 | Y |
| IVACFLU-S-0203-201-SC143 (C121) | PLACEBO | PLACEBO | 12Jun2017:10:10:00 | C121 | Y |
| IVACFLU-S-0203-201-SC144() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SC145 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |

Protocol No: IVACFLU-S-0203 714 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SC146 (C115) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:38:00 | C115 | Y |
| IVACFLU-S-0203-201-SC140 (C113) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:34:00 | C114 | Y |
| IVACFLU-S-0203-201-SC147 (C114) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:26:00 | C112 | Y |
| IVACFLU-S-0203-201-SC148 (C112) | SCREEN FAILURE | SCREEN FAILURE | 1234112017.08.20.00 | C112 | I |
| IVACFLU-S-0203-201-SC150 (C117) | IVACFLU-S | IVACFLU-S | 12Jun2017:09:17:00 | C117 | Y |
| IVACFLU-S-0203-201-SC130 (C117) | IVACELU-S IVACELU-S | IVACFLU-S | 12Jun2017:09:17:00<br>12Jun2017:08:13:00 | C109 | Y |
| IVACFLU-S-0203-201-SC131 (C109) | IVACELU-S IVACELU-S | IVACFLU-S | 12Jun2017:08:13:00<br>12Jun2017:08:28:00 | C109 | Y |
| IVACFLU-S-0203-201-SC132 (C113) | IVACELU-S IVACELU-S | IVACFLU-S | 12Jun2017:08:28:00<br>12Jun2017:08:16:00 | C110 | Y |
| IVACFLU-S-0203-201-SC133 (C110) | IVACELU-S | IVACFLU-S | 11Jun2017:09:52:00 | C074 | Y |
| IVACFLU-S-0203-201-SC154 (C0/4) | SCREEN FAILURE | SCREEN FAILURE | 1134112017.09.32.00 | C0/4 | I |
| IVACFLU-S-0203-201-SC135 () | IVACFLU-S | IVACFLU-S | 11Jun2017:16:00:00 | C104 | Y |
| IVACFLU-S-0203-201-SC130 (C104) | SCREEN FAILURE | SCREEN FAILURE | 1134112017.10.00.00 | C104 | I |
| IVACFLU-S-0203-201-SD001 ( ) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:11:00 | D071 | Y |
| IVACFLU-S-0203-201-SD002 (D071) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:07:00 | D077 | Y |
| IVACFLU-S-0203-201-SD003 (D077) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:07:00 | D076 | Y |
| IVACFLU-S-0203-201-SD004 (D076) | SCREEN FAILURE | SCREEN FAILURE | 1134112017.09.44.00 | D076 | I |
| IVACFLU-S-0203-201-SD003 ( ) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:27:00 | D074 | Y |
| IVACFLU-S-0203-201-SD000 (D074) | IVACELU-S IVACELU-S | IVACFLU-S | 12Jun2017:12:16:00 | D103 | Y |
| IVACFLU-S-0203-201-SD007 (D103) | PLACEBO | PLACEBO | 11Jun2017:12:10:00 | D103 | Y |
| IVACFLU-S-0203-201-SD008 (D073) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:40:00 | D073 | Y |
| IVACFLU-S-0203-201-SD009 (D073) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:37:00 | D073 | Y |
| IVACFLU-S-0203-201-SD010 (D008) | IVACELU-S IVACELU-S | IVACFLU-S | 08Jun2017:10:37:00 | D008 | Y |
| IVACFLU-S-0203-201-SD011 (D003) | SCREEN FAILURE | SCREEN FAILURE | 0834112017.10.11.00 | D003 | I |
| IVACFLU-S-0203-201-SD012 () | PLACEBO | PLACEBO | 08Jun2017:10:31:00 | D006 | Y |
| IVACFLU-S-0203-201-SD013 (D006) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:31:00<br>08Jun2017:10:23:00 | D006<br>D004 | Y |
| IVACFLU-S-0203-201-SD014 (D004) | SCREEN FAILURE | SCREEN FAILURE | 08Jun2017:10:23:00 | D004 | Y |
| IVACFLU-S-0203-201-SD015 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD016 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD017 ( ) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:25:00 | D108 | Y |
| IVACFLU-S-0203-201-SD018 (D108) | IVACELU-S IVACELU-S | IVACFLU-S | 08Jun2017:10:23:00 | D108<br>D001 | Y |
| · / | SCREEN FAILURE | SCREEN FAILURE | 0834112017.08.37.00 | D001 | I |
| IVACFLU-S-0203-201-SD020 ( ) IVACFLU-S-0203-201-SD021 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD021 ( ) IVACFLU-S-0203-201-SD022 (D070) | IVACFLU-S | IVACFLU-S | 11Jun2017:09:08:00 | D070 | Y |
| · / | PLACEBO | | 12Jun2017:09:08:00<br>12Jun2017:10:56:00 | D102 | Y |
| IVACFLU-S-0203-201-SD023 (D102)<br>IVACFLU-S-0203-201-SD024 (D118) | IVACFLU-S | PLACEBO<br>IVACFLU-S | 12Jun2017:10:56:00<br>12Jun2017:14:40:00 | D102<br>D118 | Y |
| IVACFLU-S-0203-201-SD024 (D118) | IVACELU-S IVACELU-S | IVACFLU-S | 08Jun2017:14:40:00<br>08Jun2017:10:28:00 | D118<br>D005 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD026 (D007) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:33:00 | D007 | Y |
| IVACFLU-S-0203-201-SD027 (D002) | IVACFLU-S | IVACFLU-S | 08Jun2017:09:57:00 | D002 | Y |
| IVACFLU-S-0203-201-SD028() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD029() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD030 (D009) | IVACFLU-S | IVACFLU-S | 08Jun2017:10:44:00 | D009 | Y |
| IVACFLU-S-0203-201-SD031() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD032 (D072) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:37:00 | D072 | Y |
| IVACFLU-S-0203-201-SD033 (D116) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:12:00 | D116 | Y |
| IVACFLU-S-0203-201-SD034() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD035() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD036 (D084) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:48:00 | C084 | Y |
| IVACFLU-S-0203-201-SD037() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD038() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD039() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD040() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD041() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD042() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD043 (D020) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:13:00 | D020 | Y |
| IVACFLU-S-0203-201-SD045() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD046() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD047 (D023) | PLACEBO | PLACEBO | 08Jun2017:15:51:00 | D023 | Y |
| IVACFLU-S-0203-201-SD048 (D019) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:05:00 | D019 | Y |
| IVACFLU-S-0203-201-SD049 (D017) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:55:00 | D017 | Y |
| IVACFLU-S-0203-201-SD050 (D016) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:52:00 | D016 | Y |
| IVACFLU-S-0203-201-SD051 (D117) | IVACFLU-S | IVACFLU-S | 12Jun2017:14:30:00 | D117 | Y |
| IVACFLU-S-0203-201-SD052 (D120) | IVACFLU-S | IVACFLU-S | 12Jun2017:14:58:00 | D120 | Y |
| IVACFLU-S-0203-201-SD053() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD054 (D013) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:35:00 | D013 | Y |
| IVACFLU-S-0203-201-SD055 (D018) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:00:00 | D018 | Y |
| IVACFLU-S-0203-201-SD056 (D022) | PLACEBO | PLACEBO | 08Jun2017:15:42:00 | D022 | Y |
| IVACFLU-S-0203-201-SD057 (D011) | PLACEBO | PLACEBO | 08Jun2017:14:18:00 | D011 | Y |
| IVACFLU-S-0203-201-SD058 (D010) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:14:00 | D010 | Y |
| IVACFLU-S-0203-201-SD059() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD060 (D014) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:42:00 | D014 | Y |
| IVACFLU-S-0203-201-SD061 (D012) | IVACFLU-S | IVACFLU-S | 08Jun2017:14:31:00 | D012 | Y |
| IVACFLU-S-0203-201-SD062() | SCREEN FAILURE | SCREEN FAILURE | | | |


Protocol No: IVACFLU-S-0203 716 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD063() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD064() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD065 (D119) | IVACFLU-S | IVACFLU-S | 12Jun2017:14:46:00 | D119 | Y |
| IVACFLU-S-0203-201-SD066 (D015) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:59:00 | D015 | Y |
| IVACFLU-S-0203-201-SD067() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD068() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD069 (D021) | IVACFLU-S | IVACFLU-S | 08Jun2017:15:30:00 | D021 | Y |
| IVACFLU-S-0203-201-SD070 (D122) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:06:00 | D122 | Y |
| IVACFLU-S-0203-201-SD071 (D044) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:36:00 | D044 | Y |
| IVACFLU-S-0203-201-SD072() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD073 (D069) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:53:00 | D069 | Y |
| IVACFLU-S-0203-201-SD074 (D066) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:11:00 | D066 | Y |
| IVACFLU-S-0203-201-SD075 (D068) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:43:00 | D068 | Y |
| IVACFLU-S-0203-201-SD076 (D065) | IVACFLU-S | IVACFLU-S | 11Jun2017:08:00:00 | D065 | Y |
| IVACFLU-S-0203-201-SD077() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD078() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD079 (D032) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:35:00 | D032 | Y |
| IVACFLU-S-0203-201-SD080 (D029) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:22:00 | D029 | Y |
| IVACFLU-S-0203-201-SD081 (D045) | PLACEBO | PLACEBO | 10Jun2017:14:40:00 | D045 | Y |
| IVACFLU-S-0203-201-SD082 (D030) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:26:00 | D030 | Y |
| IVACFLU-S-0203-201-SD083 (D067) | PLACEBO | PLACEBO | 11Jun2017:08:19:00 | D067 | Y |
| IVACFLU-S-0203-201-SD084 (D027) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:36:00 | D027 | Y |
| IVACFLU-S-0203-201-SD085() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD086 (D026) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:34:00 | D026 | Y |
| IVACFLU-S-0203-201-SD087 (D049) | PLACEBO | PLACEBO | 10Jun2017:15:05:00 | D049 | Y |
| IVACFLU-S-0203-201-SD088() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD089 (D025) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:22:00 | D025 | Y |
| IVACFLU-S-0203-201-SD090() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD091 (D031) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:31:00 | D031 | Y |
| IVACFLU-S-0203-201-SD092 (D028) | PLACEBO | PLACEBO | 10Jun2017:09:07:00 | D028 | Y |
| IVACFLU-S-0203-201-SD093 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD094() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD095() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD096() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD097 (D036) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:08:00 | D036 | Y |
| IVACFLU-S-0203-201-SD098 (D034) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:47:00 | D034 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD099 (D052) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:24:00 | D052 | Y |
| IVACFLU-S-0203-201-SD100 (D024) | IVACFLU-S | IVACFLU-S | 10Jun2017:08:30:00 | D024 | Y |
| IVACFLU-S-0203-201-SD101() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD102() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD103() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD104() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD105 (D043) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:32:00 | D043 | Y |
| IVACFLU-S-0203-201-SD106 (D041) | IVACFLU-S | IVACFLU-S | 10Jun2017:11:00:00 | D041 | Y |
| IVACFLU-S-0203-201-SD107 (D089) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:08:00 | C089 | Y |
| IVACFLU-S-0203-201-SD108() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD109 (D094) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:32:00 | D094 | Y |
| IVACFLU-S-0203-201-SD110 (D093) | PLACEBO | PLACEBO | 11Jun2017:16:29:00 | D093 | Y |
| IVACFLU-S-0203-201-SD111 (D095) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:34:00 | D095 | Y |
| IVACFLU-S-0203-201-SD112 (D085) | IVACFLU-S | IVACFLU-S | 11Jun2017:14:52:00 | D085 | Y |
| IVACFLU-S-0203-201-SD113() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD114 (D096) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:40:00 | D096 | Y |
| IVACFLU-S-0203-201-SD115() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD116 (D040) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:41:00 | D040 | Y |
| IVACFLU-S-0203-201-SD117 (D035) | IVACFLU-S | IVACFLU-S | 10Jun2017:09:56:00 | D035 | Y |
| IVACFLU-S-0203-201-SD118 (D033) | PLACEBO | PLACEBO | 10Jun2017:09:43:00 | D033 | Y |
| IVACFLU-S-0203-201-SD119 (D112) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:42:00 | D112 | Y |
| IVACFLU-S-0203-201-SD120 (D087) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:35:00 | D087 | Y |
| IVACFLU-S-0203-201-SD121() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD122 (D037) | PLACEBO | PLACEBO | 10Jun2017:10:18:00 | D037 | Y |
| IVACFLU-S-0203-201-SD123() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD124 (D097) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:37:00 | D097 | Y |
| IVACFLU-S-0203-201-SD125 (D088) | PLACEBO | PLACEBO | 11Jun2017:15:47:00 | D088 | Y |
| IVACFLU-S-0203-201-SD126 (D038) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:23:00 | D038 | Y |
| IVACFLU-S-0203-201-SD127 (D092) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:24:00 | D092 | Y |
| IVACFLU-S-0203-201-SD129() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD130 (D086) | IVACFLU-S | IVACFLU-S | 11Jun2017:15:30:00 | D086 | Y |
| IVACFLU-S-0203-201-SD131() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD132() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD133() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD134 (D042) | IVACFLU-S | IVACFLU-S | 10Jun2017:11:03:00 | D042 | Y |
| IVACFLU-S-0203-201-SD135() | SCREEN FAILURE | SCREEN FAILURE | | | |

Protocol No: IVACFLU-S-0203 718 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD136 (D039) | IVACFLU-S | IVACFLU-S | 10Jun2017:10:31:00 | D039 | Y |
| IVACFLU-S-0203-201-SD137() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD138() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD139 (D091) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:13:00 | D091 | Y |
| IVACFLU-S-0203-201-SD140() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD141() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD142 (D056) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:44:00 | D056 | Y |
| IVACFLU-S-0203-201-SD143 (D115) | IVACFLU-S | IVACFLU-S | 12Jun2017:11:16:00 | D115 | Y |
| IVACFLU-S-0203-201-SD144 (D057) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:47:00 | D057 | Y |
| IVACFLU-S-0203-201-SD145() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD146() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD147 (D051) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:18:00 | D051 | Y |
| IVACFLU-S-0203-201-SD148 (D050) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:13:00 | D050 | Y |
| IVACFLU-S-0203-201-SD149 (D047) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:53:00 | D047 | Y |
| IVACFLU-S-0203-201-SD150 (D055) | PLACEBO | PLACEBO | 10Jun2017:15:41:00 | D055 | Y |
| IVACFLU-S-0203-201-SD151 (D054) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:35:00 | D054 | Y |
| IVACFLU-S-0203-201-SD152() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD153() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD154 (D114) | PLACEBO | PLACEBO | 12Jun2017:11:12:00 | D114 | Y |
| IVACFLU-S-0203-201-SD155 (D048) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:00:00 | D048 | Y |
| IVACFLU-S-0203-201-SD156 (D059) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:56:00 | D059 | Y |
| IVACFLU-S-0203-201-SD157 (D064) | PLACEBO | PLACEBO | 10Jun2017:16:17:00 | D064 | Y |
| IVACFLU-S-0203-201-SD158 (D124) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:14:00 | D124 | Y |
| IVACFLU-S-0203-201-SD159 (D062) | IVACFLU-S | IVACFLU-S | 10Jun2017:16:13:00 | D062 | Y |
| IVACFLU-S-0203-201-SD160() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD161 (D046) | IVACFLU-S | IVACFLU-S | 10Jun2017:14:51:00 | D046 | Y |
| IVACFLU-S-0203-201-SD162 (D060) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:59:00 | D060 | Y |
| IVACFLU-S-0203-201-SD163 (D061) | IVACFLU-S | IVACFLU-S | 10Jun2017:16:05:00 | D061 | Y |
| IVACFLU-S-0203-201-SD164 (D100) | IVACFLU-S | IVACFLU-S | 12Jun2017:09:13:00 | D100 | Y |
| IVACFLU-S-0203-201-SD165 (D123) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:10:00 | D123 | Y |
| IVACFLU-S-0203-201-SD166() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD167() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD168 (D058) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:53:00 | D058 | Y |
| IVACFLU-S-0203-201-SD169 (D125) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:31:00 | D125 | Y |
| IVACFLU-S-0203-201-SD170 (D063) | IVACFLU-S | IVACFLU-S | 10Jun2017:16:11:00 | D063 | Y |
| IVACFLU-S-0203-201-SD171 (D121) | PLACEBO | PLACEBO | 12Jun2017:16:02:00 | D121 | Y |

Version 1.0 Dated: 12 March 2018

Protocol No: IVACFLU-S-0203 719

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD172() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD173 (D099) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:54:00 | D099 | Y |
| IVACFLU-S-0203-201-SD174 (D053) | IVACFLU-S | IVACFLU-S | 10Jun2017:15:31:00 | D053 | Y |
| IVACFLU-S-0203-201-SD175 (D079) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:35:00 | D079 | Y |
| IVACFLU-S-0203-201-SD176 (D101) | IVACFLU-S | IVACFLU-S | 12Jun2017:09:28:00 | D101 | Y |
| IVACFLU-S-0203-201-SD177 (D083) | IVACFLU-S | IVACFLU-S | 11Jun2017:11:18:00 | D083 | Y |
| IVACFLU-S-0203-201-SD178() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD179 (D111) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:37:00 | D111 | Y |
| IVACFLU-S-0203-201-SD180 (D106) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:13:00 | D106 | Y |
| IVACFLU-S-0203-201-SD181() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD182 (D082) | PLACEBO | PLACEBO | 11Jun2017:10:50:00 | D082 | Y |
| IVACFLU-S-0203-201-SD183 (D098) | IVACFLU-S | IVACFLU-S | 12Jun2017:08:44:00 | D098 | Y |
| IVACFLU-S-0203-201-SD184() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD185 (D110) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:34:00 | D110 | Y |
| IVACFLU-S-0203-201-SD186() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD187() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD188 (D104) | IVACFLU-S | IVACFLU-S | 12Jun2017:09:48:00 | D104 | Y |
| IVACFLU-S-0203-201-SD189() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD190 (D078) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:18:00 | D078 | Y |
| IVACFLU-S-0203-201-SD191 (D080) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:38:00 | D080 | Y |
| IVACFLU-S-0203-201-SD192 (D109) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:30:00 | D109 | Y |
| IVACFLU-S-0203-201-SD193 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD194() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD195 (D107) | IVACFLU-S | IVACFLU-S | 12Jun2017:10:22:00 | D107 | Y |
| IVACFLU-S-0203-201-SD196() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD197() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD198() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD199 (D113) | PLACEBO | PLACEBO | 12Jun2017:10:50:00 | D113 | Y |
| IVACFLU-S-0203-201-SD200 (D126) | IVACFLU-S | IVACFLU-S | 12Jun2017:16:35:00 | D126 | Y |
| IVACFLU-S-0203-201-SD201() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD202() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD203() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD204() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD205() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD206() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-201-SD207 (D081) | IVACFLU-S | IVACFLU-S | 11Jun2017:10:41:00 | D081 | Y |


Protocol No: IVACFLU-S-0203 720 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-201-SD208 (D105) | PLACEBO | PLACEBO | 12Jun2017:10:02:00 | D105 | Y |
| IVACFLU-S-0203-201-SD209 (D090) | IVACFLU-S | IVACFLU-S | 11Jun2017:16:15:00 | D090 | Y |
| IVACFLU-S-0203-203-SE001 (E025) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:42:00 | E025 | Y |
| IVACFLU-S-0203-203-SE002 (E007) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:25:00 | E007 | Y |
| IVACFLU-S-0203-203-SE003 (E038) | PLACEBO | PLACEBO | 05Jul2017:17:15:00 | E038 | Y |
| IVACFLU-S-0203-203-SE004 (E040) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:30:00 | E040 | Y |
| IVACFLU-S-0203-203-SE005() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE006 (E009) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:55:00 | E009 | Y |
| IVACFLU-S-0203-203-SE007 (E018) | PLACEBO | PLACEBO | 05Jul2017:13:57:00 | E018 | Y |
| IVACFLU-S-0203-203-SE008 (E187) | PLACEBO | PLACEBO | 10Jul2017:08:25:00 | E187 | Y |
| IVACFLU-S-0203-203-SE009() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE010() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE011 (E039) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:27:00 | E039 | Y |
| IVACFLU-S-0203-203-SE012 (E010) | PLACEBO | PLACEBO | 05Jul2017:10:08:00 | E010 | Y |
| IVACFLU-S-0203-203-SE013 (E017) | PLACEBO | PLACEBO | 05Jul2017:13:52:00 | E017 | Y |
| IVACFLU-S-0203-203-SE014 (E015) | IVACFLU-S | IVACFLU-S | 05Jul2017:13:41:00 | E015 | Y |
| IVACFLU-S-0203-203-SE015 (E005) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:03:00 | E005 | Y |
| IVACFLU-S-0203-203-SE016() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE017 (E023) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:04:00 | E023 | Y |
| IVACFLU-S-0203-203-SE018 (E014) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:49:00 | E014 | Y |
| IVACFLU-S-0203-203-SE019 (E037) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:02:00 | E037 | Y |
| IVACFLU-S-0203-203-SE020() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE021 (E013) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:41:00 | E013 | Y |
| IVACFLU-S-0203-203-SE022() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE023 (E036) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:59:00 | E036 | Y |
| IVACFLU-S-0203-203-SE024 (E012) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:27:00 | E012 | Y |
| IVACFLU-S-0203-203-SE025 (E165) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:14:00 | E165 | Y |
| IVACFLU-S-0203-203-SE026 (E029) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:01:00 | E029 | Y |
| IVACFLU-S-0203-203-SE027() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE028 (E003) | IVACFLU-S | IVACFLU-S | 05Jul2017:08:56:00 | E003 | Y |
| IVACFLU-S-0203-203-SE029 (E021) | IVACFLU-S | IVACFLU-S | 05Jul2017:14:36:00 | E021 | Y |
| IVACFLU-S-0203-203-SE030 (E030) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:16:00 | E030 | Y |
| IVACFLU-S-0203-203-SE031 (E019) | IVACFLU-S | IVACFLU-S | 05Jul2017:14:01:00 | E019 | Y |
| IVACFLU-S-0203-203-SE032 (E027) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:52:00 | E027 | Y |
| IVACFLU-S-0203-203-SE033 (E020) | IVACFLU-S | IVACFLU-S | 05Jul2017:14:06:00 | E020 | Y |
| IVACFLU-S-0203-203-SE034 (E190) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:52:00 | E190 | Y |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 721 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE035 (E028) | PLACEBO | PLACEBO | 05Jul2017:15:56:00 | E028 | Y |
| IVACFLU-S-0203-203-SE036 (E002) | IVACFLU-S | IVACFLU-S | 05Jul2017:08:51:00 | E002 | Y |
| IVACFLU-S-0203-203-SE037 (E155) | IVACFLU-S | IVACFLU-S | 09Jul2017:07:54:00 | E155 | Y |
| IVACFLU-S-0203-203-SE038 (E016) | IVACFLU-S | IVACFLU-S | 05Jul2017:13:47:00 | E016 | Y |
| IVACFLU-S-0203-203-SE039 (E001) | IVACFLU-S | IVACFLU-S | 05Jul2017:08:33:00 | E001 | Y |
| IVACFLU-S-0203-203-SE040() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE041 (E173) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:04:00 | E173 | Y |
| IVACFLU-S-0203-203-SE042 (E024) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:36:00 | E024 | Y |
| IVACFLU-S-0203-203-SE043() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE044() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE045 (E011) | PLACEBO | PLACEBO | 05Jul2017:10:14:00 | E011 | Y |
| IVACFLU-S-0203-203-SE046 (E026) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:47:00 | E026 | Y |
| IVACFLU-S-0203-203-SE047 (E035) | PLACEBO | PLACEBO | 05Jul2017:16:54:00 | E035 | Y |
| IVACFLU-S-0203-203-SE048() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE049 (E032) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:33:00 | E032 | Y |
| IVACFLU-S-0203-203-SE050 (E033) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:37:00 | E033 | Y |
| IVACFLU-S-0203-203-SE051 (E158) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:18:00 | E158 | Y |
| IVACFLU-S-0203-203-SE052 (E170) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:56:00 | E170 | Y |
| IVACFLU-S-0203-203-SE053 (E174) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:39:00 | E174 | Y |
| IVACFLU-S-0203-203-SE054() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE055 (E034) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:45:00 | E034 | Y |
| IVACFLU-S-0203-203-SE056() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE057 (E185) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:14:00 | E185 | Y |
| IVACFLU-S-0203-203-SE058 (E183) | PLACEBO | PLACEBO | 10Jul2017:08:02:00 | E183 | Y |
| IVACFLU-S-0203-203-SE059() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE060 (E022) | IVACFLU-S | IVACFLU-S | 05Jul2017:14:43:00 | E022 | Y |
| IVACFLU-S-0203-203-SE061 (E154) | IVACFLU-S | IVACFLU-S | 09Jul2017:07:50:00 | E154 | Y |
| IVACFLU-S-0203-203-SE062 (E182) | IVACFLU-S | IVACFLU-S | 09Jul2017:17:13:00 | E182 | Y |
| IVACFLU-S-0203-203-SE063 (E031) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:29:00 | E031 | Y |
| IVACFLU-S-0203-203-SE064() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE065 (E006) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:15:00 | E006 | Y |
| IVACFLU-S-0203-203-SE066 (E004) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:00:00 | E004 | Y |
| IVACFLU-S-0203-203-SE067 (E008) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:40:00 | E008 | Y |
| IVACFLU-S-0203-203-SE068() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE069 (E181) | IVACFLU-S | IVACFLU-S | 09Jul2017:17:07:00 | E181 | Y |
| IVACFLU-S-0203-203-SE070 (E171) | PLACEBO | PLACEBO | 09Jul2017:13:57:00 | E171 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE071() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE072 (E164) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:07:00 | E164 | Y |
| IVACFLU-S-0203-203-SE073 (E041) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:35:00 | E041 | Y |
| IVACFLU-S-0203-203-SE074() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE075 (E166) | PLACEBO | PLACEBO | 09Jul2017:09:42:00 | E166 | Y |
| IVACFLU-S-0203-203-SE076 (E172) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:00:00 | E172 | Y |
| IVACFLU-S-0203-203-SE077 (E178) | IVACFLU-S | IVACFLU-S | 09Jul2017:16:42:00 | E178 | Y |
| IVACFLU-S-0203-203-SE078 (E159) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:23:00 | E159 | Y |
| IVACFLU-S-0203-203-SE079() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE080 (E054) | PLACEBO | PLACEBO | 06Jul2017:09:38:00 | E054 | Y |
| IVACFLU-S-0203-203-SE081 (E053) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:19:00 | E053 | Y |
| IVACFLU-S-0203-203-SE082 (E058) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:29:00 | E058 | Y |
| IVACFLU-S-0203-203-SE083 (E046) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:42:00 | E046 | Y |
| IVACFLU-S-0203-203-SE084 (E057) | PLACEBO | PLACEBO | 06Jul2017:10:26:00 | E057 | Y |
| IVACFLU-S-0203-203-SE085 (E071) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:18:00 | E071 | Y |
| IVACFLU-S-0203-203-SE086 (E051) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:09:00 | E051 | Y |
| IVACFLU-S-0203-203-SE087() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE088 (E180) | IVACFLU-S | IVACFLU-S | 09Jul2017:17:04:00 | E180 | Y |
| IVACFLU-S-0203-203-SE089 (E061) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:01:00 | E061 | Y |
| IVACFLU-S-0203-203-SE090 (E070) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:04:00 | E070 | Y |
| IVACFLU-S-0203-203-SE091 (E064) | PLACEBO | PLACEBO | 06Jul2017:11:23:00 | E064 | Y |
| IVACFLU-S-0203-203-SE092() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE093 (E085) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:52:00 | E085 | Y |
| IVACFLU-S-0203-203-SE094 (E047) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:47:00 | E047 | Y |
| IVACFLU-S-0203-203-SE095 (E044) | PLACEBO | PLACEBO | 06Jul2017:08:42:00 | E044 | Y |
| IVACFLU-S-0203-203-SE096 (E043) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:27:00 | E043 | Y |
| IVACFLU-S-0203-203-SE097 (E060) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:57:00 | E060 | Y |
| IVACFLU-S-0203-203-SE098 (E052) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:14:00 | E052 | Y |
| IVACFLU-S-0203-203-SE099 (E056) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:15:00 | E056 | Y |
| IVACFLU-S-0203-203-SE100() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE101 (E081) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:24:00 | E081 | Y |
| IVACFLU-S-0203-203-SE102 (E065) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:27:00 | E065 | Y |
| IVACFLU-S-0203-203-SE103 (E066) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:31:00 | E066 | Y |
| IVACFLU-S-0203-203-SE104 (E048) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:53:00 | E048 | Y |
| IVACFLU-S-0203-203-SE105 (E069) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:00:00 | E069 | Y |
| IVACFLU-S-0203-203-SE106 (E045) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:37:00 | E045 | Y |

Protocol No: IVACFLU-S-0203 723 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE107 (E079) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:53:00 | E079 | Y |
| IVACFLU-S-0203-203-SE108 (E068) | IVACFLU-S | IVACFLU-S | 06Jul2017:13:57:00 | E068 | Y |
| IVACFLU-S-0203-203-SE109 (E179) | PLACEBO | PLACEBO | 09Jul2017:16:45:00 | E179 | Y |
| IVACFLU-S-0203-203-SE110 (E077) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:39:00 | E077 | Y |
| IVACFLU-S-0203-203-SE111() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE112 (E063) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:16:00 | E063 | Y |
| IVACFLU-S-0203-203-SE113 (E078) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:42:00 | E078 | Y |
| IVACFLU-S-0203-203-SE114() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE115 (E050) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:04:00 | E050 | Y |
| IVACFLU-S-0203-203-SE116() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE117() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE118 (E059) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:50:00 | E059 | Y |
| IVACFLU-S-0203-203-SE119() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE120 (E075) | PLACEBO | PLACEBO | 06Jul2017:14:32:00 | E075 | Y |
| IVACFLU-S-0203-203-SE121 (E049) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:58:00 | E049 | Y |
| IVACFLU-S-0203-203-SE122 (E073) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:24:00 | E073 | Y |
| IVACFLU-S-0203-203-SE123 (E076) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:35:00 | E076 | Y |
| IVACFLU-S-0203-203-SE124 (E080) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:20:00 | E080 | Y |
| IVACFLU-S-0203-203-SE125() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE126 (E186) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:18:00 | E186 | Y |
| IVACFLU-S-0203-203-SE127 (E189) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:35:00 | E189 | Y |
| IVACFLU-S-0203-203-SE128 (E177) | IVACFLU-S | IVACFLU-S | 09Jul2017:16:31:00 | E177 | Y |
| IVACFLU-S-0203-203-SE129 (E062) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:09:00 | E062 | Y |
| IVACFLU-S-0203-203-SE130 (E083) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:39:00 | E083 | Y |
| IVACFLU-S-0203-203-SE131() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE132() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE133() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE134 (E082) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:27:00 | E082 | Y |
| IVACFLU-S-0203-203-SE135 (E112) | PLACEBO | PLACEBO | 07Jul2017:16:59:00 | E112 | Y |
| IVACFLU-S-0203-203-SE136 (E084) | PLACEBO | PLACEBO | 06Jul2017:15:44:00 | E084 | Y |
| IVACFLU-S-0203-203-SE137 (E042) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:04:00 | E042 | Y |
| IVACFLU-S-0203-203-SE138 (E072) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:21:00 | E072 | Y |
| IVACFLU-S-0203-203-SE139 (E111) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:55:00 | E111 | Y |
| IVACFLU-S-0203-203-SE140 (E160) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:31:00 | E160 | Y |
| IVACFLU-S-0203-203-SE141 (E163) | PLACEBO | PLACEBO | 09Jul2017:08:55:00 | E163 | Y |
| IVACFLU-S-0203-203-SE142 (E184) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:06:00 | E184 | Y |

Protocol No: IVACFLU-S-0203 724 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE143 (E191) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:02:00 | E191 | Y |
| IVACFLU-S-0203-203-SE144() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE145 (E161) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:39:00 | E161 | Y |
| IVACFLU-S-0203-203-SE146 (E074) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:28:00 | E074 | Y |
| IVACFLU-S-0203-203-SE147() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE148 (E175) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:12:00 | E175 | Y |
| IVACFLU-S-0203-203-SE149 (E055) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:49:00 | E055 | Y |
| IVACFLU-S-0203-203-SE150 (E168) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:13:00 | E168 | Y |
| IVACFLU-S-0203-203-SE151 (E067) | PLACEBO | PLACEBO | 06Jul2017:13:46:00 | E067 | Y |
| IVACFLU-S-0203-203-SE152() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE153() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE154 (E100) | IVACFLU-S | IVACFLU-S | 07Jul2017:13:46:00 | E100 | Y |
| IVACFLU-S-0203-203-SE155() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE156 (E106) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:12:00 | E106 | Y |
| IVACFLU-S-0203-203-SE157 (E097) | PLACEBO | PLACEBO | 07Jul2017:11:19:00 | E097 | Y |
| IVACFLU-S-0203-203-SE158 (E093) | IVACFLU-S | IVACFLU-S | 07Jul2017:11:02:00 | E093 | Y |
| IVACFLU-S-0203-203-SE159() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE160 (E088) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:41:00 | E088 | Y |
| IVACFLU-S-0203-203-SE161 (E110) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:00:00 | E110 | Y |
| IVACFLU-S-0203-203-SE162 (E098) | IVACFLU-S | IVACFLU-S | 07Jul2017:11:23:00 | E098 | Y |
| IVACFLU-S-0203-203-SE163() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE164() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE165 (E087) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:30:00 | E087 | Y |
| IVACFLU-S-0203-203-SE166 (E104) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:18:00 | E104 | Y |
| IVACFLU-S-0203-203-SE167 (E096) | IVACFLU-S | IVACFLU-S | 07Jul2017:11:15:00 | E096 | Y |
| IVACFLU-S-0203-203-SE168 (E156) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:11:00 | E156 | Y |
| IVACFLU-S-0203-203-SE169() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE170 (E162) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:48:00 | E162 | Y |
| IVACFLU-S-0203-203-SE171 (E094) | PLACEBO | PLACEBO | 07Jul2017:11:06:00 | E094 | Y |
| IVACFLU-S-0203-203-SE172 (E101) | IVACFLU-S | IVACFLU-S | 07Jul2017:13:51:00 | E101 | Y |
| IVACFLU-S-0203-203-SE173() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE174() | SCREEN FAILURE | SCREEN FAILURE | - | | |
| IVACFLU-S-0203-203-SE175() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE176 (E099) | IVACFLU-S | IVACFLU-S | 07Jul2017:13:42:00 | E099 | Y |
| IVACFLU-S-0203-203-SE177 (E108) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:48:00 | E108 | Y |
| IVACFLU-S-0203-203-SE178 (E105) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:23:00 | E105 | Y |

Version 1.0 Protocol No: IVACFLU-S-0203 725 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE179() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE180() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE181() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE182 (E102) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:04:00 | E102 | Y |
| IVACFLU-S-0203-203-SE183() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE184 (E091) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:18:00 | E091 | Y |
| IVACFLU-S-0203-203-SE185 (E092) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:36:00 | E092 | Y |
| IVACFLU-S-0203-203-SE186 (E167) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:52:00 | E167 | Y |
| IVACFLU-S-0203-203-SE187 (E089) | PLACEBO | PLACEBO | 07Jul2017:09:46:00 | E089 | Y |
| IVACFLU-S-0203-203-SE188 (E095) | IVACFLU-S | IVACFLU-S | 07Jul2017:11:10:00 | E095 | Y |
| IVACFLU-S-0203-203-SE189 (E107) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:40:00 | E107 | Y |
| IVACFLU-S-0203-203-SE190 (E086) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:19:00 | E086 | Y |
| IVACFLU-S-0203-203-SE191() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE192 (E109) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:56:00 | E109 | Y |
| IVACFLU-S-0203-203-SE193 (E103) | PLACEBO | PLACEBO | 07Jul2017:14:09:00 | E103 | Y |
| IVACFLU-S-0203-203-SE194() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE195 (E157) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:14:00 | E157 | Y |
| IVACFLU-S-0203-203-SE196 (E090) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:51:00 | E090 | Y |
| IVACFLU-S-0203-203-SE197() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE198 (E129) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:06:00 | E129 | Y |
| IVACFLU-S-0203-203-SE199 (E148) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:31:00 | E148 | Y |
| IVACFLU-S-0203-203-SE200 (E121) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:37:00 | E121 | Y |
| IVACFLU-S-0203-203-SE201 (E147) | PLACEBO | PLACEBO | 08Jul2017:15:28:00 | E147 | Y |
| IVACFLU-S-0203-203-SE202 (E113) | IVACFLU-S | IVACFLU-S | 08Jul2017:07:55:00 | E113 | Y |
| IVACFLU-S-0203-203-SE203() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE204 (E137) | IVACFLU-S | IVACFLU-S | 08Jul2017:13:37:00 | E137 | Y |
| IVACFLU-S-0203-203-SE205 (E146) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:10:00 | E146 | Y |
| IVACFLU-S-0203-203-SE206 (E123) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:57:00 | E123 | Y |
| IVACFLU-S-0203-203-SE207 (E150) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:38:00 | E150 | Y |
| IVACFLU-S-0203-203-SE208 (E143) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:35:00 | E143 | Y |
| IVACFLU-S-0203-203-SE209 (E114) | IVACFLU-S | IVACFLU-S | 08Jul2017:07:59:00 | E114 | Y |
| IVACFLU-S-0203-203-SE210 (E135) | PLACEBO | PLACEBO | 08Jul2017:10:57:00 | E135 | Y |
| IVACFLU-S-0203-203-SE211() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE212 (E134) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:52:00 | E134 | Y |
| IVACFLU-S-0203-203-SE213 (E124) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:18:00 | E124 | Y |
| IVACFLU-S-0203-203-SE214 (E127) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:45:00 | E127 | Y |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 726 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE215 (E169) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:53:00 | E169 | Y |
| IVACFLU-S-0203-203-SE216 (E116) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:13:00 | E116 | Y |
| IVACFLU-S-0203-203-SE217() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE218 (E138) | IVACFLU-S | IVACFLU-S | 08Jul2017:13:41:00 | E138 | Y |
| IVACFLU-S-0203-203-SE219 (E119) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:29:00 | E119 | Y |
| IVACFLU-S-0203-203-SE220() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE221 (E128) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:00:00 | E128 | Y |
| IVACFLU-S-0203-203-SE222 (E144) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:39:00 | E144 | Y |
| IVACFLU-S-0203-203-SE223 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE224 (E131) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:18:00 | E131 | Y |
| IVACFLU-S-0203-203-SE225 (E151) | PLACEBO | PLACEBO | 08Jul2017:15:59:00 | E151 | Y |
| IVACFLU-S-0203-203-SE226() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE227() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE228 (E118) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:26:00 | E118 | Y |
| IVACFLU-S-0203-203-SE229() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE230 (E153) | IVACFLU-S | IVACFLU-S | 08Jul2017:16:19:00 | E153 | Y |
| IVACFLU-S-0203-203-SE231 (E149) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:35:00 | E149 | Y |
| IVACFLU-S-0203-203-SE232() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE233 (E130) | PLACEBO | PLACEBO | 08Jul2017:10:10:00 | E130 | Y |
| IVACFLU-S-0203-203-SE234() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE235 (E115) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:04:00 | E115 | Y |
| IVACFLU-S-0203-203-SE236() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE237() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE238 (E152) | IVACFLU-S | IVACFLU-S | 08Jul2017:16:10:00 | E152 | Y |
| IVACFLU-S-0203-203-SE239 (E132) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:22:00 | E132 | Y |
| IVACFLU-S-0203-203-SE240() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE241 (E122) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:49:00 | E122 | Y |
| IVACFLU-S-0203-203-SE242() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE243 (E126) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:40:00 | E126 | Y |
| IVACFLU-S-0203-203-SE244() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE245 (E145) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:43:00 | E145 | Y |
| IVACFLU-S-0203-203-SE246 (E120) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:33:00 | E120 | Y |
| IVACFLU-S-0203-203-SE247() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE248 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE249 (E125) | PLACEBO | PLACEBO | 08Jul2017:09:22:00 | E125 | Y |
| IVACFLU-S-0203-203-SE250 (E139) | PLACEBO | PLACEBO | 08Jul2017:14:01:00 | E139 | Y |

Protocol No: IVACFLU-S-0203 727 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SE251() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE252 (E176) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:19:00 | E176 | Y |
| IVACFLU-S-0203-203-SE253 (E192) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:18:00 | E192 | Y |
| IVACFLU-S-0203-203-SE254 (E141) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:12:00 | E141 | Y |
| IVACFLU-S-0203-203-SE255 (E117) | PLACEBO | PLACEBO | 08Jul2017:08:16:00 | E117 | Y |
| IVACFLU-S-0203-203-SE256() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE257 (E142) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:22:00 | E142 | Y |
| IVACFLU-S-0203-203-SE258 (E133) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:41:00 | E133 | Y |
| IVACFLU-S-0203-203-SE259() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE260() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SE261 (E140) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:08:00 | E140 | Y |
| IVACFLU-S-0203-203-SE262 (E188) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:32:00 | E188 | Y |
| IVACFLU-S-0203-203-SE263 (E136) | IVACFLU-S | IVACFLU-S | 08Jul2017:11:02:00 | E136 | Y |
| IVACFLU-S-0203-203-SG001 (G187) | PLACEBO | PLACEBO | 10Jul2017:08:49:00 | G187 | Y |
| IVACFLU-S-0203-203-SG002 (G014) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:12:00 | G014 | Y |
| IVACFLU-S-0203-203-SG003 (G004) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:29:00 | G004 | Y |
| IVACFLU-S-0203-203-SG004() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG005() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG006 (G002) | IVACFLU-S | IVACFLU-S | 05Jul2017:08:28:00 | G002 | Y |
| IVACFLU-S-0203-203-SG007() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG008 (G010) | PLACEBO | PLACEBO | 05Jul2017:14:31:00 | G010 | Y |
| IVACFLU-S-0203-203-SG009() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG010 (G020) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:10:00 | G020 | Y |
| IVACFLU-S-0203-203-SG011() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG012 (G005) | IVACFLU-S | IVACFLU-S | 05Jul2017:09:47:00 | G005 | Y |
| IVACFLU-S-0203-203-SG013() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG014 (G006) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:18:00 | G006 | Y |
| IVACFLU-S-0203-203-SG015() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG016 (G011) | IVACFLU-S | IVACFLU-S | 05Jul2017:14:59:00 | G011 | Y |
| IVACFLU-S-0203-203-SG017 (G007) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:23:00 | G007 | Y |
| IVACFLU-S-0203-203-SG018 (G016) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:25:00 | G016 | Y |
| IVACFLU-S-0203-203-SG019() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG020() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG021() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG022 (G001) | IVACFLU-S | IVACFLU-S | 05Jul2017:08:07:00 | G001 | Y |
| IVACFLU-S-0203-203-SG023() | SCREEN FAILURE | SCREEN FAILURE | | | |


| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG024 (G013) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:33:00 | G013 | Y |
| IVACFLU-S-0203-203-SG025() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG026() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG027() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG028 (G003) | PLACEBO | PLACEBO | 05Jul2017:08:46:00 | G003 | Y |
| IVACFLU-S-0203-203-SG029() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG030() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG031() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG032() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG033 (G015) | PLACEBO | PLACEBO | 05Jul2017:16:20:00 | G015 | Y |
| IVACFLU-S-0203-203-SG034 (G023) | PLACEBO | PLACEBO | 05Jul2017:17:38:00 | G023 | Y |
| IVACFLU-S-0203-203-SG035 (G022) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:22:00 | G022 | Y |
| IVACFLU-S-0203-203-SG036 (G021) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:18:00 | G021 | Y |
| IVACFLU-S-0203-203-SG037 (G145) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:35:00 | G145 | Y |
| IVACFLU-S-0203-203-SG038() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG039() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG040 (G008) | IVACFLU-S | IVACFLU-S | 05Jul2017:10:54:00 | G008 | Y |
| IVACFLU-S-0203-203-SG041 (G143) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:08:00 | G143 | Y |
| IVACFLU-S-0203-203-SG042 (G012) | IVACFLU-S | IVACFLU-S | 05Jul2017:15:11:00 | G012 | Y |
| IVACFLU-S-0203-203-SG043 (G142) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:04:00 | G142 | Y |
| IVACFLU-S-0203-203-SG044 (G147) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:03:00 | G147 | Y |
| IVACFLU-S-0203-203-SG045 (G017) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:41:00 | G017 | Y |
| IVACFLU-S-0203-203-SG046() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG047() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG048 (G140) | IVACFLU-S | IVACFLU-S | 08Jul2017:16:05:00 | G140 | Y |
| IVACFLU-S-0203-203-SG049 (G019) | IVACFLU-S | IVACFLU-S | 05Jul2017:17:06:00 | G019 | Y |
| IVACFLU-S-0203-203-SG050 (G144) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:26:00 | G144 | Y |
| IVACFLU-S-0203-203-SG051() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG052 (G155) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:09:00 | G155 | Y |
| IVACFLU-S-0203-203-SG053 (G166) | IVACFLU-S | IVACFLU-S | 09Jul2017:13:49:00 | G166 | Y |
| IVACFLU-S-0203-203-SG054 (G009) | IVACFLU-S | IVACFLU-S | 05Jul2017:11:06:00 | G009 | Y |
| IVACFLU-S-0203-203-SG055 (G183) | IVACFLU-S | IVACFLU-S | 09Jul2017:16:19:00 | G183 | Y |
| IVACFLU-S-0203-203-SG056() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG057 (G176) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:27:00 | G176 | Y |
| IVACFLU-S-0203-203-SG058 (G178) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:44:00 | G178 | Y |
| IVACFLU-S-0203-203-SG059() | SCREEN FAILURE | SCREEN FAILURE | | | |

728

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 729 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG060() | SCREEN FAILURE | SCREEN FAILURE | | Number | Flag |
| IVACFLU-S-0203-203-SG061 (G123) | PLACEBO | PLACEBO | 08Jul2017:11:07:00 | G123 | Y |
| IVACFLU-S-0203-203-SG062 ( ) | SCREEN FAILURE | SCREEN FAILURE | 003412017.11.07.00 | 0123 | 1 |
| IVACFLU-S-0203-203-SG063 (G018) | IVACFLU-S | IVACFLU-S | 05Jul2017:16:49:00 | G018 | Y |
| IVACFLU-S-0203-203-SG064 ( ) | SCREEN FAILURE | SCREEN FAILURE | 0.53412017.10.15.00 | 3010 | 1 |
| IVACFLU-S-0203-203-SG065 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG066 (G150) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:22:00 | G150 | Y |
| IVACFLU-S-0203-203-SG067 (G179) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:48:00 | G179 | Y |
| IVACFLU-S-0203-203-SG068 ( ) | SCREEN FAILURE | SCREEN FAILURE | 0,0000000000000000000000000000000000000 | 01// | |
| IVACFLU-S-0203-203-SG069 (G040) | PLACEBO | PLACEBO | 06Jul2017:10:41:00 | G040 | Y |
| IVACFLU-S-0203-203-SG070 (G043) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:06:00 | G043 | Y |
| IVACFLU-S-0203-203-SG071 (G039) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:37:00 | G039 | Y |
| IVACFLU-S-0203-203-SG072 (G025) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:08:00 | G025 | Y |
| IVACFLU-S-0203-203-SG073 (G037) | PLACEBO | PLACEBO | 06Jul2017:10:22:00 | G037 | Y |
| IVACFLU-S-0203-203-SG074 (G030) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:34:00 | G030 | Y |
| IVACFLU-S-0203-203-SG075() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG076 (G028) | PLACEBO | PLACEBO | 06Jul2017:09:24:00 | G028 | Y |
| IVACFLU-S-0203-203-SG077() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG078() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG079 (G044) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:12:00 | G044 | Y |
| IVACFLU-S-0203-203-SG080 (G032) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:55:00 | G032 | Y |
| IVACFLU-S-0203-203-SG081() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG082() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG083() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG084 (G054) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:01:00 | G054 | Y |
| IVACFLU-S-0203-203-SG085() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG086 (G042) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:53:00 | G042 | Y |
| IVACFLU-S-0203-203-SG087() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG088 (G036) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:18:00 | G036 | Y |
| IVACFLU-S-0203-203-SG089() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG090() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG091 (G052) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:49:00 | G052 | Y |
| IVACFLU-S-0203-203-SG092() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG093 (G159) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:28:00 | G159 | Y |
| IVACFLU-S-0203-203-SG094 (G035) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:09:00 | G035 | Y |
| IVACFLU-S-0203-203-SG095() | SCREEN FAILURE | SCREEN FAILURE | | | |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization | Randomization |
|---|---|---|---|---|---|
| | | | | Number | Flag |
| IVACFLU-S-0203-203-SG096 (G029) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:28:00 | G029 | Y |
| IVACFLU-S-0203-203-SG097 (G045) | NOT ASSIGNED | NOT ASSIGNED | 06Jul2017:00:00:00 | | Y |
| IVACFLU-S-0203-203-SG098 (G034) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:04:00 | G034 | Y |
| IVACFLU-S-0203-203-SG099 (G046) | IVACFLU-S | IVACFLU-S | 06Jul2017:11:20:00 | G046 | Y |
| IVACFLU-S-0203-203-SG100 (G033) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:00:00 | G033 | Y |
| IVACFLU-S-0203-203-SG101 (G041) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:47:00 | G041 | Y |
| IVACFLU-S-0203-203-SG102 (G097) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:17:00 | G097 | Y |
| IVACFLU-S-0203-203-SG103 (G100) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:30:00 | G100 | Y |
| IVACFLU-S-0203-203-SG104() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG105 (G038) | IVACFLU-S | IVACFLU-S | 06Jul2017:10:33:00 | G038 | Y |
| IVACFLU-S-0203-203-SG106 (G153) | PLACEBO | PLACEBO | 09Jul2017:10:06:00 | G153 | Y |
| IVACFLU-S-0203-203-SG107 (G031) | IVACFLU-S | IVACFLU-S | 06Jul2017:09:43:00 | G031 | Y |
| IVACFLU-S-0203-203-SG108 (G057) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:12:00 | G057 | Y |
| IVACFLU-S-0203-203-SG109 (G053) | PLACEBO | PLACEBO | 06Jul2017:14:57:00 | G053 | Y |
| IVACFLU-S-0203-203-SG110() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG111() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG112() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG113 (G141) | PLACEBO | PLACEBO | 09Jul2017:07:58:00 | G141 | Y |
| IVACFLU-S-0203-203-SG114 (G050) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:14:00 | G050 | Y |
| IVACFLU-S-0203-203-SG115 (G026) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:13:00 | G026 | Y |
| IVACFLU-S-0203-203-SG116 (G059) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:13:00 | G059 | Y |
| IVACFLU-S-0203-203-SG117 (G062) | IVACFLU-S | IVACFLU-S | 06Jul2017:16:02:00 | G062 | Y |
| IVACFLU-S-0203-203-SG118() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG119() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG120 (G027) | IVACFLU-S | IVACFLU-S | 06Jul2017:08:19:00 | G027 | Y |
| IVACFLU-S-0203-203-SG121() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG122 (G055) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:05:00 | G055 | Y |
| IVACFLU-S-0203-203-SG123 (G169) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:19:00 | G169 | Y |
| IVACFLU-S-0203-203-SG124 (G096) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:12:00 | G096 | Y |
| IVACFLU-S-0203-203-SG125() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG126 (G024) | IVACFLU-S | IVACFLU-S | 06Jul2017:07:58:00 | G024 | Y |
| IVACFLU-S-0203-203-SG127() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG128 (G051) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:46:00 | G051 | Y |
| IVACFLU-S-0203-203-SG129 (G148) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:10:00 | G148 | Y |
| IVACFLU-S-0203-203-SG130 (G058) | PLACEBO | PLACEBO | 06Jul2017:15:16:00 | G058 | Y |
| IVACFLU-S-0203-203-SG131() | SCREEN FAILURE | SCREEN FAILURE | | | |

Version 1.0 Protocol No: IVACFLU-S-0203 731 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization | Randomization |
|---|---|---|---|---|---|
| | | | | Number | Flag |
| IVACFLU-S-0203-203-SG132 (G161) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:40:00 | G161 | Y |
| IVACFLU-S-0203-203-SG133 (G095) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:08:00 | G095 | Y |
| IVACFLU-S-0203-203-SG134 (G094) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:04:00 | G094 | Y |
| IVACFLU-S-0203-203-SG135() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG136() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG137 (G102) | PLACEBO | PLACEBO | 07Jul2017:16:38:00 | G102 | Y |
| IVACFLU-S-0203-203-SG138() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG139() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG140() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG141 (G157) | PLACEBO | PLACEBO | 09Jul2017:10:21:00 | G157 | Y |
| IVACFLU-S-0203-203-SG142 (G152) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:46:00 | G152 | Y |
| IVACFLU-S-0203-203-SG143 (G189) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:59:00 | G189 | Y |
| IVACFLU-S-0203-203-SG144 (G158) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:24:00 | G158 | Y |
| IVACFLU-S-0203-203-SG145 (G146) | IVACFLU-S | IVACFLU-S | 09Jul2017:08:59:00 | G146 | Y |
| IVACFLU-S-0203-203-SG146 (G060) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:48:00 | G060 | Y |
| IVACFLU-S-0203-203-SG147() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG148 (G048) | PLACEBO | PLACEBO | 06Jul2017:14:08:00 | G048 | Y |
| IVACFLU-S-0203-203-SG149 (G156) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:17:00 | G156 | Y |
| IVACFLU-S-0203-203-SG150 (G101) | PLACEBO | PLACEBO | 07Jul2017:16:46:00 | G101 | Y |
| IVACFLU-S-0203-203-SG151() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG152 (G049) | IVACFLU-S | IVACFLU-S | 06Jul2017:14:11:00 | G049 | Y |
| IVACFLU-S-0203-203-SG153() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG154() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG155 (G138) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:51:00 | G138 | Y |
| IVACFLU-S-0203-203-SG156 (G103) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:50:00 | G103 | Y |
| IVACFLU-S-0203-203-SG157() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG158() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG159 (G174) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:43:00 | G174 | Y |
| IVACFLU-S-0203-203-SG160() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG161 (G099) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:26:00 | G099 | Y |
| IVACFLU-S-0203-203-SG162() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG163() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG164 (G047) | IVACFLU-S | IVACFLU-S | 06Jul2017:13:53:00 | G047 | Y |
| IVACFLU-S-0203-203-SG165 (G056) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:09:00 | G056 | Y |
| IVACFLU-S-0203-203-SG166() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG167() | SCREEN FAILURE | SCREEN FAILURE | | | |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG168() | SCREEN FAILURE | SCREEN FAILURE | | Number | Flag |
| IVACFLU-S-0203-203-SG169 (G181) | IVACFLU-S | IVACFLU-S | 09Jul2017:16:12:00 | G181 | Y |
| IVACFLU-S-0203-203-SG170 ( ) | SCREEN FAILURE | SCREEN FAILURE | | 0101 | |
| IVACFLU-S-0203-203-SG171 (G171) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:26:00 | G171 | Y |
| IVACFLU-S-0203-203-SG172 (G061) | IVACFLU-S | IVACFLU-S | 06Jul2017:15:56:00 | G061 | Y |
| IVACFLU-S-0203-203-SG173() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG174() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG175 (G098) | IVACFLU-S | IVACFLU-S | 07Jul2017:16:21:00 | G098 | Y |
| IVACFLU-S-0203-203-SG176() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG177 (G173) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:35:00 | G173 | Y |
| IVACFLU-S-0203-203-SG178 (G081) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:44:00 | G081 | Y |
| IVACFLU-S-0203-203-SG179() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG180 (G080) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:32:00 | G080 | Y |
| IVACFLU-S-0203-203-SG181 (G069) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:42:00 | G069 | Y |
| IVACFLU-S-0203-203-SG182 (G078) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:23:00 | G078 | Y |
| IVACFLU-S-0203-203-SG183() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG184 (G077) | PLACEBO | PLACEBO | 07Jul2017:10:12:00 | G077 | Y |
| IVACFLU-S-0203-203-SG185() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG186 (G079) | PLACEBO | PLACEBO | 07Jul2017:10:27:00 | G079 | Y |
| IVACFLU-S-0203-203-SG187() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG188() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG189 (G092) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:17:00 | G092 | Y |
| IVACFLU-S-0203-203-SG190() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG191 (G064) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:11:00 | G064 | Y |
| IVACFLU-S-0203-203-SG192() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG193 (G072) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:00:00 | G072 | Y |
| IVACFLU-S-0203-203-SG194() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG195 (G084) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:57:00 | G084 | Y |
| IVACFLU-S-0203-203-SG196() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG197 (G075) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:56:00 | G075 | Y |
| IVACFLU-S-0203-203-SG198 (G066) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:25:00 | G066 | Y |
| IVACFLU-S-0203-203-SG199 (G082) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:49:00 | G082 | Y |
| IVACFLU-S-0203-203-SG200() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG201() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG202() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG203 (G083) | IVACFLU-S | IVACFLU-S | 07Jul2017:10:53:00 | G083 | Y |

732


Protocol No: IVACFLU-S-0203 733 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG204() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG205() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG206 (G090) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:43:00 | G090 | Y |
| IVACFLU-S-0203-203-SG207 (G088) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:28:00 | G088 | Y |
| IVACFLU-S-0203-203-SG208 (G085) | IVACFLU-S | IVACFLU-S | 07Jul2017:11:26:00 | G085 | Y |
| IVACFLU-S-0203-203-SG209 (G172) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:29:00 | G172 | Y |
| IVACFLU-S-0203-203-SG210 (G068) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:37:00 | G068 | Y |
| IVACFLU-S-0203-203-SG211() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG212 (G071) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:55:00 | G071 | Y |
| IVACFLU-S-0203-203-SG213() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG214() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG215 (G063) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:05:00 | G063 | Y |
| IVACFLU-S-0203-203-SG216() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG217 (G091) | PLACEBO | PLACEBO | 07Jul2017:15:04:00 | G091 | Y |
| IVACFLU-S-0203-203-SG218() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG219() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG220() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG221() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG222 (G170) | PLACEBO | PLACEBO | 09Jul2017:14:23:00 | G170 | Y |
| IVACFLU-S-0203-203-SG223() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG224 (G093) | IVACFLU-S | IVACFLU-S | 07Jul2017:15:26:00 | G093 | Y |
| IVACFLU-S-0203-203-SG225 (G167) | IVACFLU-S | IVACFLU-S | 09Jul2017:13:53:00 | G167 | Y |
| IVACFLU-S-0203-203-SG226 (G177) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:32:00 | G177 | Y |
| IVACFLU-S-0203-203-SG227() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG228() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG229() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG230 (G115) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:53:00 | G115 | Y |
| IVACFLU-S-0203-203-SG231() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG232 (G120) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:33:00 | G120 | Y |
| IVACFLU-S-0203-203-SG233() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG234() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG235 (G188) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:56:00 | G188 | Y |
| IVACFLU-S-0203-203-SG236 (G116) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:56:00 | G116 | Y |
| IVACFLU-S-0203-203-SG237 (G135) | PLACEBO | PLACEBO | 08Jul2017:15:20:00 | G135 | Y |
| IVACFLU-S-0203-203-SG238 (G104) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:08:00 | G104 | Y |
| IVACFLU-S-0203-203-SG239 (G108) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:01:00 | G108 | Y |


Protocol No: IVACFLU-S-0203 734 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG240 (G113) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:30:00 | G113 | Y |
| IVACFLU-S-0203-203-SG241() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG242 (G112) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:26:00 | G112 | Y |
| IVACFLU-S-0203-203-SG243() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG244() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG245() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG246() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG247 (G124) | IVACFLU-S | IVACFLU-S | 08Jul2017:13:47:00 | G124 | Y |
| IVACFLU-S-0203-203-SG248 (G130) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:31:00 | G130 | Y |
| IVACFLU-S-0203-203-SG249 (G107) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:45:00 | G107 | Y |
| IVACFLU-S-0203-203-SG250() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG251() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG252 (G118) | PLACEBO | PLACEBO | 08Jul2017:10:26:00 | G118 | Y |
| IVACFLU-S-0203-203-SG253 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG254() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG255() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG256 (G121) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:37:00 | G121 | Y |
| IVACFLU-S-0203-203-SG257 (G110) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:09:00 | G110 | Y |
| IVACFLU-S-0203-203-SG258() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG259() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG260 (G164) | PLACEBO | PLACEBO | 09Jul2017:10:50:00 | G164 | Y |
| IVACFLU-S-0203-203-SG261() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG262() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG263 (G132) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:56:00 | G132 | Y |
| IVACFLU-S-0203-203-SG264 (G109) | PLACEBO | PLACEBO | 08Jul2017:09:05:00 | G109 | Y |
| IVACFLU-S-0203-203-SG265 (G128) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:05:00 | G128 | Y |
| IVACFLU-S-0203-203-SG266 (G126) | IVACFLU-S | IVACFLU-S | 08Jul2017:13:54:00 | G126 | Y |
| IVACFLU-S-0203-203-SG267 (G129) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:15:00 | G129 | Y |
| IVACFLU-S-0203-203-SG268 (G111) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:15:00 | G111 | Y |
| IVACFLU-S-0203-203-SG269 (G122) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:45:00 | G122 | Y |
| IVACFLU-S-0203-203-SG270() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG271 (G134) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:16:00 | G134 | Y |
| IVACFLU-S-0203-203-SG272() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG273 (G106) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:41:00 | G106 | Y |
| IVACFLU-S-0203-203-SG274() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG275() | SCREEN FAILURE | SCREEN FAILURE | | | |

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 735 Dated: 12 March 2018

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG276 (G127) | PLACEBO | PLACEBO | 08Jul2017:13:58:00 | G127 | Y |
| IVACFLU-S-0203-203-SG277 (G137) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:46:00 | G127 | Y |
| IVACFLU-S-0203-203-SG277 (G137) | IVACFLU-S | IVACFLU-S | 08Jul2017:13:51:00 | G125 | Y |
| IVACFLU-S-0203-203-SG278 (G123) | SCREEN FAILURE | SCREEN FAILURE | 083412017.13.31.00 | 0123 | 1 |
| IVACFLU-S-0203-203-SG280() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG280 () | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG282 (G105) | IVACFLU-S | IVACFLU-S | 08Jul2017:08:20:00 | G105 | Y |
| IVACFLU-S-0203-203-SG283 ( ) | SCREEN FAILURE | SCREEN FAILURE | 003412017.00.20.00 | 0103 | 1 |
| IVACFLU-S-0203-203-SG284 (G119) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:30:00 | G119 | Y |
| IVACFLU-S-0203-203-SG285 (G131) | IVACFLU-S | IVACFLU-S | 08Jul2017:14:52:00 | G131 | Y |
| IVACFLU-S-0203-203-SG286 ( ) | SCREEN FAILURE | SCREEN FAILURE | 003412017.11.32.00 | G151 | 1 |
| IVACFLU-S-0203-203-SG287 (G114) | IVACFLU-S | IVACFLU-S | 08Jul2017:09:49:00 | G114 | Y |
| IVACFLU-S-0203-203-SG288 ( ) | SCREEN FAILURE | SCREEN FAILURE | 000 012 017.09.19.00 | 0111 | |
| IVACFLU-S-0203-203-SG289 (G160) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:32:00 | G160 | Y |
| IVACFLU-S-0203-203-SG290 ( ) | SCREEN FAILURE | SCREEN FAILURE | | 0111 | |
| IVACFLU-S-0203-203-SG291 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG292 (G162) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:43:00 | G162 | Y |
| IVACFLU-S-0203-203-SG293 (G149) | PLACEBO | PLACEBO | 09Jul2017:09:18:00 | G149 | Y |
| IVACFLU-S-0203-203-SG294() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG295() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG296 ( ) | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG297() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG298() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG299() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG300 (G139) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:55:00 | G139 | Y |
| IVACFLU-S-0203-203-SG301 (G133) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:24:00 | G133 | Y |
| IVACFLU-S-0203-203-SG302() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG303 (G180) | PLACEBO | PLACEBO | 09Jul2017:15:51:00 | G180 | Y |
| IVACFLU-S-0203-203-SG304() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG305 (G151) | IVACFLU-S | IVACFLU-S | 09Jul2017:09:39:00 | G151 | Y |
| IVACFLU-S-0203-203-SG306() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG307 (G163) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:47:00 | G163 | Y |
| IVACFLU-S-0203-203-SG308 (G186) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:39:00 | G186 | Y |
| IVACFLU-S-0203-203-SG309 (G182) | IVACFLU-S | IVACFLU-S | 09Jul2017:16:16:00 | G182 | Y |
| IVACFLU-S-0203-203-SG310 (G136) | IVACFLU-S | IVACFLU-S | 08Jul2017:15:42:00 | G136 | Y |
| IVACFLU-S-0203-203-SG311 (G154) | IVACFLU-S | IVACFLU-S | 09Jul2017:10:03:00 | G154 | Y |

| Unique Subject Identifier | Planned Treatment | Actual Treatment | Date of Randomization | Randomization<br>Number | Randomization<br>Flag |
|---|---|---|---|---|---|
| IVACFLU-S-0203-203-SG312() | SCREEN FAILURE | SCREEN FAILURE | | 3 (3333 & 33 | |
| IVACFLU-S-0203-203-SG313() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG314 (G117) | IVACFLU-S | IVACFLU-S | 08Jul2017:10:14:00 | G117 | Y |
| IVACFLU-S-0203-203-SG315() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG316() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG317() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG318 (G089) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:37:00 | G089 | Y |
| IVACFLU-S-0203-203-SG319 (G065) | PLACEBO | PLACEBO | 07Jul2017:08:19:00 | G065 | Y |
| IVACFLU-S-0203-203-SG320 (G175) | IVACFLU-S | IVACFLU-S | 09Jul2017:15:01:00 | G175 | Y |
| IVACFLU-S-0203-203-SG321() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG322() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG323() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG324 (G074) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:35:00 | G074 | Y |
| IVACFLU-S-0203-203-SG325 (G070) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:47:00 | G070 | Y |
| IVACFLU-S-0203-203-SG326() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG327() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG328 (G067) | IVACFLU-S | IVACFLU-S | 07Jul2017:08:30:00 | G067 | Y |
| IVACFLU-S-0203-203-SG329() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG330 (G073) | IVACFLU-S | IVACFLU-S | 07Jul2017:09:24:00 | G073 | Y |
| IVACFLU-S-0203-203-SG331 (G076) | PLACEBO | PLACEBO | 07Jul2017:10:00:00 | G076 | Y |
| IVACFLU-S-0203-203-SG332() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG333 (G087) | PLACEBO | PLACEBO | 07Jul2017:14:14:00 | G087 | Y |
| IVACFLU-S-0203-203-SG334 (G168) | IVACFLU-S | IVACFLU-S | 09Jul2017:14:07:00 | G168 | Y |
| IVACFLU-S-0203-203-SG335 (G086) | IVACFLU-S | IVACFLU-S | 07Jul2017:14:00:00 | G086 | Y |
| IVACFLU-S-0203-203-SG336 (G165) | IVACFLU-S | IVACFLU-S | 09Jul2017:13:45:00 | G165 | Y |
| IVACFLU-S-0203-203-SG337 (G184) | PLACEBO | PLACEBO | 10Jul2017:07:52:00 | G184 | Y |
| IVACFLU-S-0203-203-SG338 (G193) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:21:00 | G193 | Y |
| IVACFLU-S-0203-203-SG339 (G190) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:07:00 | G190 | Y |
| IVACFLU-S-0203-203-SG340 (G192) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:14:00 | G192 | Y |
| IVACFLU-S-0203-203-SG341() | SCREEN FAILURE | SCREEN FAILURE | | | |
| IVACFLU-S-0203-203-SG342 (G185) | IVACFLU-S | IVACFLU-S | 10Jul2017:08:29:00 | G185 | Y |
| IVACFLU-S-0203-203-SG343 (G191) | IVACFLU-S | IVACFLU-S | 10Jul2017:09:11:00 | G191 | Y |
| IVACFLU-S-0203-203-SG344() | SCREEN FAILURE | SCREEN FAILURE | | | |



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

## Randomization Specification

## MINISTRY OF HEALTH

#### RESEARCH PROTOCOL OF VACCINE CLINICAL TRIAL

A PHASE 2/3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF A SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

Study Number: IVACFLU-S-0203

Author: Maria Efstathiou **Department: Biostatistics** 

QuintilesIMS QTHV

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\TVACFLU-S-0203 RandoSpec BLINDED 2017 03 31 v2 0

Author: Maria Efstathiou Version Number: 2.0 Version Date: 31MAR2017

Reference: CS\_WI\_BS002

Template No: CS\_TP\_BS025 Revision 5


Protocol No: IVACFLU-S-0203 738

QuintilesIMS

Randomization Specification

PATH / IVAC IVACFLU-S-0203 

Dated: 12 March 2018

# **Authorization**

| Randomization Biostatistician (required): | Maria Efstathiou Name | Signature Signature | 07AUG 2017<br>Date |
|---|---|---|---|
| Statistical Team Lead: | Suman Kapoor<br>Name | Signature | Date |
| Randomization Implementer (required): | <u>Dr Phan Cong Hung</u><br>Name | Signature | Date |
| Customer approval (if required): | Tushar Tewari<br>Name | Signature | Date |
| | Thang Tran Name | Signature | Date |

Document:

\\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0.docx

Author:

Maria Efstathiou

Version Number:

2.0

A - 2 2000 No.


31MAR2017

Template No: CS\_TP\_BS025 Revision 5

Effective Date: 01Nov2016

Reference: CS\_WI\_BS002

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Dated: 12 March 2018



PATH / IVAC IVACFLU-S-0203 

# Authorization

| Randomization Biostatistician (required): Statistical Team Lead: | Maria Efstathiou Name Suman Kapoor Name | Signature Surnan Lopoun. Signature | Date 3/Avg/17 Date |
|---|---|---|---|
| Randomization Implementer (required): | Dr Phan Cong Hung<br>Name | Signature | Date |
| Customer approval (if required): | Tushar Tewari Name | Signature | Date |
| | Thang Tran<br>Name | Signature | Date |

Document:

Maria Efstathiou

Version Number: 2.0

Author:


31MAR2017

Template No: CS\_TP\_BS025 Revision 5 Effective Date: 01Nov2016

Reference: CS\_WI\_BS002


740

Dated: 12 March 2018

| - | | |
|-----|-----------|------|
| (0) | Quintiles | MS |
| ~ | dan mice | 4.10 |

Randomization Specification

PATH/IVAC IVACFLU-S-0203 

## Authorization

| Randomization Biostatistician (required): | Maria Efstathiou Name | Signature | Date |
|---|---|---|---|
| Statistical Team Lead: | Suman Kapoor<br>Name | Signature | Date |
| Randomization Implementer (required): | <u>Dr Phan Cong Hung</u><br>Name | Signature | Date |
| Customer approval (if required): | <u>Tushar Tewari</u><br>Name | Signature | 03 MK 2017<br>Date |
| | Thang Tran<br>Name | Signature | Date |

Document:

Author:

Maria Efstathiou

Version Number: Version Date:

31MAR2017

Template No: CS\_TP\_BS025 Revision 5 Effective Date: 01Nov2016

Reference: CS\_WI\_BS002

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


Dated: 12 March 2018



Randomization Specification

PATH/IVAC IVACFLU-S-0203 

#### Authorization

Randomization Biostatistician Maria Efstathiou (required): Date Signature Name Statistical Team Lead: Suman Kapoor Signature Date Name Randomization Implementer Dr Phan Cong Hung (required): Signature Name Customer approval (if Tushar Tewari required): Name Signature Date Thang Tran Date Name Signature

Document:

Author: Maria Efstathiou Version Number: 2.0


31MAR2017

Template No: CS\_TP\_BS025 Revision 5

Effective Date: 01Nov2016

Reference: CS\_WI\_BS002

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 742 Dated: 12 March 2018



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

# Authorization

| Randomization Biostatistician (required): | Maria Efstathiou Name | Signature | Date |
|---|---|---|---|
| Statistical Team Lead: | Suman Kapoor<br>Name | Signature | Date |
| Randomization Implementer (required): | <u>Dr Phan Cong Hung</u><br>Name | Signature | Date |
| Customer approval (if required): | Tushar Tewari<br>Name | Signature | Date |
| | Thang Tran<br>Name | Signature | 04 Apr. 734 |

\\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03
Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0.docx Document:

Maria Efstathiou Version Number: 2.0 Author:

Version Date: 31MAR2017

Reference: CS\_WI\_BS002

Template No: CS\_TP\_BS025 Revision 5

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

743 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

#### 1. Modification History

| Unique<br>Identifie<br>r for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 0.1 | 12FEB2017 | Maria Efstathiou | N/A – First Draft Version sent for review. |
| 0.2 | 13FEB2017 | Maria Efstathiou | Minor updates and typos corrected following QI internal review. |
| 1.0 | 17FEB2017 | Maria Efstathiou | <ol> <li>Added name of randomization implementer on authorization page</li> <li>Added details for distribution to the sites in section 12.</li> </ol> |
| 2.0 | 31MAR2017 | Maria Efstathiou | 1. Authorisation page: corrected typo in Suman Kapoor's name and removed Renee Holt's name 2. Section 11, clarified that the blinded actual randomization was produced but not distributed and added reference to IVACFLU-S- 0203.SOP.04. 3. Section 11, updated block attributes to \$3. 4. Section 11, updated header in example schedule from 'block number' to 'block identifier'. 5. Section 11, updated Dummy_b labels in example to |

\\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03 Document:

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0

Maria Efstathiou Version Number: 2.0 Author: Version Date: 31MAR2017

Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002

Protocol No: IVACFLU-S-0203 744 Dated: 12 March 2018



#### Randomization Specification

PATH / IVAC IVACFLU-S-0203 

| | "DUMMY_IVACFLU-S". |
|---|---|
| 6. | Section 12, removed<br>row relating to<br>distribution of actual<br>blinded list to sites (not<br>applicable); updated |
| 7. | contact details for<br>Maria Efstathiou and<br>Suman Kapoor.<br>Section 9, removed<br>note regarding IVAC |
| | being allowed to see<br>the unblinded<br>randomization<br>specification. |

## 2. Study Details

| Protocol version and date | V3.0, 03JAN2017 |
|---------------------------|--------------------------------------|
| Study sample size | Phase 2: 252 subjects |
| | Phase 3: 636 subjects |
| | Total: $252 + 636 = 888$ subjects |
| Planned number of sites | Phase 2: 1 site (Long An) |
| | Phase 3: 2 sites (Long An; Dong Nai) |
| Study design | Parallel group |
| | Crossover |
| Number of treatment | 2 |
| groups / treatment | |
| sequences | |
| Full description of | 1 = IVACFLU-S |
| treatment groups / | 2 = PLACEBO |
| treatment sequences | |
| Ratio of subjects to | IVACFLU-S: PLACEBO: 5:1 |
| treatment groups / | |
| treatment sequences | |
| _ | |

Document: \quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

 $Rando\ specification \\ \ IVACFLU-S-0203\_Rando\ Spec\_BLINDED\_2017\_03\_31\_v2\_0$ 

Author: Maria Efstathiou Version Number: 2.0


Reference: CS\_WI\_BS002

Template No: CS\_TP\_BS025 Revision 5

Protocol No: IVACFLU-S-0203 745 Dated: 12 March 2018



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

#### 3. Randomization Requirements

| Method of randomization | Central |
|---|---|
| | □ Distributed |
| Subject or kit/component | Subject only – complete Section 4 |
| randomization schedule? | Kit/component only – complete Section 5 |
| | Subject and kit/component – complete Sections 4 and |
| | 5 |
| Stratified? | Yes – complete Section 6 |
| | No |
| Dynamic? | Yes – complete Section 7 |
| | ⊠ No |
| Is a matching schedule | Yes – complete Section 8 |
| required for replacing | ⊠ No |
| subjects who discontinue? | |
| Will randomized blocks | Yes – complete Section 9 |
| be used? | Specification must not be sent to blinded team |
| | members without redacting Section 9. |
| | □ No |
| Is a dummy | ⊠ Yes |
| randomization schedule | □ No |
| required? | |
| Is a partially unblinded | Yes – complete Section 10 |
| randomization file | ⊠ No |
| required? | |

# 4. Subject Randomization Numbers

| Number of records (randomization | Phase 2: 252 + 252 overage |
|---|---|
| numbers) to be generated: | Phase 3: 636 + 504 overage |
| Format and range of randomization | Phase 2 |
| numbers | <ul> <li>Long An, 18-45 years of age: A001 – A126 and A127 – A252 (overage)</li> <li>Long An, &gt;45 – 60 years of age: B001 – B126 and B127 – B252 (overage)</li> </ul> |
| | Phase 3 |
| | <ul> <li>Long An, 18-45 years of age: C001 –<br/>C126 and C127 – C252 (overage)</li> </ul> |
| | <ul> <li>Long An, &gt;45 – 60 years of age: D001</li> <li>D126 and D127 – D252 (overage)</li> </ul> |
| | <ul> <li>Dong Nai, 18 – 45 years of age: E001 –<br/>E192 and E193 – E318 (overage)</li> </ul> |

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

 $Rando\ specification \\ \ IVACFLU-S-0203\_Rando\ Spec\_BLINDED\_2017\_03\_31\_v2\_0$ 

Author: Maria Efstathiou Version Number: 2.0

Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002



#### Randomization Specification

PATH / IVAC IVACFLU-S-0203 

| • | Dong Nai, >45 – 60 years of age: G001 |
|---|----------------------------------------------------|
| | <ul> <li>G192 and G193 – G318 (overage)</li> </ul> |

## 5. Kit/Component Identifiers

| Generation of kit/component identifiers | ☐ Provided<br>☐ Require generation |
|---|---|
| If provided, give details of source | N/A |
| If generating, number of records (kit/component identifiers) to be generated: | Kit numbers are identical to Subject<br>Randomization Numbers (cf. Section 4 above). |
| If generating, format and range of kit/component identifiers | Kit numbers are identical to Subject<br>Randomization Numbers (cf. Section 4 above). |

#### 6. Stratification Factors

| Number of Stratification Factors | Phase 2: 1 (age group) |
|----------------------------------|---------------------------------|
| | Phase 3: 2 (age group and site) |

| Stratification Factor 1: | |
|---|---|
| Description: | Site – applies to phase 3 only.<br>Include 'Site' in the schedule for phase 2, but<br>only 1 site (Long An) is involved in phase 2. |
| Number of levels: | 2 |
| Details of levels: | Site: Long An<br>Site: Dong Nai |

| Stratification Factor 2: | |
|---|---|
| Description: | Age group – applies to phase 2 and phase 3. |
| Number of levels: | 2 |
| Details of levels: | Age group: $18-45$ years of age<br>Age group: $>45-60$ years of age |

## 7. Dynamic Randomization Methods

| N/A |
|-----|

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

 $Rando\ specification \\ \ VACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0$ 

Author: Maria Efstathiou Version Number: 2.0 Version Date: 31MAR2017

Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002


Protocol No: IVACFLU-S-0203 747 Dated: 12 March 2018



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

#### 8. Replacement Subject Numbers

| Details of randomization numbers | N/A |
|----------------------------------|-----|
| for replacement subjects | |

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0

Author: Maria Efstathiou Version Number: 2.0


Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 748 Dated: 12 March 2018



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

#### 9. Block Size

| If randomized blocks are required, | Yes |
|---|---|
| will mixed blocks be used? | No |
| Will a different block size be used | Yes |
| for any draft or dummy schedules? | □ No |
| Block size(s) | INFORMATION REMOVED FOR BLINDED |
| | SPECIFICATION |
| | ** All block sizes must be redacted before |
| | distributing to blinded team members. ** |
| Number of blocks | INFORMATION REMOVED FOR BLINDED |
| | SPECIFICATION |
| | ** Number of blocks must be redacted |
| | before distributing to blinded team |
| | members. ** |

Note: as per PATH procedures, the use of the mixed block size allows for blinded PATH / IVAC team members to review the randomisation specification, including block size. A blinded version will be created for review by the QuintilesIMS team.

#### 10. Partial Unblinding

| Partially unblinded treatment group | N/A |
|-------------------------------------|-----|
| / treatment sequence identifiers | |

## 11. Output Files

The following files will be produced:

IVACFLUS0203\_RNDSBJKIT\_ACTUAL\_U: unblinded actual randomization schedule produced for drug packaging by IVAC.

IVACFLUS0203\_RNDSBJKIT\_ACTUAL\_B: blinded actual randomization schedule produced for randomisation implementation at site. UPDATE FOR V2.0: this was produced but not distributed to the sites, as a separate instruction was issued to the sites, describing the format of the randomisation numbers for each site and stratum. Instruction reference: IVACFLU-S-0203.SOP.04.

**IVACFLUS0203\_RNDSBJKIT\_DUMMY\_B:** blinded dummy randomization schedule produced for blinded statistical programming purposes.

An example of the schedule structure is given below:

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\IVACFLU-S-0203 RandoSpec BLINDED 2017 03 31 v2 0

Author: Maria Efstathiou Version Number: 2.0

Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries Unauthorized use, disclosure or reproduction is strictly prohibited.
Protocol No: IVACFLU-S-0203 749 Dated: 12 March 2018



Randomization Specification

PATH / IVAC IVACFLU-S-0203 

Reference: CS\_WI\_BS002

Block number should be redacted before distributing to any blinded team members, even in an example

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0

Author: Maria Efstathiou Version Number: 2.0


Template No: CS\_TP\_BS025 Revision 5

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

**IVACFLU-S** 


750

QuintilesIM5

Randomization Specification

PATH / IVAC IVACFLU-S-0203 

| Protocol<br>Identifier | Schedule<br>Type | Phase | Site | Age group | Block<br>Identifier | Randomiza<br>tion<br>Number | Kit<br>Identifier | Randomiz<br>ed<br>Treatment | Numeric<br>Random<br>ized | Overage |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Group | treatmen<br>t group | |
| IVACFL<br>U-S-0203 | Actual_u | 2 | Long<br>An | 18 – 45 years<br>of age | XX | A001 | A001 | IVACFL<br>U-S | 1 | No |
| IVACFL<br>U-S-0203 | Actual_u | 2 | Long<br>An | 18 – 45 years<br>of age | XX | A126 | A126 | PLACEB<br>O | 2 | No |
| IVACFL<br>U-S-0203 | Actual_u | 2 | Long<br>An | 18 – 45 years<br>of age | XX | A252 | A252 | IVACFL<br>U-S | 1 | Yes |

- o For the PDF files, each stratum will start on a new page.
- Schedule type is 'Actual u', 'Actual b', 'Dummy b' for the actual unblinded, actual blinded and dummy blinded schedules, respectively.
- o For the Dummy b schedule, the block number will be reset to '01' for all blocks prior to sending to the recipients specified in section 12. The randomised treatment group will be preceded by 'DUMMY' (e.g. DUMMY IVACFLU-S').
- o For the Actual b schedule, Block number, randomised treatment group and numeric randomised treatment group will be removed prior to sending to the recipients specified in section 12. UPDATE FOR V2.0: this was produced but not distributed to the sites, as a separate instruction was issued to the sites, describing the format of the randomisation numbers for each site and stratum. Instruction reference: IVACFLU-S-0203.SOP.04.
- o For the PDF files, overage numbers for each stratum will start on a separate page.

\\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03 Document:

Rando specification\TVACFLU-S-0203 RandoSpec BLINDED 2017 03 31 v2 0

Maria Efstathiou Author:

Version Number: 2.0 Version Date: 31MAR2017

Template No: CS TP BS025 Revision 5 Reference: CS WI BS002

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles IMS Holdings. Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

751 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018



#### Randomization Specification

PATH / IVAC IVACFLU-S-0203 

Reference: CS\_WI\_BS002

| Variable name | Label | Attributes |
|---------------|----------------------|------------|
| PROTID | Protocol Identifier | \$16. |
| SCHEDTYP | Schedule Type | \$10. |
| PHASE | Phase | \$1. |
| SITE | Site | \$10. |
| AGEGRP | Age group | \$22. |
| BLOCK | Block Identifier | \$3. |
| RND | Randomization Number | \$4. |
| KITID | Kit Identifier | \$4. |
| RTREAT | Randomized Treatment | \$20. |
| | Group | |
| RTREATN | Numeric Randomized | 8. |
| | Treatment Group | |
| OVERAGE | Overage identifier | \$3. |

#### 12. Distribution Details For Randomization Schedule

| Authoriz ed recipient s: Hoàng Minh Hưng IVAC pharmaci st | Contact Details: Email address: hhung_nt@yahoo.com Mobile #: 84- 985.715.096 Fax #: 058 3 823 815 | Files to be distributed: IVACFLUS0203_RNDSBJKIT_ACTUAL _U.PDF IVACFLUS0203_RNDSBJKIT_ACTUAL _U.CSV | Method<br>of<br>Distribu<br>tion:<br>Passwor<br>d-<br>protected<br>email | Reason<br>for<br>Distribu<br>tion:<br>Unblinde<br>d for<br>drug<br>packagin<br>g |
|---|---|---|---|---|
| Maria<br>Efstathio<br>u,<br>Quintiles<br>IMS<br>randomis<br>ation<br>statisticia<br>n | Maria.efstathiou@quint ilesims.com | IVACFLUS0203_RNDSBJKIT_ACTUAL_U.PDF IVACFLUS0203_RNDSBJKIT_ACTUAL_U.SAS7BDAT IVACFLUS0203_RNDSBJKIT_ACTUAL_U.CSV IVACFLUS0203_RNDSBJKIT_ACTUAL_B.PDF IVACFLUS0203_RNDSBJKIT_ACTUAL_B.SAS7BDAT IVACFLUS0203_RNDSBJKIT_DUMMY_B.PDF IVACFLUS0203_RNDSBJKIT_DUMMY_B.PDF IVACFLUS0203_RNDSBJKIT_DUMMY_B.SAS7BDAT | N/A | Reviewe r and Secure storage of actual blinded and actual; unblinde d schedule s |
| Suman<br>Kapoor,<br>Quintiles<br>IMS | Suman.kapoor@quintil<br>esims.com | IVACFLUS0203_RNDSBJKIT_DUMMY_<br>B.PDF<br>IVACFLUS0203_RNDSBJKIT_DUMMY_<br>B.SAS7BDAT | Email | Blinded<br>dummy<br>schedule<br>for |

Document:

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0

Maria Efstathiou Version Number: 2.0 Author:


Template No: CS\_TP\_BS025 Revision 5 Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


Protocol No: IVACFLU-S-0203 752 Dated: 12 March 2018



PATH / IVAC IVACFLU-S-0203 

#### Randomization Specification

| STL,<br>QBAN | program<br>develop |
|--------------|--------------------|
| | ment |

Document: \\quintiles.net\Enterprise\Sites\gbthv\QTHVRANDOM\IVAC\IVACFLU-S-0203\03

Rando specification\IVACFLU-S-0203\_RandoSpec\_BLINDED\_2017\_03\_31\_v2\_0

Author: Maria Efstathiou Version Number: 2.0


Template No: CS\_TP\_BS025 Revision 5 Reference: CS\_WI\_BS002

Effective Date: 01Nov2016

Copyright © 2009, 2010, 2011, 2014, 2016 QuintilesIMS. All rights reserved. The contents of this document are confidential and proprietary to Quintiles IMS Holdings, Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 753 Dated: 12 March 2018

# 16.1.8 Audit certificates

Not Applicable


Protocol No: IVACFLU-S-0203 754 Dated: 12 March 2018

# 16.1.9 Documentation of statistical methods

| Document | Date |
|-----------------------------------------|----------------|
| Final SAP, Version 1 | 11 August 2017 |
| Table and Listing Mock Shell, Version 1 | 11 August 2017 |


Protocol No: IVACFLU-S-0203 755 Dated: 12 March 2018





STATISTICAL ANALYSIS PLAN: PROTOCOL IVACFLU-S-0203


## STATISTICAL ANALYSIS PLAN

## IVACFLU-S-0203, Phase 2/3

A PHASE 2 / 3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF A SEASONAL TRIVALENT **INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S)** PRODUCED BY IVAC

**AUTHOR: REVATHI RAYADURGAM** 

**VERSION NUMBER AND DATE: DRAFT V1.0 11AUG2017** 

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Dated: 12 March 2018






Date

Signature


## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Name

Statistical Analysis Plan V1.0 (Dated11AUG2017) for Protocol IVACFLU-S-0203 (V4.0 Dated 09FEB2017).

| Author: | Author: Revathi Rayadurgam | | (B) \$12 | 14/AUG/17 |
|---|---|---|---|---|
| Position: | Biosta | itistician 2 | | |
| Company: | Quint | ilesIMS | | K. KURINI NO SECURIO CONTROL C |
| • | | nent, the undersigned app<br>able for the reporting of th | roves this version of the Statist is study. | ical Analysis Plan, authorizing |
| T TO THE TOTAL OF | | Name | Signature | Date |
| Approved By: | | Suresh Chenji | 2- Guerrelly | - 14/AUG/2017 |
| Positi | ion: | Manager, Biostatistics | | |
| Comp | oany: | QuintilesIMS | Secretaria de Caración de Cara | THE RESERVE OF THE PROPERTY OF |
| Approved By: | | Krista Yuhas | Circille Yulia | - 14/h8/2017 |
| Posit | ion: | Biostatistician, Cente | r for Vaccine Innovation and Ad | ccess (CVIA) |
| Comp | pany: | PATH | The second secon | 4 |
| Approved By: | | Tushar Tewari | | |
| Posit | ion: | Senior Medical Office | er, Clinical and Regulatory Affai | rs |
| Company: | | PATH | | Total Commence and |

Document:

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0

Author:

Revathi Rayadurgam

Version Number: Version Date: 1.0 [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

757


Dated: 12 March 2018






## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V1.0 (Dated11AUG2017) for Protocol IVACFLU-S-0203 (V4.0 Dated 09FEB2017).

| | Name | Signature | Date |
|---|---|---|---|
| Author: | Revathi Rayadurgam | | |
| Position: | Biostatistician 2 | | * |
| Company: | QuintilesIMS | CONTROL OF ADMINISTRAÇÃO DE PRINCIPARA DE PORTA | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | | |
| Position: | Manager, Biostatistics | ; | |
| Company: | QuintilesIMS | | |
| Approved By: | Krista Yuhas | | |
| Position: | Biostatistician, Center | for Vaccine Innovation and | Access (CVIA) |
| Company: | PATH | 16 | |
| | | $\wedge$ | |
| Approved By: | Tushar Tewari | () aver | 11 AUG 2017 |
| Position: | Senior Medical Office | r, Clinical and Regulatory Aff | airs |
| Company: | PATH | | |

Document:

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0

Author:

Revathi Rayadurgam

Version Number: Version Date:

[11AUG2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005


Protocol No: IVACFLU-S-0203 758 Dated: 12 March 2018






## **MODIFICATION HISTORY**

| Unique Identifier for this Version | Date of the Document<br>Version | Author | Significant Changes<br>from Previous<br>Authorized Version |
|---|---|---|---|
| | | Revathi Rayadurgam | Not applicable. First version. |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0

Author: Revathi Rayadurgam Version Number: 1.0

Version Date: [11AUG2017]

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or

reproduction is strictly prohibited.






## **TABLE OF CONTENTS**

| Statistic | cai Analysis Plan Signature Page | Z |
|-----------|---------------------------------------------|----|
| Modifica | ation History | 3 |
| Table of | f Contents | 4 |
| List Of A | Abbreviations | 8 |
| 1. | Introduction | 10 |
| 2. | Study Objectives | 10 |
| 2.1 | Primary Objectives, Phase 2 | 10 |
| 2.2 | Primary Objectives, Phase 3 | 10 |
| 2.3 | Secondary Objective, Phase 3 | 10 |
| 2.4 | 2.3 Assessment of Objectives | 10 |
| 2.4.1 | 2.3.1 Endpoint variables | 10 |
| 2.4.1.1 | Primary Safety Endpoints, Phase 2 and 3 | 11 |
| 2.4.1.2 | Primary Immunogenicity Endpoints, Phase 3 | 11 |
| 2.4.1.3 | Secondary Immunogenicity Endpoints, Phase 3 | 12 |
| 3 | Study Design | 12 |
| 3.1 | General Description | 12 |
| 3.1.1 | Randomization and Blinding | 14 |
| 3.1.1.1 | Randomization procedures | 14 |
| 3.1.1.2 | Blinding and unblinding procedures | 14 |
| 3.2 | Schedule of Events | 15 |
| 3.3 | Changes to Analysis from Protocol | 16 |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016


Protocol No: IVACFLU-S-0203 760 Dated: 12 March 2018





#### STATISTICAL ANALYSIS PLAN: PROTOCOL IVACFLU-S-0203 

| 4 | Planned Analyses | . 1 |
|---|---|---|
| 4.1 | Data and Safety Monitoring Board | . 17 |
| 4.2 | Interim Analysis | . 17 |
| 4.3 | Final Analysis | . 17 |
| 5 | Analysis Sets | . 17 |
| 5.1 | Enrolled population | . 18 |
| 5.2 | Full Analysis [FA] POPULATION | . 18 |
| 5.3 | Per Protocol [PP] population | . 18 |
| 6. | General Considerations | . 18 |
| 6.1 | Reference Start Date and Study Day | . 19 |
| 6.2 | Baseline | . 19 |
| 6.3 | Derived Timepoints | . 19 |
| 6.4 | Retests, Unscheduled Visits and Early Termination Data | . 19 |
| 6.5 | Windowing Conventions | . 20 |
| 6.6 | Statistical Tests | . <b>2</b> ( |
| 6.7 | Common Calculations | . <b>2</b> ( |
| 6.8 | | |
| 0.0 | Software Version | . 20 |
| 7. | Software Version | |
| | | . 20 |
| 7. | Statistical Considerations | . 20 |
| 7.<br>7.1 | Statistical Considerations | . 20 |
| 7.<br>7.1<br>7.2 | Statistical Considerations | . 20 |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016


761 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018





# STATISTICAL ANALYSIS PLAN: PROTOCOL IVACFLU-S-0203


| 8. | Output Presentations |
|---|---|
| 9. | Disposition and Withdrawals |
| 10. | Demographic and other Baseline Characteristics |
| 10.1 | Derivations |
| 11. | Current medical conditions |
| 12. | Medications |
| 13. | Study Medication Exposure |
| 14. | Study Medication Compliance |
| 15. | Efficacy Outcomes |
| 16. | Immunogenicity analysis |
| 16.1 | Statistical considerations |
| 16.1.1 | Probability for demonstrating seroconversion criteria for licensure |
| 16.1.2 | Probability for demonstrating seroprotection criteria for licensure |
| 16.2 | Analysis of Immunogenicity Endpoints |
| 16.2.1 | Primary Immunogenicity Endpoints |
| 16.2.2 | Secondary Immunogenicity Endpoints |
| 16.3 | Variables & Derivations |
| 17. | Safety Outcomes |
| 17.1 | Statistical considerations:29 |
| 17.2 | Analysis of safety endpoints: |
| 17.2.1 | Solicited Local and Systemic Adverse Events |
| 17.2.1.1 | Presentation of 30-minute solicited local and systemic reactogenicity31 |
| 17.2.1.2 | Presentation of solicited local and systemic adverse events |
| Docume | ent: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203_SAP_Draft v1.0 |


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016





#### STATISTICAL ANALYSIS PLAN: PROTOCOL IVACFLU-S-0203 

| 17.2.2 | Unsolicited adverse events | 33 |
|---------|----------------------------------|----|
| 17.2.3 | Serious Adverse Events | 34 |
| 17.3 | Deaths | 35 |
| 17.4 | ECG Evaluations | 36 |
| 17.5 | Vital Signs | 36 |
| 17.6 | Physical Examination | 36 |
| 18. | Data Not Summarized or Presented | 37 |
| APPEND | IX 1 | 38 |
| APPEND | IX 2 | 39 |
| APPEND | IX 3 | 39 |
| ADDENID | IV A | 20 |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016






#### LIST OF ABBREVIATIONS

ADaM Analysis Data Model

AE Adverse Event

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

cm Centimeter

CPMP Committee for Proprietary Medicinal Products

CRF Case Report Form

DSMB Data and Safety Monitoring Board

eCRF Electronic Case Report Form

EMEA European Agency Evaluation of Medicinal Products

FA Full Analysis Population

GMFR Geometric Mean Fold Rise

GMT Geometric Mean Titer

HA Hemagglutinin

HAI Hemagglutination Inhibition

ICF Informed Consent Form

IP Investigational Product

IRB Institutional Review Board

IVAC Institute of Vaccines and Medical Biologicals

mL Milliliter

MOH Ministry of Health

PD Protocol Deviations

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016


Protocol No: IVACFLU-S-0203 764 Dated: 12 March 2018






PΕ **Physical Examination** 

ы **Principal Investigator** 

Per Protocol Population PΡ

**PSRT Protocol Safety Review Team** 

PT **Preferred Term** 

**RCD Reverse Cumulative Distribution** 

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SAS Statistical Analysis System

SOC System organ class

**SDTM** Study Data Tabulation Model

TLF Tables, Listings and Figures

WHO World Health Organization

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

765 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of safety and immunogenicity data for Protocol IVACFLU-S-0203. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on Protocol version 4.0, dated 09Feb2017.

#### 2. STUDY OBJECTIVES

#### 2.1 **PRIMARY OBJECTIVES, PHASE 2**

Safety: To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent inactivated split virion influenza vaccine in adults, 18 to 60 years of age.

#### 2.2 **PRIMARY OBJECTIVES, PHASE 3**

Safety: To evaluate the safety profile of a single intramuscular dose of IVACFLU-S seasonal trivalent split virion inactivated influenza vaccine in adults, 18 to 60 years of age.

Immunogenicity: To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single intramuscular dose of IVACFLU-S seasonal trivalent split virion, inactivated influenza vaccine in adults, 18 to 45 (inclusive) and 46-60 years of age.

#### 2.3 SECONDARY OBJECTIVE, PHASE 3

Immunogenicity: To evaluate the immune response at Day 22 to each of the three vaccine antigens after a single dose of IVACFLU-S seasonal trivalent split virion inactivated influenza vaccine in adults with and without preexisting Hemagglutination Inhibition (HAI) antibody.

#### ASSESSMENT OF OBJECTIVES

#### 2.4.1 ENDPOINT VARIABLES

Solicited local adverse events (at site of injection):

Erythema / redness - based on size in cm

Swelling / induration (hardness at site of injection) - based on size in cm

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0

Author: Revathi Rayadurgam Version Number: Version Date:

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or

reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 766 Dated: 12 March 2018






- Solicited systemic adverse events:
  - Fever-Body temperature
  - Fatigue/malaise
  - o Generalized muscle aches
  - Joint aches
  - Chills
  - o Nausea
  - Vomiting
  - Headache
- Unsolicited adverse events
- Serious adverse events
- Seroprotection
- Seroconversion
- Geometric mean titers (GMT) of serum HAI antibodies
- Geometric mean fold rises (GMFR) of serum HAI antibodies

## 2.4.1.1 PRIMARY SAFETY ENDPOINTS, PHASE 2 AND 3

The number and proportion of participants reporting the following events:

- A. Solicited local adverse events, including redness / erythema, swelling / induration, pain within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- B. Solicited systemic adverse events, including fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- C. Unsolicited Adverse Events (AEs) occurring within 21 days post vaccination.
- D. Serious Adverse Events (SAEs) occurring during the entire study period (Days 1-91).

## 2.4.1.2 Primary Immunogenicity Endpoints, Phase 3

- A. Number and percentage of participants by age groups (18-45, 46-60) with seroconversion against each of the 3 vaccine antigens post-vaccination. Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
  - pre-vaccination titer <1.:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or
  - pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day
     22

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 767 Dated: 12 March 2018






- B. Number and percentage of participants by age groups (18-45, 46-60) with a HAI antibody titer ≥1:40 to each of the 3 vaccine antigens measured on Day 22 post vaccination
- C. GMTs of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens
- D. GMFRs of serum HAI antibodies (post vaccination/prevaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens

## 2.4.1.3 Secondary Immunogenicity Endpoints, Phase 3

- A. Number and percentage of participants by age groups (18-45, 46-60) who develop at least a four-fold increase in HAI antibody titer to each of the vaccine antigen post vaccination measured on Day 22 by pre-vaccination HAI antibody titer of <1:10 or ≥1:10.
- B. GMTs of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by prevaccination HAI antibody titer of <1:10 or ≥1:10.
- C. GMFRs of serum HAI antibodies (post vaccination/prevaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by prevaccination HAI antibody titer of <1:10 or ≥1:10.

#### 3 STUDY DESIGN

#### 3.1 GENERAL DESCRIPTION

This is a phase 2/3, double-blind, randomized, placebo-controlled trial to evaluate the safety and immunogenicity of a single dose of the IVACFLU-S seasonal influenza vaccine in male and female healthy adult volunteers, aged 18 to 60 years old (inclusive). Subjects will receive a single dose of seasonal trivalent, split inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or placebo (phosphate buffered saline).

Phase 2 will be conducted at a single site, District Health Center of Ben Luc district in Long An Province. Phase 2 will involve 252 subjects randomized to receive either IVACFLU-S or placebo at a ratio of 5:1.

Following determination of "safe to proceed" based on Protocol Safety Review Team (PSRT) review of Day 8 safety data from all Phase 2 subjects and with approval from Vietnam Ministry of Health (MOH), Phase 3 enrollment will commence at 2 sites, District Health Center of Ben Luc in Long An province and District Health Center of Long Thanh in Dong Nai province.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 768 Dated: 12 March 2018






The Phase 3 components will include 636 subjects randomized to receive either IVACFLU-S or placebo at a ratio of 5:1. Randomization of Phase 2 volunteers will be stratified by age group and Phase 3 volunteers will be stratified by site and age group, as per Figure 1.

The sample size for this study was selected in response to the MOH's requirement for additional safety data from Phase 2 before proceeding to Phase 3 and for primary safety and immunogenicity analysis to satisfy the MOH licensure requirement for influenza vaccine in adults from ages 18 through 60. The sample size reflects guidance and endorsement by MOH at the MOH-IVAC Consultation Meeting held on 20 April 2016.

Figure 1: Summary of study design.



S1: Day of Screening and Enrollment

D1: Day of Vaccination

Ben Luc and Long Thanh are the two study sites at Long An and Dong Nai provinces respectively.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 769 Dated: 12 March 2018






3.1.1 RANDOMIZATION AND BLINDING

# 3.1.1.1 RANDOMIZATION PROCEDURES

This is a double-blind, randomized, controlled trial with 2 groups: vaccine and placebo. The ratio of vaccine to placebo recipients is 5:1.

This seamless design has the block randomization conducted with age group as the stratification factor for both phase 2 and phase 3, having two levels of stratification. The two age groups are:

- 1. 18-45 and
- 2. 46-60.

Block randomization for Phase 3 involves site as an additional stratification factor i.e., Phase 3 will be conducted at two sites i.e., District Health Center of Ben Luc in Long An province and District Health Center of Long Thanh in Dong Nai province.

Each participant will be assigned a unique screening number assigned by the investigator after signing the informed consent. After an individual is determined to be eligible for study participation, the participant will be randomized according to age group by assigning a unique participant identification number sequentially in ascending order from the randomization schedule, which will contain the unique participant identification number and the corresponding randomization assignment and will be produced using computer software prior to the initiation of the study.

Once a participant identification number has been assigned to a participant, it will not be used again. Additional participants may be randomized into the study at the discretion of the sponsor in the case of any participant who is randomized but does not receive any study vaccine.

## **3.1.1.2** Blinding and unblinding procedures

The randomization will be conducted by an organization or individual not involved in the conduct of the study.

The randomization lists for participants will be used by IVAC to label study vaccine and placebo vials and then will be immediately sealed. It will be opened only after the clinical trial database is declared complete and locked. In the case of any unblinding, researchers must report this in writing to the overseeing Ethics Committee.

Study product injected into each participant will be recorded on the electronic Case Report Form (eCRF) using the exact allocation code for each product received by each participant. The allocation codes link treatment identification with each participant via participant identification numbers. These will be maintained in a secure location, by an individual not involved in the conduct of the study. If any participant experiences an SAE possibly related to receipt of study treatment and the investigator determines it is necessary to unblind, treatment allocation to the participant may be communicated to the investigator.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or

reproduction is strictly prohibited.






A blinded dummy randomization schedule was produced for blinded statistical programming purposes.

An example of the schedule structure is given in Table 1.

Table 1: Example structure of randomization schedule.

| Protocol<br>Identifier | Schedule<br>Type | Phase | Site | Age<br>group | Block<br>Number | Randomization<br>Number | Kit<br>Identifier | Randomized<br>Treatment<br>Group | Numeric<br>Randomized<br>treatment<br>group | Overage |
|---|---|---|---|---|---|---|---|---|---|---|
| IVACFLU-<br>S-0203 | Actual_u | 2 | Long<br>An | 18 –<br>45<br>years<br>of<br>age | XX | A001 | A001 | IVACFLU-S | 1 | No |
| IVACFLU-<br>S-0203 | Actual_u | 2 | Long<br>An | 18 –<br>45<br>years<br>of<br>age | XX | A126 | A126 | PLACEBO | 2 | No |

## 3.2 SCHEDULE OF EVENTS

Schedule of events can be found in Table 2.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or

reproduction is strictly prohibited.






Table 2: Schedule of events of the protocol synopsis of Protocol IVACFLU-S-0203, Phase 2/3, version 4.0 dated 09Feb2017.

| | Study Day (# days from D1) | | | | | |
|---|---|---|---|---|---|---|
| Study Activities | S1/D1*<br>(up to -4/<br>D1<br>Clinic<br>Visit | D1<br>to<br>D7 | D8<br>(+/- 1)<br>Clinic<br>Visit | D9 to<br>D21 | D22<br>(+/- 1)<br>Clinic<br>Visit | D91<br>(+/- 7)<br>Telephonic<br>contact |
| Information process and written informed consent | Х | | | | | |
| Collect baseline demographic data | Х | | | | | |
| Collect/review medical history | Х | | | | | |
| Perform screening physical examination | Х | | | | | |
| Perform vital signs & targeted physical examination (symptom based & reactogenicity only) | X* | | х | | | |
| Perform urine pregnancy check (women) | X* | | | | | |
| Check/confirm inclusion/exclusion criteria | Χ* | | | | | |
| Randomization | X | | | | | |
| Collect serum for influenza serology | X** | | | | Х | |
| Administer one dose of study product (vaccine or placebo) | х | | | | | |
| Observe for 30 Minutes; record and manage immediate reactions | Х | | | | | |
| Instruct participant on use of Dairy card | Х | | | | | |
| Participant records solicited reactogenicity and unsolicited AEs in Diary cards | Х | Х | | | | |
| Clinical staff reviews interim AEs/SAEs with participant; records in CRF | | | Х | | Х | SAE only |
| Report SAEs to Sponsor, IRBs and regulatory authorities | х | Х | х | х | Х | Х |
| Participant completion of study | | | | | | Х |

<sup>\*</sup>If Day 1 is conducted on a different day from S1, eligibility must be confirmed again on Day of Injection (D1); including Targeted physical examination (PE); inclusion/exclusion; urine pregnancy test.

#### 3.3 CHANGES TO ANALYSIS FROM PROTOCOL

No changes to planned analyses in the protocol will be applied.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

<sup>\*\*</sup> Sera samples will be collected prior to vaccination in phase 3 study at one site (Ben Luc).

Protocol No: IVACFLU-S-0203 772 Dated: 12 March 2018






#### 4 PLANNED ANALYSES

The primary focus of this SAP is to describe safety analyses that will be conducted on the combined Phase 2 and Phase 3 data, as well as the immunogenicity analyses that will be conducted on the Phase 3 data.

#### 4.1 Data and Safety Monitoring Board

Given the wide global experience with seasonal influenza vaccines and the safety profile observed in the Phase 1 study, there will not be any Data Safety Monitoring Board (DSMB) for this study. The PSRT will be responsible for close safety oversight of the study.

#### 4.2 INTERIM ANALYSIS

Blinded safety data up to Day 8 for Phase 2 subjects will be analysed and reviewed by the PSRT team. In addition, all grade 3 and above unsolicited AEs and SAEs until the data cut-off date will also be part of an interim report. This report will be submitted to the Pasteur Institute Ho Chi Minh City Institutional Review Board (IRB) and Vietnam Ministry of Health (MOH) for review and approval before initiating the Phase 3 study.

## 4.3 FINAL ANALYSIS

Analyses will be conducted only after all related data have been entered, cleaned, locked and the study datasets routinely unblinded. Given the short duration of clinical follow-up and potential delays in generating immunogenicity results, analysis of safety and immunogenicity data will be conducted independently. All final, planned analyses identified in this SAP will be performed by QuintilesIMS Biostatistics following:

- 1. Sponsor authorization of the analysis sets;
- 2. Sponsor authorization of the final SAP and Tables, Listings and Figures (TLF) Shells;
- 3. Authorization of data issues log;
- 4. Authorization of data handling report;
- 5. Database lock;
- 6. Routine unblinding of study datasets for analysis; and
- 7. Identification of treatment deviations (randomized versus actual).

## 5 ANALYSIS SETS

Agreement and authorization by the sponsor of subjects included/excluded from each analysis set will be conducted prior to the unblinding of the study data.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

reproduction is strictly prohibited.

773 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018






#### 5.1 **ENROLLED POPULATION**

All screened subjects who are randomized, regardless of the subject's randomization and treatment status in the trial.

#### 5.2 **FULL ANALYSIS [FA] POPULATION**

All subjects in the enrolled population who were randomized and received a study vaccination. This population will serve as the primary analysis population for all safety objectives. The analysis based on this population will serve as the supportive results for all safety objectives. Subjects will be analyzed as randomized.

#### PER PROTOCOL [PP] POPULATION 5.3

Immunogenicity will be assessed only in Phase 3 subjects who are randomized at the Ben Luc site. All such subjects in the Full Analysis population who have valid post-vaccination immunogenicity measures with no major protocol violations that are determined to potentially interfere with the immunogenicity assessment of the study vaccine will be included. This population will serve as the primary analysis population for all immunogenicity objectives.

The criteria for exclusion of subjects from the Per Protocol Population will be established before breaking the blind and will be based on the blinded review of protocol violations, which will be identified and categorized as described in Appendix 1.

## 6. GENERAL CONSIDERATIONS

By-subject data listings, summary tables, figures and statistical tests will be performed using SAS® Version 9.4 or higher.

All clinical data, including laboratory and clinical data from an internal database will be provided as raw datasets. CDISC SDTM 3.2 compliant SAS datasets will then be generated. Coding of AEs and current medical conditions will be included in the SDTM datasets.

Appropriate SAS programs will be prepared and validated according to QuintilesIMS standard operating procedures.

The following descriptive statistics will be presented in summary tables:

Continuous variables: Number (observed cases), mean, median, standard deviation (SD), minimum, and maximum

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

774 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






Categorical variables: Summarized by treatment group using frequency tables (frequency [n] and percentage [%]). Percentages will be calculated relative to the total number of subjects in the relevant analysis set with data available, if not otherwise specified.

Two-sided exact 95% confidence intervals (CIs) will be presented unless otherwise specified.

#### 6.1 REFERENCE START DATE AND STUDY DAY

Study day will be calculated relative to the reference start date, and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of vaccination (Day 1), and will appear in every listing where an assessment date or event date appears.

- If the date of the event is on or after the reference date then: Study day = (date of event - reference date) + 1.
- If the date of the event is prior to the reference date then: Study day = (date of event - reference date).

For the derivation of study day, time of day will be considered, if applicable.

In the situation where the event date is partial or missing, Study day, and any corresponding durations will appear partial or missing in the listings i.e., Study day or any corresponding durations will not be computed.

#### 6.2 **BASELINE**

Unless otherwise specified, Baseline is defined as the last non-missing measurement taken prior to vaccination start date and time (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered pre-baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

#### **DERIVED TIMEPOINTS** 6.3

Not applicable.

#### RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA 6.4

In general, for by-visit summaries, data recorded at the nominal visit will be presented. Unscheduled measurements will not be included in by-visit summaries.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 775 Dated: 12 March 2018






In the case of a retest (same visit number assigned), the earliest available measurement for that visit will be used for by-visit summaries.

Listings will include scheduled, unscheduled, retest and early termination data.

#### 6.5 WINDOWING CONVENTIONS

No visit windowing will be performed for this study.

#### **6.6 STATISTICAL TESTS**

The default significance level will be 5%, confidence intervals will be 95%, and all tests will be two-sided, unless otherwise specified in the description of the analyses.

## 6.7 COMMON CALCULATIONS

For quantitative measurements, change from Baseline to Visit X will be calculated as:

Test Value at Visit X - Baseline Value

#### **6.8 SOFTWARE VERSION**

All analyses will be conducted using SAS version 9.4 or higher.

## 7. STATISTICAL CONSIDERATIONS

## 7.1 ADJUSTMENT FOR COVARIATES

No adjustment for covariates will be made.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 776 Dated: 12 March 2018






#### 7.2 MULTICENTER STUDIES

Phase 2 will be conducted at a single site, District Health Center of Ben Luc district in Long An Province. Phase 3 enrollment will be conducted at 2 sites, District Health Center of Ben Luc in Long An province and District Health Center of Long Thanh in Dong Nai province.

The data collected from the two study sites will be pooled together for analyses with the below exceptions:

- Subject disposition summaries will be presented both pooled and separately by study site.
- Immunogenicity measurements and analyses will be conducted only in subjects studied at the Ben Luc site during Phase 3

#### 7.3 MISSING DATA

Missing safety and immunogenicity data will not be imputed.

# 7.4 MULTIPLE COMPARISONS/ MULTIPLICITY

No multiplicity adjustment to the Type 1 probability of error, alpha, will be made for the multiple testing of immunogenicity endpoints corresponding to the three vaccine antigens under the intersection-union property. That is, the immune responses to each of the three vaccine antigens induced by IVACFLU-S seasonal trivalent split inactivated influenza vaccine need to meet Vietnam Ministry of Health licensure requirements.

#### 7.5 EXAMINATION OF SUBGROUPS

- 1. All safety and immunogenicity analyses will be conducted for subgroups of age category i.e., 18-45 and 46-60.
- 2. Analysis of secondary immunogenicity endpoints, Phase 3, will be conducted for subgroups of prevaccination HAI antibody titer i.e., <1:10 or ≥ 1:10 and subgroups of age category i.e., 18-45 and 46-60.

#### 8. OUTPUT PRESENTATIONS

The shells provided with this SAP describe the presentations for this study and therefore the format and content of the summary TLFs to be provided by QuintilesIMS Biostatistics.

Tables and figures will be presented for Phase 2 and Phase 3 subjects combined and pooled across study sites with the below exceptions:

 Subject disposition summaries will be reported separately by study site, in addition to being pooled across study sites.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 777 Dated: 12 March 2018






 Immunogenicity measurements will be from Phase 3 subjects at the Ben Luc site only; thus immunogenicity TLFs will be restricted to this subset.

All table and figure summaries will be presented by treatment group both by age group (18-45, 46-60) and pooling across age groups. Additionally, for secondary immunogenicity endpoints, outputs will be presented by pre-vaccination HAI antibody titer (<1:10 or  $\geq$  1:10).

## 9. DISPOSITION AND WITHDRAWALS

All subjects who are screened will be accounted for in this study.

Subject disposition, including the number (n) and percentage (%) of subjects in each treatment arm who completed the study and prematurely discontinued study participation (including primary reason for premature study discontinuation), will be tabulated for all subjects.

By-subject data listing of the disposition data i.e., age group, site, treatment, study status, completion/discontinuation date, and reason for discontinuation will be presented.

Frequency and percentage of subjects having critical, major and minor protocol deviations (see Appendix 1) will be presented by deviation category in vaccine, placebo and overall for all subjects in the FA Population. Subjects having multiple reasons for exclusion will be counted only once per each reason documented.

#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented both in summaries (by treatment group and overall) for the FA population and in listings for the Enrolled population.

No statistical testing will be performed for demographic or other baseline characteristics.

The following demographic and other baseline characteristics will be reported for this study:

- Age (years)
- Sex
- Ethnicity

## **10.1 DERIVATIONS**

For randomized subjects, age is calculated as the number of years from the date of birth to randomization date.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 778 Dated: 12 March 2018






## 11. CURRENT MEDICAL CONDITIONS

Current Medical Condition information will be presented for the FA population for summarising and listing the data. Current Medical Conditions will be coded using MedDRA dictionary version 20.0. The Current Medical Condition categories captured in the eCRF will be presented by system organ class (SOC) and preferred term (PT).

The summaries will be presented by primary SOC and PT for vaccine, placebo and overall for all subjects in the FA population. A subject will be counted only once within the SOC and PT if the subject has multiple medical conditions within the same SOC and PT.

A listing of current medical conditions will also be generated.

#### 12. MEDICATIONS

Medications will be presented for the FA population and are not coded.

Frequency and percentage of subjects receiving concomitant medications will be summarized by vaccine and placebo for each reported term.

A subject will be counted only once under reported term if the subject receives same concomitant medication multiple times.

By-subject listing of the data will be presented for the FA population.

#### 13. STUDY MEDICATION EXPOSURE

The date and time of vaccination and location of vaccination will be presented in the listings.

#### 14. STUDY MEDICATION COMPLIANCE

Not applicable for this study.

## 15. EFFICACY OUTCOMES

Not applicable for this study.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016






#### **16. IMMUNOGENICITY ANALYSIS**

#### 16.1 STATISTICAL CONSIDERATIONS

The Vietnam MOH guidance on serological immune response requirements for influenza vaccine is a modification of the EMEA/CPMP serological criteria for assessing seasonal influenza for licensure. The agegroup specific MOH licensure requirements for influenza vaccine in adults are shown in Table 3.

Table 3 Vietnam MOH Criteria for Evaluation of Influenza Vaccine Immune Responses

| | Age Group | |
|---|---|---|
| | 18 – 45 | 46 |
| Proportion achieving a HAI titer ≥ 1:40 (seroprotection) | ≥70% | ≥60% |
| Proportion achieving at least 4 fold rise in HAI titer (seroconversion) | ≥40% | ≥30% |
| GMT rise in HAI titer | ≥2.5 times | ≥2.0 times |

#### Null hypothesis (H<sub>0</sub>):

A single dose of IVACFLU-S seasonal trivalent split, inactivated influenza vaccine will not induce immune responses to each of the three vaccine antigens to meet one or both age group specific Vietnam Ministry of Health licensure requirements i.e., as mentioned in Table 3.

#### Alternative hypothesis (H<sub>1</sub>):

A single dose of IVACFLU-S seasonal trivalent split, inactivated influenza vaccine will induce immune responses to each of the three vaccine antigens to meet one or both age group specific Vietnam Ministry of Health licensure requirements i.e., as mentioned in Table 3.

Of the three criteria, seroconversion has been the most frequent criteria not meeting licensure threshold. Though the study assumption is based on Phase 1 immunogenicity data for adults 18-45 years of age, we anticipate the immune response in those 46 - 60 will be comparable since significant decline in antibody response is most associated with those who are ≥65 years of age.

Taken together with the immunogenicity results of the IVACFLU-S phase 1 study (refer to Section 2.1.6 in the protocol), the sample size consideration for immunogenicity for the study was based on the precision of the estimate of percent of vaccine recipients with HAI seroconversion and seroprotection responses. With a sample size of 100 evaluable vaccine recipients from each age group, the study provides the precision of immunogenicity response as estimated by width of 95% CI of ≤±10.2% around the range of estimated response rate (Table 4)

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016







Table 4: Observed Response Rate in 100 participants receiving study vaccine and Corresponding 95% CI.

| Number of responders (%) | 2-sided exact 95% CI |
|--------------------------|----------------------|
| 90 (90%) | [82.4%, 95.1%] |
| 80 (80%) | [70.8%, 87.3%] |
| 70 (70%) | [60.0%, 78.8%] |
| 60 (60%) | [49.7%, 69.7%] |
| 50 (50%) | [39.8%, 60.2%] |
| 40 (40%) | [30.3%, 50.3%] |
| 30 (30%) | [21.2%, 39.9%] |

An increase in sample size by 50% to 150 provides very limited statistical benefit as it only reduces the maximal width of 95% CI by 1.9% to  $\leq$  ±8.3%. All power calculations were made using 10000 simulations of binomial responses to each strain, based on assumed true response rates and pass/fail criteria. All calculations were made using SAS version 9.3.

# 16.1.1 PROBABILITY FOR DEMONSTRATING SEROCONVERSION CRITERIA FOR LICENSURE

For the 18-45 year old cohort, if the true seroconversion response to each strain is  $\geq$ 49%, then there is 91% probability that the point estimate for seroconversion to all three strains will be  $\geq$ 40%.

Likewise, if the true seroconversion response to each strain is  $\geq$ 60%, then there is 92% probability that the lower bound of the exact 95% CI for seroconversion to all strains will be  $\geq$ 40%. For the older age cohort (46-60 years old), if the true seroconversion response to each strain is  $\geq$ 39%, then there is 93% probability that the point estimate for seroconversion to all three strains will be  $\geq$ 30%. Given that the lowest seroconversion response in the IVAC Phase 1 trial was to B viral strain at 76.7% (95% CI, 57.7 90.1), there is high probability (Table 5) of demonstrating age group specific seroconversion requirement with a sample size of 100 evaluable participants per age group who received the study vaccine.

Table 5: Probability of demonstrating seroconversion response to all 3 viral strains by age groups and assumed true response to each viral strain.

| Age group (point | True response | | |
|---|---|---|---|
| estimate response) | Probability > 90% | Probability > 95% | Probability > 99% |
| 18-45 (≥40%) | ≥49% | ≥51% | ≥54% |
| 46- 60 (≥30%) | ≥39% | ≥40% | ≥43% |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.







# 16.1.2 PROBABILITY FOR DEMONSTRATING SEROPROTECTION CRITERIA FOR LICENSURE

For the 18-45 year old cohort there is 92% probability that the point estimate for seroprotection to all three strains will be  $\geq$  70% if the true response to each strain is  $\geq$ 78%. Likewise if the true response to each strain is  $\geq$ 87%, then there is 95% probability that the lower bound of the exact 95% CI for seroprotection to all strains will be  $\geq$ 70%. In the older age cohort (46-60 years old), if the true seroprotection response to each strain is  $\geq$ 69%, then there is 93% probability that the point estimate for seroprotection to all three strains will be  $\geq$ 60%. Given that the lowest seroprotection response in the IVAC Phase 1 trial was to B viral strain at 93.3% (95% CI 77.9; 99.2), there is high probability (Table 6) of demonstrating age group specific seroprotection requirement with a sample size of 100 evaluable participants per age group who received the study vaccine.

Table 6: Probability of demonstrating seroprotection response to all 3 viral strains by age groups and assumed true response to each viral strain.

| Ago group (point | True response | | |
|---|---|---|---|
| Age group (point estimate response) | Probability > 90% | Probability > 95% | Probability > 99% |
| 18-45 (≥70%) | ≥ 78% | ≥ 79% | ≥ 81% |
| 46- 60 (≥60%) | ≥ 69% | ≥ 70% | ≥ 72% |

#### 16.2 Analysis of Immunogenicity Endpoints

#### 16.2.1 PRIMARY IMMUNOGENICITY ENDPOINTS

- A. Number and percentage of subjects by age groups (18-45, 46-60) with seroconversion against each of the 3 vaccine antigens post-vaccination. Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
  - pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or</li>
  - pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination titer measured on Day
     22
- B. Number and percentage of subjects by age groups (18-45, 46-60) with seroprotection, defined as a HAI antibody titer ≥1:40 to each of the 3 vaccine antigens measured on Day 22 post vaccination
- C. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens
- D. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/prevaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Protocol No: IVACFLU-S-0203 782 Dated: 12 March 2018






#### 16.2.2 SECONDARY IMMUNOGENICITY ENDPOINTS

- A. Number and percentage of subjects by age groups (18-45, 46-60) who develop at least a four-fold increase in HAI antibody titer to each of the vaccine antigens post vaccination measured on Day 22 by prevaccination HAI antibody titer of <1:10 or ≥1:10.
- B. Geometric mean titers (GMTs) of serum HAI antibodies pre- (Day 1) and post vaccination (Day 22) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by prevaccination HAI antibody titer of <1:10 or ≥1:10.
- C. Geometric mean fold rises (GMFRs) of serum HAI antibodies (post vaccination/prevaccination) by age groups (18-45, 46-60) for each of the 3 vaccine antigens by prevaccination HAI antibody titer of <1:10 or ≥1:10.</p>

The following endpoints will be analyzed by age group:

- For each treatment group, the number and percentage of subjects with a serum HAI antibody titer ≥ 1:40
  to each of the 3 vaccine components measured on Day 22 post vaccination, will be presented along with
  two-sided exact 95% CIs using Clopper-Pearson method.
- 2. For each treatment group, the number and percentage of subjects with seroconversion against each of the 3 vaccine antigens post-vaccination will be presented along with two-sided exact 95% CIs using Clopper-Pearson method.
- 3. GMTs of serum HAI antibodies for each of the 3 antigens will be summarized at each time point (Day 1 and Day 22) by treatment group along with the corresponding two-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.
- 4. GMFRs of serum (HAI) antibodies (post-vaccination / pre-vaccination) for each of the 3 antigens will be summarized by treatment group along with the corresponding two-sided 95% CIs, by exponentiating the corresponding difference in log-transformed means between post-vaccination and pre-vaccination antibodies and their 95% CIs obtained via paired t-test method.

The following endpoints will be analyzed by age group and pre-vaccination HAI antibody titer of <1:10 or ≥1:10:

- For each treatment group, the number and percentage of subjects who develop at least a four-fold
  increase in HAI antibody titer to each of the 3 vaccine antigens measured on Day 22 post vaccination, will
  be presented along with two-sided exact 95% CIs using Clopper-Pearson method. (Please refer to
  Appendix 2 for sample SAS code for 95% confidence interval for single proportion using Exact ClopperPearson method).
- 2. GMTs of serum HAI antibodies for each of the 3 antigens will be summarized at each time point (Day 1 and Day 22) by treatment group along with the corresponding two-sided 95% CIs, by exponentiating the corresponding log-transformed means and their 95% CIs.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

783 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






3. GMFRs of serum (HAI) antibodies (post-vaccination / pre-vaccination) for each of the 3 antigens will be summarized by treatment group along with the corresponding two-sided 95% CIs, by exponentiating the corresponding difference in log-transformed means between post-vaccination and pre-vaccination antibodies and their 95% CIs obtained via paired t-test method.

Subject wise listing will be generated.

Graphical representation of the data will be as follows:

- 1. Geometric mean HAI titer for each of the 3 antigens at Days 1 and 22 will be plotted by vaccine group separately for each age group.
- 2. Reverse Cumulative Distribution (RCD) plot will show reverse cumulative percentages for HAI titer for each of the 3 antigens at Day 1 and Day 22 by vaccine group and by age group.

The immunogenicity analyses will be performed using PP population.

All immunogenicity analyses will also be conducted using FA population as supportive analyses.

#### 16.3 Variables & Derivations

Titers below the limit of quantification (i.e. below the starting dilution of assay reported as "< 10") will be set to half that limit (i.e. 10/2 = 5). If a titer is reported as greater or equal to the upper limit of the assay, it will be set to that limit.

#### Fold increase (rise) [FI]:

If "vpre" is a subject's pre-vaccination (baseline) immunogenicity value and "vpost" the post-vaccination value, then the "fold increase (rise)" [FI] will be calculated as:

FI = vpost / vpre

#### Seroprotection:

Taking influenza as an example, the threshold is an anti-HA antibody level of 40, and subjects with HAI antibody titre >=40 are said to be seroprotected for influenza.

#### Seroconversion:

Seroconversion is defined as

- pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40; or
- pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 22

i.e. subjects with an HAI antibody titer<10 and >=40 before vaccination and post vaccination i.e., on Day 22 respectively; or

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.






an HAI antibody titer>=10 and at least a four-fold increase in post vaccination measured on Day 22 i.e.,

#### **17. SAFETY OUTCOMES**

#### 17.1 STATISTICAL CONSIDERATIONS:

#### Null hypothesis (H<sub>0</sub>):

A single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) is not safe and well tolerated in adults 18 to 60 years of age.

#### Alternative hypothesis (H<sub>1</sub>):

A single dose of seasonal trivalent inactivated split virion influenza vaccine (IVACFLU-S) is safe and well tolerated in adults 18 to 60 years of age.

The total sample size for Phase 2 and Phase 3 combined will be 888 subjects. With subjects randomized to IVACFLU-S or placebo at a randomization ratio of 5:1, there will be 740 subjects randomized to IVACFLU-S arm in the phase 2/3 study. Accounting for a 5% dropout rate, there would be at least 700 evaluable participants for safety analysis. If no vaccine-related serious adverse events are observed in 700 vaccine recipients, the study would able to exclude events occurring at approximately 0.43% based on the upper bound of the one sided 95% Confidence Interval (CI)) using the Clopper-Pearson method.

The probability of observing at least one vaccine-related serious adverse event in 700 subjects is 90 % and >95% if the true rate of such events is 0.33 % and 0.43% respectively. The precision of the estimate of AEs judged to be related to IVACFLU-S as bounded by 95% CI is presented in Table 7.

Table 7: Exact 95% Confidence Intervals around Potential Number of Study Related Adverse Events

| Sample size | Number of events | 2-sided exact 95% CI |
|-------------|------------------|----------------------|
| | 0 | [0, 0.52*] |
| | 1 | [<0.01, 0.79] |
| 700 | 2 | [0.03, 1.02] |
| | 3 | [0.08, 1.24] |
| | 5 | [0.23, 1.65] |

<sup>\*</sup>one sided, 97.5% CI

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0

Author: Revathi Rayadurgam Version Number: Version Date: [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016
785 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






However, the full analysis population will be used for safety analysis, not the assumed number of 700 evaluable subjects.

## 17.2 ANALYSIS OF SAFETY ENDPOINTS:

The safety profile of IVACFLU-S will be evaluated by the number and proportion of subjects experiencing AEs by severity relatedness to vaccination in the following four categories for all subjects and by age group (solicited AEs will be considered related to study product):

- A. Solicited local adverse events, including redness / erythema, swelling / induration, pain within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- B. Solicited systemic adverse events, including fever, fatigue, malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache within 30 minutes of vaccination and over a 7-day period (Days 1-7) post-vaccination.
- C. Unsolicited AEs occurring within 21 days post vaccination.
- D. Serious Adverse Events occurring during the entire study period (Days 1 to 91).

## 17.2.1 SOLICITED LOCAL AND SYSTEMIC ADVERSE EVENTS

Solicited adverse events are pre-specified local and systemic adverse events that are common or known to be associated with vaccination that are actively monitored as indicators of vaccine reactogenicity. Investigators will not be required to assess causality of solicited adverse events if the onset is during the solicitation periods. If a solicited adverse event progresses beyond the solicited period, it will continue to be reported as a solicited adverse event. If the solicited adverse event occurs after the solicitation period it will be reported as an unsolicited AE.

Any solicited local or systemic reactogenicity that occurs during the 5-day period post-injection is automatically regarded as related.

Solicited local and systemic AEs will be assessed by study staff 30 minutes after vaccination then daily for 7 days by the subjects.

- Solicited local adverse event (at site of injection):
  - Erythema / redness based on size in cm
  - Swelling / induration (hardness at site of injection ) based on size in cm
  - Pain
- Systemic Reactions:
  - Fever--Body temperature (measured in degrees Celsius)
  - Fatigue/malaise
  - Generalized muscle aches
  - Joint aches
  - Chills

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


786 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






- Nausea
- Vomiting
- Headache

Solicited local and systemic adverse events will be graded by a Principal Investigator (PI) using a standardized data collection instrument. Grading will use predefined scales based on functional assessment or magnitude of reaction, where available. Where grading scales are not provided, the reaction will be graded for severity based on interference with subject functionality, as for all other AEs. Severity of redness, swelling and induration at the injection site will always be graded based on the size. Temperature will be graded according to the following criteria:

- Ungradable
- Grade 1= '38.0 <38.6°C '
- Grade 2= '38.6 <39.3°C'
- Grade 3=' 39.3 <40.0°C'
- Grade 4=' ≥ 40.0°C'

## 17.2.1.1 Presentation of 30-minute solicited local and SYSTEMIC REACTOGENICITY

The following will be presented for the FA population:

- 1. Subject-wise listing of 30-minute solicited local and systemic reactogenicity will be generated separately.
- 2. Summary of 30-minute solicited local and systemic reactogenicity will be provided separately as follows:

  - Count and percentages of participants experiencing each reaction or event, or at least one reaction or event will be calculated along with two-sided exact 95% CIs using Clopper-Pearson method (refer Appendix 2) for each treatment group, and by age group.
  - Fisher's exact test (refer Appendix 3) or Cochran-Mantel-Haenszel test (refer Appendix 4) will be used to compare the proportion of participants between the two treatment groups.
- 3. Descriptive summary (as described for continuous variables in Section 6) of the size of the solicited local reactions captured in 30-minute reactogenicity page of the eCRF will be presented by vaccine and placebo.
- 4. In addition, for all Solicited Local and Systemic Adverse Events, the following will be summarised by severity:
  - Counts of all events will be reported and summarized, as "any local AE" or "any systemic AE".

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 787 Dated: 12 March 2018






- Percentages of subjects experiencing each reaction or event, at least one reaction or event will be calculated. This will be generated separately i.e., one output for Body temperature (Oral) and one output for all other adverse events, as the severity grades will be as follows:
  - Body temperature (Oral):
    - Ungradable
    - Grade 1= '38.0 <38.6°C '</li>
    - Grade 2= '38.6 <39.3°C'</p>
    - Grade 3=' 39.3 <40.0°C'
    - Grade 4=' ≥ 40.0°C'
  - o For local and systemic adverse events:
    - None
    - Mild
    - Moderate
    - Severe
    - Potentially Life Threatening

# 17.2.1.2 PRESENTATION OF SOLICITED LOCAL AND SYSTEMIC ADVERSE EVENTS

The following will be presented for the FA population:

- 1. Subject-wise listing of solicited local and systemic adverse events will be generated separately.
- 2. Summary of solicited local and systemic adverse events will be provided separately as follows:
  - Counts and percentages of subjects experiencing each reaction or event, at least one reaction or event will be calculated.
  - Number of events for each reaction or event will also be displayed.
  - Event will be counted only one time if occurred on consecutive days.

Percentages of participants experiencing each reaction or event, or at least one reaction or event will be calculated along with two-sided exact 95% CIs using Clopper-Pearson method (refer Appendix 2) for each treatment group and by age group. Fisher's exact test (refer Appendix 3) or Cochran-Mantel-Haenszel test (refer Appendix 4) will be used to compare the proportion of participants between the two treatment groups.

3. Summary of solicited local and systemic adverse events, as described in the above point 2 will be repeated i.e., summarized by day:

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 788 Dated: 12 March 2018






- Counts and percentages of subjects experiencing each reaction or event, at least one reaction or event will be calculated.
- Number of events for each reaction or event will also be displayed.
- 4. Descriptive summary (as described for continuous variables in Section 6) of the size of the solicited local reactions captured as per the eCRF will be presented by vaccine and placebo.

In addition, for all Solicited Local and Systemic Adverse Events the following will be summarised by maximum severity until resolution:

- Counts of all events will be reported and summarized, as "any local AE" or "any systemic AE".
  - Percentages of subjects experiencing each reaction or event, at least one reaction or event will be
    calculated. This will be generated separately i.e., one output for Body temperature (Oral) and one
    output for all other adverse events, as the severity grades will be as follows:
    - o Body temperature (Oral):
    - Ungradable
    - Grade 1= '38.0 <38.6°C '</li>
    - Grade 2= '38.6 <39.3°C'
    - Grade 3=' 39.3 <40.0°C'
    - Grade 4=' ≥ 40.0°C'
    - o For local and systemic adverse events:
    - None
    - Mild
    - Moderate
    - Severe
    - Potentially Life Threatening

## 17.2.2 UNSOLICITED ADVERSE EVENTS

Unsolicited adverse events are any AEs that occur any time after the vaccine/placebo is given (temporally related to study product), whether or not deemed "related" to the product, and are not solicited (specifically asked of the participant). Unsolicited AEs can be observed by study staff while the participant is at a clinic for a study visit or reported by the participant at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination will be recorded as an unsolicited AE.

No statistical testing will be performed for unsolicited AEs. Unsolicited AEs with a missing relationship to vaccine will not be imputed.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.






Subject-wise listing will be presented.

The following will be presented for FA population:

- 1. Summary of Unsolicited Events, i.e., summary displayed for the following:
  - Total number of unsolicited AEs,
  - Subjects with at least one unsolicited AE,
  - At least one vaccine related unsolicited AE,
  - At least one serious unsolicited AE,
  - At least one severe unsolicited AE,
  - At least one life threatening unsolicited AE,
  - Subjects requiring treatment during the study,
  - Subjects with unsolicited AEs leading to withdrawal, and
  - Number of subjects died.
- 2. Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term within Day 1 to Day
- 3. Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term and severity within Day 1 to Day 22 i.e.:
  - All Adverse events are classified by severity as "Mild", "Moderate", "Severe" and "Lifethreatening".

  - Counts of all events will be reported and summarized, as "Any Unsolicited AE". Percentages of subjects experiencing each reaction or event, at least one reaction or event will be calculated.
- 4. Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term and relationship within Day 1 to Day 22
- 5. Summary of Unsolicited Adverse Events requiring treatment by System Organ Class and Preferred Term within Day 1 to Day 22

## 17.2.3 SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded as "Serious" on the Adverse Events page of the (e)CRF. A summary of serious AEs by SOC and PT will be prepared.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0

Author: Revathi Rayadurgam Version Number: Version Date: [11AUG2017]

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

790 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






No statistical testing will be performed for SAEs.

Subject-wise listing will be presented.

The following will be presented for FA population:

- 1. Summary of Serious Events, i.e., summary displayed for the following:
  - Total number of serious AEs,
  - Subjects with at least one serious AE,
  - At least one vaccine related serious AE,
  - At least one serious AE,
  - At least one severe serious AE,
  - At least one life threatening serious AE,
  - Subjects requiring treatment during the study,
  - Subjects with serious AEs leading to withdrawal, and
  - Number of subjects died.
- 2. Summary of serious Adverse Events by System Organ Class and Preferred Term within Day 1 to Day 91
- 3. Summary of serious Adverse Events by System Organ Class and Preferred Term and severity within Day 1 to Day 91 i.e.:
  - All Adverse events are classified by severity as "Mild", "Moderate", "Severe" and "Lifethreatening".
  - Adverse events with missing severity will be considered as "Severe".
  - Counts of all events will be reported and summarized, as "Any Unsolicited AE". Percentages of subjects experiencing each reaction or event, at least one reaction or event will be calculated.
- 4. Summary of Serious Adverse Events by System Organ Class and Preferred Term and relationship within Day 1 to Day 91
- 5. Summary of Serious Adverse Events requiring treatment by System Organ Class and Preferred Term within Day 1 to Day 91

#### 17.3 DEATHS

Listing of deaths will be provided.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203 SAP Draft v1.0

Author: Revathi Rayadurgam Version Number: Version Date: [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or

reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 791 Dated: 12 March 2018






## 17.4 ECG EVALUATIONS

No ECG data is collected in the study.

## 17.5 VITAL SIGNS

Vital sign measurements include body temperature (oral), blood pressure (systolic and diastolic) and heart rate collected at Screening and Day 8 of the study.

The vital signs measurements, including abnormalities (grading for body temperature and blood pressure) and heart rate associated along with clinical significance (Yes/No) will be presented in the listings.

The following summaries will be provided for vital signs data:

- Actual and change from Baseline to Day 8
- Actual and change from Baseline to Day 8 by grade
- Shift from Baseline to Day 8 by grade
- Number and percentage of subjects by clinical significance
- Number and percentage of subjects shift from Baseline to Day 8 by clinical significance

### 17.6 PHYSICAL EXAMINATION

#### **General Physical Examinations:**

Qualified study clinicians will conduct a physical examination of all participants at S1/D1. This physical examination will include the following:

- Recording of general appearance
- Physical examination of all organ systems. This includes the following:
  - o neurologic examination, including cranial nerve examination
  - o chest auscultation
  - examination of lymph nodes (axillary and cervical)
  - heart auscultation
  - abdomen palpation (to check for liver size)
- Measurement of the following vital signs:
  - o body temperature
  - blood pressure
  - o pulse/heart rate

Grade 1 elevated blood pressure (140 to < 160 mmHg systolic OR 90 to < 100 mmHg diastolic) will not be considered to be exclusionary at screening, unless judged to be clinically significant by the PI.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.


Protocol No: IVACFLU-S-0203 792 Dated: 12 March 2018






#### **Targeted Physical Examination**

The Targeted Physical Examination (PE) focuses on symptoms reported by the participant and the presence or absence of local and systemic reactogenicity. If no symptoms are reported by the participant, the Targeted PE does not need to be performed. The exam will be made by a clinician on D1 (only if D1 is on a different day from S1) and Day 8. Evaluation must be made prior to administration of injection of study product if done on Day 1.

Subject-wise listing of the data will be presented.

Summary of Shift from baseline to Day 8 by clinically significant abnormal physical examination will also be presented.

## 18. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

- Comments
- SAE narratives

These domains and/or variables will not be summarized or presented, but will be available in the clinical study database, SDTM and/or ADaM datasets.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

793 Dated: 12 March 2018 Protocol No: IVACFLU-S-0203






## **APPENDIX 1**

#### **Protocol Deviation Classifications**

| Categories | Severity |
|---|---|
| <ul> <li>Informed consent</li> <li>Eligibility and Entry Criteria</li> <li>Concomitant Medication Criteria</li> <li>Study Procedures Criteria</li> <li>Serious Adverse Event Criteria</li> <li>Randomization Criteria</li> <li>Visit Schedule Criteria</li> <li>Administrative Criteria</li> <li>Source Document Criteria</li> <li>RA or CEC Approvals Criteria</li> <li>IP Compliance</li> <li>Other Criteria</li> </ul> | Minor Deviations from accepted procedures that will not adversely affect subject/data, but should be dealt with appropriately. Major Protocol Deviation Issues that impact upon scientific, ethical, regulatory or business integrity and which, if left unattended could become critical. Such issues require timely action. Critical Protocol Deviation Issues that threaten scientific, ethical, regulatory or business integrity and could invalidate acceptability of a study (or part of it) to a customer or regulatory body, or invoke regulatory action which require immediate attention. |

Critical deviations include, but are not limited to:

Eligibility and entry criteria: subject was enrolled even though entry criteria were not satisfied

Subject did not sign ICF yet was enrolled into the study

Any study procedures on S1 day were done prior to consent being signed

## Major deviations include, but are not limited to:

Incorrect study product assigned and administered according to randomization

Incorrect version of signed ICF (not currently approved version)

ICF was not signed by either investigator or study participant

IP temperature excursion (important deviation if IP is not allowed to be used, minor deviation if IP is allowed to be used)

Subject does not complete more than 50% of subject diary card

Subject visit (D8, D22, D91) is not completed or not done Use of prohibited drugs during study period SAE not reported according to protocol requirement

Immunological sample is not collected as per protocol requirement (collected sample which cannot be analyzed is not considered as a deviation)

Loss of source documents

## Minor deviations include, but are not limited to:

Subject visit is outside of visit window

Incomplete source documents

Procedures carried out by staff not delegated in the delegation log

Temperature log is not maintained as per protocol requirement

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics Document:

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Protocol No: IVACFLU-S-0203 794 Dated: 12 March 2018






## **APPENDIX 2**

Sample SAS code for 95% confidence interval for single proportion using Exact Clopper-Pearson method:

```
proc freq data =combb order=data;
by _name_ atptn atpt mord parcat3n parcat3 cat;
tables pflg / binomial (exact) alpha = 0.05;
weight cnt/zero;
ods output BinomialCLs = bin_ci;
run;
```

## **APPENDIX 3**

Sample SAS code to compute P-value based on Chi-square or Fisher's exact test:

## **APPENDIX 4**

Sample SAS code to compute P-value based on Cochran-Mantel-Haenszel test

```
proc freq data= combb;
   tables strat1 *Treatment* strat2/ cmh;
   weight Count;
   run;
```

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics

\Documentation\SAP\IVACFLU-S-0203\_SAP\_Draft v1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.



1.0

11AUG 2017]

PROTOCOL IVACFLU-S-0203 

TABLE AND LISTING MOCK SHELL

QuintilesIMS

ANNOTATED SHELLS

## **IVACFLU-S, Phase 2/3**

A PHASE 2 / 3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF A SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA **VACCINE (IVACFLU-S) PRODUCED BY IVAC** 

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203 Mock Tables V1.0 Author:

Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

796


Dated: 12 March 2018

(Q) QuintilesIMS


(IVAC) PROTOCOL IVACFLU-S-0203 

TABLE AND LISTING MOCK SHELL

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 11AUG2017) for Protocol IVACFLU-S-0203 (Dated 09FEB2017).

| | Name | Signature | Date |
|---|---|---|---|
| Author: | Revathi Rayadurgam | (R) Her | 14/AUG/17 |
| Position: | Biostatistician 2 | V | 4 - g summer communicative management accommunication |
| Company: | QuintilesIMS | | The same transfer |

Upon review of this document, the undersigned approves this version of the Output templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | Cheesens) | 14/AUQ/2017 |
| Position: | Manager, Biostatistics | | |
| Company: | QuintilesIMS | | |
| Approved By: | Krista Yuhas | Elleur yohn | 14/Aug /2017 |
| Position: | Biostatistician, Center fo | or Vaccine Innovation and Access | (CVIA) |
| Company: | PATH | Suprama space spac | S. A. CONTROL E. L. DOMINION C. L. MINISTER, C. P. S. CONTROL C. L. MARCHANICA C. M. CONTROL C. M. C. C. C. C. |
| Approved By: | Tushar Tewari | | |
| Position: | Senior Medical Officer, ( | Clinical and Regulatory Affairs | |
| Company: | PATH | | The second secon |

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:


1.0 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS WI BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Dated: 12 March 2018

797




IVAC


TABLE AND LISTING MOCK SHELL

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 11AUG2017) for Protocol IVACFLU-S-0203 (Dated 09FEB2017).

| | Name | Signature | Date |
|-----------|--------------------|-----------|---------------|
| Author: | Revathi Rayadurgam | | |
| Position: | Biostatistician 2 | | in the second |
| Company: | QuintilesIMS | | |

Upon review of this document, the undersigned approves this version of the Output templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | | |
| Position: | Manager, Biostatistics | | |
| Company: | QuintilesIMS | 100000000000000000000000000000000000000 | THE STATE OF THE PROPERTY OF THE STATE OF |
| Approved By: | Krista Yuhas | | |
| Position: | Biostatistician, Center | for Vaccine Innovation and A | Access (CVIA) |
| Company: | PATH | | |
| Approved By: | Tushar Tewari | [luna" | 11 Aug 2017 |
| Position: | Senior Medical Office | , Clinical and Regulatory Affa | airs |
| Company: | PATH | | |

Document: Author: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Revathi Rayadurgam

Version Number: Version Date:

11AUG 2017]

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.





## QuintilesIMS

#### TABLE AND LISTING MOCK SHELL

## **MODIFICATION HISTORY**

| Unique Identifier for this Version | Date of the Document<br>Version | Author | Significant Changes from<br>Previous Authorized<br>Version |
|---|---|---|---|
| | | Revathi Rayadurgam | Not applicable. First version. |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: Version Number:

Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

799

Dated: 12 March 2018






## TABLE AND LISTING MOCK SHELL

#### Table of Contents

| Author: | Revathi Rayadurgam | Version Number:<br>Version Date: | | 1.0<br>11AUG 2017] |
|---|---|---|---|---|
| Document: | Geometric Mean Fold Rise (GMFR) for the Hemagglutina: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Doc | · | | <u> </u> |
| population | Connected a Many Bold Disc (CMBD) for the W | udan makikinin (*** | V militaria har v | 20 |
| | Geometric Mean titer (GMT) for the Hemagglutination | n inhibition (HAI) : | Titers by Age ( | |
| population | | - 1 11 1 1 1 1 1 1 1 1 1 | | 19 |
| | Geometric Mean titer (GMT) for the Hemagglutination | on innibition (HAI) | Titers by Age | |
| Full Analysis | • • | | mittage has been | |
| | Seroprotection and 95% Confidence Intervals for the | nemaggrutination inf | HIDICIOH (HAI) | Titers by Age group |
| Per-protocol po | | Homowalutinotion Inl | hibition (HAT) | |
| | Seroprotection and 95% Confidence Intervals for the | Hemaggiutination in | nibition (HAI) | Titers by Age group |
| Full Analysis | • • | H | 646444 (H7T) | 17 |
| | Seroconversion and 95% Confidence Intervals for the | Hemagglutination Inf | hibition (HAI) | 1 3 3 1 |
| Per-protocol po | | #**************************** | | |
| | Seroconversion and 95% Confidence Intervals for the | Hemagglutination Inf | hibition (HAI) | Titers by Age group |
| | Summary of Concomitant Medications Full Analysis Popu | | | 16 |
| | Summary of Current Medical Condition Full Analysis Po | - | | 15 |
| | Demographics and Other Baseline Characteristics Full | | | 13 |
| | Analysis Sets Enrolled Population | | | 12 |
| | Protocol Deviations Full Analysis Population | | | 11 |
| | Subject Disposition Enrolled Population | | | |
| m-1-1 - 14 1 1 1 | Cubinet Disperition Develop Develop | | | 9 |

Template No: CS\_TP\_BS016 Revision 4

Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

Protocol No: IVACFLU-S-0203 800

**IVACFLU-S** Version 1.0 Dated: 12 March 2018






Reference: CS\_WI\_BS005

TABLE AND LISTING MOCK SHELL

| Document:<br>Author: | \\IEEDC-NAS01A\Biosdata\Path\\VACFLU-S\IYA06804\Biostatistics \Documentation\SAP\\VACFLU-S-0203_Mock_Tables_V1.0 Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017 |
|---|---|
| Figure 14.2.1.3 | Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group 46-60 - |
| Full analysis pop | pulation 27 |
| Figure 14.2.1.2 | Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group [18-45] - |
| Per-protocol popu | alation 25 |
| Figure 14.2.1.1 | Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group [18-45] - |
| vaccination titer | group Full Analysis population 24 |
| Table 14.2.1.14 0 | Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by age group and pre- |
| vaccination titer | group Per-protocol population 23 |
| Table 14.2.1.13 0 | Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by age group and pre- |
| titer group Full | 1 Analysis population 23 |
| Table 14.2.1.12 G | eometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination |
| titer group - Per | c-protocol population 22 |
| Table 14.2.1.11 G | eometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination |
| group and pre-va | accination titer group - four-fold rise - Full Analysis population |
| Table 14.2.1.10 I: | Emmune Response Rates and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by age |
| group and pre-va | accination titer group -four-fold rise - Per-protocol population 21 |
| Table 14.2.1.9 Im | mmune Response Rates and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by age |
| population | 20 |
| Table 14.2.1.8 Ge | cometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by Age group Full Analysis |
| population | 20 |

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.


Protocol No: IVACFLU-S-0203 801 Dated: 12 March 2018





1.0

11AUG 2017]


TABLE AND LISTING MOCK SHELL

| Per-protocol population | $_{1}$ | 7 |
|---|---|---|
| Figure 14.2.1.4 Rever | se cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group 46-60 | _ |
| Full analysis population | on 2 | 7 |
| Figure 14.2.1.5 Rev | erse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Overall - Per | _ |
| protocol population | 2 | 7 |
| Figure 14.2.1.6 Revers | e cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Overall - Full analysis | S |
| population | 2 | 7 |
| Figure 14.2.1.7 Geome | tric Mean Titer (GMT) Plot for Hemagglutination Inhibition (HAI titer) at Day 1 and Day 22 by ago | е |
| group - Per-protocol po | opulation 2 | 8 |
| Figure 14.2.1.8 Geome | tric Mean Titer (GMT) Plot for Hemagglutination Inhibition (HAI titer) at Day 1 and Day 22 by ago | е |
| group - Full analysis p | population 2 | 9 |
| Table 14.3.1.1 Overview | v of Adverse Events Full Analysis Population | 0 |
| Table 14.3.2.1.1 Incide | ence of Solicited Local Adverse Events from Day 1 to Day 7 Full Analysis Population 3. | 2 |
| Table 14.3.2.1.2 Incide | ence of Solicited Systemic Adverse Events from Day 1 to Day 7 Full Analysis Population 3. | 2 |
| Table 14.3.2.1.3 Incide | ence of Solicited 30 minutes Local Adverse Event Full Analysis Population 3- | 4 |
| Table 14.3.2.1.4 Incide | ence of Solicited 30 minutes Systemic Adverse Event Full Analysis Population 3- | 4 |
| Table 14.3.2.1.5 Incide | ence of Solicited Local Adverse Event by Day Full Analysis Population | 5 |
| Table 14.3.2.1.6 Incide | ence of Solicited Systemic Adverse Event by Day Full Analysis Population | 6 |
| Table 14.3.2.1.7 Incide | ence of Solicited Local Adverse Events Captured within 30 minutes after Vaccination by severity Ful | 1 |
| Analysis Population | 3 | 6 |
| Document: \\IEEI | DC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203_Mock_Tables_V1.0 | |

Version Number:


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Author:

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Revathi Rayadurgam

Version 1.0 Protocol No: IVACFLU-S-0203 802 Dated: 12 March 2018






Reference: CS\_WI\_BS005

#### TABLE AND LISTING MOCK SHELL

| Document:<br>Author: | \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804<br>Revathi Rayadurgam | AlBiostatistics \Documentation\SAP\IVACFLU-S-0203_Mock_Tables<br>Version Number:<br>Version Date: | ;_V1.0<br>1.0<br>11AUG 2017] |
|---|---|---|---|
| Table 14.3.4.1 | .3 Summary of Serious Adverse Events by | System Organ Class and Preferred Term and So | everity Full Analysis |
| Table 14.3.4.1 | .2 Summary of Serious Adverse Events by S | ystem Organ Class and Preferred Term Full Ana | lysis Population 44 |
| Table 14.3.4.1 | .1 Summary of Serious Adverse Events Full | Analysis Population | 44 |
| Analysis Popula | ation | | 44 |
| Table 14.3.3.1 | .5 Summary of Unsolicited Adverse Events | Requiring Treatment by System Organ Class an | d Preferred Term Full |
| Analysis Popula | ation | | 43 |
| Table 14.3.3.1 | .4 Summary of Unsolicited Adverse Events | by System Organ Class and Preferred Term a | and Relationship Full |
| Population | | | 42 |
| Table 14.3.3.1 | .3 Summary of Unsolicited Adverse Events b | y System Organ Class and Preferred Term and s | everity Full Analysis |
| | | | 41 |
| Table 14.3.3.1 | .2 Summary of Unsolicited Adverse Events | by System Organ Class and Preferred Term Ful | l Analysis Population |
| Table 14.3.3.1 | .1 Summary of Unsolicited Events Full Ana | lysis Population | 40 |
| Analysis Popula | ation | | 39 |
| Table 14.3.2.2 | .2 Summary of Solicited Systemic Adverse | Event Captured by Maximum severity between | Day 1 to Day 7 Full |
| Population | | | 39 |
| Table 14.3.2.2. | .1 Summary of Solicited Local Adverse Even | t Captured by Maximum Severity between Day 1 t | to Day 7 Full Analysis |
| Analysis Popula | ation | | 38 |
| Table 14.3.2.1 | .9 Summary of the Size of the Solicited A | dverse Event Captured within 30 minutes afte | r Vaccination Full |
| Full Analysis I | Population | | 37 |

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

IVACFLU-S

Q) QuintilesIMS





#### TABLE AND LISTING MOCK SHELL

| Population | 44 |
|---|---|
| Table 14.3.4.1.4 Summary of Serious Adverse Events by System Organ Class and Preferred Term and Relationship Full Analysis | sis |
| Population | 44 |
| Table 14.3.4.1.5 Summary of Serious Adverse Events Requiring Treatment by System Organ Class and Preferred Term F | ull |
| Analysis Population | 45 |
| Table 14.3.5.1 Deaths Full Analysis Population | 46 |
| Table 14.3.6.1 Summary of Vital Signs Full Analysis Population | 47 |
| Table 14.3.6.2 Shift from Baseline to Day 8 of Vital Signs by Grade Full Analysis Population | 48 |
| Table 14.3.6.3 Shift from Baseline to Day 8 of Clinically Significant Vital Signs Parameter Full Analysis Population | 50 |
| Table 14.3.7.1 Shift from Baseline to Day 8 by Clinically Significant Abnormal Physical Examination Full Analysis Populat | ion |
| | 51 |

803

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Version Number:

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


**IVACFLU-S** Version 1.0 804 Dated: 12 March 2018






TABLE AND LISTING MOCK SHELL

Table 14.1.1.1 Subject Disposition Enrolled Population

#### Pooled sites:

| | Vaccine<br>N(=XX)<br>n(%) | Placebo<br>N(=XX)<br>n(%) | Total N(=XX) n (%) |
|---|---|---|---|
| <overall>:</overall> | | | |
| NUMBER OF SCREENED SUBJECTS | | | xx |
| NUMBER OF SUBJECTS NOT RANDOMIZED | | | xx |
| NUMBER OF SUBJECTS RANDOMIZED | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SUBJECTS COMPLETED THE STUDY | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SUBJECTS DISCONTINUED STUDY AFTER SCREENING AFTER DAY 1 AFTER DAY 8 AFTER DAY 22 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| REASON FOR DISCONTINUATION OF STUDY VOLUNTARY WITHDRAWAL LOST TO FOLLOW-UP SPONSOR DECISION INVESTIGATOR DECISION AE/SAE OTHER | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

N = Total number of subjects in each group, n = Number of subjects in each category, % = Calculated relative to the total number of subjects randomized Source Data: Listing 16.2.1.1

Programming note: Repeat the table for the following in the same table. Display each combination in separate page i.e., as shown above.

- Pooled sites: Age group: 18-45,
- Pooled Sites: Age group: 46-60,
- Site 1: Overall,

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number: Version Date:

1.0 11AUG 2017]

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** 

Protocol No: IVACFLU-S-0203 805 Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

Site 1: Age group: 18-45,Site 1: Age group: 46-60,

• Site 2: Pooled age groups,

• Site 2: Age group: 18-45,

• Site 2: Age group: 46-60

Please note that "Overall" is the pooled age groups. Not to be included in the footnotes.

Document: \|\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \|\Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Version Date: 11AUG 2017

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S

806






1.0

11AUG 2017]


TABLE AND LISTING MOCK SHELL

Table 14.1.1.2
Protocol Deviations
Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | Vaccine | Placebo | Total |
|---|---|---|---|
| | N(=XX) | N(=XX) | N(=XX) |
| | n(%) | n(%) | n (%) |
| Subjects With at Least One Protocol Deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Critical Deviations* | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxxx1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Major Deviations* | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxxx1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Minor Deviations* | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Xxxxxxxx1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population, n= Number of subjects in each category, %= Calculated relative to the total number of subjects in the relevant population

\*The same subjects with multiple protocol deviations were counted only once in that category.

The same subject meeting multiple protocol deviation criteria was counted under each criterion.

Potential Protocol Deviations for the study are categorized according to the pre-defined categories within Clinical Trial Management System (CTMS). Source Data: Listing 16.2.2.1

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Version Number:}


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** Protocol No: IVACFLU-S-0203

807






## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.1.1.3 Analysis Sets Enrolled Population

Age Group: <0verall> <18-45> <46-60>

| | Vaccine (N= XX) | Placebo (N= XX) | Total (N= XX) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Number of Subjects included in the Full Analysis Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects Excluded from the Full Analysis Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 01<br>Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects included in the Per-Protocol Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects Excluded from Per-Protocol Population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 01<br>Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population, n= Number of subjects in each category, %= Calculated relative to the total number of subjects in the relevant population


Source Data: Listing 16.2.1.3

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

1.0 11AUG 2017]

Effective Date: 01Apr2016

808





Dated: 12 March 2018


1.0

11AUG 2017]


#### TABLE AND LISTING MOCK SHELL

QuintilesIMS

#### Table 14.1.2.1 Demographics and Other Baseline Characteristics Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| /ariable (Unit) | | Vaccine | Placebo | Total |
|--------------------------|-----------|-----------|-----------|-----------|
| | Statistic | (N=XX) | (N=XX) | (N=XX) |
| (V) | | | | |
| Age (Years) | <b>n</b> | | | |
| | n | XX | XX | XX |
| | Mean | XX.X | XX.X | xx.x |
| | Median | XX.X | XX.XX | XX.XX |
| | SD | XX.XX | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Sex | | | | |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Child bearing Potential* | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | |
| Kinh | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Khmer | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hoa | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

Max: Maximum; Min; Minimum; SD: Standard Deviation

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, % = Calculated relative to the total number of subjects in the relevant population with data available


\*Percentages were based on the total number of female subjects in each group.

Source Data: Listing 16.2.4.1

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S

Protocol No: IVACFLU-S-0203 809 Dated: 12 March 2018






## TABLE AND LISTING MOCK SHELL

Programming Note: Add a "Missing" row in each category if it is applicable.

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203 Mock Tables V1.0 Version Number:

Author: 1.0 Revathi Rayadurgam 11AUG 2017] Version Date:

Template No: CS\_TP\_BS016 Revision 4

Reference: CS\_WI\_BS005 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited. IVACFLU-S Protocol No: IVACFLU-S-0203

810







#### TABLE AND LISTING MOCK SHELL

Table 14.1.2.2 Summary of Current Medical Condition Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| System organ Class/Preferred Term | Vaccine | Placebo | Total |
|-----------------------------------------|-----------|-----------|-----------|
| | (N=XX) | (N=XX) | (N=XX) |
| | n (%) | n (%) | n (%) |
| SOC 1 Preferred Term 1 Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 Preferred Term 1 Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |

...

Data is based on the combined phases 2 and 3, pooled across study sites.

MedDRA: Medical Dictionary for Regulatory Activities; SOC: System Organ Class; PT: Preferred Term

N = Total number of subjects in the relevant population (per by-group stratification level, where relevant), n = Number of subjects in each category

% = Calculated relative to the total number of subjects in the relevant population (per by-group stratification level, where relevant)

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories.

Current medical conditions were coded by System Organ Class and Preferred Term using MedDRA version 20.0.

Source Data: Listing 16.2.4.2

Programming Note: Sorted by alphabetical order of system organ class and preferred term.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0
Author: Version Number:

11AUG 2017]

Reference: CS\_WI\_BS005

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

811

**IVACFLU-S** Version 1.0 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018






Reference: CS\_WI\_BS005

#### TABLE AND LISTING MOCK SHELL

Table 14.1.3.1 Summary of Concomitant Medications Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| Reported Term | Vaccine | Placebo | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| | n (%) | n (%) | n (%) |
| Number of Subjects With at Least One Medication | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reported Term 1 Reported Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, % = Calculated relative to the total number of subjects in the relevant population

Subjects with multiple usage of the same medication within the same reported term were counted only once.

Concomitant medication: Defined as medication started on or after the day of vaccination or were ongoing on the date of vaccination or ended on or after the vaccination

Source Data: Listing 16.2.4.3

Programming Note: Sorted by alphabetical order of Reported term.

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document:

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 812 Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

Table 14.2.1.1 Seroconversion and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by Age group Per-protocol population

| Titers | Criteria | Day | Vaccine<br>(N=xx) | Placebo<br>(N=xx) |
|--------|----------------|--------|-------------------|-------------------|
| A/H1N1 | Seroconversion | | | |
| | n | Day 22 | XX | XX |
| | n/N(%) | | XX.X | XX.X |
| | 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |

Sera samples were collected in phase 3 study at one site (Ben Luc).

N= Total number of subjects in each agegroup, n= Total number of subjects meeting the event, CI= Confidence Interval

Percentages were based on the total number of subjects in each vaccine group (N).

95% confidence interval for single proportion is calculated using Exact Clopper-Pearson method.

Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:

Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or Pre-vaccination titer ≥1:10 and at least a four-fold

increase in post vaccination measured on Day 22

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups in the same table.

Table 14.2.1.2

Seroconversion and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by Age group Full Analysis population

Same layout as for 14.2.1.3

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:

1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 Protocol No: IVACFLU-S-0203 813 Dated: 12 March 2018





1.0

Reference: CS\_WI\_BS005


#### TABLE AND LISTING MOCK SHELL

Table 14.2.1.3 Seroprotection and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by Age group Per-protocol population

| Titers | Criteria | Day | Vaccine<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| A/H1N1 | Seroprotection n | Day 1 | xx | xx |
| | n/N(%)<br>95% CI | - | xx.x<br>[xx.xx, xx.xx] | xx.x<br>[xx.xx, xx.xx] |
| | | Day 22 | | |
| | | Day 1 to Day 22 | | |
| A/H3N2 | | | | |
| 3 | | | | |

Sera samples were collected in phase 3 study at one site (Ben Luc).

N= Total number of subjects in each agegroup, n= Total number of subjects meeting the event, CI= Confidence Interval

Percentages were based on the total number of subjects in each vaccine group (N).

95% confidence interval for single proportion is calculated using Exact Clopper-Pearson method.

Seroprotection: Hemagglutination Inhibition (HAI) antibody titer ≥ 1:40

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups in the same table.

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:

11AUG 2017] Version Date:

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.






1.0


#### TABLE AND LISTING MOCK SHELL

#### Table 14.2.1.4

Seroprotection and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by Age group Full Analysis population

Same layout as for 14.2.1.3

## Table 14.2.1.5 Geometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by Age group Per-protocol population

| ters | | Day | Vaccine<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| A/H1N1 | GMT | | | |
| | n | Day 1 | XX | xx |
| | Geometric mean titer | | xx.x | xx.x |
| | Geometric Standard Devi | ation | xx.x | xx.x |
| | 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| | | Day 22 | | |

A/H3N2

В

Sera samples were collected in phase 3 study at one site (Ben Luc).

Notes:

N- Total number of subjects in each agegroup; n - Total number of subjects with the titer measurement.

The confidence intervals were constructed using t distribution.

Pre-vaccination (Day 1) value is considered as baseline.

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups in the same table.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Version Number:

Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

815




1.0

11AUG 2017]


#### TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.2.1.6

Geometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by Age group Full Analysis population

Same layout as for 14.2.1.5

Table 14.2.1.7

Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by Age group Per-protocol population

Age Group: <0verall> <18-45> <46-60>

| | Day | Vaccine (N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| GMFR | | | |
| n | Day 22/Day 1 | xx | xx |
| Geometric mean fold ratio | | xx.x | xx.x |
| Geometric Standard Deviation | | XX.X | XX.X |
| 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| | n<br>Geometric mean fold ratio<br>Geometric Standard Deviation | n Day 22/Day 1<br>Geometric mean fold ratio<br>Geometric Standard Deviation | GMFR n Day 22/Day 1 xx Geometric mean fold ratio xx.x Geometric Standard Deviation xx.x |

Sera samples were collected in phase 3 study at one site (Ben Luc).

N- Total number of subjects in each agegroup; n - Total number of subjects with the titer measurements at both Day 1 and Day 22.

The confidence intervals were constructed using paired t-test.

Pre-vaccination (Day 1) value is considered as baseline.

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups in the same table.

Table 14.2.1.8

Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by Age group Full Analysis population

ruit Analysis population

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Version Number:}


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

816

Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

QuintilesIMS

Same layout as for 14.2.1.7

## Table 14.2.1.9 Immune Response Rates and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group -four-fold rise - Per-protocol population

| Titers | Pre-vaccination<br>titer group | Day | | Vaccine<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|---|
| | < <1:10 > < ≥1:10 > | | | | (== ====, |
| A/H1N1 | <1:10 | Four-fold increase | | | |
| | | n | Day 22 | xx | xx |
| | | n/N(%) | | XX.X | xx.x |
| | | 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| A/H1N1 | ≥1:10 | Four-fold increase | | | |
| | | n | Day 22 | XX | XX |
| | | n/N(%) | | xx.x | xx.x |
| | | 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| A/H3N2<br>B | | | | | |

Sera samples were collected in phase 3 study at one site (Ben Luc). N- Total number of subjects in each group; n - Total number of subjects with four-fold increase on Day 22. Percentages were based on the total number of subjects in each vaccine group (N).

95% confidence interval for single proportion is calculated using Exact Clopper-Pearson method.

Pre-vaccination (Day 1) value is considered as baseline.

Source: Listing 16.2.6.1

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Revathi Rayadurgam} \text{Version Number:} \text{Version Date:}

11AUG 2017]

Reference: CS\_WI\_BS005

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




## QuintilesIMS

#### TABLE AND LISTING MOCK SHELL

Programming note: Repeat the shell for all the three age groups and also repeat H3N2 and B for both the pre-vaccination groups i.e., <1:10, >1:10 as presented for H1N1 in the same table.

#### Table 14.2.1.10

Immune Response Rates and 95% Confidence Intervals for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group - four-fold rise - Full Analysis population

Same layout as for 14.2.1.9

#### Table 14.2.1.11

Geometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group - Per-protocol population

Age Group: <0verall> <18-45> <46-60> Titers Pre-vaccination Day Vaccine Placebo titer group (N=xx) (N=xx) < <1:10 > < ≥1:10 > H1N1 GMT <1:10 n Day 1 хx XX Geometric mean titer xx x XX X Geometric Standard xx.x XX.X Deviation 95% CI [xx.xx, xx.xx] [xx.xx, xx.xx] Day 22 H1N1 ≥1:10 GMT Day 1 XX XX XX.X XX.X Geometric mean titer XX.X xx.x Geometric Standard [xx.xx, xx.xx] [xx.xx, xx.xx] Deviation 95% CI Day 22

H3N2

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number: Version Date:

1.0 11AUG 2017]

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.



1.0

11AUG 2017]



## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Sera samples were collected in phase 3 study at one site (Ben Luc).

N- Total number of subjects in each age group; n - Total number of subjects with the titer measurement.

The confidence intervals were constructed using t distribution.

Pre-vaccination (Day 1) value is considered as baseline.

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups and also repeat H3N2 and B for both the pre-vaccination groups i.e., <1:10, >1:10 as presented for H1N1 in the same table.

Table 14.2.1.12

Geometric Mean titer (GMT) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group Full Analysis population

Same layout as for 14.2.1.11

Table 14.2.1.13

Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group Per-protocol population

Age Group: <0verall> <18-45> <46-60>

| Titers | Pre-vaccination<br>titer group<br>< <1:10 > < ≥1:10 > | | Day | Vaccine<br>(N=xx) | Placebo (N=xx) |
|---|---|---|---|---|---|
| H1N1 <1:10 | <1:10 | GMFR | | | |
| | | n | Day 22/Day 1 | xx | xx |
| | | Geometric mean fold ratio | | xx.x | xx.x |
| | | Geometric Standard Deviation | | XX.X | XX.X |
| | | 95% CI | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| H1N1 | ≥1:10 | GMFR | Day 22/Day 1 | xx | xx |
| | | n | | xx.x | xx.x |
| | | Geometric mean fold ratio | | xx.x | xx.x |
| | | Geometric Standard | | [xx.xx, xx.xx] | [xx.xx, xx.xx] |
| | | Deviation | | | |
| | | 95% CI | | | |

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 Protocol No: IVACFLU-S-0203 819 Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

H3N2

Sera samples were collected in phase 3 study at one site (Ben Luc).

N- Total number of subjects in each age group; n - Total number of subjects with the titer measurements at both Day 1 and Day 22.

The confidence intervals were constructed using t distribution.

Pre-vaccination (Day 1) value is considered as baseline.

Source: Listing 16.2.6.1

Programming note: Repeat the shell for all the three age groups and also repeat H3N2 and B for both the pre-vaccination groups i.e., <1:10, >1:10 as presented for H1N1 in the same table.

Table 14.2.1.14

Geometric Mean Fold Rise (GMFR) for the Hemagglutination Inhibition (HAI) Titers by age group and pre-vaccination titer group Full Analysis population

Same layout as for 14.2.1.13

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

1.0 11AUG 2017]

**IVACFLU-S** 


820

Dated: 12 March 2018




## TABLE AND LISTING MOCK SHELL

Q) QuintilesIMS

Figure 14.2.1.1

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group [18-45] - Per-protocol population

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203 Mock Tables V1.0 Author:

1.0 Revathi Rayadurgam Version Number: 11AUG 2017] Version Date:

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

**IVACFLU-S** 

821







## TABLE AND LISTING MOCK SHELL



Programming note: This graph is to be generated for all the three strains, each strain per page, on Day 1 and Day 22 in the same page. i.e., display H1N1 for both Day 1 and Day 22 in the same page. Repeat H3N2 and B as done for H1N1. All these to be generated in the same figure.

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Revathi Rayadurgam} \text{Version Number:} \text{Version Date:}

1.0 11AUG 2017]

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** Version 1.0 822 Dated: 12 March 2018



1.0

11AUG 2017]


## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Figure 14.2.1.2

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group [18-45] - Full analysis population

Same as 14.2.1.1

Figure 14.2.1.3

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group 46-60 - Per-protocol population

Same as 14.2.1.1

Figure 14.2.1.4

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Age group 46-60 - Full analysis population

Same as 14.2.1.1

Figure 14.2.1.5

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Overall - Per-protocol population

Same as 14.2.1.1

Figure 14.2.1.6

Reverse cumulative distribution curve for Hemagglutination Inhibition (HAI titer) - Overall - Full analysis population

Same as 14.2.1.1

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.






TABLE AND LISTING MOCK SHELL

Figure 14.2.1.7
Geometric Mean Titer (GMT) Plot for Hemagglutination Inhibition (HAI titer) at Day 1 and Day 22 by age group - Per-protocol population



Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: Revathi Rayadurgam Version Number: 

11AUG 2017]

Reference: CS\_WI\_BS005

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 Protocol No: IVACFLU-S-0203 824 Dated: 12 March 2018






## TABLE AND LISTING MOCK SHELL

Figure 14.2.1.8 Geometric Mean Titer (GMT) Plot for Hemagglutination Inhibition (HAI titer) at Day 1 and Day 22 by age group - Full analysis population Same as 14.2.1.7

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203 Mock Tables V1.0 Author: Revathi Rayadurgam Version Number:

1.0 11AUG 2017] Version Date:

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.



1.0

11AUG 2017]




**IVACFLU-S** 

TABLE AND LISTING MOCK SHELL

Table 14.3.1.1 Overview of Adverse Events Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | ( | accine<br>N=XX) | | Placebo<br>(N=XX) | | | Total<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| Variable | n (%) | [95% CI]* E | n (%) | [95% CI]* E | p-value | n (%) | [95% CI]* E |
| Solicited AE: 30 minutes | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Local AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Systemic AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Local Severe AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Systemic Severe AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited AE: Day 1 to Day 7 | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Local AEs | | x) [xx.xx, xx.xx] xx | | ) [xx.xx, xx.xx] xx | 0.xxxx | | x) [xx.xx, xx.xx] xx |
| Solicited Systemic AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Local Severe AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx. | x) [xx.xx, xx.xx] xx |
| Solicited Systemic Severe AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | 0.xxxx | xx (xx | x) [xx.xx, xx.xx] xx |
| Unsolicited AEs | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | | xx (xx. | x) [xx.xx, xx.xx] xx |
| Severe | xx (xx. | x) [xx.xx, xx.xx] xx | | ) [xx.xx, xx.xx] xx | | | x) [xx.xx, xx.xx] xx |
| Related | xx (xx. | x) [xx.xx, xx.xx] xx | | ) [xx.xx, xx.xx] xx | | | x) [xx.xx, xx.xx] xx |
| SAEs: At Any Time | vv (vv | x) [xx.xx, xx.xx] xx | v vv (vv v' | ) [xx.xx, xx.xx] xx | | vv /vv | x) [xx.xx, xx.xx] xx |
| Severe | | x) [xx.xx, xx.xx] xx | | ) [xx.xx, xx.xx] xx | | | x) [xx.xx, xx.xx] xx |
| Related | | x) [xx.xx, xx.xx] xx | | ) [xx.xx, xx.xx] xx | | | x) [xx.xx, xx.xx] xx |
| Deaths | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | | xx (xx. | x) [xx.xx, xx.xx] xx |
| Any AE leading to study | | | | | | | |
| withdrawal | xx (xx. | x) [xx.xx, xx.xx] xx | x xx (xx.x) | ) [xx.xx, xx.xx] xx | | xx (xx. | x) [xx.xx, xx.xx] xx |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Version Number:

Version Date: Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** 


Version 1.0 826 Dated: 12 March 2018





#### TABLE AND LISTING MOCK SHELL

QuintilesIMS

Data is based on the combined phases 2 and 3, pooled across study sites.

AE: Adverse Events, SAE: Serious Adverse Events

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population

Any solicited local or systemic reactogenicity that occurs during the 5-day period post-injection is automatically regarded as related.

Solicited AEs captured within 30 minutes and between day 1 to day 7 after administration of treatment were considered.

\*95% confidence interval (CI) for single proportion: Calculated using Clopper-Pearson method for a single binomial proportion.

p-value: Calculated using Fisher's exact test

Source Data: Listing 16.2.7.1, 16.2.7.2, 16.2.7.4, 16.2.7.5

Programming Note: Please note that p-value calculated using Fisher's exact test should be displayed for solicited AEs only.

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document:

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Reference: CS\_WI\_BS005 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited. Protocol No: IVACFLU-S-0203 827 Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

Table 14.3.2.1.1 Incidence of Solicited Local Adverse Events from Day 1 to Day 7 Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | Vaccine<br>(N=XX) | Placebo<br>(N=XX) | Total (N=XX) |
|---|---|---|---|
| | n (%) [95% CI]* E | n (%) [95% CI]* E P-value | n (%) [95% CI]* E |
| <br>Solicited Local Adverse<br>Events | xx (xx.x) [xx.xx, xx.xx] xx | xx (xx.x) [xx.xx, xx.xx] xx 0.xxxx | Xx (xx.x) [xx.xx, xx.xx] xx |
| Subjects with at least one solicited Local AE | xx (xx.x) [xx.xx, xx.xx] xx | xx (xx.x) [xx.xx, xx.xx] xx 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| Redness | xx (xx.x) [xx.xx, xx.xx] xx | xx (xx.x) [xx.xx, xx.xx] xx 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| Swelling | xx (xx.x) [xx.xx, xx.xx] xx | xx (xx.x) [xx.xx, xx.xx] xx 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| | xx (xx.x) [xx.xx, xx.xx] xx | xx (xx.x) [xx.xx, xx.xx] xx 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population

\*95% confidence interval (CI) for single proportion: Calculated using Clopper-Pearson method for a single binomial proportion.

P-value: Calculated using Fisher's exact test or Cochran-Mantel-Haenszel test comparing vaccine groups.

Event will be counted only one time if occurred on consecutive days.

Source Data: Listing 16.2.7.1

Table 14.3.2.1.2

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:


Reference: CS\_WI\_BS005

11AUG 2017]

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S

Protocol No: IVACFLU-S-0203 828 Dated: 12 March 2018






## TABLE AND LISTING MOCK SHELL

Incidence of Solicited Systemic Adverse Events from Day 1 to Day 7 Full Analysis Population

Source Data: Listing 16.2.7.2.

Programming Note: Repeat the template of Table 14.3.2.1.1 with appropriate changes.

Document: \(\text{IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0}\)

Version Date: 11AUG 2017

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Protocol No: IVACFLU-S-0203 829 Dated: 12 March 2018





1.0

11AUG 2017]


### TABLE AND LISTING MOCK SHELL

#### Table 14.3.2.1.3 Incidence of Solicited 30 minutes Local Adverse Event Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | n (%) | Vaccine<br>(N=XX)<br>[95% CI]* E | n (%) | Placebo<br>(N=XX)<br>[95% CI]* E | P-value | Total<br>(N=XX)<br>n (%) [95% CI]* E |
|---|---|---|---|---|---|---|
| 30 Minutes Local<br>Reactogenicity | xx (xx.x | ) [xx.xx, xx.xx] xx | xx (xx.x) | [xx.xx, xx.xx] xx | 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| Subjects with at<br>least<br>one solicited Local<br>AE | xx (xx.x | ) [xx.xx, xx.xx] xx | xx (xx.x) | [xx.xx, xx.xx] xx | 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| Redness | xx (xx.x | ) [xx.xx, xx.xx] xx | xx (xx.x) | [xx.xx, xx.xx] xx | 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| Swelling | xx (xx.x | ) [xx.xx, xx.xx] xx | xx (xx.x) | [xx.xx, xx.xx] xx | 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |
| <br> | xx (xx.x | ) [xx.xx, xx.xx] xx | xx (xx.x) | [xx.xx, xx.xx] xx | 0.xxxx | xx (xx.x) [xx.xx, xx.xx] xx |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population

Solicited local AEs captured within 30 minutes after administration of treatment were considered.

\*95% confidence interval (CI) for single proportion: Calculated using Clopper-Pearson method for a single binomial proportion.

P-value: Calculated using Fisher's exact test or Cochran-Mantel-Haenszel test comparing vaccine groups.

Source Data: Listing 16.2.7.1

Table 14.3.2.1.4 Incidence of Solicited 30 minutes Systemic Adverse Event Full Analysis Population

Source Data: Listing 16.2.7.2.

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:

Version Date: Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




## TABLE AND LISTING MOCK SHELL

Q) QuintilesIMS

Programming Note: Repeat the template of Table 14.3.2.1.3 with appropriate changes.

# Table 14.3.2.1.5 Incidence of Solicited Local Adverse Event by Day Full Analysis Population

| | Day | Vaccine<br>(N=XX)<br>n (%) E | Placebo<br>(N=XX)<br>n (%) E | Total<br>(N=XX)<br>n (%) E |
|---|---|---|---|---|
| Solicited Local Adverse<br>Events | | xx (xx.x) xx | xx (xx.x) xx | Xx (xx.x) xx |
| Subjects with at least one solicited Local AE | Day 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Redness | | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Swelling | | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| <br> | | xx (xx.x) xx | xx (xx.x) xx | xx (xx,x) xx |
| | Day 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| | | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Version Number:


Reference: CS\_WI\_BS005

1.0 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.





1.0

11AUG 2017]


### TABLE AND LISTING MOCK SHELL

QuintilesIMS

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population
Solicited local AEs captured from Day 1 to Day 7 after administration of treatment were considered.

Source Data: Listing 16.2.7.1

Table 14.3.2.1.6
Incidence of Solicited Systemic Adverse Event by Day
Full Analysis Population

Source Data: Listing 16.2.7.2.

Programming Note: Repeat the template of Table 14.3.2.1.5 with appropriate changes.

# Table 14.3.2.1.7 Incidence of Solicited Local Adverse Events Captured within 30 minutes after Vaccination by severity Full Analysis Population

| | | Vaccine<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|
| Solicited Adverse Event | Severity | n (%) E | n (%) E | n (%) E |
| Swelling | None | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| | Mild | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| | Moderate | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| | Severe | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| | Life Threatening | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| Redness | None | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| | Mild | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Version Number:}


Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

\_ \_ \_

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S


832

Dated: 12 March 2018




Reference: CS\_WI\_BS005

## TABLE AND LISTING MOCK SHELL

QuintilesIMS

| Moderate | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
|------------------|--------------|--------------|--------------|
| Severe | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |
| Life Threatening | Xx (xx.x) xx | Xx (xx.x) xx | Xx (xx.x) xx |

...

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level, N= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population

Source Data: Listing 16.2.7.1

Table 14.3.2.1.8

Incidence of Solicited Systemic Adverse Event Captured within 30 minutes after Vaccination by severity
Full Analysis Population

Source Data: Listing 16.2.7.1

Programming Note: Repeat the template of Table 14.3.2.1.7 with corresponding Solicited Systemic events.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Version Number:}

Version Date: 11AUG 2017

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.






Dated: 12 March 2018


Reference: CS\_WI\_BS005

### TABLE AND LISTING MOCK SHELL

#### Table 14.3.2.1.9 Summary of the Size of the Solicited Adverse Event Captured within 30 minutes after Vaccination Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| Solicited Adverse Event | Vaccine<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Swelling (cm) | | | |
| n | XX | xx | xx |
| Mean | xx.x | XX.X | xx.x |
| Median | xx.x | XX.X | xx.x |
| SD | XX.XX | XX.XX | XX.XX |
| Min, Max | xx, xx | xx, xx | xx, xx |

Erythema/Redness (cm) Induration (cm) Temperature (°C)

Data is based on the combined phases 2 and 3, pooled across study sites.

Max: Maximum; Min: Minimum; SD: Standard Deviation

N= Total number of subjects in the relevant population per by-group stratification level.; n= Number of subjects with the event.

Solicited local AEs captured within 30 minutes after administration of treatment were considered.

Source Data: Listing 16.2.7.1

Programming Note: Present temperature also in addition to solicited local adverse events including in the data.

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Version Number:

Revathi Rayadurgam 1.0 11AUG 2017] Version Date:

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.






## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.3.2.2.1

Summary of Solicited Local Adverse Event Captured by Maximum Severity between Day 1 to Day 7 Full Analysis Population

Source Data: Listing 16.2.7.3

Programming Note: Repeat the template of Table 14.3.2.1.7

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Table 14.3.2.2.2

Summary of Solicited Systemic Adverse Event Captured by Maximum severity between Day 1 to Day 7 Full Analysis Population

Source Data: Listing 16.2.7.3

Programming Note: Repeat the template of Table 14.3.2.1.7 with corresponding Solicited Systemic events.

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author:

Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

IVACFLU-S

835








TABLE AND LISTING MOCK SHELL

#### Table 14.3.3.1.1 Summary of Unsolicited Events Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | Vaccine | Placebo | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Unsolicited event | n (%) E | n (%) E | n (%) E |
| Total number of unsolicited AEs | xx | xx | xx |
| Subjects with at least one unsolicited AE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| At least one vaccine related unsolicited AE | xx (xx.x) xx | Xx (xx.x) xx | xx (xx.x) xx |
| At least one serious unsolicited AE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| At least one severe unsolicited AE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| At least one life threatening unsolicited AE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Subjects requiring treatment during the study | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Subjects with unsolicited AEs leading to withdrawal | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Number of subjects died | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

Data is based on the combined phases 2 and 3, pooled across study sites.

AE: Adverse Events

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, E= Number of Adverse Events, % = Calculated relative to the total number of subjects in the relevant population

AEs captured through day 22 were considered.

Any AE or solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Source Data: Listing 16.2.7.4

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: \text{Revathi Rayadurgam} \text{Version Number:} \text{Version Date:}

11AUG 2017]

Reference: CS\_WI\_BS005

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** Version 1.0 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018





1.0

11AUG 2017]


### TABLE AND LISTING MOCK SHELL

Table 14.3.3.1.2 Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term Full Analysis Population

| | Vaccine | Placebo | Total |
|----------------------------------------|-----------|-----------|-----------|
| ystem Organ Class/ | (N=xx) | N=xx) | (N=xx) |
| Preferred term | n (%) | n (%) | n (%) |
| umber of Subjects with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ystem Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ystem Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

AE: Adverse Events; MedDRA: Medical Dictionary for Regulatory Activities;

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, % = Calculated relative to the total number of subjects in the relevant population

Adverse Event terms were coded by System Organ Class and Preferred term using MedDRA version 20.0.

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories.

Any AE or solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Source Data: Listing 16.2.7.4

Programming Note: Sorted by alphabetical order of system organ class and preferred term.

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document: Author: Revathi Rayadurgam Version Number:


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

837

Dated: 12 March 2018



1.0

11AUG 2017]


## TABLE AND LISTING MOCK SHELL

QuintilesIMS

#### Table 14.3.3.1.3 Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term and severity Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| System Organ | | | .ccine<br>N=xx) | | | | lacebo<br>N=xx) | | | | otal<br>(=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class/<br>Preferred<br>Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Life<br>Threatening<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Life<br>Threatening<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Life<br>Threatening<br>n (%) |
| Number of<br>Subjects with<br>at least one<br>AE | xx<br>(xx.x) | xx (xx.x) | xx<br>(xx.x) | xx (xx.x) | xx<br>(xx.x) | xx (xx.x) | xx<br>(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx<br>(xx.x) | Xx(xx.x) |
| System Organ<br>Class 1<br>Preferred<br>Term 1 | xx<br>(xx.x)<br>xx<br>(xx.x) | xx (xx.x)<br>xx (xx.x) | xx<br>(xx.x)<br>xx<br>(xx.x) | xx (xx.x)<br>xx (xx.x) | xx<br>(xx.x)<br>xx<br>(xx.x) | xx (xx.x)<br>xx (xx.x) | (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx<br>(xx.x)<br>xx<br>(xx.x) | xx (xx.x)<br>xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

AE: Adverse Events; MedDRA: Medical Dictionary for Regulatory Activities;

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, % = Calculated relative to the total number of subjects in the relevant population

Adverse Event terms were coded by System Organ Class and Preferred term using MedDRA version 20.0.

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories.

Any AE or solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories and the subjects were counted for the maximum


Source Data: Listing 16.2.7.4

Programming Note: Sorted by alphabetical order of system organ class and preferred term.

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Tables V1.0 Document: Author: Revathi Rayadurgam Version Number:

Reference: CS WI BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


Reference: CS\_WI\_BS005






## TABLE AND LISTING MOCK SHELL

QuintilesIMS

### 

838

Age Group: <0verall> <18-45> <46-60>

| | 7 | Vaccine<br>(N=xx) | | lacebo<br>(N=xx) | Total<br>(N=xx) | |
|---|---|---|---|---|---|---|
| System Organ Class/ | Related | Not Related | Related | Not Related n (%) | Related | Not Related |
| Preferred Term | n (%) | n (%) | n (%) | | n (%) | n (%) |
| Number of Subjects with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

AE: Adverse Events; MedDRA: Medical Dictionary for Regulatory Activities;

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects in each category, % = Calculated relative to the total number of subjects in the relevant population.

Adverse Event terms were coded by System Organ Class and Preferred term using MedDRA version 20.0.

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories.

Any AE or solicited sign or symptom starting after 7 days post-vaccination will be recorded as an Unsolicited AE.

Subjects experiencing multiple events within the same SOC or preferred term were counted only once under those categories and the subjects were counted worst case relationship to study medication.

Source Data: Listing 16.2.7.4

Programming Note: Sorted by alphabetical order of system organ class and preferred term.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Version Number:

Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 Protocol No: IVACFLU-S-0203 839 Dated: 12 March 2018






### TABLE AND LISTING MOCK SHELL

Table 14.3.3.1.5

Summary of Unsolicited Adverse Events Requiring Treatment by System Organ Class and Preferred Term Full Analysis Population

Source Data: Listing 16.2.7.4

Programming Note: Repeat the template of Table 14.3.3.1.2

Table 14.3.4.1.1

Summary of Serious Adverse Events Full Analysis Population

Source Data: Listing 16.2.7.5

Programming Note: Repeat the template of Table 14.3.3.1.1

Table 14.3.4.1.2

Summary of Serious Adverse Events by System Organ Class and Preferred Term Full Analysis Population

Source Data: Listing 16.2.7.5

Programming Note: Repeat the template of Table 14.3.3.1.2

Table 14.3.4.1.3

Summary of Serious Adverse Events by System Organ Class and Preferred Term and Severity Full Analysis Population

Source Data: Listing 16.2.7.5

Programming Note: Repeat the template of Table 14.3.3.1.3

Table 14.3.4.1.4

Summary of Serious Adverse Events by System Organ Class and Preferred Term and Relationship Full Analysis Population

Source Data: Listing 16.2.7.5

Programming Note: Repeat the template of Table 14.3.3.1.4

\\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Document:

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** 

Protocol No: IVACFLU-S-0203 840 Dated: 12 March 2018






TABLE AND LISTING MOCK SHELL

Table 14.3.4.1.5

Summary of Serious Adverse Events Requiring Treatment by System Organ Class and Preferred Term Full Analysis Population

Source Data: Listing 16.2.7.5

Programming Note: Repeat the template of Table 14.3.3.1.2

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Version Date: 11AUG 2017

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

841






## TABLE AND LISTING MOCK SHELL

Q) QuintilesIMS

# Table 14.3.5.1 Deaths Full Analysis Population

| | | | ruii imarysi | D TOPULUCION | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Subject<br>ID/ Site<br>ID/ Age<br>group | Date/Study<br>Day<br>of Death | Days since Vaccination | Primary Cause<br>of Death (eCRF) | Death certificate<br>Obtained | Autopsy<br>Performed<br>(Yes/No) | Report Available (Yes/No) |
| Vaccine | Xxxxx/<br>xxxxx/<br>xxxxx | DDMMMYYYY | XX | xxxxxxxxxxx | Yes | Yes | Yes |

Days: Derived relative to administration date/time of vaccination.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: \Revathi Rayadurgam \Version \Number:

Version Date: 11A

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

1.0 11AUG 2017]

Reference: CS\_WI\_BS005





1.0

Reference: CS\_WI\_BS005


# TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.3.6.1 Summary of Vital Signs Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | | | | | nccine<br>N=xx) | | lacebo<br>N=xx) | Total (N=xx) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessment<br>(Unit) | Visit | Outcome | Statistic | Actual | CFB | Actual | CFB | Actual | CFB | p-value^ |
| Body | | | | | | | | | | |
| Temperature(°C) | Screening | Result | n | XX | | XX | | XX | | |
| | | | Mean | XX.X | | XX.X | | XX.X | | |
| | | | Median | XX.X | | XX.X | | XX.X | | |
| | | | SD | XX.XX | | XX.XX | | XX.XX | | |
| | | | Min, Max | XX, XX | | XX, XX | | XX, XX | | |
| | | | Missing | XX | | XX | | XX | | |
| | Day 8 | Result | n | xx | XX | xx | xx | XX | xx | |
| | | | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxxxx |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| | | | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | |
| | | | missing | XX | XX | XX | XX | XX | XX | |
| | | | p-value* | 0.xxxxx | | 0.xxxxx | | | | |

Data is based on the combined phases 2 and 3, pooled across study sites.

CFB: Change From Baseline; Max: Maximum; Min; Minimum; SD: Standard Deviation

N= Total number of subjects in relevant population per by-group stratification level. n= Number of subjects with an assessment.

Source Data: Listing 16.2.8.2

Programming Note: Summarize for the parameters systolic blood pressure (mmHq), diastolic blood pressure (mmHq) and pulse rate (beats/min).

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:

Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved. The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

<sup>^</sup>P-value was computed using or 2-sample t test comparing vaccine groups.

<sup>\*</sup> P-value was computed using paired t test comparing vaccine groups.






## TABLE AND LISTING MOCK SHELL

QuintilesIMS

# Table 14.3.6.2 Shift from Baseline to Day 8 of Vital Signs by Grade Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | | | | | | Day 8 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Vaccine<br>(N=xx)<br>n (%) | : | | | Placebo<br>(N=xx)<br>n (%) | | | | Total (N=xx) n (%) | | |
| Parameter<br>(Unit) | Baseline | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 |
| Body<br>Temperature<br>(Oral)(°C)* | 1 | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) |
| | 2 | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) | Xx<br>(xx.xx) |
| | 3 | | | | | | | | | | | | |
| | 4 | | | | | | | | | | | | |

Data is based on the combined phases 2 and 3, pooled across study sites.

N= Total number of subjects in the relevant population per by-group stratification level. n= Number of subjects with available response under each group at both visit. % = Calculated relative to the total number of subjects have measurable assessment for analysis in each group at both time points. Grades: 1- Mild; 2 - Moderate; 3 - Severe; 4 - Life-Threatening;

\*Body temperature collected in vital signs.

Source Data: Listing 16.2.8.2

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0
Author: \text{Revathi Rayadurgam} \text{Version Number:}


Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** 

Protocol No: IVACFLU-S-0203 844 Dated: 12 March 2018






## TABLE AND LISTING MOCK SHELL

Programming Note: Summarize for the parameters systolic blood pressure (mmHg), diastolic blood pressure (mmHg) and pulse rate (beats/min).

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0

Author: Revathi Rayadurgam Version Number: 1.0 Version Date: 11AUG 2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

845 Dated: 12 March 2018

xx (xx.x) xx (xx.x)



1.0

11AUG 2017]




xx (xx.x)

## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.3.6.3

Shift from Baseline to Day 8 of Clinically Significant Vital Signs Parameter
Full Analysis Population

| Age Group: <overall></overall> | <18-45> <46-60> | | | D | ay 8 | | |
|---|---|---|---|---|---|---|---|
| | | | Vaccine<br>(N=xx)<br>n (%) | | | Placebo<br>(N=xx)<br>n (%) | |
| Parameter (Unit) | Baseline | Normal | Abnormal, NCS | Abnormal, CS | Normal | Abnormal, NCS | Abnormal, CS |
| Body Temperature (°C) | 1 | | | | | | |
| | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal, NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

xx (xx.x)

Data is based on the combined phases 2 and 3, pooled across study sites.

CS: Clinically Significant; NCS: Not Clinically Significant;

Abnormal, CS

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects with available response under each group at both time point, % = Calculated relative to the total number of subjects have measurable assessment for analysis in each group at both visit Percentages were based on the total number of subjects have measurable assessment for analysis in each group.

Source Data: Listing 16.2.8.2

Programming Note: Add Total Column also i.e., in addition to Vaccine and Placebo.

xx (xx.x)

Summarize for the parameters systolic blood pressure (mmHq), diastolic blood pressure (mmHq) and pulse rate (beats/min).

xx (xx.x)

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Tables\_V1.0
Author: Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.





1.0

11AUG 2017]



## TABLE AND LISTING MOCK SHELL

QuintilesIMS

Table 14.3.7.1 Shift from Baseline to Day 8 by Clinically Significant Abnormal Physical Examination Full Analysis Population

Age Group: <0verall> <18-45> <46-60>

| | | | Day 8 | | |
|---|---|---|---|---|---|
| Area/ System | | Vaccine (N=xx) n (%) | | Placebo<br>(N=xx)<br>n (%) | |
| | Baseline | Abnormal, NCS | Abnormal, CS | Abnormal, NCS | Abnormal, CS |
| XXXXXXXX | | | | | |
| | Abnormal, NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal, CS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Data is based on the combined phases 2 and 3, pooled across study sites.

CS: Clinically Significant; NCS: Not Clinically Significant;

N= Total number of subjects in the relevant population per by-group stratification level, n= Number of subjects with available response under each group at both time points, % = Calculated relative to the total number of subjects have measurable assessment for analysis in each group at both visit Programming Note: Add Total Column also i.e., in addition to Vaccine and Placebo.

Source Data: Listing 16.2.8.3

Document: \\IEEDC-NAS01A\Biosdata\Path\\IVACFLU-S\\IYA06804\Biostatistics \Documentation\SAP\\IVACFLU-S-0203\_Mock\_Tables\_V1.0 Author: Revathi Rayadurgam Version Number:


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.






TABLE AND LISTING MOCK SHELL

ANNOTATED SHELLS

## **IVACFLU-S, Phase 2/3**

A PHASE 2 / 3 DOUBLE BLINDED, RANDOMIZED, PLACEBO-CONTROLLED STUDY IN HEALTHY ADULT VOLUNTEERS IN VIETNAM TO EXAMINE THE SAFETY AND IMMUNOGENICITY OF A SEASONAL TRIVALENT INACTIVATED SPLIT VIRION INFLUENZA VACCINE (IVACFLU-S) PRODUCED BY IVAC

Document: Author: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0 Revathi Rayadurgam Version Number:

ayadurgam Version Numb Version Date:

[11AUG2017]

Reference: CS WI BS005

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


(Q) Quintiles MS

848


Dated: 12 March 2018

Page 2 of 26



TABLE AND LISTING MOCK SHELL

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 11AUG2017) for Protocol IVACFLU-S-0203 (Dated 09FEB2017).

| | Name | Signature | Date |
|---|---|---|---|
| Author: | Revathi Rayadurgam | ( ) TI | 14 Aug 117 |
| Position: | Biostatistician 2 | ma (200 mily) confortes communication (200 mily) | and the many of the second |
| Company: | Quintiles IMS | | Control of the state of the sta |

Upon review of this document, the undersigned approves this version of the Output templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | a freed | 14/AUC/2017 |
| Position: | Manager, Biostatistic | S - | The state of the s |
| Company: | QuintilesIMS | ELECTRONIC CONTROL OF CONTROL | |
| Approved By: | Krista Yuhas | Merch Yeller | u 14/Aug/2017 |
| Position: | Biostatistician, Center | for Vaccine Innovation and Acc | ess (CVIA) |
| Company: | PATH | THE COMMON AND REPORT OF THE PARTY OF THE PA | The state of the s |
| Approved By: | Tushar Tewari | | |
| Position: | Senior Medical Office | r, Clinical and Regulatory Affairs | NET CONTROL OF THE CO |
| Company: | PATH | | |

Document:

\\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0

Author:

Revathi Rayadurgam

Version Number:


[11AUG2017]

1.0

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Dated: 12 March 2018



PROTOCOL IVACFLU-S-0203 Page 2 of 26

## TABLE AND LISTING MOCK SHELL

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 11AUG2017) for Protocol IVACFLU-S-0203 (Dated 09FEB2017).

| | Name | Signature | Date |
|-----------|--------------------|-----------|------|
| Author: | Revathi Rayadurgam | | |
| Position: | Biostatistician 2 | | |
| Company: | Quintiles IMS | | |

Upon review of this document, the undersigned approves this version of the Output templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | | |
| Position: | Manager, Biostatistics | i | |
| Company: | QuintilesIMS | | |
| Approved By: | Krista Yuhas | | |
| Position: | Biostatistician, Center | for Vaccine Innovation and A | Access (CVIA) |
| Company: | PATH | | |
| A | Tushar Tewari | f | |
| Approved By: | Tustiar Tewari | News | 11 AUG 2017 |
| Position: | Senior Medical Officer | , Clinical and Regulatory Affa | irs |
| Company: | PATH | | |

Document: Author: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0

Version Number:


1.0 [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Revathi Rayadurgam

IVACFLU-S

Protocol No: IVACFLU-S-0203 850 Dated: 12 March 2018






TABLE AND LISTING MOCK SHELL

Please note that listing shells for immunogenicity endpoints are only needed for Phase 3 and all the listing shells other than immunogenicity are needed for both Phase 2 and Phase 3.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0

Author: Version Number:


Reference: CS WI BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.







## TABLE AND LISTING MOCK SHELL

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 11AUG2017) for Protocol IVACFLU-S-0203 (Dated 09FEB2017).

| | Name | Signature | Date |
|-----------|--------------------|-----------|------|
| Author: | Revathi Rayadurgam | | |
| Position: | Biostatistician 2 | | |
| Company: | Quintiles IMS | | |

Upon review of this document, the undersigned approves this version of the Output templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Suresh Chenji | | |
| Position: | Manager, Biostatistics | <u>'</u> | <u>'</u> |
| Company: | QuintilesIMS | | |
| Approved By: | Krista Yuhas | | |
| Position: | Biostatistician, Center fo | r Vaccine Innovation and | Access (CVIA) |
| Company: | PATH | | |
| Approved By: | Tushar Tewari | | |
| Position: | Senior Medical Officer, C | linical and Regulatory Af | fairs |
| Company: | PATH | | |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock\_Listings\_V1.0


Template No: CS TP BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Q) QuintilesIMS




## TABLE AND LISTING MOCK SHELL

## **MODIFICATION HISTORY**

| Unique Identifier for | Date of the Document | Author | Significant Changes from |
|---|---|---|---|
| this Version | Version | | Previous Authorized<br>Version |
| | | Revathi Rayadurgam | Not applicable. First version. |

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


852

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


Protocol No: IVACFLU-S-0203 853 Dated: 12 March 2018





1.0

[11AUG2017]


TABLE AND LISTING MOCK SHELL

Table of Contents

| Listing 16.1.1.1 Eligibility Criteria All subjects | 7 |
|---|---|
| Listing 16.2.1.1 Subject Disposition All subjects | 8 |
| Listing 16.2.1.2 Subject Randomization Enrolled Population | 9 |
| Listing 16.2.1.3 Subject Population Enrolled Population | 10 |
| Listing 16.2.2.1 Protocol Deviations Full Analysis Population | 11 |
| Listing 16.2.4.1 Demographics and Baseline Characteristics Enrolled Population | 12 |
| Listing 16.2.4.2 Current Medical Condition Full Analysis Population | 13 |
| Listing 16.2.4.3 Concomitant Medication Full Analysis Population | 14 |
| Listing 16.2.5 Study Medication Full Analysis Population | 15 |
| Listing 16.2.6.1 Immunogenicity Result Per-Protocol Population | 16 |
| Listing 16.2.6.2 Immunogenicity Result- Antigens Per-Protocol Population | 17 |
| Listing 16.2.7.1 Solicited Local Reactogenicity Full Analysis Population | 18 |
| Listing 16.2.7.2 Solicited Systemic Reactogenicity Full Analysis Population | 19 |
| Listing 16.2.7.3 Local and Systemic Solicited Reactogenecity by Maximum Severity between Day 1 to Day 7 Full A | malysis |
| Population | 20 |
| Listing 16.2.7.4 Unsolicited Adverse Events Full Analysis Population | 21 |

Document: Author: Version Number: Revathi Rayadurgam

Reference: CS\_WI\_BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S


Protocol No: IVACFLU-S-0203 854 Dated: 12 March 2018



| | IVAC |
|-----------------|----------------|
| <b>PROTOCOL</b> | IVACFLU-S-0203 |

1.0

[11AUG2017]


## TABLE AND LISTING MOCK SHELL

| Listing 16.2.7.5 Serious Adverse Events Full Analysis Population | 22 |
|---|---|
| Listing 16.2.8.1 Serum Collection Full Analysis Population | 23 |
| Listing 16.2.8.2 Physical Examination - Vital Signs Full Analysis Population | 24 |
| Listing 16.2.8.3 Physical Examination - Abnormal Findings Full Analysis Population | 25 |
| Listing 16.2.8.4 Pregnancy Report Full Analysis Population | 26 |

Document: \IEEDC-NAS01a\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0

Author: Version Number:

Reference: CS WI BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Q) QuintilesIMS

855






1.0

[11AUG2017]


## TABLE AND LISTING MOCK SHELL

Listing 16.1.1.1 Eligibility Criteria All subjects

| Subject ID/ Site<br>ID/ Age Group | Consent Given<br>(Yes/No) | Date of Informed<br>Consent/Study Day | Met Eligibility (Yes/No) | If Not Met, Specification (eCRF) |
|---|---|---|---|---|
| Xxxxx/ xxxx/ xxxx | Yes | DDMMMYYYY | Yes | |
| xxxxx/ xxxx/ xxxx | Yes | DDMMMYYYY | No | Refused to come for screening |
| xxxxx/ xxxx/ xxxx | Yes | DDMMMYYYY | Yes | |
| xxxxx/ xxxx/ xxxx | Yes | DDMMMYYYY | Yes | |

Study day: Derived relative to administration date/time of vaccination.

Programming Note: Sort by Subject ID.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0

Author: Version Number:

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005


Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.


QuintilesIMS




Reference: CS WI BS005

## TABLE AND LISTING MOCK SHELL


Listing 16.2.1.1 Subject Disposition All subjects

| Treatment | Subject ID/ Site<br>ID/ Age Group | Subject Study Status | Completion/<br>Discontinuation Date<br>Study Day | Reason for Discontinuation | Other/AE/SAE/Specification (eCRF) |
|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | Completed | DDMMMYYYY | | |
| Vaccine | xxxxx/ xxxx/ xxxx | Completed | DDMMMYYYY | | |
| Placebo | xxxxx/ xxxx/ xxxx | Completed | DDMMMYYYY | | |
| Placebo | xxxxx/ xxxx/ xxxx | Discontinued | DDMMMYYYY | Other | xxxxxxxxxxx |

AE: Adverse Event. SAE: Serious Adverse Event.

Study day: Derived relative to administration date/time of vaccination.

Programming Note: Sort by Treatment and Subject ID


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.





## TABLE AND LISTING MOCK SHELL

Listing 16.2.1.2
Subject Randomization

| Subject ID/<br>Site ID/ Age<br>Group | Subject Randomized<br>(Yes/No) | Date of<br>Randomization/Study Day | Randomization Number | Treatment Description | Reason If Not Randomized |
|---|---|---|---|---|---|
| xxxxx/ xxxx/<br>xxxx | Yes | DDMMMYYYY/ xx | xxxxx | Vaccine | |
| xxxxx/ xxxx/<br>xxxx | No | | xxxxx | | Lost to follow-up |
| xxxxx/ xxxx/<br>xxxx | Yes | DDMMMYYYY/ xx | xxxxx | Placebo | |
| xxxxx/ xxxx/<br>xxxx | Yes | DDMMMYYYY/ xx | xxxxx | Placebo | |

Enrolled Population

Study day: Derived relative to administration date/time of vaccination.

Programming Note: Sort by Subject ID.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Reference: CS WI BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

858






## TABLE AND LISTING MOCK SHELL


Listing 16.2.1.3 Subject Population Enrolled Population

| Treatment | Subject ID/ Site ID/ Age<br>Group | All Enrolled<br>Population | Full Analysis<br>Population | Per-Protocol Population | Reason for Exclusion from the population |
|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | Yes | Yes | Yes | xxxxxxxxxxxxx |
| Vaccine | xxxxx/ xxxx/ xxxx | Yes | No | No | xxxxxxxxxxxxx |

Programming Note: Sort by Treatment and Subject ID

Document: 

Author: Version Number: 1.0 Revathi Rayadurgam Version Date: [11AUG2017]

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS WI BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




(IVAC)


### TABLE AND LISTING MOCK SHELL

Listing 16.2.2.1 Protocol Deviations Full Analysis Population

Site ID: xxxxxx

| Treatment | Subject ID/ Site ID/<br>Age Group | Category | Severity | Protocol Deviation Term | Deviation Description |
|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | Informed Consent<br>Criteria | Critical | xxxxxxx | xxxxxxx |

Potential Protocol Deviations for the study and categorize according to the pre-defined categories within the Clinical Trial Management System (CTMS).

Programming Note: Sort by Treatment and Subject ID

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS TP BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS WI BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Reference: CS WI BS005



Dated: 12 March 2018




## TABLE AND LISTING MOCK SHELL

#### Listing 16.2.4.1 Demographics and Baseline Characteristics Enrolled Population

860

| Treatment | Subject ID/ Site<br>ID/ Age Group | Date of Birth/<br>Age(Years) | Sex | Ethnicity | Child Bearing<br>Potential [a] | Urine Pregnancy Test<br>Result[a] |
|---|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ | DDMMMYYYY/ xx | Male | Kinh | Yes | Negative |

[a]: Applicable only for female subjects.

Programming Note: Sort by Treatment and Subject ID.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




## TABLE AND LISTING MOCK SHELL

Listing 16.2.4.2 Current Medical Condition Full Analysis Population

| Treatment | Subject ID/ Site ID/ Age<br>Group | System Organ Class/ Preferred<br>Term/Verbatim Term [a] | Condition | Medication Taken for this Current<br>Condition (Yes/No) |
|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | xxxx/ xxxxxx/ xxxxxxx | xxxxx | No |
| Placebo | xxxxx/ xxxx/ xxxx | xxxx/ xxxxxx/ xxxxxxx | xxxx | Yes |

e-CRF: Electronic Case Report Form. MedDRA: Medical Dictionary for Regulatory Activities. [a]: Medical History terms (including other systems): Coded using MedDra version 20.0.

Programming Note: Sort by Treatment, Subject ID and SOC

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS TP BS016 Revision 4

Reference: CS WI BS005 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Version 1.0 Protocol No: IVACFLU-S-0203 862 Dated: 12 March 2018






#### TABLE AND LISTING MOCK SHELL

Listing 16.2.4.3 Concomitant Medication Full Analysis Population

| Treatment | Subject ID/ Site<br>ID/Age Group | Medication<br>Name | Start Date/ Stop<br>Date/Study Day | Ongoing | Dose/Unit/<br>Frequency | Route of<br>Administration | Indication | Specification (eCRF) |
|---|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY/<br>DDMMMYYYY/ xx | No | Xx/xx/xx | Oral | Unsolicited AE | xxxxxx |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY/<br>DDMMMYYYY/ xx | No | Xx/xx/xx | xxxx | xxxxxx | xxxxxx |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY/<br>DDMMMYYYY/ xx | No | Xx/xx/xx | xxxx | xxxxxxx | xxxxxxx |

AE: Adverse Event.

Study day: Derived relative to administration date/time of vaccination.

Concomitant medication: Defined as medication started on or after the day of vaccination or were ongoing on the date of vaccination or ended on or after the vaccination.

Programming Note: Sort by Treatment Subject ID and Start date.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS TP BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS WI BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

QuintilesIMS

**IVACFLU-S** Version 1.0 863 Dated: 12 March 2018




Reference: CS WI BS005



Listing 16.2.5 Study Medication Full Analysis Population

| Actual<br>Treatment | Randomized<br>Treatment | Subject ID/ Site<br>ID/Age Group | Visit | Vaccination Date/Time<br>(HH:MM)/Study Day | Arm of<br>Administration | Treatment Deviation |
|---|---|---|---|---|---|---|
| Vaccine | Vaccine | xxxxx/ xxxx/ xxxx | Day 1 | DDMMMYYYY/HH:MM/ xx | Left | No |
| Vaccine | Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY/HH:MM/ xx | Left | No |
| Vaccine | Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY/HH:MM/ xx | Right | No |

Study day: Derived relative to administration date/time of vaccination. Please ensure that for all shells footnotes are relevant and complete

NOTE: in eCRF is Product Code which means that we will be able to check "actual" treatment. We have the RND number so we can check RND treatment if not as part of DS then at least here we need to show actual and randomized treatment and flag any deviations. Also please ensure this is clarified in the SAP.

Programming Note: Sort by Actual Treatment, Subject ID and Visit.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0

Version Number: 1.0 Author: Revathi Rayadurgam Version Date: [11AUG2017]

Template No: CS TP BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

**IVACFLU-S** 

QuintilesIMS


864





## TABLE AND LISTING MOCK SHELL

Listing 16.2.6.1 Immunogenicity Result Per-Protocol Population

| | Subject ID/ | | | | HAI | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Site ID/Age<br>Group | Visit | Collection<br>Date/Study Day | Antigens | Titer | Fold Increase<br>(Day 22/Day 1) | >=1:40 Titer<br>(Yes/No) | Seroconversion (Yes/No) |
| Vaccine | xxxxx/ xxxx/<br>xxxx | Day 1 | DDMMMYYYY/ xx | H1N1 | xx | xx | Yes | Yes |
| | | Day 22 | | | | | | |
| | xxxxx/ xxxx/<br>xxxx | | | | | | | |
| | xxxxx/ xxxx/<br>xxxx | | | | | | | |

HAI: Hemagglutination Inhibition

Study day: Derived relative to administration date/time of vaccination.

Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:

- Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40 or
- Pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 22

Programming Note: Sort by Treatment, Subject ID and Visit.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS TP BS016 Revision 4

Reference: CS WI BS005 Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S

Q) QuintilesIMS


865





## TABLE AND LISTING MOCK SHELL

#### Listing 16.2.6.2 Immunogenicity Result- Antigens Per-Protocol Population

| | | | | | HAI(Titer) | | |
|---|---|---|---|---|---|---|---|
| Treatment | | H1N1 | | H3N2 | | В | |
| | Subject ID | Day 1 | Day22 | Day1 | Day 22 | Day 1 | Day 22 |
| Vaccine | xxxxx/ xxxx/ xxxx | xxx | xxx | xxx | xxx | xxx | xxx |

HAI: Hemagglutination Inhibition

Programming Note: Sort by Treatment, Subject ID and Visit.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS WI BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




Protocol No: IVACFLU-S-0203 866 Dated: 12 March 2018



TABLE AND LISTING MOCK SHELL

Listing 16.2.7.1 Solicited Local Reactogenicity Full Analysis Population

| Treatment | Subject ID/<br>Site ID/ Age<br>Group | Temperature (°C)/<br>Finding | Grade of<br>Temperature | Time Point | Solicited Local Adverse Events | Result |
|---|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/<br>xxxx | Xx/Normal | | 30 Minute After<br>Vaccination | Redness (cm)/ Grade Swelling (cm)/ Grade Induration (Hardness) (cm)/ Grade Pain Tenderness | Xx/ xx<br>Xx/ xx<br>Xx/ xx<br>Xx<br>Xx |
| | | | | Day 1 | Redness<br>Swelling<br>Hardness<br>Pain<br>Tenderness | Mild<br>None<br>Moderate<br>xx<br>xx |
| | | | | Day 2 | | |

CS: Clinically Significant; NCS: Not Clinically Significant;

Programming Note: Sort by Treatment, Subject ID and Time point.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Reference: CS WI BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S Protocol No: IVACFLU-S-0203

867







## TABLE AND LISTING MOCK SHELL

#### Listing 16.2.7.2 Solicited Systemic Reactogenicity Full Analysis Population

| Treatment | Subject ID/ Site<br>ID/ Age Group | Time Point | Solicited Systemic Adverse Events | Result |
|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | 30 Minute After Vaccination | Fatigue/ Malaise<br>Generalized Muscle Aches<br>Joint Aches | Mild<br>Mild<br>Moderate |
| | | | Chills<br>Nausea<br>Vomiting<br>Headache | Xxxx<br>Xxx<br>Xxx<br>xxxx |
| | | Day 1 | Temperature (°C) Fatigue/ Malaise Generalized Muscle Aches Joint Aches Chills Nausea Vomiting Headache | xxx Mild Mild Moderate Xxxx Xxx Xxx Xxx |
| | | Day 2 | Temperature (°C)<br>Fatigue/ Malaise<br>Generalized Muscle Aches<br> | xxx<br>Mild<br>Mild |

Programming Note: Sort by Treatment, Subject ID and Time point.

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

Protocol No: IVACFLU-S-0203 868 Dated: 12 March 2018






Reference: CS WI BS005

## TABLE AND LISTING MOCK SHELL

#### Listing 16.2.7.3 Local and Systemic Solicited Reactogenecity by Maximum Severity between Day 1 to Day 7 Full Analysis Population

| Treatment | Subject<br>ID/<br>Site<br>ID/ Age<br>Group | Pain | Tenderness | Redness | Swelling | Hardness | Temperature (°C) | Fatigue/<br>Malaise | Muscle<br>Aches | Joint<br>Aches | Chills | Nausea | Vomiting | Headache |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/<br>xxxx/<br>xxxx | Mild | xxxx | xxx | xxxx | xxxx | Grade 0 | Severe | xxx | xxx | xxx | xxx | xxxx | xxxx |

Programming Note: Sort by Treatment and Subject ID.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

QuintilesIMS

869





Reference: CS WI BS005

## TABLE AND LISTING MOCK SHELL

Listing 16.2.7.4 Unsolicited Adverse Events Full Analysis Population

| Treatment | Subject<br>ID/ Site<br>ID/ Age<br>Group | SOC/<br>Preferred<br>Term/<br>Verbatim<br>Term | Start Date/<br>End Date/<br>Study Day | Duration of<br>AE (Days) | Severity/<br>Serious<br>(Yes/No) | Relationship to<br>Study Product | Action Taken/<br>Specification(e-<br>CRF) | Outcome | Treatment Required (Yes/No) |
|---|---|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/<br>xxxx/ | Xxx/ xxxxx/ | DDMMMYYYY/ | xx | Moderate/No | Not Related | None | Resolved | No |

e-CRF: Electronic Case Report Form; MedDRA: Medical Dictionary for Regulatory Activities; SOC: System Organ Class Adverse Event terms were coded by SOC and Preferred Term using MedDRA version xx.x. Study day: Derived relative to administration date/time of vaccination. Duration is calculated based on start date and end date of AE.

Programming Note: Sort by Treatment, Subject ID, SOC and Preferred Term.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

870







Listing 16.2.7.5 Serious Adverse Events Full Analysis Population

| Treatment | Subject ID/<br>Site ID/Age<br>Group | SOC/ Preferred<br>Term/ Verbatim Term | Start Date/ End<br>Date/ Study Day | Duration<br>of AE | Resolved<br>Date | Serious<br>Criteria | Severity | Relationship to<br>Study Product | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/<br>xxxx/ xxxx | Xxx/ xxxxx/ xxxx | DDMMMYYYY/<br>DDMMMYYYY/ xx | xx | DDMMMYYYY | Death/<br>DDMMMYYYY | Moderate | No | Resolved |

SOC: System Organ Class;

Adverse Event terms were coded by SOC and Preferred Term using MedDRA version xx.x. Study day: Derived relative to administration date/time of vaccination.

Duration is calculated based on start date and end date of AE.

Programming Note: Sort by Treatment, Subject ID, SOC and Preferred Term.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203 Mock Listings V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Revision 4 Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




Reference: CS WI BS005

## TABLE AND LISTING MOCK SHELL

Listing 16.2.8.1 Serum Collection Full Analysis Population

| Treatment | Subject ID/ Site ID/Age Group | Visit | Sample Collected | Collection Date and Time/ Study Day |
|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | xxxx | Yes | DDMMMYYYY/HH:MM/ xx |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | Yes | DDMMMYYYY/HH:MM/ xx |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | Yes | DDMMMYYYY/HH;MM/ xx |

Study day: Derived relative to administration date/time of vaccination.

Programming Note: Sort by Treatment and Subject ID.

Document: \IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

872




TABLE AND LISTING MOCK SHELL


Reference: CS WI BS005

#### Listing 16.2.8.2 Physical Examination - Vital Signs Full Analysis Population

| Treatment | Subject ID/<br>Site ID/Age<br>Group | Visit | Assessment Date | Vital Signs | Result | PE Finding/<br>Specify(e-CRF) | Grading Scale<br>[a] |
|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/<br>xxxx | Screening | DDMMMYYYY | Body Temperature (°C) | Xxx* | Normal | |
| Vaccine | xxxxx/ xxxx/<br>xxxx | xxxxx | DDMMMYYYY | Systolic Blood<br>Pressure(mmHg) | Xxx | Abnormal-NCS | |
| Vaccine | xxxxx/ xxxx/<br>xxxx | xxxxx | DDMMMYYYY | Systolic Blood<br>Pressure(mmHg) | Xxx | Abnormal-CS | 3 |
| Vaccine | xxxxx/ xxxx/<br>xxxx | xxxxx | DDMMMYYYY | Pulse Rate (beats/min) | Xxx | Abnormal-CS/<br>xxxxxxxx | |

CS: Clinically Significant; e-CRF: Electronic Case Report Form; PE: Physical Examination; NCS: Not Clinically Significant; [a]: Applicable only for Abnormal-Clinically significant PE findings.

\*denotes the baseline result.

Programming Note: Sort by Treatment, Subject ID and Visit.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.




Reference: CS WI BS005

## TABLE AND LISTING MOCK SHELL

## Listing 16.2.8.3 Physical Examination - Abnormal Findings Full Analysis Population

| Treatment | Subject ID/ Site<br>ID/Age Group | Visit | Assessment Date | Area/System/<br>Specify(e-CRF) | Finding | Description of<br>Finding |
|---|---|---|---|---|---|---|
| Vaccine | xxxxx/ xxxx/ xxxx | Screening | DDMMMYYYY | Xxxxx | Abnormal-NCS | |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY | xxxxx | Abnormal-NCS | |
| Vaccine | xxxxx/ xxxx/ xxxx | xxxxx | DDMMMYYYY | xxxxx | Abnormal-CS | xxxxxxx |

e-CRF: Electronic Case Report Form; CS: Clinically Significant; PE: Physical Examination; NCS: Not Clinically Significant;

Programming Note: Sort by Treatment, Subject ID and Visit.

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S Protocol No: IVACFLU-S-0203

874







## TABLE AND LISTING MOCK SHELL

Listing 16.2.8.4 Pregnancy Report Full Analysis Population

| Treatment | Subject<br>ID/<br>Site<br>ID/Age<br>Group | Test Date | Date of Last<br>Menstrual<br>Period/<br>Estimated Date<br>of Delivery | Pregnancy<br>History | History of Fatal<br>Anomalies/<br>History of<br>Premature<br>Births/ History<br>of Fatal Deaths | History of Still<br>Births/ History<br>of Miscarriage/<br>Other/<br>Specify(e-CRF) | Medication Taken During Time of Contraception or During Pregnancy | Additional<br>Information/<br>Specify(e-CRF) | Subject<br>Willing to<br>Contact After<br>Delivery |
|---|---|---|---|---|---|---|---|---|---|
| Vaccine | xxxxx/<br>xxxx/<br>xxxx | DDMMMYYYY | DDMMMYYYY/<br>DDMMMYYYY | Yes | No/ No/ No | No/ Yes/ No | No | Yes/ xxxxxx | Yes |
| Vaccine | xxxxx/<br>xxxx/<br>xxxx | DDMMMYYYY | DDMMMYYYY/<br>DDMMMYYYY | Yes | Yes/ No/ No | Yes/ No/ No | No | No | Yes |
| Vaccine | xxxxx/<br>xxxx/<br>xxxx | DDMMMYYYY | DDMMMYYYY/<br>DDMMMYYYY | No | | | | No | Yes |

Programming Note: Sort by Treatment and Subject ID.

Document: 


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Reference: CS\_WI\_BS005

Copyright © 2009, 2010, 2012, 2016 Quintiles Transnational Corp. All rights reserved.

IVACFLU-S

Protocol No: IVACFLU-S-0203 875 Dated: 12 March 2018



**IVAC** 


1.0

[11AUG2017]


TABLE AND LISTING MOCK SHELL

Document: \\IEEDC-NAS01A\Biosdata\Path\IVACFLU-S\IYA06804\Biostatistics \Documentation\SAP\IVACFLU-S-0203\_Mock\_Listings\_V1.0
Author: Revathi Rayadurgam Version Number:

Reference: CS\_WI\_BS005


Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

 $\label{thm:copyright} \ @\ 2009,\ 2010,\ 2012,\ 2016\ \ Quintiles\ Transnational\ Corp.\ All\ rights\ reserved.$ 

IVACFLU-S Version 1.0 Protocol No: IVACFLU-S-0203 876 Dated: 12 March 2018

# 16.1.10 Documentation of inter-laboratory standardization methods and quality assurance procedures

## **Certifications of Accreditation**

| Document | <b>Expiration Date</b> |
|---|---|
| Quality report by Vietnam Bureau of Accreditation (English Version) | 14 October 2016 |
| Quality report by Vietnam Bureau of Accreditation (Vietnamese Version) | 14 October 2016 |
| Pasteur Institute of Hochiminh City - Laboratory Respiratory Virus | 24 January 2017 |
| Pasteur Institute of Hochiminh City - Laboratory Respiratory Virus | 17 October 2020 |
| VidMederi Srl - Testing Laboratory | 17 December 2017 |
| VidMederi Srl - Medical Laboratory | 21 May 2019 |
| Criteria for Marked Vital Signs Abnormalities | NA |

Protocol No: IVACFLU-S-0203 877 Dated: 12 March 2018

# MINISTRY OF SCIENCE AND TECHNOLOGY BUREAU OF ACCREDITATION

**SOCIALIST REPUBLIC OF VIETNAM Independence - Freedom - Happiness** 

No.: 2271/VPCNCL Regarding the conformity assessment results Hanoi, date 14 month 10 year 2016

# To: LABORATORY OF RESPIRATORY VIRUS DEPARTMENT OF MICROBIOLOGY AND IMMUNOLOGY - PASTEUR INSTITUTE IN HO CHI MINH CITY

Based on the surveillance visit report dated 12 - 13 July 2016, Based on the requests of the Certification Audit Team and the Review Committee dated 22 September 2016.

### DIRECTOR OF BEREAU OF ACCREDITATION INFORMS THAT:

Name of the organization recognized:

## LABORATORY OF RESPIRATORY VIRUS

Of

# DEPARTMENT OF MICROBIOLOGY AND IMMUNOLOGY - PASTEUR INSTITUTE IN HO CHI MINH CITY

Accreditation No. VILAS Med 012 according to the Decision No.: 520.2015 QD/VPCNCL dated 14 December 2015: Found to conform with the requirements for maintaining certification.

Sincerely.

Recipients: DIRECTOR

- As mentioned above;
- Filling: Office;
- Laboratory Records.

Signed and stamped

**VU XUAN THUY** 

881 Protocol No: IVACFLU-S-0203 Dated: 12 March 2018





## **CERTIFICATO DI ACCREDITAMENTO** Accreditation Certificate

Accreditamento nº Accreditation no

1411

Rev. **1** 

Si dichiara che We declare that

VisMederi Srl

Sede/Headquarters:

Strada Petriccio e Belriguardo, 35 - 53100 Siena SI

è conforme ai requisiti della norma

UNI CEI EN ISO/IEC 17025:2005 "Requisiti generali per la competenza dei

Laboratori di prova e taratura"

meets the requirements of the standard EN ISO/IEC 17025:2005 "General Requirements for the Competence of Testing

and Calibration Laboratories" standard

quale

Laboratorio di Prova

**Testing Laboratory** as

L'accreditamento attesta la competenza tecnica del Laboratorio relativamente allo scopo riportato nelle schede allegate al presente certificato. Le schede possono variare nel tempo. I requisiti gestionali della ISO/IEC 17025:2005 (sezione 4) sono scritti in un linguaggio idoneo all'attività dei Laboratori di Prova, sono conformi ai principi della ISO 9001:2008 ed allineati con i suoi requisiti applicabili. Il presente certificato non è da ritenersi valido se non accompagnato dalle schede allegate e può essere sospeso o revocato in qualsiasi momento nel caso di inadempienza accertata da parte di ACCREDIA. La vigenza dell'accreditamento può essere verificata sul sito WEB (www.accredia.it) o richiesta direttamente ai singoli Dipartimenti .

The accreditation certifies the technical competence of the laboratory limited to the scope detailed in the attached Enclosure. The scope may vary in the time. The management system requirements in ISO/IEC 17025:2005 (Section 4) are written in a language relevant to Testing Laboratories operations and meet the principles of ISO 9001:2008 and are aligned with its pertinent requirements. The present certificate is valid only if associated to the annexed schedule, and can be suspended or

withdrawn at any time in the event of non fulfilment as ascertained by ACCREDIA.

The in force status of the accreditation may be checked in the WEB site (www.accredia.it) or on direct

request to appointed Department.

Data di 1ª emissione 1st issue date 2013-12-18

Data di modifica Modification date 2016-06-23

Data di scadenza Expiring date 2017-12-17

Il Direttore Generale The General Director (Dr. Filippo Trifiletti)

Il Direttore di Dipartimento Department Director (Dr.ssa Silvia Tramontin)

II Presidente The President (Ing. Giuseppe Rossi)

**ACCREDIA** 

Pag. 1 di 1


Dated: 12 March 2018





## CERTIFICATO DI ACCREDITAMENTO Accreditation Certificate

Accreditamento n° Accreditation n°

0002

Rev. 1

Si dichiara che We declare that VisMederi Srl Sede/Headquarters:

Via Fiorentina 1 - 53100 Siena SI

è conforme ai requisiti della norma UNI EN ISO 15189:2013 "Laboratori medici - Requisiti riguardanti la qualità e la competenza"

meets the requirements

ISO 15189:2012 "Medical Laboratories - Requirements for Quality and Competence" standard

of the standard

----**,** 

quale

Laboratorio medico

as Medical Laboratory

L'accreditamento attesta la competenza tecnica del Laboratorio relativamente allo scopo riportato nelle schede allegate al presente certificato. Le schede possono variare nel tempo. I requisiti gestionali della ISO 15189:2012 (sezione 4) sono scritti in un linguaggio idoneo all'attività dei Laboratori medici, sono conformi ai principi della ISO 9001:2008 ed allineati con i suoi requisiti applicabili.

Il presente certificato non è da ritenersi valido se non accompagnato dalle schede allegate e può essere sospeso o revocato in qualsiasi momento nel caso di inadempienza accertata da parte di ACCREDIA. La vigenza dell'accreditamento può essere verificata sul sito WEB (www.accredia.it) o richiesta direttamente ai singoli Dipartimenti .

The accreditation certifies the technical competence of the laboratory limited to the scope detailed in the attached Enclosure. The scope may vary in the time. The management system requirements in ISO 15189:2012 (Section 4) are written in a language relevant to Medical Laboratories operations and meet the principles of ISO 9001:2008 and are aligned with its pertinent requirements.

principles of ISO 9001:2008 and are aligned with its pertinent requirements.

The present certificate is valid only if associated to the annexed schedule, and can be suspended or withdrawn at any time in the event of non fulfilment as ascertained by ACCREDIA.

The in force status of the accreditation may be checked in the WEB site (www.accredia.it) or on direct request to appointed Department.

Data di 1ª emissione 1st issue date 2015-05-22

Data di modifica Modification date 2016-02-18 Data di scadenza Expiring date 2019-05-21

Direttore Generale
The General Director
(Dr. Filippo Trifiletti)

Il Direttore di Dipartimento Department Director (Dr.ssa Silvia Tramontin)

Il Presidente The President (Ing. Giuseppe Rossi)

Mod. CA-01 rev. 01

ACCREDIA

Pag. 1 di 1

Protocol No: IVACFLU-S-0203 883 Dated: 12 March 2018

## Criteria for Marked Vital Signs Abnormalities

| Vital sign | Assessment criteria |
|---|---|
| Body | • Normal: 36.4 - 37.2 °C. |
| temperature | • Abnormal - NCS: $37.3 - 37.9^{\circ}$ C; OR < $36.4^{\circ}$ C and there are no clinical |
| (oral) | signs or symptoms which require intervention. |
| | • <b>Abnormal - CS:</b> $\geq 38.0^{\circ}$ C OR $< 36.4^{\circ}$ C and there are clinical signs or |
| | symptoms which need intervention |
| Blood | • Normal: 90 - 120 mmHg systolic OR 60 - 85 mmHg diastolic. |
| pressure | Abnormal - NCS: |
| (mmHg) | Upward trend |
| | - <b>121 - 139</b> mmHg systolic AND/OR |
| | - <b>86 - 89</b> mmHg diastolic |
| | Downward trend |
| | - 85-89 mmHg systolic AND/OR 50 - 59 mmHg diastolic |
| | <ul> <li>For the participants who have grade 1 elevated blood pressure, the Investigator will judge if it is clinically significant or not based on the medical history and physical examination, e.g., history of elevated blood pressure, blood pressure monitoring and treatment, presence of clinical signs or symptoms which need intervention, presence of risk factors (obesity, too much alcohol, tobacco use); the Investigator should also refer to the local guideline for diagnosis and treatment of high blood pressure. If the findings are clinical significant, they should be graded according to the DAIDS Table For Grading the Severity in the protocol and MOP 04.</li> <li>Similarly, if the participants have &lt; 85 mmHg systolic OR &lt; 50mmHg diastolic; the Investigator will judge it is clinically significant when the participants have clinical signs or symptoms which need intervention.</li> </ul> |
| | • For the 2 cases above, the Investigator should record the reason for his |
| | assessment in the subject binders. |
| | <ul> <li>Grade 2 elevated blood pressure will be judged to be clinically<br/>significant.</li> </ul> |
| | • Note: |
| | • For those who have history of elevated blood pressure, they will be judged to be non-clinically significant and enrolled according to the criterium #4 if they are stable for the past 3 months and the medication dose is stable for at least 1 month preceding vaccination. |
| | • For those who have clinically significant abnormalities, the study doctor will consult and refer the participants to the health facilities for diagnosis and treatment. |

Protocol No: IVACFLU-S-0203 884 Dated: 12 March 2018

| Vital sign | Assessment criteria |
|---|---|
| | Life-threatening blood presure is defined to be grade 3 elevated blood pressure along with one of the following symptoms which |
| | require hospitalization indicated, e.g., headache, breathing difficulty, |
| | blurred vision, chest pain. |
| Pulse rate | Normal: 60 - 90 beats/min. |
| | • <b>Abnormal - NCS: 55 - &lt; 60</b> beats/min or <b>91-100</b> beats/min. |
| | <ul> <li>Abnormal - CS: &lt; 55 beats/min, or &gt; 100 beats/min and there are clinical signs or symptoms which need intervention or there are abnormal cardiac findings after examination. For this case, the Investigator should record the reason for his assessment in the subject binder.</li> <li>Note: There is no grading scale for pulse rate.</li> </ul> |

## Protocol No: IVACFLU-S-0203 885 Dated: 12 March 2018

In Progression

16.1.11 Publications based on the study

Protocol No: IVACFLU-S-0203 886 Dated: 12 March 2018

## 16.1.12 Important publications referenced in the report

Available Upon Request.